Supplemental Clinical Study Report: 20130411


# 16.1.1 Protocol and Amendments

Protocol Amendment 3, dated 07 March 2018 was generated and approved. Shortly thereafter, a decision was made to terminate the study program, the amendment was not implemented. The last version of the protocol, under which the study was active, was Amendment 2, dated 2014 March 20.



Supplemental Clinical Study Report: 20130411


Onyx Therapeutics Oprozomib ER Tablets Clinical Study Protocol No. OPZ007 

# **CLINICAL STUDY PROTOCOL**

**Protocol Title:** Phase 1b Multicenter Study of Oprozomib, Pomalidomide,

and Dexamethasone in Primary Refractory or Relapsed

and Refractory Multiple Myeloma Subjects

**Protocol Number:** OPZ007

Name of Investigational

**Product:** Oprozomib ER Tablets

**IND Number:** 117,851

NCT Number: NCT01999335

**Sponsor:** Onyx Therapeutics, **Inc.** 

One Amgen Center Drive

Thousand Oaks, CA 91320, USA

Phone: (805) 447-1000

**Study Medical Monitor:** MD

**Medical Director, Early Development** 

1120 Veterans Blvd

South San Francisco, CA 94080 USA

Phone: Email:

Investigator(s):

MD

Assistant Professor

Department of Lymphoma/Myeloma MD Anderson Cancer Center 1515 Holcombe Blvd., Unit 429

Houston, Texas 77030

Office:

Email:

**Date of Original Protocol:** 15 August 2013

**Date of Amendment 1.0:** 21 March 2014

**Date of Amendment 2.0:** 08 July 2014

Date of Amendment 3.0: 07 March 2018

**Confidentiality Statement:** This material is the property of Onyx Therapeutics (a

wholly owned subsidiary of Onyx Pharmaceuticals, an Amgen subsidiary). The material is highly confidential and is to be used only in connection with matters





Supplemental Clinical Study Report: 20130411


Onyx Therapeutics Clinical Study Protocol No. OPZ007
Oprozomib ER Tablets 

authorized by a senior representative of Onyx

Therapeutics, and no part of it is to be disclosed to a third party without the express prior written permission of Onyx

Therapeutics.

Compliance Statement: This study will be conducted in accordance with

Protocol OPZ007, the International Council for Harmonisation (ICH), Good Clinical Practice (GCP) guidelines, and the applicable country and regional

regulatory requirements.

Approved



Supplemental Clinical Study Report: 20130411


| PROTOCOL ACCEPTANCE PA | AGE |
|---|---|
| Issue/Date: OPZ007 (07 March 2018) | |
| I have read this protocol for Study OPZ007 entitled: | |
| Phase 1b Multicenter Study of Oprozomib, Pomalidomide, an<br>Refractory or Relapsed and Refractory Multiple Myeloma Su | • |
| As Investigator, I understand and agree to conduct this study | as outlined herein. |
| Investigator Name (print) | |
| Investigator Signature | Date |

Signature on this page assures the sponsor that, to the best of the investigator's knowledge, the affiliated Institutional Review Board (IRB)/Independent Ethics Committee (IEC) operates in accordance with the governing regulations, and that the investigator understands, and agrees to abide by, all governing regulatory obligations and the International Council for Harmonisation (ICH) Guideline for Good Clinical Practice (GCP) while conducting this clinical investigation. Once signed, the original of this form should be detached from the protocol and returned to Onyx Therapeutics or its designee (please retain a copy for your files).

Approved




Clinical Study Protocol No. OPZ007 

# 1 <u>SYNOPSIS</u>

| Name of | |
|---|---|
| sponsor/compan<br>y: | Onyx Therapeutics |
| Name of | Oprozomib |
| product: | • |
| Title of study<br>and protocol<br>number and<br>phase: | Protocol Number: OPZ007 Phase 1b Multicenter Study of Oprozomib, Pomalidomide, and Dexamethasone in Primary Refractory or Relapsed and Refractory Multiple Myeloma Subjects |
| Study objective( | Primary Objectives |
| s): | <ul> <li>To determine the maximum tolerated dose (MTD) and identify the recommended Phase 3 dose (RP3D) and schedule of oprozomib in combination with pomalidomide and dexamethasone (OPomd) in subjects with primary refractory or relapsed and refractory multiple myeloma</li> <li>To evaluate the safety and tolerability of the OPomd combination in subjects with</li> </ul> |
| | primary refractory or relapsed and refractory multiple myeloma |
| | Secondary Objectives |
| | <ul> <li>To estimate the overall response rate (ORR) of OPomd, defined as the proportion of<br/>subjects with an overall response of stringent complete response (scR), complete<br/>response (CR), very good partial response (VGPR), or partial response (PR) as<br/>determined by investigator according to the International Myeloma Working<br/>Group - Uniform Response Criteria (IMWG-URC)</li> </ul> |
| | <ul> <li>To estimate the clinical benefit rate (CBR) of OPomd, defined as the proportion of subjects with an overall response of minimal response (MR) or better as determined by investigator according to the IMWG-URC and modified European Group for Blood and Marrow Transplantation (EBMT) criteria</li> </ul> |
| | To characterize the pharmacokinetics (PK) of oprozomib in the OPomd regimen |
| | Exploratory Objectives |
| | <ul> <li>To evaluate the pharmacodynamic (PDn) biomarkers that may correlate with<br/>antitumor activity</li> </ul> |
| | <ul> <li>To evaluate genomic biomarkers that may correlate with antitumor activity and<br/>resistance following treatment with proteasome inhibitors</li> </ul> |
| | <ul> <li>To evaluate (in the dose-expansion portion only) the patient-reported outcomes (PRO) using the tools listed below:</li> </ul> |
| | <ul> <li>Bone pain and the impact of bone pain measured with the Brief Pain<br/>Inventory - Short Form (BPI-SF)</li> </ul> |
| | <ul> <li>Health-related quality of life (HRQoL) measured by the global health<br/>status/QoL scale of the European Organization for Research and Treatment of<br/>Cancer (EORTC) Quality of Life Core Module (QLQ-C30) questionnaire</li> </ul> |
| | <ul> <li>Health status assessed by the EQ-5D-5L</li> </ul> |
| | <ul> <li>Disease symptoms as measured by the disease symptoms subscale of the<br/>EORTC Multiple Myeloma Module (QLQ-MY20) questionnaire</li> </ul> |
| | <ul> <li>Neurotoxicity symptoms as measured by the neurotoxicity subscale of the<br/>Functional Assessment of Cancer Therapy / Gynecological Oncology<br/>Group - Neurotoxicity (FACT/GOG-Ntx4 [(Version 4]) questionnaire</li> </ul> |





Date: 30 July 2019


# Study design:

This is a Phase 1b study of oprozomib in combination with pomalidomide and dexamethasone in subjects with primary refractory or relapsed and refractory multiple myeloma. This study includes an open-label, Phase 1b, dose-escalation and dose-expansion portion (equivalent to a small Phase 2), during which the RP3D will be identified. Further evaluation of safety and activity will be assessed during the dose-expansion portion. During this study, subjects will receive Oprozomib extended release (ER) Tablets according to their assigned dose cohort.

This study will include subjects with primary refractory or relapsed and refractory multiple myeloma, ie, those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy (including bortezomib and lenalidomide and/or thalidomide, and in the dose-expansion portion of the study only, been treated with adequate alkylator therapy). Subjects whose last therapy was bortezomib and who were not refractory but developed bortezomib intolerance, as defined by the development of Grade 2 peripheral neuropathy with pain or ≥ Grade 3 peripheral neuropathy after  $\geq 2$  consecutive cycles, are eligible.

Treatment cycles are 28 days in duration. Two (2) oprozomib dosing schedules will be assessed during dose escalation. All study subjects will receive oprozomib once daily either on Days 1–5 and 15–19, referred to hereafter as the 5/14 schedule, or an alternate schedule of once daily on Days 1, 2, 8, 9, 15, 16, 22, and 23, referred to hereafter as the 2/7 schedule. Pomalidomide will be given on Days 1–21 and dexamethasone will be given on Days 1, 2, 8, 9, 15, 16, 22, and 23 of every 28-day cycle.

# 5/14 Schedule Study Dosing Schema



Approved



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019




The safety, MTD, PK/PDn, and RP3D of oprozomib when given in combination with pomalidomide and dexamethasone will be assessed using a standard 3+3 dose-escalation design. For each of the 2 schedules being studied, groups of 3 to 6 subjects will be enrolled into dose-escalation cohorts. As long as fewer than 33% of subjects experience a dose-limiting toxicity (DLT) in a given cohort, escalation will continue by 30-mg increments of oprozomib onto the next designated cohort(s). A minimum of 6 subjects must be treated at the MTD to establish the dose as the MTD. If the starting dose of oprozomib cannot be safely administered with the labeled pomalidomide dose, or at sponsor discretion, then up to 2 possible alternative paths for oprozomib with lower pomalidomide doses will be explored. (See tables below for primary and alternative dose-escalation paths.) Dose escalation will continue until sponsor discretion, the maximum planned dose of pomalidomide is reached, or  $\geq 2$  DLTs occur in a cohort, whichever occurs first. The prior cohort will be expanded to at least 6 subjects if not previously done to establish that dose as the MTD. There may be more than 1 MTD for oprozomib if more than 1 dose level of pomalidomide is studied. The MTD of oprozomib associated with each dose level of pomalidomide assessed will be the dose level where < 2 DLTs in 6 subjects are observed. There is no planned maximum dose of oprozomib to be studied as it is being added to the FDA-approved regimen of pomalidomide/dexamethasone, however, this could be imposed at any time during the course of the study, based on Sponsor discretion. The starting dose of oprozomib for the 5/14 schedule is 150 mg, 3 dose levels below the established 5/14 single-agent MTD of 240 mg. The starting dose of oprozomib for the 2/7 schedule is 210 mg, 3 dose levels below the established 2/7 single-agent MTD of 300 mg. Following

dose escalation, the sponsor has the option of expanding 1 or both schedules in order to

establish the RP3D and schedule.




# Study design (cont'd):

# Dose-Escalation Schema for the 5/14 Oprozomib Dosing Schedule

The starting dose for the 5/14 schedule will be 150 mg of oprozomib and 4 mg of pomalidomide. The 5/14 primary and alternate paths are summarized below; these are examples, and are not inclusive of all possible dose-escalation paths.

# 5/14 Schedule Primary Study Dose-Escalation Paths<sup>a</sup>



5/14 = Dosing on Days 1–5 and 15–19; Dex = dexamethasone; OPZ = oprozomib; Pom = pomalidomide.

Approved



<sup>&</sup>lt;sup>a</sup> There is no predefined maximum dose level of oprozomib being studied.


# Study design (cont'd):

# Primary Dose-Escalation Path for Oprozomib on 5/14 Schedule with Pomalidomide 4mg in Phase 1b

| Cohort | Oprozomib Dose<br>(mg/day) | Pomalidomide Dose<br>(mg/day) |
|---|---|---|
| 1a (initial cohort) | 150 | 4 |
| 2a | 180 | 4 |
| 3a | 210 | 4 |

5/14 = Dosing on Days 1–5 and 15–19; MTD = maximum tolerated dose.

Note: This is an example of the primary dose-escalation cohort. Dose escalation will continue in 30-mg increments of oprozomib at sponsor discretion or until the MTD has been identified.

# Alternative Dose-Escalation Path 1 for Oprozomib on 5/14 Schedule with Pomalidomide in Phase 1b if Cohort 1a Exceeds the MTD, or at Sponsor Discretion

| Cohort | Oprozomib Dose<br>(mg/day) | Pomalidomide Dose<br>(mg/day) |
|--------|----------------------------|-------------------------------|
| 1b | 150 | 3 |
| 2b | 180 | 3 |
| 3b | 210 | 3 |

5/14 = Dosing on Days 1–5 and 15–19; MTD = maximum tolerated dose.

# Alternative Dose-Escalation Path 2 for Oprozomib on 5/14 Schedule with Pomalidomide in Phase 1b if Cohort 1b Exceeds the MTD, or at Sponsor Discretion

| Cohort | Oprozomib Dose<br>(mg/day) | Pomalidomide Dose<br>(mg/day) |
|--------|----------------------------|-------------------------------|
| 1c | 150 | 2 |
| 2c | 180 | 2 |
| 3c | 210 | 2 |

5/14 = Dosing on Days 1–5 and 15–19; MTD = maximum tolerated dose.

Approved



Supplemental Clinical Study Report: 20130411


# Study design (cont'd):

# Dose-Escalation Schema for the 2/7 Oprozomib Dosing Schedule

The starting doses for the 2/7 oprozomib dosing schedule will be 210 mg of oprozomib and 4 mg of pomalidomide. The 2/7 primary and alternate paths are summarized below; these are examples, and are not inclusive of all possible dose-escalation paths.

# 2/7 Schedule Primary Study Dose-Escalation Paths<sup>a</sup>



2/7 = Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23; Dex = dexamethasone; OPZ = oprozomib; Pom = pomalidomide.

# Primary Dose-Escalation Path for Oprozomib on 2/7 Schedule with Pomalidomide 4 mg in Phase 1b

| Cohort | Oprozomib Dose<br>(mg/day) | Pomalidomide Dose<br>(mg/day) |
|---|---|---|
| 101a (initial cohort) | 210 | 4 |
| 201a | 240 | 4 |
| 301a | 270 | 4 |

2/7 = Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23; MTD = maximum tolerated dose.

Note: This is an example of the primary dose-escalation cohort. Dose escalation will continue in 30-mg increments of oprozomib at sponsor discretion or until the MTD has been identified.



<sup>&</sup>lt;sup>a</sup> There is no predefined maximum dose level of oprozomib being studied.

Supplemental Clinical Study Report: 20130411


# Study design (cont'd):

# Alternative Dose-Escalation Path 1 for Oprozomib on 2/7 Schedule with Pomalidomide in Phase 1b if Cohort 101a Exceeds the MTD, or at Sponsor Discretion

| Cohort | Oprozomib Dose<br>(mg/day) | Pomalidomide Dose<br>(mg/day) |
|--------|----------------------------|-------------------------------|
| 101b | 210 | 3 |
| 201b | 240 | 3 |
| 301b | 270 | 3 |

2/7 = Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23; MTD = maximum tolerated dose

# Alternative Dose-Escalation Path 2 for Oprozomib on 2/7 Schedule with Pomalidomide in Phase 1b if Cohort 101b Exceeds the MTD, or at Sponsor Discretion

| Cohort | Oprozomib Dose<br>(mg/day) | Pomalidomide Dose<br>(mg/day) |
|--------|----------------------------|-------------------------------|
| 101c | 210 | 2 |
| 201c | 240 | 2 |
| 301c | 270 | 2 |

2/7 = Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23; MTD = maximum tolerated

At the sponsor's discretion, once the MTD for oprozomib is reached on 1 or both schedules, or if the initial cohort exceeds the MTD, additional dose escalation with oprozomib may continue with lower doses of pomalidomide down to the 2-mg dose level.

The sponsor, with input from the Cohort Safety Review Committee ([CSRC] consisting of investigators, sponsor's medical monitor, and sponsor's drug safety representative), will determine which dose and schedule of oprozomib in combination with Pomd to use for the dose-expansion (ie, the RP3D) portion of the study. The sponsor has the option of expanding 1 or both schedules in order to establish the RP3D and schedule. The RP3D may differ from the MTD, but will not be higher than the MTD, and will be selected based upon the assessment of the safety, tolerability, PK, PDn, preliminary activity, and other variables to be observed across multiple cycles of combination therapy.

# **Dose-Limiting Toxicities**

During this study, assessment of DLTs will occur during the 28-day period of Cycle 1 combination therapy. For the purposes of this study, a DLT is defined as any of the study drug-related events listed below occurring within the 4 weeks after the first dose of combination therapy. Study drug is defined as the combination of oprozomib, pomalidomide, and dexamethasone. Study drug-related is defined as a reasonable likelihood of clinical causality based on time of event, biology, dechallenge improvement, and that the adverse event (AE) was not likely explained by the subject's clinical state, underlying disease, concomitant medication, or study/nonstudy procedure.

- Any toxicity requiring a dose reduction or requiring that a dose of oprozomib or pomalidomide be held in Cycle 1 that does not meet the criteria for DLT will be discussed by the CSRC to determine whether the subject should be considered evaluable for DLT determination. If it is determined that the subject is not evaluable for DLT, the subject will be replaced.
- A delay in ability to receive Day 1 dose of Cycle 2 due to a hematologic or nonhematologic drug-related toxicity persisting beyond 14 days from Cycle 1 Day 28 will be considered a DLT



Supplemental Clinical Study Report: 20130411


# Study design (cont'd):

- For a nonhematologic DLT, any ≥ Grade 3 toxicity will be considered a DLT with exceptions as described below:
  - Grade 3 asymptomatic electrolyte abnormalities will not be considered a DLT
  - Asymptomatic Grade 3 hypophosphatemia lasting less than 24 hours will not be considered a DLT
  - Grade 3 nausea and vomiting will not be considered a DLT unless persisting longer than 3 days despite optimal supportive care, which at a minimum must include a 5-hydroxytryptamine type-3 (5-HT<sub>3</sub>) antagonist and aprepitant
  - Grade 3 diarrhea will not be considered a DLT unless persisting longer than 3 days despite optimal supportive care, which at a minimum must include loperamide (Imodium) and atropine diphenoxylate (Lomotil)
  - Grade 3 fatigue lasting < 14 days is not considered a DLT
  - ≥ Grade 3 hyperglycemia or toxicity attributed to dexamethasone is not considered a DLT
  - ≥ Grade 3 rash attributed specifically to pomalidomide is not considered a DLT
- Hematologic DLTs consist of the following:
  - Grade 4 neutropenia:
    - Absolute neutrophil count (ANC) <  $0.5 \times 10^9$ /L lasting ≥ 7 days despite adequate growth factor support (eg, granulocyte-colony stimulating factor [G-CSF])
    - Febrile neutropenia: Any single temperature ≥ 38.3°C or a sustained temperature of ≥ 38.0°C for over 1 hour with ≥ Grade 3 neutropenia  $(ANC < 1.0 \times 10^9/L)$
  - Thrombocytopenia:
    - Grade 4 lasting  $\geq 7$  days, or
    - Grade 4 lasting < 7 days with Grade 2 clinically significant bleeding or < 10,000 platelets requiring platelet transfusion, or
    - Grade 3 with clinically significant bleeding or requiring platelet transfusion

Note: Grade 4 anemia is not considered a DLT

# **Subject Replacement**

Subjects must meet the following criteria to be considered evaluable for MTD determination during the 4-week DLT evaluation period unless a DLT occurs before the subject receives all planned doses of oprozomib for both the 5/14 and 2/7 dosing schedules:

- A minimum of 17 of 21 planned doses of pomalidomide must be received
- A minimum of 6 of 8 planned doses of dexamethasone must be received
- All planned doses of oprozomib must be received

Subjects not meeting all of the above criteria or assessed as unevaluable by the CSRC will be replaced. Each subject in the cohort under review will be discussed and assessed. Once all data have been presented, the CSRC will decide on the most appropriate course of action regarding dose escalation based on guidance in Section 5.1.



Supplemental Clinical Study Report: 20130411


# Study design (cont'd):

# Dose Expansion

The criteria for selecting the RP3D for 1 or both schedules of oprozomib at the sponsor's discretion will include assessment of the safety, tolerability, and preliminary activity observed across multiple cycles of therapy. In addition, both PK and PDn assessments to demonstrate adequate exposure and proteasome inhibition will be a key factor. Therefore, the RP3D may differ from the MTD. Once the MTD(s) has been determined and the recommended dose for the expansion phase has been selected, a minimum of 20 additional subjects for 1 or both schedules of oprozomib at the sponsor's discretion will be enrolled in the dose-expansion portion **of the study** in order to continue the evaluation of the safety and efficacy of the regimen. The safety of subjects in the Dose Expansion will be monitored on an ongoing basis by the CSRC during regularly scheduled calls. This information will inform the selection of a RP3D and schedule by the sponsor and CSRC.

# Number of investigational sites:

Approximately 35 study sites will participate in **this** study (15 sites for the dose-escalation and 20 additional sites for the dose-expansion portions of the study).

# Planned number of subjects:

A total enrollment of approximately 82 subjects is planned for this study. During the Dose-Escalation portion, approximately 21 subjects will be enrolled for each schedule. The estimate assumes the need to enroll up to 6 subjects in 3 different dose cohorts and the need for replacement of 1 in 6 subjects in order to enable MTD determination. The RP3D may differ from the MTD depending on observed safety and activity data during dose escalation. A minimum of 20 additional subjects are planned for enrollment for each schedule at the sponsor's discretion and treatment at the RP3D during the Dose-Expansion portion of the study.

# Sample size justification:

The estimated sample size for the dose-escalation part of the study is based on standard 3+3 dose-escalation rules, with the expectation that 2–3 dosing cohorts of 3–6 subjects per cohort will be required to establish the MTD.

A minimum of 20 additional subjects will be enrolled for each schedule at the sponsor's discretion during the dose expansion to acquire additional safety and efficacy experience for the RP3D in the population before initiation of the Phase 3 portion of the study. In the dose-expansion portion of the study, if the true  $ORR \ge 40\%$  then the probability of seeing at least 7 responses among the 26 subjects (6 treated at the MTD during escalation + 20 in the expansion) in either schedule is approximately 94%.

# Study populatio

The study population will consist of subjects with primary refractory or relapsed and refractory, multiple myeloma, ie, those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy (including bortezomib and lenalidomide and/or thalidomide, and in the dose-expansion portion of the study only, been treated with adequate alkylator), and who are considered to be appropriate for this clinical study by their treating physicians.

# Test product, dose, and mode of administration:

Oprozomib ER Tablet in strengths of 150, 180, 210, 240, and 270 mg Oral pomalidomide with capsule strengths of 1, 2, 3, and 4 mg Oral dexamethasone with tablet strengths of 4 and 6 mg

# Reference therapy, dose, and mode of administration:

# Active control

Oral pomalidomide with capsule strengths of 1, 2, 3, and 4 mg Oral dexamethasone with tablet strengths of 4 and 6 mg



Supplemental Clinical Study Report: 20130411


| Oprozonno EK | 1 age 13 01 223 |
|---|---|
| Treatment regimen(s): | Oral oprozomib taken Days 1–5 and 15–19 or Days 1, 2, 8, 9, 15, 16, 22, and 23, pomalidomide taken on 21 of 28 days, and oral dexamethasone taken on Days 1, 2, 8, 9, 15, 16, 22, and 23 |
| Inclusion | Disease Related |
| criteria: | 1. Multiple myeloma that is primary refractory, relapsed and refractory, or intolerant after at least 2 lines of standard therapy for multiple myeloma including: |
| | <ul> <li>a. ≥2 consecutive cycles of both bortezomib and lenalidomide or thalidomide<br/>(alone or in combination)</li> </ul> |
| | <ul> <li>In the dose-expansion portion of the study only: In addition to the above,<br/>treatment with adequate alkylator therapy, defined as:</li> </ul> |
| | <ul> <li>High-dose melphalan or other alkylating agent as conditioning for<br/>autologous or allogeneic stem cell transplant (SCT), or</li> </ul> |
| | ii. $\geq 6$ cycles of induction therapy, or |
| | iii. Progressive disease after $\geq 2$ cycles |
| | 2. Measurable disease as indicated by 1 or more of the following: |
| | a. Serum M-protein ≥ 500 mg/dL |
| | b. Urine M-protein ≥ 200 mg/24 h |
| | c. Only for subjects without measurable M-protein by serum protein electrophoresis<br>(SPEP) and urine protein electrophoresis (UPEP), involved free light chain (FLC)<br>concentration ≥ 10 mg/dL provided serum free light chain (SFLC) ratio is<br>abnormal |
| | 3. Disease progression on or within 60 days of completion of the last therapy, or intolerance to bortezomib if received as their last therapy |
| | <ul> <li>a. Patients who received bortezomib as their last therapy who were not refractory<br/>but developed bortezomib intolerance, as defined by the development of<br/>Grade 2 peripheral neuropathy with pain or ≥ Grade 3 peripheral neuropathy<br/>after ≥ 2 consecutive cycles, are eligible</li> </ul> |
| | 4. Prior carfilzomib is allowed if a subject was not removed from carfilzomib therapy due to toxicity, unless approved by the <b>Sponsor's</b> study medical monitor. |
| | Demographic |
| | 5. Males and females ≥ 18 years old |
| | 6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0–2 |
| | Laboratory |
| | 7. Adequate hepatic function, with bilirubin $\leq 1.5$ times the upper limit of normal (ULN) |
| | in the absence of Gilbert's disease or hemolysis, and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) $\leq$ 3 times ULN |
| | <ol> <li>ANC ≥ 1500/mm<sup>3</sup>. Screening ANC should be independent of myeloid growth factor<br/>support for at least 1 week or 2 weeks for pegylated growth factors.</li> </ol> |
| | <ol> <li>Hemoglobin ≥ 8.0 g/dL. Patients may receive red blood cell (RBC) transfusions or<br/>receive erythropoietin or darbepoetin alfa in accordance with institutional guidelines<br/>up to 1 week before Screening.</li> </ol> |
| | 10. Platelet count ≥ 75,000 mm³. Patients should not have received platelet transfusions for at least 1 week before Screening. |
| | 11 TT: 11:01 41 41 44 14:11 4 1 1 0 1 1 |

11. Uric acid, if elevated, must be correct to within laboratory normal range before dosing 12. Calculated or measured creatinine clearance (CrCl) ≥ 30 mL/min calculated using the

formula of Cockcroft and Gault [(140 – age)  $\times$  mass (kg) / (72  $\times$  serum

creatinine mg/dL)]. Multiply result by 0.85 if female.



Supplemental Clinical Study Report: 20130411


# Inclusion criteria (cont'd):

# Ethical/Other

- 13. Patient must sign a written informed consent form in accordance with federal, local, and institutional guidelines
- 14. Female patients of childbearing potential must have a negative pregnancy test (with a sensitivity of at least 50 mIU/mL) within 1 day of the first dose of study drug, and agree to use 2 effective methods of contraception during the study and for 28 days following the last dose of study drug. Postmenopausal females (> 45 years old and without menses for  $\geq 2$  years) and surgically sterilized females are exempt from these requirements.
- 15. Male patients, including those with prior vasectomy, must use an effective barrier method of contraception during the study and for 3 months following the last dose if sexually active with a female of childbearing potential. Additionally, they must agree not to donate sperm while being treated and for up to 3 months after discontinuing treatment.

# **Exclusion** criteria:

## Disease Related

- 1. Systemic chemotherapy with approved or investigational anticancer therapeutics, intended to treat underlying malignancy, within 3 weeks before the first dose of study treatment or 6 weeks for antibody therapy
- 2. Dexamethasone at cumulative doses greater than 160 mg or equivalent within 21 days prior to the first dose of study treatment is not allowed. Use of topical or inhaled steroids is acceptable.
- Radiation therapy within 3 weeks before first dose of study drug. Radioimmunotherapy within 8 weeks before first dose of study drug.
- Plasmapheresis is not permitted at any time during the Screening period or while the subject is receiving study treatment. If a subject has started Screening procedures requiring plasmapheresis, or is anticipated to require plasmapheresis during or after the Screening period, this patient will be considered ineligible and should not be enrolled.
- Autologous SCT within 8 weeks and allogeneic SCT within 16 weeks prior to initiation of study treatment. Patients with prior allogeneic SCT should not have evidence of moderate-to-severe graft-versus-host disease (as defined in Filipovich 2005) and must be approved by the Sponsor's study medical monitor.
- 6. Known hypersensitivity to any immunomodulatory drugs (IMiDs), including rash
- 7. Prior pomalidomide exposure
  - a. For the Dose-Escalation portion of the study: Subjects requiring pomalidomide dose reduction or removal due to toxicity
  - b. For the Dose-Expansion portion of the study: Prior pomalidomide treatment of any duration
- 8. Known hypersensitivity/toxicity or intolerance to dexamethasone
- Prior exposure to oprozomib
- 10. Hypersensitivity, intolerance, or inability to take antithrombotic prophylaxis

# **Concurrent Conditions**

- 11. Major surgery within 3 weeks before first dose of study drug
- 12. Congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months before first dose of study drug
- 13. Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks before first dose of study drug
- 14. History of previous clinically significant gastrointestinal (GI) bleed in the 6 months prior to first dose of study drug



Supplemental Clinical Study Report: 20130411


| Exclusion criteria (cont'd): | <ol> <li>Known or suspected human immunodeficiency virus (HIV) infection or patients who<br/>are HIV seropositive</li> </ol> |
|---|---|
| | 16. Active hepatitis A, B, or C infection |
| | 17. Significant neuropathy (Grade 2 with pain or ≥ Grade 3) at the time of the first dose of study drug |
| | 18. Other malignancy within the past 3 years, except those considered cured by surgical resection; examples include some cases of: |
| | a. Adequately treated basal or squamous cell carcinoma of the skin |
| | b. Thyroid cancer |
| | c. Carcinoma in situ of the cervix or breast |
| | <ul> <li>d. Prostate cancer with Gleason Score of 6 or less with stable prostate-specific<br/>antigen levels</li> </ul> |
| | 19. Plasma cell leukemia |
| | <ol> <li>POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal<br/>protein, and skin changes)</li> </ol> |
| | 21. Known amyloidosis |
| | 22. Female patients who are pregnant or nursing |
| | <ul> <li>23. Uncontrolled diabetes or hypertension</li> <li>24. Inability to swallow medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal condition that could interfere with the oral absorption or tolerance of treatment</li> </ul> |
| | <ol> <li>Any contraindication to oral hydration (e.g., preexisting cardiac impairment or fluid<br/>restriction)</li> </ol> |
| | 26. Any clinically significant psychiatric, social, or medical condition that, in the opinion<br>of the investigator, could increase patient risk, interfere with protocol adherence, or<br>affect a patient's ability to give informed consent |
| Overview of treatment and assessments: | Treatment cycles will last 28 days. Disease response assessments will be performed at the end of every 4-week cycle for the first 18 months on study, and at the end of every other cycle (every 8 weeks) thereafter, beginning with Month 20. |
| | Details are provided in Appendices A1, A2, B1, and B2 (Schedule of Assessments). |
| Criteria for evaluation: | |
| Efficacy<br>variables: | Disease response assessments will be performed at the end of every 4-week cycle for the first 18 months of study treatment, and at the end of every other cycle (every 8 weeks) thereafter, beginning with Month 20, according to the IMWG-URC and modified EBMT criteria. |
| Safety<br>variables: | Safety assessments will include monitoring and assessment of all AEs, clinical laboratory parameters, electrocardiograms (ECGs), and vital signs. Safety assessments will begin after the subject has signed the informed consent form and will continue until 30 days after the End of Study Treatment. The safety and tolerability of the study treatment will be assessed through documentation of AEs graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events ([NCI-CTCAE] Version 4.03). |



Supplemental Clinical Study Report: 20130411


# Other:

## **Pharmacokinetics**

In the Dose-Escalation and Dose-Expansion portions of the study, blood samples will be collected from all subjects for determination of plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose) and 1 predose time point on Day 2 of Cycle 1 for both schedules.

Population PK parameter estimates and variability in these estimates will be determined using a population-based analysis method.

# **Pharmacodynamics**

Blood samples for quantitation of proteasome inhibition by oprozomib will be collected from all subjects in this study.

Analysis of genomic biomarkers that may predict response and resistance following treatment with proteasome inhibitors will be conducted for all subjects receiving oprozomib who consent to optional genomic biomarker analysis. These analyses will be performed on the required bone marrow aspirate obtained at Baseline (within 45 days prior to Cycle 1 Day 1 dosing; a portion of the bone marrow aspirate sample obtained at Baseline will be used; no additional sample is required), as well as a sample of blood and saliva also collected at Baseline. Bone marrow aspirate or biopsy collection does not need to be repeated if previously completed within 45 days prior to Cycle 1 Day 1 dosing. Additional bone marrow samples for biomarkers may be collected at disease progression (End of Study Treatment due to progressive disease [PD]) from all subjects who consent.

# Statistical methods and analyses:

# **Safety Population (All Subjects)**

The safety population includes all subjects receiving any amount of study treatment (oprozomib, pomalidomide, or dexamethasone).

# **Efficacy Population**

For this study, the efficacy population is equivalent to the safety population.

# Endpoints

# **Primary Endpoints**

- **DLTs**
- Adverse events and laboratory abnormalities graded according to NCI-CTCAE,
- Vital signs and clinical laboratory results during and following study drug administration

# Secondary Endpoints

- Overall response, defined as the best response of sCR, CR, VGPR, or PR, as determined by investigator according to the IMWG-URC
- Clinical benefit, defined as the best response of MR or better, as determined by the investigator, according to the IMWG-URC and modified EBMT criteria
- Pharmacokinetic parameters, including maximum plasma concentration (C<sub>max</sub>), time to maximum concentration (T<sub>max</sub>), area under the plasma concentration time curve from time 0 to last time point (AUC $_{0-\tau}$ ), and area under the plasma concentration time curve from time 0 to time infinity (AUC $_{0-\infty}$ ) using noncompartmental methods




# Statistical methods and analyses (cont'd):

# **Exploratory Endpoints**

- Pharmacodynamic biomarkers that may be correlated with antitumor activity
- Genomic biomarkers that may be correlated with antitumor activity and resistance following treatment with proteasome inhibitors
- Change over time in bone pain and the impact of bone pain measured with the BPI-SF (Dose Expansion only)
- Change over time in the global health status/QoL scale of the EORTC QLQ-C30 (Dose Expansion only)
- Change over time in health status assessed by EQ-5D-5L (Dose Expansion only)
- Change over time in the disease symptoms subscale of the EORTC QLQ-MY20 (Dose Expansion only)
- Change over time in neurotoxicity symptoms measured by the FACT/GOG-Ntx4 score (Version 4) (Dose Expansion only)

# **Efficacy Analyses**

Progression-free survival and duration of response will be listed for all subjects by dose level and schedule. Overall response rate and clinical benefit rate will be estimated for all subjects treated at the RP3D along with the associated 95% exact binomial confidence intervals (CIs).

# Safety Analyses

For this study, safety will be assessed through summaries of DLTs, AEs, changes in laboratory test results, ECGs, vital signs, and oprozomib, pomalidomide, and dexamethasone exposure. All AE data collected will be listed by study site, cohort, subject number, and study day.

Approved



Product: Oprozomib Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


# TABLE OF CONTENTS

| | | | | <u>Page</u> |
|---|---|---|---|---|
| CLI | INICAL | STUDY | PROTOCOL | 1 |
| PRO | отосо | L ACCE | PTANCE PAGE | 3 |
| 1 | SYN | OPSIS | | 4 |
| TAl | BLE OF | CONTE | ENTS | 18 |
| 2 | LIST | T OF AB | BREVIATIONS AND DEFINITIONS OF TERMS | 25 |
| 3 | BAC | KGROU | UND INFORMATION | 29 |
| | 3.1 | Introdu | action | 29 |
| | 3.2 | Multip | le Myeloma Background | 30 |
| | 3.3 | Proteas | some Background | 31 |
| | 3.4 | Oprozo | omib Background | 31 |
| | | 3.4.1 | Relevant Nonclinical Background | 32 |
| | | 3.4.2 | Relevant clinical Background | 32 |
| | 3.5 | Dose F | Rationale | 36 |
| | | 3.5.1 | Oprozomib | 36 |
| | | 3.5.2 | Dexamethasone | 37 |
| | | 3.5.3 | Pomalidomide | 38 |
| | 3.6 | Study 1 | Rationale | 40 |
| 4 | STU | DY OBJ | ECTIVES | 43 |
| | 4.1 | Primary Objectives | | 43 |
| | 4.2 | Secondary Objectives | | |
| | 4.3 | 4.3 Exploratory Objectives | | 43 |
| 5 | STU | STUDY DESIGN | | |
| | 5.1 | 5.1 Dose-Escalation and Dose-Expansion Portions of the Study | | 45 |
| | | 5.1.1 | Dose-Escalation Schema for the 5/14 Oprozomib Dosing Schedule | 46 |
| | | 5.1.2 | Dose-Escalation Schema for the 2/7 Oprozomib Dosing Schedule | 48 |
| | | 5.1.3 | Dose-Limiting Toxicities | 51 |
| | | 5.1.4 | Subject Replacement | 51 |
| | | 5.1.5 | Dose Expansion | 51 |





Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

| | zomib ER | | Cimical Su | |
|---|---|---|---|---|
| | 5.2 | Estimat | ed Study Duration and Study Closure | 52 |
| | 5.3 | Minimi | zing Bias | 52 |
| | | 5.3.1 | Blinding | 52 |
| 6 | SUBJ | JECT SE | LECTION | 52 |
| | 6.1 | Inclusio | on Criteria | 52 |
| | 6.2 | Exclusi | on Criteria | 54 |
| 7 | SUBJ | JECT SC | REENING | 56 |
| 8 | SUBJ | JECT EN | ROLLMENT | 56 |
| 9 | STUI | DY DRU | G | 57 |
| | 9.1 | Oprozo | mib | 57 |
| | | 9.1.1 | Oprozomib Physical Description | 57 |
| | | 9.1.2 | Oprozomib Formulation | 57 |
| | | 9.1.3 | Oprozomib Packaging and Labeling | 58 |
| | | 9.1.4 | Oprozomib Storage | 58 |
| | 9.2 | Pomalio | domide | 58 |
| | | 9.2.1 | Pomalidomide Physical Description | 58 |
| | | 9.2.2 | Pomalidomide Packaging and Labeling | 58 |
| | | 9.2.3 | Pomalidomide Storage | 58 |
| | 9.3 | Dexame | ethasone | 59 |
| | | 9.3.1 | Dexamethasone Packaging and Labeling | 59 |
| | | 9.3.2 | Dexamethasone Storage | 59 |
| | 9.4 | Study I | Orug Accountability | 59 |
| 10 | OPR | OZOMII | B TREATMENT ADMINISTRATION | 60 |
| | 10.1 | Oprozo | mib Treatment Administration | 60 |
| | 10.2 | Pomalio | domide Treatment Administration | 60 |
| | 10.3 | Dexame | ethasone Treatment Administration | 61 |
| | 10.4 | Dose M | Iodification Guidelines | 61 |
| | | 10.4.1 | Dose Reductions | 61 |
| | | 10.4.2 | Dose Modification Guidelines | 64 |
| | 10.5 | Definiti | on of Dose-limiting Toxicity | 71 |
| | 10.6 | Concon | nitant Medications | 72 |
| | | 10.6.1 | Required Concomitant Medications | 72 |
| | | 10.6.2 | Optional and Allowed Concomitant Medication | s76 |




**Product: Oprozomib** 

Onyx Therapeutics

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019

| Oproz | omib ER | Tablets P | age 20 of 223 |
|---|---|---|---|
| | | 10.6.3 Excluded Concomitant Medications | 76 |
| 11 | STUI | DY PROCEDURES | 77 |
| | 11.1 | Study-Specific Procedures | 78 |
| | | 11.1.1 Vital Signs | 78 |
| | | 11.1.2 Complete Physical Examination | 78 |
| | | 11.1.3 Electrocardiogram | 78 |
| | 11.2 | Laboratory Evaluations for Safety | 78 |
| | | 11.2.1 Chemistry | 79 |
| | | 11.2.2 Hematology | 79 |
| | | 11.2.3 Coagulation | 80 |
| | | 11.2.4 Pregnancy | 80 |
| | 11.3 | Disease Response Assessments | 80 |
| | 11.4 | Correlative Studies | 82 |
| | | 11.4.1 Pharmacokinetic Measurements | 82 |
| | | 11.4.2 Pharmacodynamic Measurements | 82 |
| | | 11.4.3 Genomic Measurements | 82 |
| | 11.5 | Patient-Reported Outcomes Assessments | 83 |
| 12 | STUI | DY AND STUDY TREATMENT DISCONTINUATION | 84 |
| | 12.1 | Study Treatment Discontinuation | 84 |
| | 12.2 | Study Discontinuation | 85 |
| | 12.3 | Long-term Follow-up | 86 |
| | 12.4 | Study Termination | 86 |
| 13 | ADV | ERSE EVENTS AND SERIOUS ADVERSE EVENTS | 86 |
| | 13.1 | Adverse Event Reporting | 86 |
| | | 13.1.1 Definitions | 86 |
| | 13.2 | Causality | 88 |
| | 13.3 | Adverse Events Reporting Procedures | 89 |
| | | 13.3.1 General | 89 |
| | | 13.3.2 Disease Progression | 90 |
| | 13.4 | Serious Adverse Events Definitions | 90 |
| | 13.5 | Serious Adverse Event Reporting and Documentation Requirement | s91 |
| | 13.6 | Pregnancy Reporting | 92 |
| 14 | STAT | TISTICS | 94 |



| Product: | Oprozomi | t |
|----------|----------|---|
|----------|----------|---|

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

| Oprozor | nib ER T | | Page | 21 of 223 |
|---|---|---|---|---|
| | 14.1 | Study E | ndpoints | 95 |
| | | 14.1.1 | Primary Endpoints | 95 |
| | | 14.1.2 | Secondary Endpoints | 95 |
| | | 14.1.3 | Exploratory Endpoints | 95 |
| | 14.2 | Analysis | s of the Conduct of the Study | 95 |
| | 14.3 | Data Mo | onitoring Committee | 96 |
| | 14.4 | Analysis | s of Treatment Group Comparability | 96 |
| | | 14.4.1 | Treatment Exposure and Medication Compliance | 96 |
| | 14.5 | Statistic | al Methods | 97 |
| | | 14.5.1 | Analysis Populations | 97 |
| | | 14.5.2 | Efficacy Analyses | 97 |
| | | 14.5.3 | Safety Analysis | 98 |
| | | 14.5.4 | Pharmacokinetic Analyses | 98 |
| | 14.6 | Handlin | g of Missing Data | 99 |
| | 14.7 | Determi | nation of Sample Size | 99 |
| 15 | ETHI | CAL AN | D ADMINISTRATIVE CONSIDERATIONS | 101 |
| | 15.1 | Complia | ince Statement | 101 |
| | 15.2 | Institution | onal Review Board or Independent Ethics Committee | 101 |
| | 15.3 | Informe | d Consent and Human Subject Protection | 101 |
| | 15.4 | Direct A | access to Source Data, Source Documents, and Study Records. | 102 |
| | 15.5 | Data Co | llection and Handling | 102 |
| | 15.6 | Confide | ntiality | 103 |
| 16 | REFE | RENCE | S | 105 |
| APPE | | | SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B<br>ATION 5/14 SCHEDULE | 109 |
| APPE | NDIX . | <b>A2</b> | SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B<br>ATION 2/7 SCHEDULE | |
| APPE | NDIX 1 | <b>B</b> 1 | SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B SION 5/14 SCHEDULE | |
| APPE | NDIX 1 | <b>B2</b> | SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B<br>SION 2/7 SCHEDULE | |
| APPE | | | RESPONSE CRITERIA FOR MULTIPLE MYELOMA. | |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

| Onyx Therapeutics Oprozomib ER Tablets | Clinical Study Protocol No. OPZ007<br> |
|---|---|
| TREATMEN | EUROPEAN ORGANIZATION FOR RESEARCH AND T OF CANCER (EORTC) CORE MODULE (QLQ-C30) CMULTIPLE MYELOMA MODULE (QLQ-MY20)132 |
| <b>FUNCTION</b> | NEUROTOXICITY SUBSCALE OF THE OGIC ONCOLOGY GROUP'S AL ASSESSMENT OF CANCER THERAPY -NTX4 [VERSION 4])133 |
| APPENDIX F | EQ-5D-5L (V.2)134 |
| | EASTERN COOPERATIVE ONCOLOGY GROUP<br>FORMANCE SCALE135 |
| APPENDIX H<br>OPROZOMI | DRUG-DRUG INTERACTION POTENTIAL OF B AND POMALIDOMIDE136 |
| | POMALIDOMIDE RISKS OF FETAL EXPOSURE, Y TESTING GUIDELINES, AND ACCEPTABLE BIRTH METHODS138 |
| | POMALIDOMIDE EDUCATION AND COUNSELLING DOCUMENT143 |
| | POMALIDOMIDE INFORMATION SHEET FOR ENROLLED IN CLINICAL RESEARCH STUDIES147 |
| APPENDIX L<br>SCREENING | ACTG BRIEF PERIPHERAL NEUROPATHY G TOOL150 |
| APPENDIX M<br>SHORT FOR | SAMPLE BRIEF PAIN INVENTORY – 2M (BPI-SF)153 |
| | EXAMPLE ELECTRONIC SERIOUS ADVERSE EVENT NCY REPORT FORM155 |
| APPENDIX O<br>NOTIFICAT | EXAMPLE AMGEN PREGNANCY ION WORKSHEET158 |
| APPENDIX P | EXAMPLE AMGEN LACTATION ION WORKSHEET159 |
| | SUMMARY OF CHANGES IN STUDY OPZ007<br>NT 3.0160 |




Onyx Therapeutics

Product: Oprozomib Supplemental Clinical Study Report: 20130411


| Oprozomib | Oprozomib ER Tablets Page 23 of 2 | |
|---|---|---|
| | LIST OF TABLES | |
| Table 1 | Phase 1 Response Rates for Subjects with Multiple Myeloma, by Schedule and Formulation | 33 |
| Table 2 | Phase 1 Response Rates for Subjects with Waldenström macroglobulinemia, by Schedule and Formulation | 34 |
| Table 3 | Primary Dose-Escalation Path for Oprozomib on 5/14 Schedule with Pomalidomide 4 mg in Phase 1b | 47 |
| Table 4 | Alternative Dose-Escalation Path 1 for Oprozomib on 5/14 Schedule with Pomalidomide in Phase 1b if Cohort 1a Exceeds the MTD or at Sponsor Discretion | 48 |
| Table 5 | Alternative Dose-Escalation Path 2 for Oprozomib on 5/14 Schedule with Pomalidomide in Phase 1b if Cohort 1b Exceeds the MTD or at Sponsor Discretion | 48 |
| Table 6 | Primary Dose-Escalation Path for Oprozomib on the 2/7 Schedule with Pomalidomide 4 mg in Phase 1b | 50 |
| Table 7 | Alternative Dose-Escalation Path 1 for Oprozomib on 2/7 Schedule with Pomalidomide in Phase 1b if Cohort 101a Exceeds the MTD or at Sponsor Discretion | 50 |
| Table 8 | Alternative Dose-Escalation Path 2 for Oprozomib on 2/7 Schedule with Pomalidomide in Phase 1b if Cohort 101b Exceeds the MTD or at Sponsor Discretion | 50 |
| Table 9 | Dose Decrements for Oprozomib – 5/14 Schedule | 62 |
| Table 10 | Dose Decrements for Oprozomib – 2/7 Schedule | 62 |
| Table 11 | Dose Decrements for Pomalidomide | 63 |
| Table 12 | Dose Decrements for Dexamethasone | 63 |
| Table 13 | Guidelines for Dose Modification of Oprozomib/Placebo and Pomalidomide for Hematologic Toxicities | 65 |
| Table 14 | Guidelines for Dose Modification of Oprozomib/Placebo and Pomalidomide for Nonhematologic Toxicities | 67 |
| Table 15 | Treatment Guidelines for Dexamethasone-Related Toxicity | 70 |
| Table 16 | Full Chemistry Panel | 79 |
| Table 17 | Toxicity Grading for Adverse Events Not Covered in the NCI-CTCAE (Version 4.03) | 87 |
| Table 20 | Properties of the Dose-Escalation Rules for Different Underlying DLT Rates | .100 |



# Approved

| Product: Oprozomib | |
|--------------------------------------------|---------|
| <b>Supplemental Clinical Study Report:</b> | 2013041 |


| Oprozomib ER Tablets | | |
|---|---|---|
| | LIST OF FIGURES | |
| Figure 1 | Study Dosing Schema for the 5/14 Dosing Schedule. | 46 |
| Figure 2 | 5/14 Schedule Primary Study Dose-Escalation Paths <sup>a</sup> | 47 |
| Figure 3 | Study Dosing Schema for the 2/7 Dosing Schedule | 49 |
| Figure 4 | 2/7 Schedule Primary Study Dose-Escalation Paths <sup>a</sup> . | 49 |




# 2 <u>LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS</u>

| Abbreviation | Definition |
|---|---|
| 5-HT <sub>3</sub> | 5-hydroxytryptamine type-3 |
| ADCC | antibody-dependent cytotoxic T-cell activity |
| ADL | activities of daily living |
| AE | adverse event |
| ALT | alanine aminotransferase |
| ANC | absolute neutrophil count |
| APEX trial | Assessment of Proteasome Inhibition for Extending Remissions Investigators trial |
| ASCO | American Society of Clinical Oncology |
| AST | aspartate aminotransferase |
| AUC | area under the plasma concentration-time curve |
| AUC <sub>0-∞</sub> | area under the plasma concentration time curve from time 0 to time infinity |
| AUC <sub>0-t</sub> | area under the curve at the last measurable time point |
| BPI-SF | Brief Pain Inventory – Short Form |
| С | Cycle |
| CBC | complete blood count |
| CBR | clinical benefit rate |
| СНМР | Committee for Medicinal Products for Human Use |
| CI | confidence interval |
| $C_{max}$ | maximum plasma concentration |
| CPomd | carfilzomib + pomalidomide + dexamethasone |
| CR | complete response |
| CrCl | creatinine clearance |
| CRF | case report form |
| CSRC | Cohort Safety Review Committee |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CT-L | chymotrypsin-like |
| CYP1A2 | cytochrome P450, 1A2 (enzyme) |
| CYP3A | cytochrome P450 3A (enzyme) |
| D | Day |
| D/C | discontinue |
| DLT | dose-limiting toxicity |
| DOR | duration of response |
| DVT | deep vein thrombosis |
| EBMT | European Group for Blood and Marrow Transplantation |
| ECG | electrocardiogram |






| Abbreviation | Definition |
|---|---|
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| ELISA | enzyme-linked immmunosorbent assay |
| EORTC | European Organization for Research and Treatment of Cancer |
| ER | Extended Release |
| EU | European Union |
| EQ-5D-5L | European Quality of Life – Descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) |
| FACT/GOG-Ntx | Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity subscale questionnaire |
| FCBP | females of childbearing potential |
| FDA | Food and Drug Administration |
| FISH | fluorescence in situ hybridization |
| FLC | free light chain |
| GCP | Good Clinical Practice |
| G-CSF | granulocyte-colony stimulating factor |
| GFR | glomerular filtration rate |
| GI | gastrointestinal |
| GLP | Good Laboratory Practices |
| $H_2$ | histamine 2 blocker |
| HIV | human immunodeficiency virus |
| HR | hazard ratio |
| HRQoL | health-related quality of life |
| IB | Investigator's Brochure |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IMiDs | immunomodulatory drug(s) |
| IMWG-URC | International Myeloma Working Group-Uniform Response Criteria |
| IND | Investigational New Drug |
| IP | investigational product |
| IRB | Institutional Review Board |
| IUD | intrauterine device |
| IV | intravenous(ly) |
| Κ/λ | kappa lambda |
| MAD | maximum administered dose |



Date: 30 July 2019


| Abbreviation | Definition |
|---|---|
| MedDRA | Medical Dictionary for Regulatory Activities |
| MR | minimal response |
| MTD | maximum tolerated dose |
| NA | not applicable or not available |
| NCI-CTCAE | National Cancer Institute – Common Terminology Criteria for Adverse Events |
| NF-Kappa B | nuclear factor kappa light chain enhancer of activated B cells |
| NHL | non-Hodgkin lymphoma |
| OPomd | oprozomib + pomalidomide + dexamethasone |
| ORR | overall response rate |
| OS | overall survival |
| PBMC | peripheral blood mononuclear cell |
| PD | progressive disease |
| PDn | pharmacodynamic(s) |
| PFS | progression-free survival |
| P-gp | P-glycoprotein |
| PK | pharmacokinetic(s) |
| PN | peripheral neuropathy |
| POEMS | polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes |
| Pomd | pomalidomide + dexamethasone |
| PR | partial response |
| PRO | patient-reported outcomes |
| QLQ-C30 | Quality of Life Core Module |
| QOL | quality of life |
| QT <sub>c</sub> | corrected QT interval |
| RBC | red blood cell |
| RP3D | recommended Phase 3 dose |
| SAE | serious adverse event |
| SAH | subachnoid hemorrhage |
| SAP | Statistical Analysis Plan |
| sCR | stringent complete response |
| SCT | stem cell transplant |
| SD | stable disease |
| SFLC | serum free light chain |
| SPEP | serum protein electrophoresis |
| TLS | tumor lysis syndrome |
| $T_{\text{max}}$ | time to maximum plasma concentration |
| ULN | upper limit of normal |



Approved

Product: Oprozomib Supplemental Clinical Study Report: 20130411


| Abbreviation | Definition |
|--------------|-------------------------------|
| UPEP | urine protein electrophoresis |
| US | United States |
| VGPR | very good partial response |
| WBC | white blood cell |
| WES | whole exome sequencing |
| WGS | whole genome sequencing |
| WM | Waldenström macroglobulinemia |

Supplemental Clinical Study Report: 20130411


#### 3 **BACKGROUND INFORMATION**

#### INTRODUCTION 3.1

This is a Phase 1b clinical trial of the oral proteasome inhibitor, oprozomib, in subjects with primary refractory or relapsed and refractory multiple myeloma. See Section 5 for a complete description of the study design.

The protocol has been amended with changes to the study design as new data became available from other ongoing oprozomib studies, and based on review of safety results from these studies. A summary of changes for each amendment is included in the appendix of each version of the protocol. The main purposes for each amendment are summarized below.

# **Amendment 1:**

- 1. Added an alternative oprozomib dosing schedule consisting of 2 consecutive days every 7 days (2/7), as preliminary data suggest that a 2/7 schedule has single-agent activity, and may be better tolerated than the existing schedule of 5 consecutive days every 14 days (5/14 schedule).
- 2. Clarified that plasmapheresis is not permitted at any time during the study.
- 3. The starting dose of oprozomib was changed from 210 mg to 150 mg to provide increased margin of safety for subjects participating in this study. This dose (150 mg) is 3 dose levels below the single-agent MTD and was selected due to the overlapping toxicities of oprozomib with pomalidomide.
- 4. Additional dose modification text was added to the dose modification table for nonhematologic toxicities and guidance to investigators to mitigate Grade 4 gastrointestinal (GI) hemorrhage.

# **Amendment 2:**

- 1. To allow subjects with prior carfilzomib exposure to be considered for inclusion in the study, if carfilzomib was not withdrawn due to toxicity.
- 2. To allow subjects with prior pomalidomide exposure to be considered for inclusion in the dose-escalation portion of the study, if pomalidomide was neither dose-reduced nor withdrawn due to toxicity.
- 3. To specify that only subjects who have been treated with adequate alkylator therapy are eligible to be considered for inclusion in the Phase 1b dose-escalation portion and Phase 3 portion of the study.
- 4. Additional safety guidance regarding Grade 3 or 4 GI hemorrhage (see Section 10.4.2.1.2), mandatory proton-pump inhibitors (see Section 10.6.1.5), and the addition of an exclusion criterion for patients with prior clinically significant





Approved

Supplemental Clinical Study Report: 20130411


bleed in the 6 months prior to first dose of study treatment, because of toxicities observed in Study 2011-001.

5. Revisions in synopsis, statistical sections, objectives, and endpoints for accuracy, clarity, and consistency within the protocol.

# **Amendment 3:**

1. Data collection for subjects on active treatment is being pared down due to both the completion of this study's analysis and its abbreviated clinical study report.

#### 3.2 MULTIPLE MYELOMA BACKGROUND

Multiple myeloma, a clonal neoplastic proliferation of plasma cells, is the second most common hematologic malignancy and is responsible for approximately 11,000 deaths per year in the United States (US) and more than 19,000 deaths per year in Europe (American Cancer Society 2005; Boyle 2005). Multiple myeloma is characterized by anemia, bone destruction, monoclonal gammopathy, renal failure, hypercalcemia, and increased susceptibility to infections. The disease is systemic, and chemotherapy or novel agents are indicated for management of symptomatic myeloma. Current treatment options for relapsed/refractory myeloma commonly include single-agent or combination regimens using alkylators such as melphalan (Alkeran) or cyclophosphamide (Cytoxan), bortezomib (Velcade), carfilzomib (Kyprolis), an immunomodulatory drug (IMiD) such as thalidomide (Thalomid), lenalidomide (Revlimid), or pomalidomide (Pomalyst) with and without corticosteroids such as dexamethasone or prednisone, and other agents. Subjects aged 65 to 70 years or younger frequently undergo consolidation therapy with myeloablative chemotherapy or radiation followed by autologous stem cell transplantation (SCT). Carflizomib and pomalidomide received accelerated approval in the US to treat this patient population in 2012 and 2013, respectively. In the European Union (EU), pomalidomide has received a positive opinion from the Committee for Medicinal Products for Human Use (CHMP) for the treatment of patients with advanced myeloma and was approved in August 2013. Although improvements in progression-free survival (PFS) and overall survival (OS) have occurred in the past 5 years, even with the best available approved agents, essentially all patients eventually relapse. Median OS from diagnosis was reported at 3 years for high-risk patients, 4 to 5 years for intermediate-risk patients, and 8 to 10 years for standard-risk patients (Mikhael 2013).




Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


#### 3.3 PROTEASOME BACKGROUND

The proteasome is a multicatalytic proteinase complex that is responsible for degradation of a wide variety of protein substrates within normal and transformed cells. Intracellular proteins targeted for degradation by the proteasome are first ubiquitinated via the ubiquitin conjugation system. Ubiquitinated proteins are cleaved within the proteasome by 1 or more of 3 separate N-terminal threonine protease activities: a chymotrypsin-like (CT-L) activity, a trypsin-like activity, and a caspase-like activity.

Proteasome inhibitors have been shown to have antiproliferative, proapoptotic, antiangiogenic, and antitumor activities across multiple tumor models. Treatment with oprozomib, carfilzomib, or bortezomib results in an increase in the accumulation of proapoptotic proteins, promotion of autophagy, and an increase in the stability of negative regulators of the cell cycle (Boccadoro 2005; Shen 2013; Zang 2012).

#### 3.4 OPROZOMIB BACKGROUND

Oprozomib (formerly ONX 0912) is a tripeptide epoxyketone proteasome inhibitor and structural analogue of carfilzomib (Kyprolis) that primarily targets the CT-L activity of the 20S proteasome. Carfilzomib received accelerated approval in the US for the treatment of patients with multiple myeloma who have received at least 2 prior therapies, including bortezomib and an immunomodulatory agent, and have demonstrated disease progression on or within 60 days of completion of the last therapy (Kyprolis Prescribing Information [Onyx Pharmaceuticals 2012]). Similar to carfilzomib, oprozomib is a potent, selective, and irreversible inhibitor of the CT-L activity of the constitutive proteasome (the form of proteasome found in most cell types) and the immunoproteasome (the form of proteasome found in many hematopoietic cells) (Zhou 2009). In addition, when measured against a broad panel of proteases containing metallo-, aspartyl, cysteine, and serine proteases, oprozomib demonstrated minimal reactivity against nonproteasomal proteases.

Exposure to oprozomib is associated with potent pro-apoptotic activity across a broad panel of tumor-derived cell lines in culture. The antitumor efficacy of oprozomib has been tested in immunocompromised mice implanted with a variety of human tumor cell lines, including models of both solid (colorectal adenocarcinoma, non-small cell lung carcinoma) and





Supplemental Clinical Study Report: 20130411


hematologic (multiple myeloma, non-Hodgkin lymphoma [NHL]) tumors, where its activity was equivalent to carfilzomib (Zhou 2009).

#### 3.4.1 RELEVANT NONCLINICAL BACKGROUND

Oprozomib is orally bioavailable in plasma following solution administration in rodents and dogs. Pharmacodynamic (PDn) determinations demonstrate that proteasome inhibition of > 80% was readily achieved in blood and a wide variety of tissues at tolerated doses in rodents and in whole blood in dogs.

The safety of oprozomib has been established in Good Laboratory Practices (GLP)-compliant toxicity studies in rats and dogs. In 28-day repeat-dose studies, a suspension formulation of oprozomib was administered orally, once daily, for 5 consecutive days with 9 days rest (5 consecutive days bimonthly) for 2 complete 14-day cycles. Oprozomib was administered to rats at doses of 20, 30, and 40 mg/kg (120, 180, and 240 mg/m<sup>2</sup>) and to dogs at 3, 6, and 10 mg/kg (60, 120, and 200 mg/m<sup>2</sup>). A GLP-compliant, single-dose cardiovascular safety pharmacology study in dogs was also performed. The results of these studies show that oprozomib can be safely administered at doses that result in > 80% proteasome inhibition. This level of proteasome inhibition with carfilzomib has been shown to correlate with antitumor activity in subjects with malignancies.

Further information about the preclinical pharmacology and toxicology of oprozomib is presented in the Oprozomib Investigator's Brochure (IB).

#### 3.4.2 RELEVANT CLINICAL BACKGROUND

#### 3.4.2.1 Study 2009-003: Solid Tumors

# **Efficacy**

In Study 2009-003, oprozomib, dosed as powder in capsule, was studied in solid tumor subjects. In the Phase 1 study in refractory solid tumors (n = 44), no subject achieved an objective response. Stable disease (SD) was observed in 6 subjects (30%) in the once daily dosing group and 4 subjects (23.5%) in the split daily dosing group.





Date: 30 July 2019


# Safety

The majority of adverse events (AEs) were Grade 1 and 2, manageable, and there were no apparent cumulative toxicities. The most common AEs were in the GI system organ class. This was consistent with preclinical animal studies with oprozomib. Dose-limiting toxicities for the once daily dose group in Study 2009-003 included Grade 3 dehydration/vomiting and Grade 3 hypophosphatemia in the 180 mg cohort. The maximum tolerated dose (MTD) for the once daily x5 days dose group is 150 mg. Dose-limiting toxicities for the split daily x5 days dosing group in Study 2009-003 included Grade 3 hypophosphatemia at 180 mg and Grade 5 upper GI hemorrhage and Grade 3 hallucinations at 210 mg. The MTD for the split dosing is 180 mg.

#### 3.4.2.2 Study 2011-001: Hematologic Malignancies

# **Efficacy**

As of 21 January 2014, the Phase 1b portion of Study 2011-001 has completed enrollment; 61 response-evaluable subjects with hematologic malignancies have received Oprozomib in Capsules in split dosing, or Oprozomib Tablets with daily dosing, on a 5 consecutive day bimonthly (5/14) schedule or a 2 consecutive day weekly (2/7) schedule in Phase 1. Response rates for subjects with multiple myeloma (n = 43) and subjects with Waldenström macroglobulinemia (WM; n = 18) by schedule and formulation are summarized in Table 1 and Table 2, respectively.

Table 1 Phase 1 Response Rates for Subjects with Multiple Myeloma, by Schedule and Formulation

| Formulation/Schedule (n) | Dose Range (mg) | ORR | Clinical Benefit Rate |
|--------------------------|-----------------|-------|-----------------------|
| PIC 5/14 (10) | 120–210 | 40% | 50% |
| Tablets 5/14 (18) | 150–270 | 27.8% | 38.9% |
| Tablets 2/7 (15) | 150–330 | 20.0% | 46.7% |

ORR = overall response rate; PIC = powder in capsule.

Approved




Table 2 Phase 1 Response Rates for Subjects with Waldenström macroglobulinemia, by Schedule and Formulation

| Formulation/Schedule (n) | Dose Range (mg) | ORR <sup>a</sup> | Major Responseb |
|---|---|---|---|
| Tablets 5/14 (11) | 150–270 | 63.6% | 54.5% |
| Tablets 2/7 (7) | 150-330 | 42.9% | 14.3% |

MR = minimal response; ORR = overall response rate; PR = partial response.

The Phase 2 portion of Study 2011-001 is ongoing. Eight (8) response-evaluable subjects have received Oprozomib Tablets on the 5/14 schedule with once daily dosing in Phase 2; 7 subjects had SD, and 1 subject was off study prior to any disease response assessment.

# Safety

In the Phase 1 portion of the study (as of 21 January, 2014):

- Thirty-two (32) subjects have been enrolled on the 5/14 schedule. Dose-limiting toxicities for the 5/14 schedule observed at the maximum administered dose (MAD) of 270 mg were tumor lysis syndrome (TLS) and Grade 3 vomiting. The MTD was defined as 240 mg, and this was initially selected for the Phase 2 portion for the 5/14 schedule. Due to toxicities, including fatal GI bleeding in 2 subjects, and a high rate of discontinuations observed at this dose level, the dose under evaluation in Phase 2 has been reduced. The Phase 2 portion of the study will reopen using a step-up dose approach starting with 150 mg as the initial dose level, with an increase to 180 mg in Cycle 2.
- Twenty-nine (29) subjects have been enrolled on the 2/7 schedule. Dose-limiting toxicities for the 2/7 schedule observed at the MAD of 330 mg were Grade 3 diarrhea and Grade 4 thrombocytopenia. The MTD was defined as 300 mg. With the opening of Amendment 6, a step-up dosing regimen using 240 mg as the initial dose level, with an increase to 300 mg in Cycle 2, was selected for Phase 2 portion for the 2/7 schedule.

In the Phase 2 portion of the study (as of 21 January 2014):

- A total of 13 subjects have been enrolled in the 5/14 schedule
- No subjects have been enrolled in the 2/7 schedule

Nineteen subjects (19) experienced serious adverse events (SAEs) across both schedules. The 11 treatment-related SAEs comprised 4 GI events (diarrhea, nausea/vomiting,

fatigue/dehydration/nausea, and dehydration), 2 hematological events (anemia and neutropenia), 2 cases of TLS, 1 infection (pneumonia), and 1 general event





<sup>&</sup>lt;sup>a</sup> ORR is defined as > MR.

<sup>&</sup>lt;sup>b</sup> Major response is defined as  $\geq$  PR.

Approved

Supplemental Clinical Study Report: 20130411


(fatigue/dehydration/nausea; events could be counted in more than 1 category). All of these are expected events based on the Oprozomib IB (Version 6). There were 2 cases of renal failure. There were also 2 Grade 5 GI hemorrhages at the 240 mg dose level on the 5/14 schedule.

## 3.4.2.3 Study 2012-001: Oprozomib in Combination with Dexamethasone in Multiple Myeloma

# **Efficacy**

For the 2012-001 Phase 1b/2 study, as of 31 March 2014, 5 response-evaluable relapsed and/or refractory multiple myeloma subjects received Oprozomib Tablets on a 5 consecutive day bimonthly (5/14) schedule with daily dosing; 1 subject had MR and 4 subjects had SD as their best response. As of 31 March 2014, 8 response-evaluable subjects have received Oprozomib Tablets administered orally, once daily, on Days 1, 2, 8, and 9 of a 14-day cycle (2/7) in combination with 20 mg of dexamethasone; 1 subject had a VGPR (unconfirmed), 2 subjects had a partial response ([PR] confirmed or unconfirmed), 1 subject had a MR, and 4 subjects had SD as the best response.

# Safety

The 2012-001 Phase 1b/2 study assessing safety and activity of Oprozomib Tablets in combination with dexamethasone is currently enrolling in the Phase 1b portion of the study.

- As of May 2014, 12 subjects have been enrolled and treated at doses of 180 mg (n = 5) to 210 mg (n = 7) on the 5/14 schedule, and 4 subjects remain on study. Three (3) subjects have experienced DLTs at the 210 mg dose, including 1 subject with a subarachnoid hemorrhage (SAH), 1 subject with Grade 3 transaminitis, and 1 subject with Grade 4 thrombocytopenia. In addition, 1 subject had 3 SAEs (esophagitis, urinary tract infection, and pneumonia). Data suggest that the 180-mg dose level will be the tolerable dose in combination with dexamethasone. This dose level exceeds the starting dose for the combination of oprozomib, pomalidomide, and dexamethasone (OPomd) of 150 mg.
- As of May 2014, 13 subjects have been enrolled and treated at doses of 180 mg (n = 3), 210 mg (n = 3), 240 mg (n = 3), to 270 mg (n = 4) on the 2/7 schedule, and 7 subjects remain on study. One DLT of Grade 4 thrombocytopenia has been observed. Dose escalation is ongoing at the 300-mg dose level, suggesting that doses of 270 mg in combination with dexamethasone are tolerable. Current doses explored in this schedule exceed the starting dose for the combination of OPomd of 210 mg.


**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411


As of 31 March 31 2014, ten (10) subjects experienced serious adverse events (SAEs) across both schedules. The 3 treatment-related SAEs were 1 subject with a SAH, hypertension, and headache, 1 subject with thrombocytopenia, pneumonia, and sepsis, and 1 subject with delirium. Thrombocytopenia and infection were expected events based on the Oprozomib IB (Version 6), but the SAH, hypertension, headache, and delirum were not.

### 3.4.2.4 Study OPZ003: Oprozomib in Combination with Lenalidomide and **Dexamethasone in Multiple Myeloma**

# **Efficacy**

No efficacy data are available at this time.

### Safety

The OPZ003 Phase 1b/2 study, assessing oprozomib in combination with lenalidomide and dexamethasone, is currently enrolling in the Phase 1b portion of the study in newly diagnosed subjects with multiple myeloma. As of 21 January 2014, 3 subjects have been enrolled. Two (2) subjects remain on study. One subject, a wear old a treatment-related SAE of Grade 3 syncope during treatment at the 210 mg dose level. The subject discontinued treatment, and the SAE resolved. Subsequently, the subject experienced a second event of syncope. The dose level in this study has since been de-escalated to 180 mg and syncope has been identified as an event of interest for oprozomib.

### 3.5 DOSE RATIONALE

### 3.5.1 **OPROZOMIB**

Early development of oprozomib focused on the 5 consecutive day bimonthly (either once or twice daily) (5/14) and 2 consecutive days weekly (2/7) schedules, both on 14-day treatment cycles. The MAD for Oprozomib Tablets administered once daily on a 5 consecutive day bimonthly schedule has been reached with a total daily dose of up to 270 mg in subjects with hematologic malignancies, with 1 dose-limiting toxicity (DLT) of TLS and 1 Grade 3 vomiting out of 6 subjects. At the 240-mg dose, 6 subjects were dosed with 1 DLT of TLS, therefore 240 mg was the declared as the MTD. For the 5/14 schedule, the starting dose of 150 mg of oprozomib will be added to the Food and Drug Administration (FDA)-approved






Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


regimen of pomalidomide/dexamethasone, 3 dose levels below the MTD in the single-agent study.

For the 2/7 schedule, the MAD was reached with a total daily dose of 330 mg with 1 DLT of Grade 3 diarrhea and 1 DLT of Grade 4 thrombocytopenia. One DLT of Grade 3 orthostatic hypotension was reported in the 300-mg cohort, therefore 300 mg was declared the MTD. The starting dose for the 2/7 schedule in combination with Pomd will be 210 mg, 3 dose levels below the single agent MTD of 300 mg.

This study will assess both schedules in this study, as oprozomib has demonstrated preliminary activity in subjects with hematologic malignancies on both schedules (Kaufman, 2013).

### 3.5.2 **DEXAMETHASONE**

Dexamethasone will be administered in this study based on data from the SUMMIT trial (Richardson, 2003) and an expanded access trial (Mikhael, 2009), in which dexamethasone was shown to have improved efficacy when administered with proteasome inhibitors. Preclinical studies also suggest the potential therapeutic advantage of dexamethasone combined with carfilzomib (Kuhn, 2007) and bortezomib (Hideshima, 2001) in multiple myeloma.

In a previous study, the addition of steroids to a proteasome inhibitor reduced GI toxicity when compared with single-agent bortezomib (Jagannath, 2006). The addition of low doses of 4 mg of dexamethasone to oprozomib appears to reduce GI toxicity in Study 2011-001. Given that GI AEs have been the most frequent events observed in subjects treated with oprozomib, it is anticipated that Oprozomib ER Tablets will have even less GI toxicity in combination with antimyeloma doses of 20 to 40 mg of dexamethasone once weekly, and therefore may be safely dosed at the same level as or higher than oprozomib monotherapy.

Approved




### 3.5.3 **POMALIDOMIDE**

Pomalidomide (Pomalyst), a thalidomide analogue, is an IMiD that displays similar antiangiogenic activity but far greater antiproliferative and immunomodulatory activity compared with the parent drug (Bartlett, 2007; Payvandi, 2004). Pomalidomide has also been shown to stimulate antibody-dependent cytotoxic T-cell activity (ADCC) (Bartlett, 2007).

Pomalidomide received accelerated approval in the EU in August 2013 and in the US in February 2013. The European Commission has granted approval for pomalidomide in combination with dexamethasone, for the treatment of relapsed and refractory multiple myeloma who received at least two prior therapies and have demonstrated disease progression on the last drug taken and the US FDA granted accelerated approval for patients with multiple myeloma with 2 prior therapies including both bortezomib and lenalidomide and who are refractory to their last therapy or progressed within 60 days. The approved dose of pomalidomide is 4 mg given 21 days of a 28-day cycle until progressive disease (PD).

Approval was based on Study MM002, a randomized Phase 2 comparison of pomalidomide in combination with low-dose therapeutic dexamethasone (POM + LoDex) to pomalidomide alone (Jagannath, 2012). The overall response rate (ORR) was 34%, with a median PFS of 4.6 months and median OS of 16.5 months. Grade 3 or 4 AEs reported in > 5% of subjects were neutropenia (41%), anemia (22%), pneumonia (22%), thrombocytopenia (19%), fatigue (14%), dyspnea (13%), leukopenia (10%), back pain (10%), and urinary tract infection (9%). Grade 3 or 4 neutropenia occurred in 46% of subjects aged ≤ 65 years and in 35% of subjects aged > 65 years. Febrile neutropenia was observed in only 1 subject in each age group (2%). Overall, 78% of subjects who developed Grade 3 or 4 neutropenia were treated with granulocyte-colony stimulating factor (G-CSF) during study treatment. There was no Grade 3 or 4 peripheral neuropathy (PN) reported, although Grade 1 or 2 PN occurred in 7% of subjects treated with POM + LoDex. Deep vein thrombosis (DVT) occurred in 2 subjects (2%). Pomalidomide appears to provide an efficacious option with a manageable toxicity profile for subjects with refractory or relapsed and refractory multiple myeloma.

Approved



Date: 30 July 2019


The MM003 randomized Phase 3 study was designed to assess relapsed and/or refractory subjects with multiple myeloma who had been previously treated with bortezomib and lenalidomide or thalidomide, and progressed on or within 60 days of the last therapy. A regimen of pomalidomide and dexamethasone was compared to high-dose dexamethasone.

Subjects were randomized 2:1 to receive 28-day cycles of pomalidomide 4 mg on Days 1-21 + dexamethasone 40 mg (20 mg for subjects more than 75 years old) weekly or dexamethasone 40 mg (20 mg for subjects more than 75 years old) on Days 1–4, 9–12, and 17–20. Treatment continued until PD or unacceptable toxicity. The primary endpoint was PFS. Secondary endpoints included OS, ORR (≥ PR), and safety. Analyses were based on intent-to-treat. A total of 455 subjects were randomized to pomalidomide + low-dose dexamethasone (n = 302) or high-dose dexamethasone (n = 153). The median number of prior therapies was 5 (range: 1-17). Seventy-two percent (72%) of subjects were refractory to lenalidomide and bortezomib. Median follow-up was 4 months.

Pomalidomide + low-dose dexamethasone significantly extended median PFS (3.6 versus 1.8 months, hazard ratio [HR] = 0.45, p < 0.001) and OS (not reached versus 7.8 months, HR = 0.53, p < 0.001) compared with high-dose dexamethasone. The OS benefit was observed despite 29% of high-dose dexamethasone subjects receiving pomalidomide after PD (Jagannath, 2012). With updated data, the ORR was 21% for pomalidomide + low-dose dexamethasone versus 3% for high-dose dexamethasone (p < 0.001) and 24% versus 3% for subjects randomized  $\geq 6$  months after enrollment (p < 0.001). Median OS was 12.7 months for pomalidomide + low-dose dexamethasone and 8.1 months for high-dose dexamethasone; HR = 0.74 (p = 0.28). The most frequent Grade 3/4 AEs for pomalidomide + low-dose dexamethasone versus high-dose dexamethasone were neutropenia (42% versus 15%), anemia (27% versus 29%), and infection (24% versus 23%). Discontinuation due to AEs was infrequent (7% versus 6%) (San Miguel, 2013).

Lacy et al. (2011) conducted a study to assess efficacy and toxicity of 2- and 4-mg doses of pomalidomide. Pomalidomide was given orally on Days 1–28 of a 28-day cycle at a dose of 2 or 4 mg, with dexamethasone administered at 40 mg weekly. Thirty-five (35) subjects were enrolled in each cohort. Based on confirmed responses, the ORR was 49% in the 2-mg cohort and 43% in the 4-mg cohort. Overall survival at 6 months was 78% and 67% in




the 2- and 4-mg cohorts, respectively. Myelosuppression was the most common toxicity. Grade 3 or 4 hematologic toxicity, regardless of attribution, occurred in 83% (2-mg cohort) and 80% (4-mg cohort) of subjects, and was considered to be at least possibly related to the regimen in 71% (2-mg cohort) and 74% (4-mg cohort). Grade 3 or 4 neutropenia (regardless of attribution) was seen in 51% (2-mg cohort) and 66% (4-mg cohort) of subjects. Grade 3 or 4 nonhematologic toxicity, regardless of attribution, occurred in 69% (2-mg cohort) and 54% (4-mg cohort) of subjects, and was considered to be at least possibly related to the regimen in 26% (2-mg cohort) and 26% (4-mg cohort). These data obtained from nonrandomized subjects suggest no advantage for 4 mg over the 2 mg daily dose. This is the basis for the dose de-escalation to 2 mg of pomalidomide in the event the initial dose level of 4 mg or the first dose de-escalation to 3 mg is not tolerated (Lacy, 2011).

#### 3.6 STUDY RATIONALE

The clinical activity of proteasome inhibition in hematologic malignancies has been demonstrated in multiple myeloma in the clinical setting. Specifically, bortezomib, which is a covalent, slowly reversible proteasome inhibitor that primarily targets the CT-L activity of the proteasome, was the first approved proteasome inhibitor. Because of the benefit of bortezomib observed in subjects with relapsed or refractory myeloma in Phase 1 and 2 trials, the drug received accelerated approval by the US FDA, and was made available to subjects with advanced myeloma in May 2003 (Dispenzieri, 2005). Full approval of bortezomib for multiple myeloma was based on the results of the Assessment of Proteasome Inhibition for Extending Remissions (APEX) trial (Richardson, 2005).

Carfilzomib (Kyprolis) is an irreversible inhibitor of the epoxyketone class (proteasome) that received accelerated approval in the US for the treatment of patients with multiple myeloma who have received at least 2 prior therapies, including bortezomib and an immunomodulatory agent, and have demonstrated disease progression on or within 60 days of completion of the last therapy (Kyprolis Prescribing Information [Onyx Pharmaceuticals, 2012]). Carfilzomib is selective and structurally distinct from bortezomib (O'Connor, 2009). Proteasome inhibition by bortezomib is slowly reversible. Consequently, proteasome inhibition is more sustained with carfilzomib than with bortezomib (Demo, 2007; Suzuki, 2011). In comparison to bortezomib, carfilzomib exhibits





Date: 30 July 2019


equal potency, but greater selectivity for the CT-L activity of the proteasome. In cell culture, carfilzomib is more cytotoxic than bortezomib following brief treatments that mimic the in vivo PK of both molecules (Demo, 2007).

Phase 1 development of carfilzomib included 2 studies, PX-171-001 and PX-171-002, that explored 2 different dosing schedules (daily dosing for 5 consecutive days within Week 1 and 9 days rest; and daily dosing for 2 consecutive days for 3 weeks [Days 1, 2, 8, 9, 15, and 16] and 12 days rest). Prolonged proteasome inhibition was believed to have greater antitumor activity and would be pursued if tolerable.

Data collected in these 2 trials suggested that the 2 consecutive day weekly schedule was better tolerated and demonstrated clinically meaningful response rates. Subsequent Phase 2 and Phase 3 carfilzomib studies have utilized this dose and schedule and have provided data indicating both tolerability and efficacy in advanced stage, heavily pretreated multiple myeloma subjects. Both schedules will be assessed with oprozomib to determine which schedule provides an advantage in tolerability and efficacy.

Oprozomib, a structural analogue of carfilzomib, is a synthetic small-molecule peptide that specifically functions as an irreversible and highly selective inhibitor of the CT-L activity of the 20S proteasome, which leads to the accumulation of protein substrates within the cell and induction of apoptosis. The studies discussed above demonstrate the treatment potential for proteasome inhibition in multiple myeloma. There is also a continued need for more effective agents and those that can be administered orally, which would improve compliance, patient convenience, and potentially prolong treatment duration.

Preclinical studies show that lenalidomide sensitizes multiple myeloma to the proteasome inhibitor bortezomib, suggesting combination therapy may enhance clinical activity. The combination of a proteasome inhibitor and an IMiD is attractive, as the expected overlapping toxicities would be manageable. This concept was confirmed in Phase 1 and 2 studies of lenalidomide, high-dose dexamethasone, and bortezomib, which demonstrated synergistic effects in relapsed and refractory multiple myeloma (Richardson, 2006a; Anderson, 2009), although treatment-emergent peripheral neuropathy (observed in 35% of subjects) may limit the utility of that combination (Richardson, 2006b). An ongoing,



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411


Phase 1/2 study of carfilzomib in combination with lenalidomide and low-dose dexamethasone in subjects with newly diagnosed multiple myeloma has demonstrated excellent activity and tolerability, with 62% of 53 subjects achieving near complete response or better and with only Grade 1/2 peripheral neuropathy in 23% of the subjects (Jakubowiak, 2012).

Stadtmauer et al. (2013) demonstrated the activity of carfilzomib in combination with pomalidomide and dexamethasone (CPomd) in a Phase 1b/2 study. In this ongoing 82-subject trial, the primary objective is to assess the safety, tolerability, and MTD of carfilzomib in combination with pomalidomide and low-dose therapeutic dexamethasone. Secondary objectives include a preliminary assessment of efficacy as measured by best ORR, PFS, and OS. All subjects were refractory to prior lenalidomide and relapsed and refractory to their most recent therapy at the time of enrollment. The MTD of carfilzomib was determined to be 20/27 mg/m² in combination with 4 mg of pomalidomide per day on Days 1–21, and 40 mg/week of dexamethasone. Drug-related AEs occurring in > 20% of subjects included fatigue, anemia, thrombocytopenia, neutropenia, diarrhea, dyspnea, skin rash/pruritis, elevated creatinine, and hypocalcemia. Notable SAEs were Grade 3 pneumonia (n = 3), pulmonary embolism (n = 1), and congestive heart failure (n = 1). The ORR was 50% and the 6-month PFS was 71%. The OS at 12 months was 90%. The authors concluded that this regimen was safe and adequately tolerated and led to compelling improvements in outcome for subjects with advanced myeloma.

The rationale for this study is based on the results of the previously described study (Stadtmauer, 2013), as well as the similarities between carfilzomib and oprozomib in mechanism of action, preclinical toxicity profile, clinical profile, and the non-overlapping toxicity profile of oprozomib and pomalidomide. Subjects treated with carfilzomib have demonstrated an ORR of 23% and an OS of 15.6 months (Siegel, 2012), while subjects treated with pomalidomide in combination with dexamethasone have demonstrated an ORR of 30% and an OS of 16.5 months (Jagannath, 2012). The proposed study of oprozomib in combination with pomalidomide and dexamethasone will assess whether this triplet can confer improvements in outcome as measured by PFS when compared with pomalidomide and dexamethasone alone.






### 4 **STUDY OBJECTIVES**

#### 4.1 PRIMARY OBJECTIVES

- To determine the maximum tolerated dose (MTD) and identify the recommended Phase 3 dose (RP3D) and schedule of oprozomib in combination with pomalidomide and dexamethasone (OPomd) in subjects with primary refractory or relapsed and refractory multiple myeloma
- To evaluate the safety and tolerability of the OPomd combination in subjects with primary refractory or relapsed and refractory multiple myeloma

### 4.2 SECONDARY OBJECTIVES

- To estimate the overall response rate (ORR) of OPomd, defined as the proportion of subjects with an overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) as determined by investigator according to the International Myeloma Working Group- Uniform Response Criteria (IMWG-URC)
- To estimate the clinical benefit rate (CBR) of OPomd, defined as the proportion of subjects with an overall response of minimal response (MR) or better as determined by investigator according to the IMWG-URC and modified European Group for Blood and Marrow Transplantation (EBMT) criteria
- To characterize the pharmacokinetics (PK) of oprozomib in the OPomd regimen

### 4.3 **EXPLORATORY OBJECTIVES**

- To evaluate the pharmacodynamic (PDn) biomarkers that may correlate with antitumor activity
- To evaluate genomic biomarkers that may correlate with antitumor activity and resistance following treatment with proteasome inhibitors
- To evaluate (in the dose-expansion portion only) the patient-reported outcomes (PRO) using the tools listed below:
  - Bone pain and the impact of bone pain measured with the Brief Pain Inventory- Short Form (BPI-SF)
  - Health-related quality of life (HRQoL) measured by the global health status/QoL scale of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Module (QLQ-C30) questionnaire
  - Health status assessed by the EO-5D-5L
  - Disease symptoms as measured by the disease symptoms subscale of the EORTC Multiple Myeloma Module (QLQ-MY20) questionnaire
  - Neurotoxicity symptoms as measured by the neurotoxicity subscale of the Functional Assessment of Cancer Therapy / Gynecological Oncology Group-Neurotoxicity (FACT/GOG-Ntx4 [Version 4]) questionnaire






Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


### 5 **STUDY DESIGN**

This is a Phase 1b study of oprozomib in combination with pomalidomide and dexamethasone in subjects with primary refractory or relapsed and refractory multiple myeloma. This study includes an open-label, Phase 1b, dose-escalation and dose-expansion portion (the equivalent of a small Phase 2) during which the RP3D will be identified. Further evaluation of safety and efficacy will be assessed during the dose-expansion portion. During this study, subjects will receive Oprozomib ER Tablets according to their assigned dose cohort.

This study will include subjects with primary refractory or relapsed and refractory multiple myeloma, ie, those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy (including bortezomib and lenalidomide and/or thalidomide, and in the dose-expansion portion of the study only, been treated with adequate alkylator therapy). Subjects whose last therapy was bortezomib and who were not refractory but developed bortezomib intolerance, as defined by the development of Grade 2 peripheral neuropathy with pain or ≥ Grade 3 peripheral neuropathy after  $\geq 2$  consecutive cycles, are eligible.

Treatment cycles are 28 days in duration. Two (2) oprozomib dosing schedules will be assessed during dose escalation. Subjects will receive oprozomib once daily either on Days 1–5 and 15–19, referred to hereafter as the 5/14 schedule, or an alternate schedule of once daily on Days 1, 2, 8, 9, 15, 16, 22, and 23, referred to hereafter as the 2/7 schedule. Pomalidomide will be given on Days 1–21 and dexamethasone will be given on Days 1, 2, 8, 9, 15, 16, 22, and 23 of every 28-day cycle.

Approximately 35 study sites will participate in this study (15 sites for the dose-escalation and 20 additional sites for the dose-expansion portions of the study).

Disease assessments will be performed every 4 weeks for subjects in both arms for 18 months. Further disease assessments will be conducted every 8 weeks after this period, beginning with Month 20. Details of the study assessments required for this study are provided in Appendices A1, A2, B1, and B2.






### 5.1 DOSE-ESCALATION AND DOSE-EXPANSION PORTIONS OF THE **STUDY**

In this study, the safety, MTD, PK/PDn, and RP3D of oprozomib when given in combination with pomalidomide and dexamethasone will be assessed using a standard 3 + 3 dose-escalation design. For each of the 2 schedules being studied, groups of 3 to 6 subjects will be enrolled into dose-escalation cohorts. As long as fewer than 33% of subjects experience a DLT in a given cohort, escalation will continue by 30-mg increments of oprozomib onto the next designated cohort(s). A minimum of 6 subjects must be treated at the MTD to establish the dose as the MTD. If the starting dose of oprozomib cannot be safely administered with the labeled pomalidomide dose or at sponsor discretion, then up to 2 possible alternative dose-escalation paths for oprozomib with lower pomalidomide doses will be explored (See tables below for primary and alternative dose-escalation paths). Dose escalation will continue until until sponsor discretion, the maximum planned dose of pomalidomide is reached, or  $\geq 2$  DLTs occur in a cohort, whichever occurs first. The prior cohort will be expanded to at least 6 subjects if not previously done to establish it as the MTD. There may be more than 1 MTD of oprozomib if more than 1 dose level of pomalidomide is studied. The MTD for oprozomib associated with each dose level of pomalidomide assessed will be the dose level where < 2 DLTs in 6 subjects are observed.

There is no planned maximum dose of oprozomib to be evaluated as it is being added to the FDA-approved regimen of pomalidomide/dexamethasone, however, this could be imposed at any time during the course of the study, based on sponsor discretion. The starting dose of oprozomib for the 5/14 schedule is 150 mg, 3 dose levels below the established single-agent MTD of 240 mg. The starting dose of oprozomib for the 2/7 schedule is 210 mg, 3 dose levels below the established 2/7 single-agent MTD of 300 mg. The MTD will be determined as outlined in the protocol for each schedule. Following dose escalation, the sponsor has the option of expanding 1 or both schedules in order to establish the RP3D and schedule.

The sponsor, with input from the Cohort Safety Review Committee ([CSRC] consisting of investigators, sponsor's medical monitor, and sponsor's drug safety representative), will determine which dose and schedule of oprozomib in combination with Pomd to use for the dose-expansion (ie, the RP3D) portion of the study. The sponsor has the option of expanding






Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets

1 or both schedules in order to establish the RP3D and schedule. The RP3D may differ from the MTD, but will not be higher than the MTD, and will be selected based upon the assessment of the safety, tolerability, PK, PDn, preliminary activity, and other variables to be observed across multiple cycles of combination therapy.

### *5.1.1* DOSE-ESCALATION SCHEMA FOR THE 5/14 OPROZOMIB DOSING **SCHEDULE**

The study dosing schema for the 5/14 schedule is displayed in Figure 1. The potential doses to be evaluated on the 5/14 dosing schedule are displayed in Figure 2. The primary and alternative pathways for dose escalation of oprozomib and pomalidomide for the 5/14 Schedule are summarized in Table 3 through Table 5; these are examples, and are not inclusive of all possible dose-escalation paths.

Figure 1 Study Dosing Schema for the 5/14 Dosing Schedule






Figure 2 5/14 Schedule Primary Study Dose-Escalation Paths<sup>a</sup>



5/14 = Dosing on Days 1–5 and 15–19; Dex = Dexamethasone; OPZ = oprozomib; Pom = pomalidomide

**Primary Dose-Escalation Path for Oprozomib** Table 3 on 5/14 Schedule with Pomalidomide 4 mg in Phase 1b

| Cohort 5/14 Schedule | Oprozomib Dose<br>(mg/day) | Pomalidomide Dose<br>(mg/day) |
|---|---|---|
| 1a (initial cohort) | 150 | 4 |
| 2a | 180 | 4 |
| 3a | 210 | 4 |

5/14 = Dosing on Days 1–5 and 15–19; MTD = maximum tolerated dose.

Note: This is an example of the primary dose-escalation cohort. Dose escalation will continue in 30-mg increments of oprozomib until the MTD is identified.

If Cohort 1a exceeds the MTD, or at the sponsor's discretion, the alternative path 1 described in Table 4 may be followed.

Approved



<sup>&</sup>lt;sup>a</sup> There is no predefined maximum dose level of oprozomib being studied.


Alternative Dose-Escalation Path 1 for Oprozomib on 5/14 Schedule with Pomalidomide in Phase 1b if Cohort 1a Exceeds the MTD or at Sponsor Discretion

| Cohort 5/14 Schedule | Oprozomib Dose<br>(mg/day) | Pomalidomide Dose<br>(mg/day) |
|---|---|---|
| 1b | 150 | 3 |
| 2b | 180 | 3 |
| 3b | 210 | 3 |

5/14 = Dosing on Days 1–5 and 15–19; MTD = maximum tolerated dose.

If Cohort 1b exceeds the MTD, or at the sponsor's discretion, the alternative path 2 described in Table 5 may be followed.

Alternative Dose-Escalation Path 2 for Oprozomib on 5/14 Schedule with Pomalidomide in Phase 1b if Cohort 1b Exceeds the MTD or at Sponsor Discretion

| Cohort 5/14 Schedule | Oprozomib Dose<br>(mg/day) | Pomalidomide Dose<br>(mg/day) |
|---|---|---|
| 1c | 150 | 2 |
| 2c | 180 | 2 |
| 3c | 210 | 2 |

5/14 = Dosing on Days 1–5 and 15–19; MTD = maximum tolerated dose.

### DOSE-ESCALATION SCHEMA FOR THE 2/7 OPROZOMIB DOSING 5.1.2 **SCHEDULE**

The study dosing schema for the 2/7 schedule is displayed in Figure 3. The potential doses to be evaluated on the 2/7 dosing schedule are displayed in Figure 4. The primary and alternative pathways for dose escalation of oprozomib and pomalidomide in the Phase 1b portion of the study for the 2/7 schedule are summarized in Table 6 through Table 8; these are examples, and are not inclusive of all possible dose-escalation paths.

Approved



Oprozomib ER Tablets


Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Clinical Study Protocol No. OPZ007 Onyx Therapeutics

Figure 3 Study Dosing Schema for the 2/7 Dosing Schedule



Figure 4 2/7 Schedule Primary Study Dose-Escalation Paths<sup>a</sup>



2/7 = Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23; Dex = Dexamethasone; OPZ = oprozomib; Pom = pomalidomide



<sup>&</sup>lt;sup>a</sup> There is no predefined maximum dose level of oprozomib being studied.

Date: 30 July 2019


Onyx Therapeutics

Oprozomib ER Tablets

Supplemental Clinical Study Report: 20130411

Table 6 Primary Dose-Escalation Path for Oprozomib on the 2/7 Schedule with Pomalidomide 4 mg in Phase 1b

| Cohort 2/7 Schedule | Oprozomib Dose (mg/day) | Pomalidomide Dose (mg/day) |
|-----------------------|-------------------------|----------------------------|
| 101a (initial cohort) | 210 | 4 |
| 201a | 240 | 4 |
| 301a | 270 | 4 |

2/7 = Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23; MTD = maximum tolerated dose.

Note: This is an example of the primary dose-escalation cohort. Dose escalation will continue in 30-mg increments of oprozomib until the MTD is identified.

If Cohort 101a exceeds the MTD, or at the sponsor's discretion, the alternative path 1 described in Table 7 may be followed.

Table 7 Alternative Dose-Escalation Path 1 for Oprozomib on 2/7 Schedule with Pomalidomide in Phase 1b if Cohort 101a Exceeds the MTD or at Sponsor Discretion

| Cohort 2/7 Schedule | Oprozomib Dose (mg/day) | Pomalidomide Dose (mg/day) |
|---------------------|-------------------------|----------------------------|
| 101b | 210 | 3 |
| 201b | 240 | 3 |
| 301b | 270 | 3 |

2/7 = Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23; MTD = maximum tolerated dose.

If Cohort 101b exceeds the MTD, or at the sponsor's discretion, the alternative path 2 described in Table 8 may be followed.

Table 8 Alternative Dose-Escalation Path 2 for Oprozomib on 2/7 Schedule with Pomalidomide in Phase 1b if Cohort 101b Exceeds the MTD or at Sponsor Discretion

| Cohort 2/7 Schedule | Oprozomib Dose (mg/day) | Pomalidomide Dose (mg/day) |
|---------------------|-------------------------|----------------------------|
| 101c | 210 | 2 |
| 201c | 240 | 2 |
| 301c | 270 | 2 |

2/7 = Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23; MTD = maximum tolerated dose.

Approved



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411


### 5.1.3 **DOSE-LIMITING TOXICITIES**

Subjects in both dosing schedules will be evaluated for DLTs according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03 during the 28-day period of Cycle 1 combination therapy. Intrasubject dose escalation to the RP3D may be permitted once that dose has been determined and after a discussion has occurred between the treating physician and the Sponsor's study medical monitor. The decision to escalate to the next higher dose of oprozomib in this study will be based on an assessment of study drug-related DLTs during Cycle 1 by the CSRC. The CSRC consists of investigators, the **Sponsor's study** medical monitor, and **the Sponsor's drug** safety representative. Each subject in the cohort under review will be discussed and assessed. Once all data have been presented, the CSRC will decide on the most appropriate course of action regarding dose escalation based on guidance in Section 5.1.

Study drug is defined as the combination of oprozomib, pomalidomide, and dexamethasone. Study drug-related is defined as a reasonable likelihood of clinical causality based on time of event, biology, dechallenge improvement and that the AE was not likely explained by the subject's clinical state, underlying disease, concomitant medication, or study/nonstudy procedure. Definition of DLTs and additional details are provided in Section 10.5.

#### 5.1.4 SUBJECT REPLACEMENT

Subjects must meet the following criteria to be considered evaluable for MTD determination during the 4-week DLT evaluation period unless a DLT occurs before the subject receives all planned doses of oprozomib for both the 5/14 and 2/7 dosing schedules:

- A minimum of 17 of 21 planned doses of pomalidomide must be received
- A minimum of 6 of 8 planned doses of dexamethasone must be received
- All planned doses of oprozomib must be received

Subjects not meeting all of the above criteria or assessed as unevaluable by the CSRC will be replaced.

#### 5.1.5 DOSE EXPANSION

The criteria for selecting the RP3D for 1 or both schedules of oprozomib at the sponsor's discretion will include assessment of the safety, tolerability, and preliminary activity






observed across multiple cycles of therapy. In addition, both PK and PDn assessments to demonstrate adequate exposure and proteasome inhibition will be a key factor. Therefore, the RP3D may differ from the MTD. Once the MTD and the recommended dose for the expansion phase have been determined, a minimum of 20 additional subjects at 1 or both schedules of oprozomib at the sponsor's discretion will be enrolled in the dose-expansion portion of the study in order to continue the evaluation of the safety and efficacy of the regimen. The safety of subjects in the Dose Expansion will be monitored on an ongoing basis by the CSRC during regularly scheduled calls.

### 5.2 ESTIMATED STUDY DURATION AND STUDY CLOSURE

The total study duration is expected to be approximately 12-13 months.

- The Phase 1b portion of the study will take approximately 7–8 months to complete
- Approximately 5 months will be required to enroll and evaluate response status of subjects in the dose-expansion portion of the study

#### 5.3 **MINIMIZING BIAS**

#### 5.3.1 BLINDING

Both the dose-escalation and dose-expansion portions of **this study** are open-label.

### 6 **SUBJECT SELECTION**

### 6.1 **INCLUSION CRITERIA**

### **Disease Related**

- 2. Multiple myeloma that is primary refractory, relapsed and refractory, or intolerant after at least 2 lines of standard therapy for multiple myeloma, including:
  - a.  $\geq 2$  consecutive cycles of both bortezomib and lenalidomide or thalidomide (alone or in combination)
  - b. In the dose-expansion portion of the study only: In addition to the above, treatment with adequate alkylator therapy, defined as:
    - i. High-dose melphalan or other alkylating agent as conditioning for autologous or allogeneic SCT, or
    - ii.  $\geq 6$  cycles of induction therapy, or
    - iii. Progressive disease after  $\geq 2$  cycles

Approved




- 3. Measurable disease as indicated by 1 or more of the following:
  - a. Serum M-protein ≥ 500 mg/dL
  - b. Urine M-protein  $\geq$  200 mg/24 h
  - c. Only for subjects without measurable M-protein by serum protein electrophoresis (SPEP) and urine protein electrophoresis (UPEP), involved free light chain (FLC) concentration ≥ 10 mg/dL provided serum free light chain (SFLC) ratio is abnormal
- 4. Disease progression on or within 60 days of completion of the last therapy, or intolerance to bortezomib if received as their last therapy
  - a. Patients who received bortezomib as their last therapy who were not refractory but developed bortezomib intolerance, as defined by the development of Grade 2 peripheral neuropathy with pain or  $\geq$  Grade 3 peripheral neuropathy after  $\geq 2$  consecutive cycles, are eligible
- 5. Prior carfilzomib is allowed if a subject was not removed from carfilzomib therapy due to toxicity, unless approved by the **Sponsor's** study medical monitor.

# **Demographic**

- 6. Males and females  $\geq$  18 years old
- 7. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0–2 (Appendix H)

## Laboratory

- 8. Adequate hepatic function, with bilirubin  $\leq 1.5$  times the upper limit of normal (ULN) in the absence of Gilbert's disease or hemolysis, and alanine aminotransferase (ALT) and aspartate aminotransferase (AST)  $\leq$  3 times ULN
- 9. Absolute neutrophil count (ANC)  $\geq 1500/\text{mm}^3$ . Screening ANC should be independent of myeloid growth factor support for at least 1 week or 2 weeks for pegylated growth factors.
- 10. Hemoglobin  $\geq 8.0$  g/dL. Patients may receive red blood cell (RBC) transfusions or receive erythropoietin or darbepoetin alfa in accordance with institutional guidelines up to 1 week before screening.
- 11. Platelet count  $\geq$  75,000 mm<sup>3</sup>. Patients should not have received platelet transfusions for at least 1 week before screening.
- 12. Uric acid, if elevated, must be corrected to within laboratory normal range before dosing.
- 13. Calculated or measured creatinine clearance (CrCl) ≥ 30 mL/min calculated using the formula of Cockcroft and Gault  $[(140 - age) \times mass (kg) / (72 \times serum)]$ creatinine mg/dL)]. Multiply result by 0.85 if female.




### Ethical/Other

- 14. Patient must sign a written informed consent form in accordance with federal, local, and institutional guidelines.
- 15. Female patients of childbearing potential must have a negative pregnancy test (with a sensitivity of at least 50 mIU/mL) within 1 day of the first dose of study drug and agree to use 2 effective methods of contraception during the study and for 28 days following the last dose of study drug. Postmenopausal females (> 45 years old and without menses for ≥2 years) and surgically sterilized females are exempt from these requirements.
- 16. Male patients, including those with prior vasectomy, must use an effective barrier method of contraception during the study and for 3 months following the last dose if sexually active with a female of childbearing potential. Additionally, they must agree not to donate sperm while being treated and for up to 3 months after discontinuing treatment.

### 6.2 **EXCLUSION CRITERIA**

# **Disease Related**

- 1. Systemic chemotherapy with approved or investigational anticancer therapeutics, intended to treat underlying malignancy, within 3 weeks before the first dose of study treatment or 6 weeks for antibody therapy.
- 2. Dexamethasone at cumulative doses of greater than 160 mg or equivalent within 21 days prior to the first dose of study treatment is not allowed. Use of topical or inhaled steroids is acceptable.
- 3. Radiation therapy within 3 weeks before first dose of study drug. Radioimmunotherapy within 8 weeks before first dose of study drug.
- 4. Plasmapheresis is not permitted at any time during the Screening period or while the subject is receiving study treatment. If a subject has started Screening procedures requiring plasmapheresis, or is anticipated to require plasmapheresis during or after the Screening period, this patient will be considered ineligible and should not be enrolled.
- 5. Autologous SCT within the prior 8 weeks or allogeneic SCT within 16 weeks prior to initiation of study treatment. Patients with prior allogeneic SCT should not have evidence of moderate-to-severe graft-versus-host disease (as defined in Filipovich 2005) and must be approved by the **Sponsor's** study medical monitor.
- 6. Known hypersensitivity to any IMiDs, including rash

Approved




- 7. Prior pomalidomide exposure
  - a. For the dose-escalation portion of the study: Subjects requiring pomalidomide dose reduction or removal due to toxicity
  - b. For the dose-expansion portion of the study: Prior pomalidomide treatment of any duration
- 8. Known hypersensitivity/toxicity or intolerance to dexamethasone
- 9. Prior exposure to oprozomib
- 10. Hypersensitivity, intolerance, or inability to take antithrombotic prophylaxis

## **Concurrent Conditions**

- 11. Major surgery within 3 weeks before first dose of study drug
- 12. Congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months before first dose of study drug
- 13. Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 2 weeks before first dose of study drug
- 14. History of previous clinically significant GI bleed in the 6 months prior to first dose of study drug
- 15. Known or suspected human immunodeficiency virus (HIV) infection or patients who are HIV seropositive
- 16. Active hepatitis A, B, or C infection
- 17. Significant neuropathy (Grade 2 with pain or ≥ Grade 3) at the time of the first dose of study drug
- 18. Other malignancy within the past 3 years except those considered cured by surgical resection; examples include some cases of:
  - a. Adequately treated basal or squamous cell carcinoma of the skin
  - b. Thyroid cancer
  - c. Carcinoma in situ of the cervix or breast
  - d. Prostate cancer with Gleason Score of 6 or less with stable prostate-specific antigen levels
- 19. Plasma cell leukemia
- 20. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
- 21. Known amyloidosis

Approved



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411


- 22. Female patients who are pregnant or nursing
- 23. Uncontrolled diabetes or hypertension
- 24. Inability to swallow medication, inability or unwillingness to comply with the drug administration requirements, or GI condition that could interfere with the oral absorption or tolerance of treatment
- 25. Any contraindication to oral hydration (eg, preexisting cardiac impairment or fluid restriction)
- 26. Any clinically significant psychiatric, social, or medical condition that, in the opinion of the investigator, could increase patient risk, interfere with protocol adherence, or affect a patient's ability to give informed consent

# 7 **SUBJECT SCREENING**

A signed and dated informed consent form will be obtained before any screening procedures are performed. Evaluations obtained as part of routine medical care and performed during the screening period may be used in place of the study-specific evaluations, provided they meet the time windows described below. Subjects will acknowledge and agree to the possible use of this information for the study by giving informed consent. The screening period for a particular subject commences at the point, after informed consent is signed, at which the subject undergoes the first study-specific screening assessment, and must be completed within 28 days of receiving the first dose of study drug.

# 8 SUBJECT ENROLLMENT

All subjects who sign consent will be assigned a unique study number. This number will be used to identify the subject throughout the clinical study and must be used on all study documentation related to that subject. The **Sponsor's** study medical monitor or designee will review the subject's information before enrollment. Only subjects who are approved by the **Sponsor's** study medical monitor will be allowed to enroll into the study. A minimum time of 24 hours during weekdays (Monday through Friday) will be required for the **Sponsor's** study medical monitor or designee to approve a subject for enrollment, and additional time may be required when approval is sought during a weekend or holiday. Subjects are only considered enrolled when the **Sponsor's** study medical monitor or designee approves the patient for enrollment.






## **STUDY DRUG**

No changes in drug product, dosage, or treatment-regimen occurred in this protocol amendment from the previous version.

### 9.1 **OPROZOMIB**

#### 9.1.1 OPROZOMIB PHYSICAL DESCRIPTION

Oprozomib is a synthetic small molecule peptide bearing the chemical name N-((S)-3-methoxy-1-((S)-3-methoxy-1-((S)-1-((R)-2-methyloxiran-2-yl)-1-oxo-3-phenylpropan-2-ylamino)-1-oxopropan-2-ylamino)-1-oxopropan-2-yl)-2-methylthiazole-5-carboxamide. The molecular formula is C<sub>25</sub>H<sub>32</sub>N<sub>4</sub>O<sub>7</sub>S and the molecular weight is 532.61. It specifically functions as an inhibitor of the CT-L activity of the 20S proteasome, which leads to the accumulation of protein substrates within the cell and induction of apoptosis.

### 9.1.2 **OPROZOMIB FORMULATION**

Oprozomib will be provided as a tablet for oral administration. Oprozomib ER Tablets are intended to release greater than or equal to 75% (Quantity) of the total dose of oprozomib over approximately 8 hours.

Oprozomib ER Tablets are white to off-white tablets manufactured at 5 dosage strengths:

- Oprozomib 150 mg oval shape tablets are debossed with "H" on one side and contain 150 mg of oprozomib
- Oprozomib 180 mg oval shape tablets are debossed with "I" on one side and contain 180 mg of oprozomib
- Oprozomib 210 mg oval shape tablets are debossed with "J" on one side and contain 210 mg of oprozomib
- Oprozomib 240 mg oval shape tablets are debossed with "K" on one side and contain 240 mg of oprozomib
- Oprozomib 270 mg oval shape tablets are debossed with "L" on one side and contain 270 mg of oprozomib

The excipients for the drug product are lactose monohydrate, microcrystalline cellulose, sodium lauryl sulfate, magnesium stearate, hydroxy propyl methyl cellulose, and Opadry II White. The drug substance-to-excipient ratio is the same in all 5 dosage strengths.




Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


### 9.1.3 OPROZOMIB PACKAGING AND LABELING

The Oprozomib ER Tablets will be available in 150, 180, 210, 240, and 270 mg of oprozomib. Details are provided in the Pharmacy Manual.

## 9.1.4 OPROZOMIB STORAGE

Oprozomib must be stored at room temperature (15°C–30°C; 59°F–86°F) in a secured area to which access is limited to appropriate study personnel.

## 9.2 **POMALIDOMIDE**

Pomalidomide is available as a capsule containing 1, 2, 3, and 4 mg of pomalidomide drug substance for oral administration. Additional product information is provided in the Pomalidomide Prescribing Information (Celgene Corporation, 2013).

# 9.2.1 POMALIDOMIDE PHYSICAL DESCRIPTION

POMALYST is available in 1-mg, 2-mg, 3-mg, and 4-mg capsules for oral administration. Each capsule contains pomalidomide as the active ingredient and the following inactive ingredients: mannitol, pregelatinized starch, and sodium stearyl fumarate. The 1-mg capsule shell contains gelatin, titanium dioxide, FD&C blue 2, yellow iron oxide, white ink, and black ink. The 2-mg capsule shell contains gelatin, titanium dioxide, FD&C blue 2, yellow iron oxide, FD&C red 3, and white ink. The 3-mg capsule shell contains gelatin, titanium dioxide, FD&C blue 2, yellow iron oxide, and white ink. The 4-mg capsule shell contains gelatin, titanium dioxide, FD&C blue 1, FD&C blue 2, and white ink.

# 9.2.2 POMALIDOMIDE PACKAGING AND LABELING

Pomalidomide is commercially available as capsules for oral administration.

## 9.2.3 POMALIDOMIDE STORAGE

Store at 20°C–25°C (68°F–77°F); excursions permitted to 15°C–30°C (59°F–86°F). See USP Controlled Room Temperature.

Approved



Date: 30 July 2019


### 9.3 **DEXAMETHASONE**

Dexamethasone, a synthetic adrenocortical steroid, is available as tablets containing 4 or 6 mg of dexamethasone drug substance for oral administration.

### 9.3.1 DEXAMETHASONE PACKAGING AND LABELING

Dexamethasone is commercially available both as tablets for oral administration and as various sterile formulations for parenteral administration. Additional information is provided in the Dexamethasone Prescribing Information (Pfizer Laboratories, 2012).

#### 9.3.2 DEXAMETHASONE STORAGE

Dexamethasone is not to be stored above 30°C (86°F). Additional storage and usage instructions are provided in the Dexamethasone Prescribing Information (Pfizer Laboratories, 2012).

### 9.4 STUDY DRUG ACCOUNTABILITY

The Sponsor (or designee) and the investigator will maintain records of each shipment of investigational product (IP). Upon receipt of IP, the designated recipient at the study site will inspect the shipment, verify the number and condition of the bottles or blister packs, and prepare an inventory or drug accountability record. The records will document shipment dates, method of shipment, batch numbers, product presentation, quantity of bottles or blister packs contained in the shipment, and dispensation to individual subjects using the subject identification number.

Sites will be required to record and document subject compliance with oprozomib, pomalidomide, and dexamethasone dosing.

Additional details for oprozomib are provided in the Pharmacy Manual.

Approved




### 10 **OPROZOMIB TREATMENT ADMINISTRATION**

It is recommended that oprozomib not be taken on an empty stomach. Subjects will be instructed to take the oprozomib doses after eating with approximately 8 ounces of water. On the PK collection days, dosing of oprozomib in relation to the meal intake (within 2 hours before and 1 hour after dose) will be recorded.

#### 10.1 OPROZOMIB TREATMENT ADMINISTRATION

Oprozomib ER Tablets will be administered in single daily doses. Oprozomib will be administered orally, once daily for 5 consecutive days every other week ([5/14 schedule] ie, on Days 1–5 and 15–19) or once daily for 2 consecutive days of every week ([2/7 schedule] ie, on Days 1, 2, 8, 9, 15, 16, 22, and 23) of each 28-day treatment cycle. Treatment with oprozomib will continue until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason. On days on which oprozomib and dexamethasone are administered concurrently, dexamethasone should be taken at least 30 minutes before oprozomib. Subjects are to be informed not to break, chew, or crush the Oprozomib ER Tablets.

In the dose-escalation and dose-expansion portions of the study, subjects who permanently discontinue pomalidomide or oprozomib may continue on study. If both pomalidomide and oprozomib are permanently discontinued, study treatment will be discontinued but the subject will be followed until disease progression.

### 10.2 POMALIDOMIDE TREATMENT ADMINISTRATION

Pomalidomide will be administered at 4 mg, orally, in the fasted condition (2 hours before or after meals) according to the Prescribing Information (Celgene Corporation, 2013) on Days 1–21. Pomalidomide may be taken with water. Subjects are to be informed not to break, chew, or open the capsules.

The starting dose of pomalidomide for this study is 4 mg once daily, orally, on Days 1–21 of repeated 28-day cycles until disease progression. Pomalidomide may be given at the same time as dexamethasone; however, dexamethasone must be given at least 30 minutes prior to oprozomib.





Date: 30 July 2019


### 10.3 DEXAMETHASONE TREATMENT ADMINISTRATION

Dexamethasone will be administered at 20 mg, orally, on Days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day cycle. On days of concurrent oprozomib and dexamethasone administration, dexamethasone should be taken at least 30 minutes prior to oprozomib. Subjects may take dexamethasone with or without food. Dexamethasone may be given at the same time as pomalidomide; however, dexamethasone must be given at least 30 minutes prior to oprozomib.

Dexamethasone may be administered intravenously (IV), if needed, at the investigator's discretion, but IV dexamethasone will not be provided by the sponsor.

### 10.4 DOSE MODIFICATION GUIDELINES

This section provides dose reduction and other modification guidelines for oprozomib, pomalidomide, and dexamethasone to manage possible toxicity. Administration of oprozomib or pomalidomide will be discontinued in the event of a treatment-related toxicity that, in the opinion of the investigator, warrants permanent discontinuation.

Monotherapy with dexamethasone is not allowed in the dose-escalation and dose-expansion portions of the study.

Exceptions to the dose modification guidelines are permitted with written approval from the **Sponsor's** study medical monitor.

### 10.4.1 **DOSE REDUCTIONS**

For this study, the initial cohort will start at an oprozomib dose level of 150 mg for the 5/14 schedule and 210 mg for the 2/7 schedule. For these subjects, oprozomib or pomalidomide or dexamethasone dose reductions are discouraged during the DLT assessments. Subjects requiring dose reductions in Cycle 1 will be referred to the CSRC for determination if the subject is considered evaluable and for DLT assessment per Section 5.1.4. Dose reduction levels for oprozomib subsequent to Cycle 1 for the 5/14 and 2/7 dosing schedules are provided in Table 9 and Table 10, respectively. Modifications of the dose of oprozomib will occur in up to three 30-mg decrements down to a minimum dose of 150 mg. Additional reductions will be managed by schedule change.




Table 9 Dose Decrements for Oprozomib – 5/14 Schedule

| Nominal | Reduced Oprozomib Doses | | |
|---|---|---|---|
| Dose Level | First Dose Reduction | Second Dose Reduction | Third Dose Reduction |
| 150 mg | Continue 150 mg AND change to 3/14 <sup>a</sup> schedule (Days 1, 2, 3, 15, 16, 17 of 28-day schedule) | D/C oprozomib | NA |
| 180 mg | Dose – 30 mg | Dose – 30 mg AND change<br>to 3/14 schedule<br>(Days 1, 2, 3, 15, 16, 17 of<br>28-day schedule) | D/C oprozomib |
| 210 mg | Dose – 30 mg | Dose – 60 mg | Dose – 60 mg AND change<br>to 3/14 schedule<br>(Days 1, 2, 3, 15, 16, 17 of<br>28-day schedule) |
| ≥ 240 mg | Dose – 30 mg | Dose – 60 mg | Dose – 90 mg |

<sup>5/14 =</sup> Dosing on Days 1–5 and 15–19; D/C = discontinue; NA = not applicable.

Table 10 Dose Decrements for Oprozomib – 2/7 Schedule

| Nominal | | Reduced Oprozomib Doses | |
|---|---|---|---|
| Dose Level | First Dose Reduction | Second Dose Reduction | Third Dose Reduction |
| 210 mg | Dose – 30 mg | Dose – 60 mg | Dose – 60 mg AND change<br>to 1/7 <sup>a</sup> schedule<br>(Days 1, 8, 15, 22 of 28-day<br>schedule) |
| ≥ 240 mg | Dose – 30 mg | Dose – 30 mg | Dose – 90 mg |

<sup>2/7 =</sup> Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23.

**The** dose reduction levels for pomalidomide are provided in Table 11. Dose adjustments should, in general, follow the instructions provided in the Pomalidomide Prescribing Information 2013 (Celgene Corporation, 2013).



<sup>&</sup>lt;sup>a</sup> The minimum oprozomib dose is 150 mg; thus, additional reductions will be managed by schedule change to the 3/14 schedule where doses of oprozomib will be skipped on Days 4, 5, 18, and 19.

<sup>&</sup>lt;sup>a</sup> The minimum oprozomib dose is 150 mg; thus, additional reductions will be managed by schedule change to the 1/7 schedule where doses of oprozomib will be skipped on Days 2, 9, 16, and 23.


**Table 11 Dose Decrements for Pomalidomide** 

| | Reduced Pomalidomide Doses | | |
|---|---|---|---|
| Dose | First Dose Reduction Second Dose Reduction Third Dose Reduction | | |
| 4 mg | 3 mg | 2 mg | 1 mg |

If the dose of either the pomalidomide or oprozomib is reduced during the previous cycle, the reduced dose level will be continued on Day 1 of the next cycle. If the reduced dose level is well tolerated for a complete cycle, the subject may, at the investigator's discretion, be rechallenged with the dose level prior to the reduction at the start of the next cycle.

Treatment guidelines for specific hematologic toxicities are outlined in Section 10.4.2.1.1 and nonhematologic toxicities in Section 10.4.2.1.2. In addition to dose reductions, administration of oprozomib, pomalidomide, and dexamethasone may be temporarily interrupted for a maximum of 4 weeks in the event of a treatment-related toxicity. If the dose delay because of toxicity is longer than 4 weeks, the subject will be discontinued from study treatment. If a subject misses more than 4 consecutive weeks for reasons other than toxicity after completing Cycle 1, the subject will be discontinued from study treatment unless it is determined that the subject was benefiting from therapy and the Sponsor's study medical monitor permits the subject to resume therapy.

Dose reduction levels for dexamethasone are provided in Table 12.

**Table 12** Dose Decrements for Dexamethasone

| | Reduced Dexamethasone Doses | |
|---|---|---|
| Nominal Dose | Dose -1 | Dose -2 |
| 20 mg | 12 mg | 8 mg |
| Cycle 2 +: Age > 75 yrs per investigator discretion 10 mg | 8 mg | 4 mg |

For subjects over 75 years old, after the first cycle and at the investigator's discretion, dexamethasone can be reduced to 10 mg. Dexamethasone will be permanently discontinued after 2 dose reductions for either nominal dose in the event of additional dexamethasone-related toxicity. At the investigator's discretion, dexamethasone may be



Date: 30 July 2019


Clinical Study Protocol No. OPZ007 Onyx Therapeutics Oprozomib ER Tablets 

tapered prior to complete discontinuation according to institutional practice. If the dexamethasone dose is reduced during the previous cycle, the reduced dose level will be continued on Day 1 of the new cycle. If the reduced dose level is well tolerated for a complete cycle, the subject may, at the investigator's discretion, be rechallenged with the dose level prior to the reduction at the start of the next cycle.

If dexamethasone dosing is permanently stopped due to toxicity in accordance with the dose modification guidelines described in Table 15, the subject should stay on oprozomib and/or pomalidomide, depending on the arm to which they are randomized, and continue to follow protocol required therapy, procedures, and assessments. Subjects may continue to take antiemetic doses of dexamethasone (4 mg) on days of oprozomib dosing, if tolerated, at the investigator's discretion.

### 10.4.2 **DOSE MODIFICATION GUIDELINES**

### 10.4.2.1 **Oprozomib Dose Modification Guidelines**

### 10.4.2.1.1 **Hematologic Toxicities**

Dose modification guidelines for oprozomib/placebo and pomalidomide for hematologic toxicities are summarized in Table 13.

Approved




Table 13 Guidelines for Dose Modification of Oprozomib/Placebo and Pomalidomide for Hematologic Toxicities

| Findings | Oprozomib | Pomalidomide |
|---|---|---|
| Findings on Day 1 of Cycle | Recommended Action | |
| Platelets $< 25 \times 10^9 / L$ | Hold dose <sup>a</sup> until recovery<br>≥ 25 × 10 <sup>9</sup> /L; restart at previous<br>dose. | Not applicable. |
| Platelets < 30 x 10 <sup>9</sup> /L | Not Applicable. | Hold dose <sup>a</sup> , follow CBCs.<br>Hold prophylactic<br>anticoagulation until platelets<br>return to $\geq 30 \times 10^9/L^a$ , then<br>resume at 1 dose decrement. |
| ANC < $0.5 \times 10^9$ /L or febrile neutropenia (fever $\geq 38.5$ °C and ANC < $1.0 \times 10^9$ /L) | Hold dose <sup>a</sup> . Add colony stimulating factor <sup>b</sup> With resolution to $\geq 1.0 \times 10^9/L$ , restart at previous dose. | Hold dose <sup>a</sup> . Add colony stimulating factor <sup>b</sup> With resolution to ≥ 0.5 × 10 <sup>9</sup> /L, restart at 1 dose decrement. |
| Findings on Subsequent Days of Cycle | Recommend | |
| Platelets 25 to < 50 × 10 <sup>9</sup> /L without<br>≥ Grade 2 bleeding/hemorrhage | Full dose. | Full dose. |
| Platelets 25 to < 50 × 10 <sup>9</sup> /L with ≥ Grade 2 bleeding/hemorrhage | Hold dose <sup>a</sup> until platelets return to $\geq 50 \times 10^9$ /L and/or bleeding is controlled, then resume at 1 dose decrement. | Hold dose until platelets<br>return to $\geq 50 \times 10^9$ /L and/or<br>bleeding is controlled, then<br>resume at 1 dose decrement. |
| Platelets < 25 × 10 <sup>9</sup> /L or thrombocytopenia with ≥ Grade 2 bleeding/hemorrhage | Hold dose <sup>a</sup> until recovery to<br>≥ 25 × 10 <sup>9</sup> /L; restart at 1 dose decrement. | Hold dose <sup>a</sup> .<br>Hold prophylactic<br>anticoagulation until platelets<br>return to $\geq 30 \times 10^9/L^a$ , then<br>resume at 1 dose decrement. |
| Neutropenic fever (ANC $< 1.0 \times 10^9$ /L and single temperature $> 38.3^{\circ}$ C or temperature $> 38.0^{\circ}$ C sustained for more than 1 hour) ANC $< 0.5 \times 10^9$ /L | Hold dose <sup>a</sup> ; follow CBC at least 3 times per week. Add colony stimulating factor. <sup>b</sup> With resolution of fever and ANC ≥ 1.0 × 10 <sup>9</sup> /L, restart at 1 dose decrement. Hold dose <sup>a</sup> ; follow CBC at least 3 times per week; administration of colony stimulating factor <sup>b</sup> is permitted. Resume at full dose if ANC | Hold dose <sup>a</sup> ; follow CBCs. Add colony stimulating factor <sup>b</sup> . With resolution of fever and ANC ≥ 1.0 × 10 <sup>9</sup> /L, restart at 1 dose decrement. Hold dose <sup>a</sup> until ANC increases to ≥ 0.5 × 10 <sup>9</sup> /L. Administer colony stimulating growth factor <sup>b</sup> . Resume at 1 dose decrement |
| | $\geq 0.5 \times 10^9/L$ within < 7 days.<br>Resume at 1 dose decrement if ANC returns to $\geq 0.5 \times 10^9/L$ $\geq 7$ days. | each subsequent decrease to $< 0.5 \times 10^9/L$ ). |

ANC = absolute neutrophil count; CBC = complete blood count.

Approved



<sup>&</sup>lt;sup>a</sup> The maximum allowed dose interruption is 4 weeks for treatment-related toxicity.

<sup>&</sup>lt;sup>b</sup> Colony stimulating factors such as filgrastim or sargramostim as examples.

**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411


Additional guidance regarding hematologic toxicities and dosing actions is as follows:

- To initiate a new cycle of pomalidomide, the neutrophil count must be at least 500 per μL and the platelet count must be at least 50,000 per μL. If toxicities continue to occur after dose reductions down to 1 mg, then discontinue pomalidomide.
- Nontreatment-related events: If the toxicity resolves to ≤ Grade 1 or baseline and the toxicity is not treatment-related, oprozomib may be restarted at the same dose level
- If required by continued or recurrent toxicity, a second or third dose reduction of
  oprozomib may be permitted after discussion with the **Sponsor's** study medical monitor.
  No more than 3 dose reductions down to a minimum of 150 mg will be permitted for an
  individual subject on study and additional reductions will be managed by schedule
  change. If toxicity continues, oprozomib should be discontinued.

# 10.4.2.1.2 Nonhematologic Toxicities

Table 14 provides oprozomib dosing actions that should be taken for nonhematologic toxicities.

Approved




Table 14 Guidelines for Dose Modification of Oprozomib/Placebo and Pomalidomide for Nonhematologic Toxicities

| | | Recommended Action <sup>a</sup> | |
|---|---|---|---|
| Symptom | Findings | Oprozomib | Pomalidomide |
| Tumor Lysis<br>Syndrome | Generally recognized in at least 3 or more of the following categories: (1) Increase in creatinine, uric acid, or phosphate of ≥ 50% (2) Increase in potassium of ≥ 30% (3) Decrease in calcium of ≥ 20%, or (4) Increase in LDH ≥ 2-fold from baseline | Hold both oprozomib and pomalidomide until all abnormalities in serum chemistries have resolved baseline; resume at full doses. | |
| Neuropathy | Grade 2 neuropathy with pain or ≥ Grade 3 neuropathy | Hold dose until toxicity resolves to ≤ Grade 1 or has returned to baseline. Resume study drug at 1 dose decrement. | Hold dose until toxicity resolves to ≤ Grade 1 or has returned to baseline. Resume study drug 1 dose decrement from previous dose. |
| Infection | Grade 3 or 4 | Hold both oprozomib and pomalidomide until systemic treatment for infection complete. If ANC $\geq 1.0 \times 10^9$ /L, resume both drugs at full dose. If ANC $< 1.0 \times 10^9$ /L, follow hematologic toxicities dose reduction guidelines (Table 13). | |
| Nausea,<br>vomiting,<br>diarrhea, or<br>constipation | ≥ Grade 3 without optimal supportive care as defined by use of both a 5-HT <sub>3</sub> antagonist and aprepitant | Oprozomib-related: Full dose oprozomib but institute optimal supportive care. | Pomalidomide-related:<br>Hold dose until toxicity<br>resolves to ≤ Grade 1 or<br>has returned to baseline. |
| | ≥ Grade 3 with optimal supportive care as defined by use of both a 5-HT <sub>3</sub> antagonist and aprepitant | Oprozomib-related: Hold dose until toxicity resolves to ≤ Grade 1 or has returned to baseline. Resume study drug at 1 dose decrement. | Resume study drug at 1 dose decrement from previous dose. |
| Fatigue | Grade 3 fatigue lasting < 14 days | Full dose. | Hold dose until toxicity |
| | Grade 3 fatigue lasting ≥ 14 days | Hold dose until toxicity resolves to ≤ Grade 1 or has returned to baseline. Resume study drug at 1 dose decrement. | resolves to ≤ Grade 1 or<br>has returned to baseline.<br>Resume study drug at<br>1 dose decrement from<br>previous dose. |

Approved



Date: 30 July 2019


Approved


Table 14 Guidelines for Dose Modification of Oprozomib/Placebo and Pomalidomide for Nonhematologic Toxicities (cont'd)

| | | Recommended Actiona | |
|---|---|---|---|
| Symptom | Findings | Oprozomib | Pomalidomide |
| Renal | CrCl 30 to < 50 mL/min (Grade 2) | Full dose. | Full dose. |
| Dysfunction | CrCl 15 to < 30 mL/min (Grade 3) | Hold dose. When CrCl recovers to ≤ Grade 2, resume at 1 dose decrement. | Hold dose. When CrCl recovers to ≤ Grade 2, resume dose at 1 dose decrement. If Grade 3 CrCl reappears, then hold dose until CrCl recovers to ≤ Grade 2 and reduce dose an additional 1 dose decrement. |
| | CrCl 0 to < 15 mL/min (Grade 4) | Discontinue. | Discontinue. |
| Elevation in<br>Liver Function<br>Tests | ≥ Grade 3 (AST, ALT, or total bilirubin) <sup>b</sup> | Hold until resolves to baseline. Resume at 1 dose decrement. | Hold pomalidomide and restart treatment at 1 dose decrement less than the previous dose when toxicity has resolved to ≤ Grade 2 at physician discretion. |
| Other<br>Nonhematologic<br>Toxicity | Assessed as oprozomib-related and $\geq$ Grade 3° | Hold oprozomib dose until toxicity resolves to ≤ Grade 1 or baseline; restart at 1 dose decrement. | Full dose. |
| Other<br>Nonhematologic<br>Toxicity | Assessed as pomalidomide-related and $\geq$ Grade $3^{c,d}$ | Full dose. | Hold pomalidomide and restart treatment at 1 dose decrement less than the previous dose when toxicity has resolved to ≤ Grade 2 at physician discretion. |
| Grade 1 or 2 GI<br>hemorrhage | Assessed as oprozomib-related | DELAY until Grade 0<br>DECREASE one dose<br>level for Grade 2 | Full dose at physician discretion |
| Grade 3 or 4 GI<br>Hemorrhage | Assessed as oprozomib-related | Discontinue. | Full dose when AE resolves to ≤ Grade 2 at physician discretion. |

5-HT<sub>3</sub> = 5-hydroxytryptamine type-3; AE = adverse event; ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; CrCl = creatinine clearance; eCRF = electronic case report form; GI = gastrointestinal; LDH = lactate dehydrogenase; ULN = upper limit of normal.



<sup>&</sup>lt;sup>a</sup> The maximum allowed dose interruption is 4 weeks for treatment-related toxicity.

b If AST or ALT is ≥ 3 × ULN, the "evaluation of treatment emergent liver abnormalities" eCRF should be completed.

c If cardiac or pulmonary treatment-emergent toxicities occur, the "cardiopulmonary AE" eCRF should be completed.

<sup>&</sup>lt;sup>d</sup> See Celgene Corporation, 2013.

**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411


Additional guidance regarding nonhematologic toxicities and dosing actions is as follows:

- Nontreatment-related events: If the toxicity resolves to ≤ Grade 1 or baseline and the toxicity is not treatment-related, oprozomib may be restarted at the same dose level
- If the subject tolerates the reduced dose for 1 cycle, the subject's dose may be re-escalated to the dose being taken prior to the dose reduction
- If required by continued or recurrent toxicity, a second or third dose reduction of oprozomib may be permitted after discussion with the **Sponsor's** study medical monitor. No more than 3 dose reductions down to a minimum of 150 mg will be permitted for an individual subject on study and additional reductions will be managed by schedule change. If toxicity continues, oprozomib should be discontinued.
- Subjects who develop Grade 3 or 4 GI hemorrhage should not be rechallenged with oprozomib. Oprozomib should be permanently discontinued. Endoscopy should be strongly considered for any subject with GI hemorrhage.

# 10.4.2.2 **Dexamethasone Dose Modification Guidelines**

Guidelines for dexamethasone dose modifications and treatment are summarized in Table 15.

Approved




Table 15 Treatment Guidelines for Dexamethasone-Related Toxicity

| Body System | Symptom | Recommended Action |
|---|---|---|
| Gastrointestinal | Dyspepsia, gastric or<br>duodenal ulcer, or gastritis<br>Grade 1 or 2 (requiring<br>medical management) | Continue dexamethasone at same dose and treat with therapeutic doses of H <sub>2</sub> blockers, or proton pump inhibitor. May consider adding sucralfate or other antiulcer treatment as clinically indicated. If symptoms persist despite above measures, decrease dexamethasone dose by 1 dose level. |
| Gastrointestinal | Dyspepsia, gastric or<br>duodenal ulcer, or gastritis<br>≥ Grade 3 (requiring<br>hospitalization or surgery) | Hold dexamethasone until symptoms return to baseline. Restart dexamethasone at 1 dose decrement along with concurrent therapy with $H_2$ blockers, sucralfate, or omeprazole. If symptoms persist despite above measures, discontinue dexamethasone permanently. |
| Gastrointestinal | Acute pancreatitis | Discontinue dexamethasone permanently. |
| General Disorders | Edema > Grade 3 (> 30% limb discrepancy in volume; gross deviation from normal anatomic contour; limiting self-care activities of daily living ) | Hold dexamethasone until symptoms return to baseline. Administer diuretics as needed, and restart dexamethasone at 1 dose decrement; if edema persists despite above measures, decrease dose another level. Discontinue dexamethasone permanently if symptoms persist despite second reduction. |
| Psychiatric<br>Disorders | Confusion or mood alteration<br>≥ Grade 2 (interfering with<br>function ± interfering with<br>activities of daily living) | Hold dexamethasone until symptoms return to baseline. Restart dexamethasone at 1 dose decrement. If symptoms persist despite above measures, reduce by another dose decrement. |
| Musculoskeletal | Muscle weakness ≥ Grade 2 (symptomatic and interfering with function ± interfering with activities of daily living) | Hold dexamethasone until symptoms return to baseline. Restart dexamethasone at 1 dose decrement. If weakness persists, decrease dose by 1 more dose level. Discontinue dexamethasone permanently if symptoms persist. |
| Metabolism and<br>Nutrition<br>Disorders | Hyperglycemia ≥ Grade 3<br>(fasting glucose<br>> 250 mg/dL) | Hold dexamethasone until glucose is ≤ Grade 2 (< 250 mg/dL) and treat with insulin or other hypoglycemic agents as needed. If uncontrolled despite above measures, decrease dose by 1 dose level until ≤ Grade 2 (< 250 mg/dL) |
| All Other | Other nonhematologic toxicity ≥ Grade 3 felt related to dexamethasone | Hold dexamethasone dose. Resume at 1 dose decrement when toxicity has resolved to Grade 2 or less or to baseline. If toxicity recurs, hold dexamethasone dose until toxicity has resolved to Grade 2 or less or to baseline and resume dexamethasone dose by 1 more dose decrements. If toxicity recurs despite 2 dose decrements, discontinue dexamethasone permanently. |

 $H_2$  = histamine 2 blocker.

Approved




Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


#### 10.5 **DEFINITION OF DOSE-LIMITING TOXICITY**

During this study, assessment of DLTs will occur during the 28-day period of Cycle 1 combination therapy. For the purposes of this study, a DLT is defined as any of the study drug-related events listed below occurring within the 4 weeks after the first dose of combination therapy. Study drug-related is defined as a reasonable likelihood of clinical causality based on time of event, biology, dechallenge improvement and that the AE was not likely explained by the subject's clinical state, underlying disease, concomitant medication, or study/nonstudy procedure.

- Any toxicity requiring a dose reduction or requiring that a dose of oprozomib or pomalidomide be held in Cycle 1 that does not meet the criteria for DLT will be discussed by the CSRC to determine whether the subject should be considered evaluable for DLT determination. If it is determined that the subject is not evaluable for DLT, the subject will be replaced.
- A delay in ability to receive Day 1 dose of Cycle 2 due to a hematologic or nonhematologic drug-related toxicity persisting beyond 14 days from Cycle 1 Day 28 will be considered a DLT
- For a nonhematologic DLT, any  $\geq$  Grade 3 toxicity will be considered a DLT with exceptions as described below:
  - Grade 3 asymptomatic electrolyte abnormalities will not be considered a DLT
  - Asymptomatic Grade 3 hypophosphatemia lasting less than 24 hours will not be considered a DLT
  - Grade 3 nausea and vomiting will not be considered a DLT unless persisting longer than 3 days despite optimal supportive care, which at a minimum must include a 5-hydroxytryptamine type-3 (5-HT<sub>3</sub>) antagonist and aprepitant
  - Grade 3 diarrhea will not be considered a DLT unless persisting longer than 3 days despite optimal supportive care, which at a minimum must include loperamide (Imodium) and atropine diphenoxylate (Lomotil)
  - Grade 3 fatigue lasting < 14 days is not considered a DLT
  - ≥ Grade 3 hyperglycemia or toxicity attributed to dexamethasone is not considered a DLT (see dose reduction guidelines for dexamethasone in Section 10.4.1)
  - Second a DLT

Approved




- Hematologic DLTs consist of the following:
  - o Grade 4 neutropenia:
    - Absolute neutrophil count (ANC) <  $0.5 \times 10^9$ /L lasting ≥ 7 days despite adequate growth factor support (eg, G-CSF)
    - Febrile neutropenia: Any single temperature ≥ 38.3°C or a sustained temperature of  $\geq 38.0^{\circ}$ C for over 1 hour with  $\geq$  Grade 3 neutropenia  $(ANC < 1.0 \times 109/L)$
  - Thrombocytopenia:
    - Grade 4 lasting  $\geq$  7 days, or
    - Grade 4 lasting < 7 days with Grade 2 clinically significant bleeding or < 10,000 platelets requiring platelet transfusion, or
    - Grade 3 with clinically significant bleeding or requiring platelet transfusion.

Note: Grade 4 anemia is not considered a DLT

#### 10.6 CONCOMITANT MEDICATIONS

A concomitant medication is defined as any prescription or over-the-counter preparation, including vitamins and supplements. All concomitant medications from 30 days before Day 1 until 30 days after the subject's last dose of study drug or before start of subsequent anticancer treatment (whichever occurs first) must be recorded on the electronic case report form (eCRF). Blood or blood products are not considered concomitant medications and must be recorded on the appropriate eCRF.

#### 10.6.1 REQUIRED CONCOMITANT MEDICATIONS

#### 10.6.1.1 **Contraception**

Females of reproductive potential must commit either to abstain continuously from heterosexual sexual intercourse or to use 2 methods of effective contraception simultaneously (1 highly effective form of contraception—tubal ligation, intrauterine device [IUD], hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy and 1 additional effective contraceptive method—male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to initiating treatment and continue during therapy, dose interruptions, and for 28 days after discontinuation of therapy. Reliable contraception is indicated even where there has been



Supplemental Clinical Study Report: 20130411


a history of infertility, unless this is due to hysterectomy. Females of reproductive potential should be referred to a qualified provider of contraceptive methods, if needed. Additional details are provided in Pomalidomide Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods (Appendix J), Pomalidomide Education and Counseling Guidance Document (Appendix K), and Pomalidomide Information Sheet for Subjects Enrolled in Clinical Research Studies (Appendix L).

Females of reproductive potential must have 2 negative pregnancy tests before initiating study treatment. The first test should be performed within 10–14 days of study treatment and the second test should be performed within 24 hours before study treatment. Once treatment has started and during dose interruptions, pregnancy testing for female subjects of reproductive potential should occur weekly during the first 4 weeks of treatment. Pregnancy testing should be repeated every 4 weeks thereafter for female subjects with regular menstrual cycles. For female subjects with irregular menstrual cycles (± 7 days of a 28-day cycle), pregnancy testing should be performed every 2 weeks. Pregnancy testing and counseling should be performed if a subject misses her period or if there is any abnormality in her menstrual bleeding. Study treatment must be discontinued during this evaluation.

Postmenopausal females (> 45 years old and without menses for > 2 years) and surgically sterilized females are exempt.

Male subjects must use an effective barrier method of contraception during the study and for 3 months following the last dose if sexually active with a female of childbearing potential.

Because pomalidomide is present in the semen of male subjects who receive it, they must always use a latex or synthetic condom during any sexual contact with females of reproductive potential and for up to 3 months after discontinuation of study treatment, even if they have undergone a successful vasectomy. Male subjects must agree not to donate sperm while being treated and for up to 3 months after discontinuing treatment.

# 10.6.1.2 **Antinausea and Antiemetics**

It is strongly recommended that subjects be premedicated with a 5-HT<sub>3</sub> inhibitor, such as ondansetron or granisetron, prior to administration of the first dose of oprozomib each day





Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


and throughout the day as needed to prevent nausea and vomiting. If nausea/vomiting at any grade persists, aprepitant or fosaprepitant is recommended. Additional antiemetics may be used per investigator discretion.

#### 10.6.1.3 **Antidiarrheals**

For subjects developing any grade of diarrhea, loperamide (Imodium) is strongly recommended at the first onset of symptoms. For subjects with persistent diarrhea despite the use of Imodium, the use of diphonoxylate/atropine (Lomotil) is strongly recommended. Other antidiarrheal agents may be used if necessary; a work-up for other etiologies is suggested if diarrhea continues despite the prior 2 agents.

#### 10.6.1.4 **Antivirals**

Valacyclovir or an equivalent antiviral is recommended for the duration of treatment to prevent Herpes zoster (additional prophylaxis is at the investigator's discretion).

#### 10.6.1.5 **Acid-related Medications**

Lansoprazole or another oral proton-pump inhibitor is required (unless subject has intolerance or hypersensitivity) for the duration of treatment to prevent peptic disease or other GI toxicities.

#### 10.6.1.6 Thrombo-prophylaxis

Aspirin (or other anticoagulant or antiplatelet medication such as clopixisdogrel bisulfate, low-molecular-weight heparin, or warfarin based on subject risk factors for deep vein thrombosis) while taking pomalidomide is required to prevent thrombosis (refer to the Pomalidomide Prescribing Information [Celgene Corporation, 2013] for more information).

#### 10.6.1.7 **Tumor Lysis Syndrome**

Monitoring and Prophylaxis Guidelines: Oral hydration of 1.5–2 liters per 24 hours must be instituted in all subjects 24–48 hours prior to initiation of therapy for every cycle and continued throughout every day of oprozomib dosing. Premedication with allopurinol or other approved uric acid-lowering agents is highly recommended for subjects with high tumor burden (i.e., for multiple myeloma: Durie-Salmon or International Staging System




Stage II/III, or rapidly increasing M-protein or light chains) or compromised renal function (CrCl < 50 cc/min). These subjects may be at elevated risk for TLS and should be closely monitored. Uric acid levels should be normalized prior to initiation of treatment, if appropriate.

### **Tumor Lysis Syndrome Laboratory Abnormalities**

Subjects with laboratory abnormalities prior to dosing that are consistent with lysis of tumor cells (e.g., as defined by abnormalities in at least 3 of the following 4 categories: [1] a 2-fold increase of lactate dehydrogenase above the ULN; [2] increases in serum creatinine, uric acid, or phosphorus > 50% over baseline; [3] potassium increases > 30% above the ULN; or [4] calcium decreases from baseline of > 20% in the absence of concomitant bisphosphonate therapy) (Sezer, 2006). Subjects must not receive the scheduled dose prior to institution of the aforementioned preventive measures.

# **Tumor Lysis Syndrome Treatment Guidelines**

If TLS occurs as defined by the laboratory abnormalities described above, cardiac rhythm, fluid, and serial laboratory monitoring should be instituted. Correction of electrolyte abnormalities, monitoring of renal function and fluid balance, and administration of therapeutic and supportive care, including dialysis, should be done as clinically indicated. In the setting of TLS, oprozomib treatment will be interrupted until resolution of all clinical and laboratory abnormalities consistent with TLS. Once TLS has resolved, the subject can resume treatment at the initial dose level. The **Sponsor's** study medical monitor should be consulted if there is a treatment delay > 4 weeks.

All cases of TLS must be reported to **the Sponsor** as an SAE as outlined in Section 13.5.

#### 10.6.1.8 **Orthostatic Hypotension**

Orthostatic hypotension has been reported in subjects taking oprozomib. The following guidelines should be employed in the management of subjects exhibiting orthostatic hypotension. An etiology should be sought for the orthostatic hypotension to determine if its cause is neurogenic, non-neurogenic or iatrogenic. Dose modifications should be taken in accordance with Table 13 and Table 14.





Supplemental Clinical Study Report: 20130411


- For those subjects with orthostatic hypotension who are taking antihypertensives, the subject's dosage and use of antihypertensive agents should be evaluated and reassessed on an ongoing basis while on study
- Fluid intake should be assessed to confirm the subject is getting appropriate hydration in accordance with protocol requirements of 6–8 eight ounce glasses of fluids in the 24–48 hours prior to dosing and on every day of oprozomib dosing
- Fluid status should be repleted to normal levels in subjects with orthostatic hypotension
- If protocol requirements for oral intake of fluids are already being met, additional measures should be taken to increase blood pressure per investigator discretion, such as increased oral intake, florinef or midodrine, others depending on the etiology. Holding the dose and dose reduction upon resolution may be a consideration.
- Ongoing monitoring of fluid status is warranted and should be managed per investigator discretion
- In addition, vital signs monitoring may be extended beyond the time periods specified in the Schedules of Assessments (Appendices A1, A2, B1, and B2)

### 10.6.2 OPTIONAL AND ALLOWED CONCOMITANT MEDICATIONS

The following medications are optional and are allowed during the study:

- Mycostatin or oral fluconazole to prevent oral thrush is optional and may be given at the investigator's discretion
- Additional antiemetics, antidiarrheal agents, and/or laxatives as necessary
- Myeloid growth factors (eg, G-CSF) may be used if neutropenia occurs, in accordance with American Society of Clinical Oncology (ASCO) Guidelines (Smith, 2006), but are not to be given prophylactically.
- Red blood cell transfusions, erythropoietic stimulating agents, or platelet transfusions, if clinically indicated in accordance with institutional guidelines
- Bisphosphonates
- Palliative radiation for pain management is permitted with the written approval of the Sponsor's study medical monitor

### 10.6.3 EXCLUDED CONCOMITANT MEDICATIONS

In vitro tests indicate that the time-dependent inhibitory effect of oprozomib on human cytochrome P450 3A (CYP3A) is weak (Kinact to KI was only 1.4 mL/min/µmol). However, as a precaution, concomitant use of drugs that are CYP3A substrates with narrow therapeutic range should be avoided within 2 weeks of Day 1 of Cycle 1 and during treatment with oprozomib. Cytochrome P450 3A substrates with narrow therapeutic range are drugs






whose exposure response indicates that increases in their exposure levels by the concomitant use of CYP3A inhibitors may lead to serious safety concerns. Examples of sensitive CYP3A substrates with narrow therapeutic range are provided in Appendix I. Investigators should consider switching to an alternative drug, or be alert to the need for dose adjustment.

In accordance with the Pomalidomide Prescribing Information, use of concomitant medications including CYP3A, cytochrome P450 1A2 (CYP1A2) and P-glycoprotein (P-gp) inhibitors and inducers are to be carefully monitored and substituted for others if necessary (Appendix I).

Glucocorticoid therapy that exceeds a cumulative dose of 160 mg of dexamethasone is not permitted within 21 days prior to randomization. During the study, glucocorticoid therapy (in addition to dexamethasone) is only permitted at the discretion of the **Sponsor's** study medical monitor to treat a concurrent medical condition (eg, asthma, inflammatory bowel disease, emesis, etc.).

Other antimyeloma or investigational agents are not permitted prior to the subject developing confirmed progressive disease.

Plasmapheresis is not permitted at any time during the screening period or while the subject is receiving study treatment. If a subject has started screening procedures requires plasmapheresis, or is anticipated to require plasmapheresis during or after the screening period, this patient will be considered ineligible and should not be enrolled. Subjects requiring plasmapheresis while on study treatment should have every attempt made to document progressive disease by IMWG criteria first, and then will discontinue study treatment and will enter Long Term Follow-up for survival. Subjects requiring plasmapheresis must have 2 serum samples (for SPEP and immunofixation) and at least one 24-hour urine sample (for UPEP and immunofixation) obtained prior to the procedure.

#### 11 **STUDY PROCEDURES**

All protocol-required tests and observations, along with their chronology, are outlined in the Schedules of Assessments (Appendices A1, A2, B1, and B2). A general summary of on-treatment tests and observations is provided below.




#### 11.1 STUDY-SPECIFIC PROCEDURES

#### 11.1.1 **VITAL SIGNS**

All vital sign assessments will include measurement of orthostatic blood pressure, pulse rate, respiration rate, and temperature. Subjects should lie down for 5 minutes and then have blood pressure and pulse measured consistently in either arm. Following the supine blood pressure/pulse reading, the subject should stand and the blood pressure and pulse should be repeated after 1 and 3 minutes. Any drop of 20 mmHg systolic, 10 mmHg diastolic or lightheadedness/dizziness between supine and standing blood pressures would indicate orthostatic hypotension. Usually an increase in pulse of 10 beats/min is associated with but not required for identification of orthostatic hypotension. For time points where PK and vital signs are to be done together, vital signs should be obtained first as the act of phlebotomy may impact vital sign measurement results.

#### 11.1.2 COMPLETE PHYSICAL EXAMINATION

A complete physical examination will include examination of the skin, head and neck, chest (heart and lungs), abdomen, extremities, and a brief neurological examination including an assessment for peripheral neuropathy. Rectal and pelvic examinations are optional. Eastern Cooperative Oncology Group (ECOG) performance status (assessed at the time of the physical examination) will be conducted (Appendix H).

A limited physical examination will include an examination of the chest (heart and lungs) and abdomen, with additional examinations as clinically indicated or directed by AEs.

#### 11.1.3 ELECTROCARDIOGRAM

Twelve-lead electrocardiograms (ECGs), including corrected QT interval (QTc), will be performed locally.

#### 11.2 LABORATORY EVALUATIONS FOR SAFETY

Laboratory tests, including hematology, blood chemistries, and coagulation tests during scheduled visits, will be performed locally. Unscheduled or additional laboratory samples may be collected and analyzed by local laboratories if results are necessary for management of treatment-emergent AEs or dose modification.






The schedule for laboratory evaluations for safety is outlined in Appendices A1, A2, B1, and B2. The laboratory tests included in the full chemistry panel are defined in Table 16.

### 11.2.1 CHEMISTRY

**Table 16 Full Chemistry Panel** 

| Full Chemistry Panel | |
|-----------------------------------------------|-----------------------|
| Alanine aminotransferase | Glucose |
| Albumin | Lactate dehydrogenase |
| Alkaline phosphatase | Magnesium |
| Aspartate aminotransferase | Phosphorous |
| Bicarbonate | Potassium |
| Blood urea nitrogen | Sodium |
| Calcium | Total bilirubin |
| Chloride | Total protein |
| Creatinine | Uric acid |
| Creatinine clearance (calculated or measured) | |

### 11.2.2 HEMATOLOGY

The complete blood count (CBC) with differential includes the following:

- Hemoglobin
- Hematocrit
- White blood cell (WBC) count with complete manual or automated differential (reported as absolute counts)
  - o Total neutrophils
  - Lymphocytes
  - Monocytes
  - Eosinophils
  - o Basophils
- Red blood cell count
- Platelet count

Approved




#### 11.2.3 **COAGULATION**

- Prothrombin time
- Activated partial thromboplastin time
- International normalized ratio

#### PREGNANCY 11.2.4

For females of childbearing potential (FCBP), both a serum pregnancy test that is confirmed negative at Screening and a serum pregnancy test that is confirmed negative within 24 hours prior to Day 1 of each cycle is required prior to dosing. For the first cycle, negative pregnancy tests are required weekly. Starting with the second cycle, a negative pregnancy test monthly is required. For FBCP subjects with irregular menses (ie, other than  $28 \pm 7$  days) or whose menses are not present, a negative pregnancy test every other week is required. More frequent pregnancy tests may be conducted if required according to local regulations.

#### 11.3 DISEASE RESPONSE ASSESSMENTS

The schedule of disease assessments for treated subjects is provided in Appendices A1, A2, B1, and B2. Disease response will be assessed by the investigator. Beginning with Cycle 1, assessments are to be completed at the end of every 4-week cycle for the first 18 months of study treatment, and then at the end of every other cycle (every 8 weeks), beginning with Month 20, for the remainder of study treatment. Response assessment will be according to the IMWG-URC and modified EBMT guidelines (Appendix C). Disease response and progression assessments include:

- Serum protein electrophoresis (SPEP)
- Urine protein electrophoresis (UPEP)
- Serum immunofixation, serum free light chain (SFLC)
- Urine immunofixation
- Serum calcium
- Bone marrow sample as clinically indicated to confirm CR
- Radiographic assessments including plasmacytoma evaluation if baseline assessments were positive and as clinically indicated per the response criteria





Date: 30 July 2019


Skeletal survey if baseline assessments were positive and as clinically indicated per the response criteria

Serum protein electrophoresis and immunofixation assessments will be conducted according to the schedule outlined in Appendices A1, A2, B1, and B2, Schedule of Assessments. Immunofixation will only be required after Screening, Baseline (Day -7 to 1), and End of Study Treatment, if results of the previous SPEP are zero/undetectable.

Urine protein electrophoresis and immunofixation will be performed on a 24-hour urine specimen collected from all subjects during the Screening period, Baseline (Day -7 to 1), and at the End of Study Treatment visit. The UPEP with 24-hour urine collection will be conducted according to the schedule outlined in Appendices A1, A2, B1, and B2, Schedule of Assessments, and is required: 1) only if Baseline UPEP was  $\geq 200 \text{ mg}/24 \text{ hours}$ , and 2) to confirm a disease response or disease progression. If the Baseline UPEP was negative, spot urine is required at each time point. If positive for paraprotein, a 24-hour urine collection with UPEP must be done at the next assessment and at each subsequent assessment unless the UPEP shows an absence of paraprotein.

Serum free light chain assay and kappa:lambda  $(K/\lambda)$  ratio will be conducted according to the schedule outlined in the Schedule of Assessments, Appendices A1, A2, B1, and B2. Only in subjects without measurable serum and urine M-protein levels (serum M-protein < 0.5 g/dL or urine M-protein < 200 mg/24 hours) at Baseline will SFLC assays be used to determine eligibility and response. In subjects with measurable SPEP and/or UPEP, SFLC may be used in conjunction with those assessments to determine response per disease response criteria but only SPEP and/or UPEP will be used to determine eligibility.

All response categories (CR, sCR, VGPR, PR, MR, PD) require 2 consecutive assessments made at any time before the institution of any new therapy. All subjects will be followed until disease progression (confirmed by 2 consecutive measurements that are also verified by the **Sponsor's** medical monitor prior to treatment discontinuation), unacceptable toxicity, or withdrawal of consent, whichever occurs first.

Disease progression will be determined and confirmed with the medical monitor by two consecutive assessments using the IMWG-URC (Appendices A1, A2, B1, and B2).



Supplemental Clinical Study Report: 20130411


Serum M component increases of  $\geq 1.0$  g/dL are sufficient to define progression if the starting component is  $\geq 0.5$  g/dL according to these criteria. However, it is understood from these criteria that a single measurement is adequate in cases of clear increased bone marrow plasma cell percentage, development of new or worsened bone lesions from a skeletal survey, or development of new or worsened soft tissue plasmacytomas.

# 11.4 CORRELATIVE STUDIES

### 11.4.1 PHARMACOKINETIC MEASUREMENTS

In the dose-escalation and dose-expansion portions of the study, blood samples will be collected from all subjects from both schedules to measure plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose) and 1 predose time point on Day 2 of Cycle 1. Estimates of oprozomib PK parameters will be determined when possible.

# 11.4.2 PHARMACODYNAMIC MEASUREMENTS

In the dose-escalation and dose-expansion portions of the study, blood samples for the quantitation of proteasome inhibition by oprozomib will be collected from all subjects for both schedules at 1 predose time point, up to 2 postdose time points (4 and 6 hours postdose) on Day 1 of Cycle 1 and Cycle 2, and 1 predose timepoint on Day 2 of Cycle 1. These timepoints are also specified in the Laboratory Manual. Details about collection times and volumes, and processing and shipping of PDn samples, are provided in the Laboratory Manual. Measurement of proteasome activity in whole blood and peripheral blood mononuclear cells (PBMCs) will be performed using a fluorogenic substrate assay and/or enzyme-linked immunosorbent assay.

### 11.4.3 GENOMIC MEASUREMENTS

Analysis of genomic biomarkers that may predict for response and resistance following treatment with proteasome inhibitors will be conducted for all subjects **in** the study who consent to optional genomic biomarker analysis. These analyses will be performed on the required bone marrow aspirate obtained at Baseline (within 45 days prior to Cycle 1 Day 1 dosing; a portion of the bone marrow aspirate sample obtained at Baseline will be used; no





Supplemental Clinical Study Report: 20130411


additional sample is required), as well as a sample of blood and saliva, also collected at Baseline. Bone marrow aspirate or biopsy collection does not need to be repeated if previously completed within 45 days prior to Cycle 1 Day 1 dosing. Additional bone marrow samples for biomarkers may be collected at disease progression (End of Study Treatment due to PD) from all subjects who consent.

Whole genome sequencing (WGS), whole exome sequencing (WES), whole transcriptome sequencing, and/or other methods of nucleic acid quantification will be conducted on isolated tumor (CD138<sup>+</sup>) cells from bone marrow samples taken at Baseline and disease progression. In addition, WGS or WES will be performed on a normal tissue sample (eg, saliva or peripheral blood) in order to determine the presence of somatic mutations in tumor cell samples. Data will be analyzed to examine specific hypotheses about whether drug response is related to alterations in genes regulated by or involved in activation of nuclear factor kappa light chain enhancer of activated B cell (NF-κB) transcription factors as well as genes involved in immunoglobulin production and plasma cell protein homeostasis. Immunoglobulin levels in tumor cells will be quantified by enzyme-linked immmunosorbent assay (ELISA) and/or other protein quantification methods. These data will also be used to derive new hypotheses about mechanisms of drug response, resistance, and safety.

The schedule for genomic sampling is provided in the Laboratory Manual and in the Schedule of Assessments (Appendices A1, A2, B1, and B2).

#### 11.5 PATIENT-REPORTED OUTCOMES ASSESSMENTS

Beginning with Cycle 1, HRQoL/PRO assessments are to be completed at the beginning of every cycle prior to drug administration through End of Study Treatment/Early Discontinuation visit during the dose-expansion portion of the trial, and at the beginning of every cycle prior to drug administration through End of Study Treatment/Early Discontinuation visit. The HRQoL/PRO assessments include:

- BPI-SF (See Appendix M for a sample Brief Pain Inventory Short Form)
- EORTC QLQ-C30 (Appendix D)
- EORTC QLQ-MY20 (Appendix D)





Supplemental Clinical Study Report: 20130411


• Neurotoxicity subscale of the FACT/GOG-Ntx4 (Version 4; Appendix E)

• EQ-5D-5L (Appendix F)

# 12 STUDY AND STUDY TREATMENT DISCONTINUATION

Early discontinuation and End of Study Treatment assessments must be performed within 30 days following the subject's last dose of study drug and prior to initiation of any other treatment.

All subjects must complete a visit approximately 4 weeks after the last cycle of treatment to allow for safety follow-up 30 days after the last dose of oprozomib. An individual subject who discontinues study treatment for PD will be followed for OS in long-term follow-up. Any subject who withdraws without PD will **no longer** be followed with long-term assessments every 4 weeks through 18 months on study, and then every 8 weeks thereafter, beginning with Month 20, until progression or initiation of next therapy **under**Amendment 3. The study will be completed once the last subject completes the last required follow-up visit. The same methods of disease assessment must be used throughout the study. If 2 prior disease assessments show disease progression, assessments do not need to be repeated with End of Study Treatment assessments.

### 12.1 STUDY TREATMENT DISCONTINUATION

For this study, subjects may withdraw from study treatment at any time.

The investigator may remove a subject from study treatment for the following reasons:

- Disease progression
- Unacceptable toxicity
- Noncompliance with study procedures
- Need of treatment with medications not allowed by the study protocol
- Subject no longer consents to participate in the study
- Intercurrent illness that interferes with study assessments
- Suspected pregnancy

The primary reason for treatment discontinuation will be documented in the eCRF.





Supplemental Clinical Study Report: 20130411


If the reason for treatment discontinuation is the occurrence of an AE, the subject will be followed by the investigator until such event(s) resolve, stabilize, or, according to the investigator's judgment, there is no need of further follow-up.

Subjects who discontinue from study treatment will be monitored for AEs for 30 days after the last dose of oprozomib or immediately before the start of subsequent anticancer treatment (whichever occurs first). Treatment discontinuation due to progression should be recorded on the Study Drug Completion/Discontinuation eCRF as "Disease Progression." Verbatim terms such as "disease progression," "progressive disease," etc. should not be reported as AEs or SAEs as outlined in Section 13.3.2 unless the investigator considers the progression to be atypical, accelerated, or caused by the study drug, in which case it should also be recorded as an SAE in the AE eCRF.

**The Sponsor**, or designee must be notified within 24 hours if a subject is withdrawn from treatment for any reason (ie, disease progression, toxicity, etc.). Disease progression with 2 consecutive disease assessments must be confirmed by the medical monitor before any subject is discontinued from study treatment.

For dose escalation and expansion, subjects who withdraw from treatment before completing adequate safety or efficacy evaluations, or Cycle 1 dosing, will be considered unevaluable and may be replaced. Additional subjects may be enrolled to account for subjects who have not had adequate safety or efficacy evaluations.

### 12.2 STUDY DISCONTINUATION

Each subject will be followed until death or study closure. The reason for discontinuation from the study will be documented on the eCRF.

Reasons for complete withdrawal from the study (treatment and all follow-up) before documentation of subject death include:

- Withdrawal of consent
- Lost to follow-up
- Sponsor decision


Approved



Supplemental Clinical Study Report: 20130411


### 12.3 LONG-TERM FOLLOW-UP

After completion of the End of Study Treatment visit, subjects will be followed for OS. Subjects will be followed based on their disease progression status at End of Study Treatment.

### **Progression and Overall Survival**

- For subjects who have not progressed at end of study treatment, disease response assessments will **no longer** be performed every 4 weeks through 18 months on study, and then every 8 weeks thereafter, beginning with Month 20, until progression or initiation of next therapy **under Amendment 3**
- Subjects who have progressed at end of study treatment or long-term follow-up will be followed for survival status approximately every 3 months, or as needed

Long-term follow-up will continue until the subject has withdrawn consent for further participation, is lost to follow-up, has died, or the sponsor makes a decision to close the study. For any subject who is lost to follow-up, the study site will attempt to ascertain survival information via public database search.

### 12.4 STUDY TERMINATION

**The Sponsor** has the right to terminate this study, either schedule, or a study site from participating in a study at any time. Reasons for terminating the study overall or at a specific study site may include, but are not limited to, the following:

- The incidence or severity of AEs in this or other studies indicates a potential health hazard to subjects
- Subject enrollment is unsatisfactory
- Data recording is inaccurate or incomplete
- Investigator does not adhere to the protocol or applicable regulatory requirements in conducting the study

### 13 ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS

### 13.1 ADVERSE EVENT REPORTING

# 13.1.1 DEFINITIONS

An AE is any untoward medical occurrence in a study subject administered an investigational product(s) regardless of the causal relationship with treatment.






An AE, therefore, can be any unfavorable and unintended sign (including laboratory finding), symptom, or disease temporally associated with participation in an investigational study, whether or not considered drug-related. In addition to new events, any increase in the severity or frequency of a preexisting condition that occurs after the subject signs the informed consent form (ICF) for participation is considered an AE. This includes any side effect, injury, toxicity, or sensitivity reaction. All reported AEs will be coded using the current version of Medical Dictionary for Regulatory Activities (MedDRA).

Whenever possible, the NCI-CTCAE Version 4.03 should be used to describe the event and for assessing the severity of AEs. For AEs not adequately addressed in the NCI-CTCAE Version 4.03, Table 17 below should be used.

Table 17 Toxicity Grading for Adverse Events Not Covered in the NCI-CTCAE (Version 4.03)

| Severity | Description |
|---|---|
| GRADE 1 - Mild | Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| GRADE 2 – Moderate | Minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL) |
| GRADE 3 – Severe | Medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL |
| GRADE 4 – Life-threatening | Life-threatening consequences; urgent intervention indicated |
| GRADE 5 – Fatal | Death |

NCI-CTCAE = National Cancer Institute-Common Terminology Criteria for Adverse Events

An AE or suspected adverse reaction is considered "unexpected" if it is not listed in the current IB or is not listed at the specificity or severity that has been observed. Adverse events or suspected adverse reactions that are mentioned in the IB as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with a particular study drug, are considered "unexpected." For example, an event more specific or more severe than described in the IB would be considered "unexpected." Any condition, laboratory abnormality, or physical finding with an onset date prior to the subject signing the ICF is considered to be preexisting in nature and part of the subject's medical history.





Supplemental Clinical Study Report: 20130411


Abnormal laboratory findings should be reported as AEs if medical intervention or corrective action (eg, transfusions, initiation of antibiotics or other treatment regimens, hydration, study drug placed on hold) is required or the event is deemed clinically significant by the treating physician.

### 13.2 CAUSALITY

A suspected adverse event means any AE for which there is reasonable possibility that the study drug caused the AE. "Reasonable possibility" means that there is evidence to suggest a causal relationship between the drug and the AE.

The relationship of the AE to the study drug should be assessed using the following criteria:

YES; the event is suspected to be related if:

- There is a clinically plausible time sequence between the AE onset and administration of study treatment; and/or
- There is a biologically plausible mechanism for the study treatment to cause or contribute to the AE; and/or
- The event improves or diminishes upon withdrawal of the study drug without the initiation of any specific treatment for the event (dechallenge) and/or recurs or worsens with rechallenge (when clinically feasible); and/or
- The AE cannot be reasonably attributed to concurrent or underlying illness, other drugs, or procedures

NO; the event is not suspected to be related if:

- The AE is more likely to be explained by the subject's clinical state, underlying disease, or concomitant medical, study, or nonstudy procedure; and/or
- The time of occurrence of the AE is not reasonably related to administration of study treatment; and/or
- The event is not related to the investigational product(s)

In the event of a possible drug-related AE, the investigator should to the best of his/her ability assess its relationship to each of the study drugs: oprozomib, pomalidomide, and dexamethasone.

Approved




#### 13.3 ADVERSE EVENTS REPORTING PROCEDURES

#### 13.3.1 **GENERAL**

All AEs (eg, any new event or worsening in severity or frequency of a preexisting condition or laboratory finding) with an onset date after the subject signs the informed consent for participation in the clinical trial must be promptly documented on the AE eCRF via the electronic data capture (EDC) system. Details of the event must include severity, relationship to study drug(s), duration, action taken, and outcome. Whenever possible, reporting a specific diagnosis is preferred when reporting AEs in the AE eCRF rather than reporting individual signs and symptoms.

All AEs will be collected from the time the subject signs informed consent through 30 days after receiving the last dose of study drug or before start of subsequent anticancer treatment (whichever occurs first). If initiation of new anticancer therapy occurs following the last dose of study drug(s), the date of new anticancer therapy will be recorded on the appropriate eCRF. In addition, the investigator should report any AEs that may occur after this time period that are assessed to have a reasonable possibility of being associated with study drug. If the subject is randomized but discontinues participation in the study prior to receiving study drug, AEs must be reported through the End of Study Treatment visit.

All AE severity changes will be recorded on the AE case report form (CRF) as separate events. All AEs that are considered related to study drug and all SAEs regardless of relationship to study drug must be followed to resolution or to stabilization if improvement is not expected. Adverse events that completely resolve and then recur should be recorded as a new AE. For subjects who complete the End of Study Treatment visit less than 30 days following the last dose of study drug, a follow-up of ongoing AEs should be attempted by telephone and documented in the subject's source file. Adverse events continuing at 30 days after the last dose of study treatment should have a comment in the source file by the investigator that the event has stabilized or is not expected to improve.

Approved



Supplemental Clinical Study Report: 20130411


The investigator is responsible for evaluating all AEs, obtaining supporting source documents, and determining that documentation of the event is adequate. The investigator may delegate these duties to subinvestigators and must ensure that these subinvestigators are qualified to perform these duties under the supervision of the investigator and that they are listed on the FDA Form 1572.

### 13.3.2 DISEASE PROGRESSION

Disease progression will be documented on an eCRF intended to capture PD information and will be analyzed as a study endpoint. Signs and symptoms related to disease progression (eg, pathologic fracture in a subject with progressive multiple myeloma) should be reported in the appropriate case report form as an AE or as a SAE (if the event in question meets the criteria for seriousness) while the cause of study treatment discontinuation should be reported as progression of disease. Verbatim terms such as "disease progression," "progressive disease," etc. should not be reported as AEs or SAEs unless the investigator considers the progression to be atypical, accelerated, or caused by the study drug. Similarly, deaths occurring as a result of disease progression should be reported on the eCRF intended to capture death information and should not be reported as SAEs.

### 13.4 SERIOUS ADVERSE EVENTS DEFINITIONS

An SAE is an AE that meets 1 or more of the following criteria:

- Death
- Life-threatening experience, defined as any adverse experience that places the subject, in the view of the sponsor or investigator, at immediate risk of death at the time of occurrence; ie, it does not include a reaction that, had it occurred in a more severe form, might have caused death
- Requires inpatient hospitalization or prolongation of an existing hospitalization (except scheduled hospitalizations for a nonacute, unrelated cause such as elective surgery)
- Results in persistent or significant disability/incapacity (ie, substantial disruption in a subject's ability to conduct normal activities of daily living)
- Is a congenital anomaly/ birth defect in the offspring of an exposed female subject or offspring of a female partner of a male subject





Supplemental Clinical Study Report: 20130411


Important medical events that may not result in death, be life-threatening, or require
hospitalization may be considered an SAE when, based on appropriate medical judgment,
the event jeopardizes the subject and may require medical or surgical intervention to
prevent 1 of the outcomes listed in this definition

# 13.5 SERIOUS ADVERSE EVENT REPORTING AND DOCUMENTATION REQUIREMENTS

Amgen Global Patient Safety must be notified of the occurrence of any SAE within 24 hours of the investigator, designee, or site personnel's knowledge of the event. The SAE will be reported by completing and submitting the SAE report form through the EDC system. In the event that the EDC system is not available, paper SAE report forms may be used to report the SAE to Amgen Global Patient Safety. Please refer to the SAE Reporting Guidelines below.

The primary mechanism for reporting serious adverse events will be the EDC via the Safety Report Form. If the EDC system is unavailable for more than 24 hours, then the site will report the information to Amgen using an electronic Serious Adverse Contingency Report Form (see Appendix N) within 24 hours of the investigator's knowledge of the event. The site will enter the serious adverse event data into the electronic system as soon as it becomes available.

After the study is completed at a given site, the EDC system will be taken off line to prevent the entry of new data or changes to existing data.

If a site receives a report of a new serious adverse event from a study subject or receives updated data on a previously reported serious adverse event after the EDC has been taken off line, then the site can report this information on a paper Serious Adverse Event Report Form (see Appendix N).

If a subject is permanently withdrawn from protocol-required therapies because of a serious adverse event, this information must be submitted to Amgen.

New or updated information will be recorded in the originally completed Event CRF.





Supplemental Clinical Study Report: 20130411


The investigator will submit any updated serious adverse event data to Amgen Global Patient Safety within 24 hours of receipt of the information.

The investigator is responsible for notifying the Institutional Review Board (IRB) or Independent Ethics Committees (IEC), in accordance with local regulations, of all SAEs. The sponsor may request additional source documentation pertaining to the SAE from the investigational site. If a subject is permanently withdrawn from the study due to an SAE, this information must be included in the initial or follow-up SAE report in the eCRF.

The sponsor is responsible for notifying the appropriate global health authorities of SAEs, when required, and in accordance with applicable laws and regulations.

### 13.6 PREGNANCY REPORTING

Pregnancy occurring in a female subject, or in a male subject's partner, while enrolled in this clinical trial through 30 days after the subject's last dose of study drug, although not considered an SAE, must be reported to **Amgen Global Patient** Safety on an **Amgen** Pregnancy **Notification Worksheet (Appendix O)** within 24 hours of the investigator, designee, or site personnel learning of the event. If the subject is pregnant, all study treatment must be discontinued immediately and the pregnancy must be reported to the investigator and sponsor within 24 hours. **To report a pregnancy to Amgen Global Patient Safety, please refer to the pregnancy reporting guidelines below.** 

### **Collection of Pregnancy Information**

### Female Subjects Who Become Pregnant

- Investigator will collect pregnancy information on any female subject who becomes pregnant while taking protocol-required therapies through 30 days after stopping oprozomib.
- Information will be recorded on the Pregnancy Notification Worksheet (Appendix O). The worksheet must be submitted to Amgen Global Patient Safety within 24 hours of learning of a subject's pregnancy. Note: Sites are not required to provide any information on the Pregnancy Notification Worksheet that violates the country or regions local privacy laws.
- After obtaining the female subject's signed authorization for release of pregnancy and infant health information, the investigator will collect pregnancy





Supplemental Clinical Study Report: 20130411


and infant health information and complete the pregnancy questionnaire for any female subject who becomes pregnant while taking protocol-required therapies through 30 days after stopping oprozomib. This information will be forwarded to Amgen Global Patient Safety. Generally, infant follow-up will be conducted up to 12 months after the birth of the child (if applicable).

- Any termination of pregnancy will be reported to Amgen Global Patient Safety, regardless of fetal status (presence or absence of anomalies) or indication for procedure.
- While pregnancy itself is not considered to be an adverse event or serious adverse event, any pregnancy complication or report of a congenital anomaly or developmental delay, fetal death, or suspected adverse reactions in the neonate will be reported as an adverse event or serious adverse event. Note that an elective termination with no information on fetal congenital malformation or maternal complication is generally not considered an adverse event, but still must be reported to Amgen as a pregnancy exposure case.
- If the outcome of the pregnancy meets a criterion for immediate classification as a serious adverse event (eg, female subject experiences a spontaneous abortion, stillbirth, or neonatal death or there is a fetal or neonatal congenital anomaly) the investigator will report the event as a serious adverse event.
- Any serious adverse event occurring as a result of a post-study pregnancy which
  is considered reasonably related to the study treatment by the investigator will
  be reported to Amgen Global Patient Safety as described in Section 13.5. While
  the investigator is not obligated to actively seek this information in former study
  subjects, he or she may learn of a serious adverse event through spontaneous
  reporting.
- Any female subject who becomes pregnant while participating will discontinue study treatment.

Male Subjects With Partners Who Become Pregnant or Were Pregnant at the Time of Enrollment

- In the event a male subject fathers a child during treatment, and for an additional 90 days after discontinuing protocol-required therapies, the information will be recorded on the Pregnancy Notification Worksheet (Appendix O). The worksheet must be submitted to Amgen Global Patient Safety within 24 hours of the site's awareness of the pregnancy. Note: Sites are not required to provide any information on the Pregnancy Notification Worksheet that violates the country or regions local privacy laws.
- The investigator will attempt to obtain a signed authorization for release of pregnancy and infant health information directly from the pregnant female partner to obtain additional pregnancy information.





Supplemental Clinical Study Report: 20130411


- After obtaining the female partner's signed authorization for release of pregnancy and infant health information, the investigator will collect pregnancy outcome and infant health information on the pregnant partner and her baby and complete the pregnancy questionnaires. This information will be forwarded to Amgen Global Patient Safety.
- Generally, infant follow-up will be conducted up to 12 months after the birth of the child (if applicable).
- Any termination of the pregnancy will be reported to Amgen Global Patient Safety regardless of fetal status (presence or absence of anomalies) or indication for procedure.

### **Collection of Lactation Information**

- Investigator will collect lactation information on any female subject who breastfeeds while taking protocol-required therapies through 30 days after stopping oprozomib.
- Information will be recorded on the Lactation Notification Worksheet (Appendix P) and submitted to Amgen Global Patient Safety within 24 hours of the investigator's knowledge of event.
- Study treatment will be discontinued if female subject breastfeeds during the study as described in exclusion criterion 22.

With the female subjects signed authorization for release of mother and infant health information, the investigator will collect mother and infant health information and complete the lactation questionnaire on any female subject who breastfeeds while taking protocol-required therapies through 30 days after discontinuing protocol-required therapies.

### 14 STATISTICS

This section outlines the statistical analysis strategy and procedures for the study. Specific details of the primary and key secondary analyses will be provided in the Statistical Analysis Plan (SAP). If, after the study has begun but prior to the final analysis, important changes are made to the protocol that affect principal features of the primary and/or key secondary analyses, then the protocol and/or SAP will be amended, as appropriate. Any other changes made to the planned analyses after the protocol and SAP have been finalized, along with an explanation as to when and why they occurred, will be described in the Clinical Study Report, in which any post hoc exploratory analyses also will be clearly identified.





Supplemental Clinical Study Report: 20130411


### 14.1 STUDY ENDPOINTS

### 14.1.1 PRIMARY ENDPOINTS

- DLTs
- Adverse events and laboratory abnormalities graded according to NCI-CTCAE, Version 4.03
- Vital signs and clinical laboratory results during and following study drug administration

### 14.1.2 SECONDARY ENDPOINTS

- Overall response, defined as the best response of sCR, CR, VGPR, or PR, as determined by investigator according to the IMWG-URC
- Clinical benefit, defined as defined as the best response of MR or better, as determined by investigator according to the IMWG-URC and modified EBMT criteria
- Pharmacokinetic parameters, including maximum plasma concentration (C<sub>max</sub>), time to maximum concentration (T<sub>max</sub>), area under the plasma concentration time curve from time 0 to last time point (AUC<sub>0-τ</sub>), and area under the plasma concentration time curve from time 0 to time infinity (AUC<sub>0-∞</sub>) using noncompartmental methods

# 14.1.3 EXPLORATORY ENDPOINTS

- Pharmacodynamic biomarkers that may be correlated with antitumor activity
- Genomic biomarkers that may be correlated with antitumor activity and resistance following treatment with proteasome inhibitors
- Change over time in bone pain and the impact of bone pain measured with the BPI-SF (Dose Expansion only)
- Change over time in the global health status/QoL scale of the EORTC QLQ-C30 (Dose Expansion only)
- Change over time in health status assessed by EQ-5D-5L (Dose Expansion only)
- Change over time in the disease symptoms subscale of the EORTC QLQ-MY20 (Dose Expansion only)
- Change over time in neurotoxicity symptoms measured by the FACT/GOG-Ntx4 score (Version 4) (Dose Expansion only)

### 14.2 ANALYSIS OF THE CONDUCT OF THE STUDY

Enrollment, subject disposition, study treatment administration, and discontinuation from the study will be summarized. Eligibility exceptions and important protocol deviations will be summarized.






#### 14.3 **DATA MONITORING COMMITTEE**

In this study, safety will be monitored by a CSRC for both the dose-escalation and dose-expansion portions of the study.

#### 14.4 ANALYSIS OF TREATMENT GROUP COMPARABILITY

Descriptive statistics will be used to summarize baseline subject characteristics. Summaries of discrete data will include number of subjects and incidence as a frequency and as a percentage. Summaries of continuous data will include mean, standard deviation, median, minimum, maximum, and sample size.

#### 14.4.1 TREATMENT EXPOSURE AND MEDICATION COMPLIANCE

Extent of exposure to all study treatments (oprozomib, pomalidomide, and dexamethasone) will be evaluated by summary statistics (N, mean, standard deviation, median, and range). Percentage of subjects and cycles with dose delays and reductions will be calculated by treatment group.

The dose intensity of oprozomib, pomalidomide, and dexamethasone (ie, the amount of drug delivered to a subject per week of treatment) will be calculated according to standard methodology (Hryniuk, 1990; Longo, 1991) that accounts for treatment delays on the calculated dose intensity result. For each subject, the relative dose intensity (actual versus planned) of each treatment will be calculated. The average relative dose intensity for each treatment group will be calculated by summarizing the average relative dose intensity for individual subjects. The results for pomalidomide and dexamethasone will be provided to determine the presence of any major differences between the treatment groups for the planned versus actual dose and schedule of these two (2) study medications.




#### 14.5 STATISTICAL METHODS

#### 14.5.1 ANALYSIS POPULATIONS

#### 14.5.1.1 **Safety Population**

All subjects receiving any amount of study treatment (oprozomib, pomalidomide, or dexamethasone) will be included in safety analyses. A baseline measurement and at least 1 laboratory, vital sign, or ECG measurement obtained after any amount of study treatment is required for inclusion in the analysis of a specific safety parameter when applicable.

#### 14.5.1.2 **Efficacy Population**

For this study, the efficacy population is equivalent to the safety population.

#### 14.5.1.3 **PK-Evaluable Population**

Subjects evaluable for PK are defined as those who have adequate oprozomib plasma concentration-versus-time data to allow proper estimation of PK parameters.

#### 14.5.2 EFFICACY ANALYSES

Overall response rate is defined as the proportion of subjects with a best response of sCR, CR, VGPR, or PR as determined by investigator according to the IMWG-URC.

Clinical benefit rate is defined as the proportion of subjects with a best response of PR or better according to IMWG-URC or a best response of MR according to the EBMT criteria, as determined by the investigator. A point estimate and 95% exact binomial confidence interval (CI) will be calculated for both ORR and CBR for all subjects treated at the RP3D (during dose escalation and expansion for each schedule). A descriptive summary of ORR and responses will also be provided by dose cohort.

Progression-free survival and duration of response (DOR) will be listed for all subjects in the efficacy population by dose cohort level and schedule.

Approved



Supplemental Clinical Study Report: 20130411


#### 14.5.3 SAFETY ANALYSIS

The safety population will be used in all safety analyses (see Section 14.5.1.1).

For this study, safety data will be summarized for each cohort and for the pooled cohorts. Safety will be assessed through summaries of DLTs, AEs, changes in laboratory test results, ECGs, vital signs, and oprozomib, pomalidomide, and dexamethasone exposure. Subgroup Analyses and Effects of Baseline Factors

To determine whether the treatment effect is consistent across various subgroups, the estimate of the hazard ratio (or odds ratio) for treatment group (with 95% CI) will be provided for the primary and selected secondary efficacy endpoints and plotted within each of the following baseline variables, provided there is a reasonable sample size in the subgroups of interest:

- Number of prior therapies: 2 versus 3 or more (stratification factor)
- Age (< 75 years versus  $\ge 75$  years) (stratification factor)
- Prior carfilzomib (naïve/sensitive versus refractory) (stratification factor)
- Refractory status: Primary refractory versus relapsed-refractory versus bortezomib-intolerant
- Refractory to lenalidomide
- Refractory to bortezomib
- Double refractory (refractory to lenalidomide and bortezomib)
- FISH risk status: High-risk group versus standard-risk group.
- No prior transplant versus prior transplant
- Bone marrow infiltration by plasma cells  $\leq 50\%$  versus > 50% at baseline
- Renal function  $\leq 60 \text{ mL/min versus} > 60 \text{ mL/min at baseline}$
- Age (< 65 years versus  $\ge 65$  years)
- Race (Caucasian versus all others)
- Sex (male versus female)

#### 14.5.4 PHARMACOKINETIC ANALYSES

In the Dose-Escalation and Dose-Expansion portions of the study, blood samples will be collected from all subjects for determination of plasma concentrations of oprozomib at


Approved



Supplemental Clinical Study Report: 20130411


1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose) and 1 predose time point on Day 2 of Cycle 1 for both schedules. Individual and mean plasma-concentration-versus time data will be tabulated and plotted by dose level.

The PK parameter estimates for oprozomib will be summarized, including total plasma exposure (AUC), maximum plasma concentration (C<sub>max</sub>), time to maximum concentration  $(T_{max})$ , total plasma clearance, and plasma terminal half-life  $(t_{1/2}$ , as appropriate for data collected). Estimates for these parameters will be tabulated and summarized (mean, standard deviation).

Unless otherwise specified, the PK parameter will be estimated based on noncompartmental methods. These estimates will be summarized descriptively by dose cohort. Exploratory analyses may be performed to evaluate the relationship between the estimate PK parameters and selected safety, biomarker, or clinical effect endpoints.

#### 14.6 HANDLING OF MISSING DATA

Missing data for partial dates on AEs or concomitant medication may be imputed according to prespecified, conservative imputation rules. Censoring rules for PFS, OS, and DOR and details about the handling of missing data are explained in the SAP.

#### 14.7 **DETERMINATION OF SAMPLE SIZE**

A total enrollment of approximately 82 subjects is planned for this study. During the dose-escalation portion of the study, approximately 21 subjects are expected to be enrolled for each schedule. The estimated sample size for the dose-escalation part of the study is based on standard 3 + 3 dose-escalation rules, with expectations that 2-3 dosing cohorts of 3–6 subjects per cohort will be required to establish the MTD. A minimum of 6 subjects must be treated at the MTD. For each schedule, more than 1 MTD for oprozomib may be established if additional dose levels of pomalidomide are assessed. The MTD for oprozomib in combination with each dose level of pomalidomide will be the dose(s) where < 2 DLTs in 6 subjects are observed.





Date: 30 July 2019


The actual number of required subjects will depend on both the total number of cohorts, and the need to expand a given cohort from 3 to 6 subjects in order to identify the MTD. Properties of the dose-escalation rules for different underlying DLT rates are provided in Table 18.

Table 18 Properties of the Dose-Escalation Rules for Different Underlying DLT Rates

| Underlying Rate<br>of DLT | Probability of Enrolling<br>3 Additional Subjects | Probability that Dose is<br>Determined to be Tolerated |
|---|---|---|
| 0.10 | 0.24 | 0.91 |
| 0.20 | 0.38 | 0.71 |
| 0.33 | 0.44 | 0.43 |
| 0.40 | 0.43 | 0.31 |
| 0.50 | 0.38 | 0.17 |
| 0.60 | 0.29 | 0.08 |

DLT = dose-limiting toxicity.

The criteria for selecting the RP3D for each schedule at the sponsor's discretion will include assessment of the safety, tolerability, and preliminary activity of oprozomib observed across multiple cycles. In addition, both PK and PDn assessments to demonstrate adequate exposure and proteasome inhibition will be a key factor. The CSRC will review the data and provide guidance in selection of the RP3D. Therefore the RP3D may differ from the MTD, but will not be higher than the MTD. A minimum of 20 additional subjects are planned for enrollment and treatment for 1 or both schedules at the sponsor's discretion at the RP3D during the dose-expansion portion of the study. In the dose-expansion portion of the study, if the true  $ORR \ge 40\%$ , then the probability of seeing at least 7 responses among the 26 subjects (6 treated at the MTD during escalation + 20 in the expansion) is approximately 94%.



Date: 30 July 2019

#### 15 ETHICAL AND ADMINISTRATIVE CONSIDERATIONS

#### 15.1 **COMPLIANCE STATEMENT**

This study will be conducted in accordance with the protocol and with International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines, as well as all applicable country and regional legal and regulatory requirements. The investigator is responsible for ensuring that this protocol, the site's informed consent form, and any other information that will be presented to potential subjects are reviewed and approved by the appropriate IRB or IEC prior to the enrollment of any study subjects.

#### 15.2 INSTITUTIONAL REVIEW BOARD OR INDEPENDENT ETHICS **COMMITTEE**

The investigator will submit this protocol, the informed consent, IB, and any other relevant supporting information to the appropriate IRB or IEC for review and approval prior to study initiation.

Amendments to the protocol must also be approved by the IRB/IEC and the local regulatory agency, as appropriate, prior to the implementation of changes in this study. No protocol deviations are allowed. However, the investigator may implement a deviation from, or a change of, the protocol to eliminate an immediate hazard(s) to the study subjects without prior IRB/IEC/Sponsor approval/favorable opinion. As soon as possible, the implemented deviation or change, the reasons for it, and, if appropriate, the proposed protocol amendment, should be submitted to the IRB/IEC/Sponsor. Any deviations from the protocol must be fully explained and documented by the investigator.

#### 15.3 INFORMED CONSENT AND HUMAN SUBJECT PROTECTION

No investigator may involve a human being as a subject in research unless the investigator has obtained the legally effective informed consent of the subject or the subject's legally authorized representative. An investigator shall seek such consent only under circumstances that provide the prospective subject or the subject's legally authorized representative sufficient opportunity to consider whether or not to participate, and that minimize the possibility of coercion or undue influence. The information that is given to the subject or the representative shall be in a language understandable to the subject or representative.





Supplemental Clinical Study Report: 20130411


The Sponsor or its designated representative will provide the investigator with a sample consent form. Local and/or institutional requirements may require disclosure of additional information in the ICF. Any changes to the consent form must be submitted to the sponsor or its designated representative for approval, prior to submission to the IRB/IEC. The IRB/IEC will review the consent form for approval. A copy of the approved form must be submitted to the sponsor or its designated representative for its approval prior to initiation of the study. Before implementing any study procedure on a particular subject, informed consent shall be documented in such subject's case histories and by the use of a written consent form approved by the Sponsor and the IRB/IEC and signed and dated by the subject or the subject's legally authorized representative at the time of consent. A copy of the signed informed consent will be given to the subject or subject's legally authorized representative. The original signed consent must be maintained by the investigator and available for inspection by the Sponsor, its designated representative, or regulatory authority at any time.

# 15.4 DIRECT ACCESS TO SOURCE DATA, SOURCE DOCUMENTS, AND STUDY RECORDS

The study will be carried out in keeping with applicable local laws and regulations. This may include an inspection by Onyx representatives/designees, and/or regulatory authority representatives at any time. The investigator/institution must agree to the inspection of study-related records by the regulatory authority/Onyx representatives/designees, and must allow direct access to source documents to the regulatory authority/Onyx representatives/designees/IRB/IEC. The investigator must allocate time (investigator and study staff) to discuss findings and relevant issues with the regulatory authority/Onyx representatives.

### 15.5 DATA COLLECTION AND HANDLING

As part of the responsibilities assumed by participating in the study, the investigator agrees to maintain adequate case histories for the subjects treated as part of the research under this protocol. The investigator agrees to maintain accurate eCRFs and source documentation as part of the case histories. These source documents may include subject diaries, laboratory reports, and other documents. Onyx will supply the eCRF, which will be completed in English.


Approved



Supplemental Clinical Study Report: 20130411


Data collection will involve the use of the EDC system, to which only authorized personnel will have access.

The investigator or designee must enter all results collected during the clinical study into eCRFs (or CRFs). Guidelines for completion of eCRFs will be reviewed with study site personnel at the site initiation visits. Investigators are responsible for approval of the entered/corrected data. Detailed instructions may be found in the other study-specific documents.

All entries made on the eCRF must be verifiable against source documents. In addition to periodic monitoring occurring within the system by study monitors, programmatic edit checks and data listings will be used to review the data for completeness, logic, and adherence to study protocol. As a result of this monitoring and these checks, queries may be electronically issued to the clinical study sites and electronically resolved by those sites.

All data collected in the context of this study will be stored and evaluated according to regulatory requirements and applicable guidance for electronic records. Also, data will be stored and evaluated in such a way as to assure subject confidentiality in accordance with the legal and regulatory requirements applying to protected health information. Study records (eg, copies of eCRFs, regulatory documents) will be retained at the study site, along with adequate source documentation. The study file and all source data should be retained for the time period required by applicable regulatory requirements and will not be destroyed until written notification is given by the sponsor or designee for destruction.

### 15.6 CONFIDENTIALITY

All records identifying the subject will be kept confidential and, in accordance with the applicable laws and/or regulations, will not be made publicly available.

Subject names will not be supplied to the sponsor. Only the subject number will be recorded on the CRF. If the subject name appears on any other document or study materials, then that information must be redacted before a copy of the document is supplied to the sponsor. Study data stored on a computer will be stored in accordance with local data protection laws and regulations. Subjects will be informed in writing that representatives of the sponsor,





Supplemental Clinical Study Report: 20130411


IRB/IEC, or regulatory authorities may inspect their medical records to verify the information collected, and that all personal information made available for inspection will be handled in strictest confidence and in accordance with local data protection laws and regulations.

If the results of the study are published, the subject's identity will remain confidential.

The investigator will maintain a list to enable subjects' records to be identified in accordance with applicable laws and regulations and according to the terms agreed upon in such subjects' signed consent forms.

Approved




#### 16 **REFERENCES**

American Cancer Society. Cancer Facts & Figures 2005. Atlanta, GA: American Cancer Society, 2005.

Anderson KC, Jagannath A, Jakubowiak A, et al. Lenalidomide, bortezomib, and dexamethasone in relapsed/refractory multiple myeloma (MM): Encouraging outcomes and tolerability in a phase II study. J Clin Oncol. 2009;27(15 suppl). ASCO Annual Meeting 2009. Abstract 8536.

Aaronson NK, Ahmedzai S, Bergman B, et al. The European Organization for Research and Treatment of Cancer QLQ C30: a quality of life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993;85(5):365-76.

Bartlett JB, Wu L, Adams M, et al. Lenalidomide and pomalidomide strongly enhance tumor cell killing in vitro during antibody-dependent cellular cytotoxicity (ADCC) mediated by trastuzumab, cetuximab and rituximab. J Clin Oncol. 2007;25(18 suppl). ASCO Annual Meeting 2007. Abstract 3023.

Bladé J, Samson D, Reece D, et al. Criteria for evaluating disease response and progression in patients with multiple myeloma treated by high-dose therapy and haemopoietic stem cell transplantation. European Group for Blood and Marrow Transplant. Myeloma Subcommittee of the EBMT. Br J Haematology. 1998;102(5):1115–23.

Boccadoro M, Morgan G, Cavenagh J. Preclinical evaluation of the proteasome inhibitor bortezomib in cancer therapy. Cancer Cell Int. 2005;5(1):18.

Boyle P, Ferlay J. Cancer incidence and mortality in Europe, 2004. Ann Oncol. 2005;16(3):481-88.

Brookmeyer R, Crowley J. A confidence interval for the median survival time. Biometrics 1982;38:29-41.

Celgene Corporation. Pomalyst (pomalidomide) full prescribing information. February 2013.

Cleeland CS. The measurement of pain from metastatic bone disease: capturing the patient's experience. Clin Cancer Res. 2006;12(20 Pt 2):6236s-42s.

Cocks K, Cohen D, Wisløff F, et al. EORTC Quality of Life Group. An international field study of the reliability and validity of a disease specific questionnaire module (the QLQ MY20) in assessing the quality of life of patients with multiple myeloma. Eur J Cancer. 2007;43(11):1670-78.

Demo SD, Kirk CJ, Aujay MA, et al. Anti-tumor activity of PR-171, a novel irreversible inhibitor of the proteasome. Cancer Res. 2007;67(13):6383–91.

Dispenzieri A. Bortezomib for myeloma—much ado about something. N Engl J Med. 2005;352(24):2546–48.





Supplemental Clinical Study Report: 20130411


Durie BG, Harousseau JL, Miguel JS, et al. International Myeloma Working Group. International uniform response criteria for multiple myeloma. Leukemia. 2006;20(9): 1467–73. Erratum in: Leukemia 2006;20(12):2220. Leukemia 2007;21(5):1134.

Fayers PM, Aaronson NK, Bjordal K, Groenvold M, Curran D, and Bottomley A, on behalf of the EORTC Quality of Life Group. The EORTC QLQ C30 Scoring Manual (3rd Edition). Brussels, Belgium: European Organisation for Research and Treatment of Cancer; 2001.

Filipovich AH, Weisdorf D, Pavletic S, et al. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005;11(12):945–56.

Hideshima T, Richardson P, Chauhan D, et al. The proteasome inhibitor PS-341 inhibits growth, induces apoptosis, and overcomes drug resistance in human multiple myeloma cells. Cancer Res. 2001;61(7):3071-76.

Hryniuk W, Goodyear M. The calculation of received dose intensity. J Clin Oncol. 1990;8(12):1935–37.

Jagannath S, Hofmeister C, Siegel D, et al. Pomalidomide (POM) with low-dose dexamethasone (LoDex) in patients (pts) with relapsed and refractory multiple myeloma who have received prior therapy with lenalidomide (LEN) and bortezomib (BORT): updated phase 2 results and age subgroup analysis. Blood. 2012;120(21). ASH Annual Meeting 2012. Abstract 450.

Jagannath S, Richardson RG, Barlogie B, et al. Bortezomib in combination with dexamethasone for the treatment of patients with relapsed and/or refractory multiple myeloma with less than optimal response to bortezomib alone. Haematologica. 2006;91(7):929–34.

Jakubowiak AJ, Dytfeld D, Griffith KA, et al. A phase 1/2 study of carfilzomib in combination with lenalidomide and low-dose dexamethasone as a frontline treatment for multiple myeloma. Blood. 2012;120(9):1801–09.

Kaufman JL, Seigel D, Vij R, et al. Clinical profile of once-daily, modified release oprozomib tablets in patients with hematologic malignancies: results of a phase 1b/2 trial. 14th Annual International Myeloma Workshop (IMW2013). April 3–7, 2013; Kyoto, Japan. Abstract P-771.

Kuhn DJ, Chen Q, Voorhees PM, et al. Potent activity of carfilzomib, a novel, irreversible inhibitor of the ubiquitin proteasome pathway, against preclinical models of multiple myeloma. Blood. 2007;110(9):3281–90.

Kyle RA, Rajkumar SV. Criteria for diagnosis, staging, risk stratification and response assessment of multiple myeloma. Leukemia. 2009;23(1):3–9.


Approved



Date: 30 July 2019


Lacy M, Jacob A, Gertz M. Pomalidomide plus low-dose dexamethasone in myeloma refractory to both bortezomib and lenalidomide: comparison of two dosing strategies in dual refractory disease. Blood. 2011;118(11):2970–75.

Longo D, Duffey P, DeVita V, et al. The calculation of actual or received dose intensity: a comparison of published methods. J Clin Oncol. 1991;9(11):2042–51.

Mikhael JR, Belch AR, Prince HM, et al. High response rate to bortezomib with or without dexamethasone in patients with relapsed or refractory multiple myeloma: results of a global phase 3b expanded access program. Br J Haematol. 2009;144(2):169-75.

Mikhael JR, Dingli D, Roy V, et al. Management of newly diagnosed symptomatic multiple myeloma: updated Mayo stratification of myeloma and risk-adapted therapy (mSMART) consensus guidelines 2013. Mayo Clin Proc. 2013;88(4):360–76.

National Cancer Institute. Common Terminology Criteria for Adverse Events (CTCAE) v4.0. May 29, 2009 (v4.03 June 14, 2010). NCI, NIH, DHHS. NIH publication # 09-7473.

O'Connor OA, Stewart AK, Vallone M, et al. A phase 1 dose escalation study of the safety and pharmacokinetics of the novel proteasome inhibitor carfilzomib (PR-171) in patients with hematologic malignancies. Clin Cancer Res. 2009;15(22):7085–91.

Oken MM, Creech RH, Tormey DC, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982;5(6):649–55.

Onyx Pharmaceuticals. Kyprolis (carfilzomib) for Injection full prescribing information. 2012.

Payvandi F, Wu L, Haley M, et al. Immunomodulatory drugs inhibit expression of cyclooxygenase-2 from TNF-alpha, IL-1 beta, and LPS-stimulated human PBMC in a partially IL-10-dependent manner. Cell Immunol. 2004;230(2):81–8.

Pfizer Laboratories, Div Pfizer, Inc. Dexamethasone sodium phosphate full prescribing information. October 2012.

Rajkumar SV, Harousseau JL, Durie B. Consensus recommendations for the uniform reporting of clinical trials: report of the International Myeloma Workshop Consensus Panel 1.Blood. 2011;117(18):4691–95.

Richardson PG, Barlogie B, Berenson J, et al. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003;348(26):2609–17.

Richardson PG, Blood E, Mitsiades CS, et al. A randomized phase 2 study of lenalidomide therapy for patients with relapsed or relapsed and refractory multiple myeloma. Blood. 2006a;108(10):3458-64.


Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


Richardson PG, Jagannath S, Avigan DE, et al. Lenalidomide plus bortezomib (Rev-Vel) in relapsed and/or refractory multiple myeloma (MM): final results of a multicenter phase 1 trial. Blood. 2006b;108(11). ASH Annual Meeting 2006. Abstract 405.

Richardson PG, Sonneveld P, Schuster MW, et al. Bortezomib or high dose dexamethasone for relapsed multiple myeloma. N Engl J Med. 2005;352(24):2487–98.

San Miguel SJ, Weisel K, Moreau P. Updated survival for pomalidomide plus low-dose dexamethasone in relapsed refractory multiple myeloma. J Clin Oncol. 2013; 31(15 suppl). ASCO Annual Meeting 2013. Abstract 8510.

Schemper M, Smith TL. A note on quantifying follow-up in studies of failure time. Control Clin Trials. 1996;17(4):343–46.

Sezer O, Vesoleb DH, Singhal S, et al. Bortezomib-induced tumor lysis syndrome in multiple myeloma. Clin Lymphoma Myeloma. 2006;7(3)233–35.

Shen M, Schmitt S, Buac D, et al. Targeting the ubiquitin-proteasome system for cancer therapy. Expert Opin Ther Targets. 2013;17(9):1091–108.

Siegel D, Martin T, Wang M, et al. A phase 2 study of single-agent carfilzomib (PX-171-003-A1) in patients with relapsed and refractory multiple myeloma. Blood. 2012; 120(14):2817-25.

Smith TJ, Khatcheressian J, Lyman GH, et al. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol. 2006;24(19):3187-205.

Stadtmauer J, Shah R, Abonour A, et al. Carfilzomib, pomalidomide and dexamethasone (CPomd) for relapsed/refractory multiple myeloma (RRMM): a phase I/II trial. 14th Annual International Myeloma Workshop (IMW2013). April 3–7, 2013; Kyoto, Japan. Abstract P-250.

Suzuki E, Demo S, Deu E, et al. Molecular mechanisms of bortezomib resistant adenocarcinoma cells. PLoS One. 2011;6(12):e27996.

Zang Y, Thomas SM, Chan ET, et al. The next generation proteasome inhibitors carfilzomib and oprozomib activate prosurvival autophagy via induction of the unfolded protein response and ATF4. 2012;8(12):1873-74.

Zhou HJ, Aujay MA, Bennett MK, et al. Design and synthesis of an orally bioavailable and selective peptide epoxyketone proteasome inhibitor (PR-047). J Med Chem. 2009;52(9): 3028-38.



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


Onyx Therapeutics Oprozomib ER Tablets


#### APPENDIX A1 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE ESCALATION 5/14 SCHEDULE

| | Screening | Baseline | | | | | Cy | cle 1 | | | | | | | Cycle 2 | 2 | | Cycl | le 3 + | End of Study | Long- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Day<br>-28 to -1 | (Pre-<br>C1D1<br>dose) | Day 1 | Day 2 | Day 3-4 | Day 5 | Day<br>6-7 | Day 8 | Day<br>9–14 | Day<br>15 | Day<br>16–21 | Day<br>22-28 | Day<br>1 | Day 2–14 | Day<br>15 | Day<br>16–21 | Day<br>22-28 | Day<br>1 | Day<br>22-28 | Treatment/<br>Early | term<br>Follow<br>-up |
| Written Informed<br>Consent | X | | | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | Х | | | | | | | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | | | | | | | |
| Previous Treatment<br>History | Х | | | | | | | | | | | | | | | | | | | | |
| Physical Examination <sup>b</sup> | X | | X | | | | | | | | | | X | | | | | X | | X | |
| Height | X | | | | | | | | | | | | | | | | | | | | |
| Weight | X | | X | | | | | | | | | | X | | | | | X | | X | |
| Neurological<br>Assessment (BPNS and<br>NCI-CTCAE Grading) <sup>c</sup> | X | | | | | | | | | | | | X | | | | | X | | X | |
| Vital Signs <sup>d,e,f</sup> | X | | X | X | X | X | | X | | X | X | | X | X | X | X | | X | | X | |
| 12-lead ECGg (Local) | X | | X | | | | | | | | | | X | | | | | X | | X | |
| Urinalysis <sup>h</sup> | X | | | | | | | | | | | | | | | | | | | X | |
| Serum Chemistry <sup>i,j</sup> | X | | X | | X | X | | X | | X | X | | X | X | X | X | | X | | X | |
| CBC with Diff and<br>Platelets <sup>j,k</sup> | Х | | Х | | X | X | | X | | Х | X | | X | X | X | X | | X | | X | |
| Coagulation Tests <sup>1</sup> | X | | | | | | | | | | | | | | | | | | | | |
| Pregnancy Test <sup>m</sup> | X | | X | | | | | X | | X | | X | X | | X | | | X | | X | |
| SPEP/UPEP/Serum FLC<br>Immunofixation <sup>n</sup> | X | X<br>Day -7<br>to 1 | | | | | | | | X<br>sFLC<br>only | | | X | | | | | X | | X | |

Footnotes are defined on next page


Approve



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019 **Page 111** 

Onyx Therapeutics Oprozomib ER Tablets


#### APPENDIX A1 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE ESCALATION 5/14 SCHEDULE (CONT'D)

| | Screening | Baseline | | | | | Cyc | cle 1 | | | | | | | Cycle 2 | 2 | | Cyc | le 3 + | End of Study | Long- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Day<br>-28 to -1 | (Pre-<br>C1D1<br>dose) | Day 1 | Day 2 | Day 3-4 | Day 5 | Day 6-7 | Day<br>8 | Day<br>9–14 | Day<br>15 | Day<br>16-21 | Day 22-28 | Day<br>1 | Day 2-14 | Day<br>15 | Day<br>16-21 | Day 22-28 | Day<br>1 | Day 22-28 | Treatment/<br>Early | term<br>Follow<br>-up |
| β2 Microglobulin | X | | | | | | | | | | | | | | | | | | | | |
| Skeletal Survey <sup>o</sup> | | X | | | | | | | | | | | | | | | | | | X | |
| Plasmacytoma<br>Evaluation <sup>p</sup> | | X | | | | | | | | | | | | | | | | | | X | |
| Bone Marrow Aspirate<br>and FISH Analyses <sup>q,</sup> | | X | | | | | | | | | | | | | | | | | | X | |
| Optional – Genomic<br>Biomarker Assessment:<br>Blood <sup>r</sup> | | Х | | | | | | | | | | | | | | | | | | | |
| Optional – Genomic<br>Biomarker Assessment:<br>Saliva <sup>r</sup> | | х | | | | | | | | | | | | | | | | | | | |
| Blood for PKs | | | X | X | | | | | | | | | X | | | | | | | | |
| Blood for PDn Assays | | | X | X | | | | | | | | | X | | | | | | | | |
| Oprozomib Dosing <sup>t</sup> | | | X | X | X | X | | | | X | X | | X | X | X | X | | X | | | |
| Dexamethasone<br>Dosing <sup>u</sup> | | | X | X | | | | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Pomalidomide Dosing <sup>v</sup> | | | X | X | X | X | X | X | X | X | X | | X | X | X | X | | X | | | |
| AEs and Concomitant<br>Medications <sup>w</sup> | | | | • | • | | | | | • | • | | | | | • | • | | | <b></b> | |
| Telephone or other<br>contact for disease and<br>survival status <sup>x</sup> | | | | | | | | | | | | | | | | | | | | | X |

Footnotes are defined on next page





Supplemental Clinical Study Report: 20130411


> Onvx Therapeutics Oprozomib ER Tablets


#### APPENDIX A1 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE ESCALATION 5/14 SCHEDULE (CONT'D)

AE = adverse event; BPNS = Brief Peripheral Neuropathy Screen; C = Cycle; CBC = complete blood count; D = Day; Discon. = discontinuation; EBMT = European Group for Blood and Marrow Transplantation; ECG = electrocardiogram; FISH = fluorescence in situ hybridization; FLC = free light chain; IMWG-URC = International Myeloma Working Group-Uniform Response Criteria; NCI-CTCAE = National Cancer Institute - Common Terminology Criteria for Adverse Events; PDn = pharmacodynamic(s); PK = pharmacokinetic(s); SFLC = serum free light chain; SPEP = serum protein electrophoresis; UPEP = urine protein electrophoresis

- a All End of Study Treatment/Early Discontinuation Assessments must be performed within 30 days following the subject's last administration of study drug and prior to initiation of any other treatment, whichever comes first.
- b Complete physical examinations will be performed during Screening and at the End of Study Treatment/Early Discontinuation visits. All other physical examinations will be limited physical examinations only if clinically indicated. A complete physical examination will include examination of the skin, head and neck, chest (heart and lungs), abdomen, extremities, and a brief neurological examination including an assessment for peripheral neuropathy. Rectal and pelvic examinations are optional. Eastern Cooperative Oncology Group (ECOG) performance status (assessed only at the time of the Screening and End of Study Treatment/Early Discontinuation physical examination) will be conducted. A limited physical examination will include an examination of the chest (heart and lungs) and abdomen, with additional examinations as clinically indicated or directed by AEs. Screening physicals may be used for Cycle 1 Day 1 if done within 7 days prior to Day 1. Physical exams for additional cycles can be conducted within 3 days of Day 1 of the next cycle prior to dosing.
- c Neurological assessments (BPNS and if applicable record AEs with CTCAE grading) will be performed at Screening and on Day 1 of every cycle starting from Cycle 2 if clinically indicated and at the End of Study Treatment/Early Discontinuation (See Appendix M).
- d Vital signs: On Cycle 1 Days 1–5, 8, 15, and 19. On days when oprozomib is administered, measure vitals within 1 hour prior to oprozomib dose and approximately 1 hour after each oprozomib dose. Include measurement of orthostatic blood pressure, temperature, respiration rate, and pulse on every study visit, including Screening and End of Study Treatment/Early Discontinuation. Subject should lie down for 5 minutes and then have blood pressure and pulse measured consistently in either arm. This should be followed by having the subject stand and repeating the blood pressure and pulse at 1 and 3 minutes. A drop of 20 mmHg systolic, 10 mmHg diastolic, or lightheadedness/dizziness between supine and standing blood pressures would indicate orthostatic hypotension. Usually an increase in pulse of 10 beats/min is associated but not required. Subject's dosage and use of antihypertensive agents in the setting of orthostatic hypotension should be evaluated and reassessed on an ongoing basis while on study. Fluid intake should be assessed to confirm the subject is acting in accordance with protocol requirements. Re-education should occur if subject is not adhering to protocol requirements. Fluid status should be repleted to normal levels. If protocol requirements for oral intake of fluids are being met, additional measured should be taken to increase volume status, and ongoing monitoring is warranted and can be managed per investigator discretion. For time points where PK and vital signs are to be done together, vital signs should be obtained first as the act of phlebotomy may impact vital sign measurement results.
- <sup>e</sup> At the investigator's medical discretion, vital signs monitoring may be extended beyond the time periods specified above (d).
- For Cycle 2, if clinically indicated, vital signs are required within approximately 1 hour prior to oprozomib administration on Days 1, 5, 15, and 19. For Cycles 3 and higher, if clinically indicated, vital signs are required within approximately 1 hour prior to oprozomib administration on Day 1.
- g Perform ECG approximately within 1 hour before (predose) and approximately 1 hour after (postdose) administration of oproxomib for Cycles 1, 2, 3, 4, 6, 8, 12, 18, 24 and then every 6 months solely if clinically indicated, until progression or unacceptable toxicity. Perform standard ECG assessment at Screening and End of Study Treatment/Early Discontinuation visit.
- h Subjects with urine positive for protein (> than trace) will need to collect a 24-hour urine sample for creatinine and protein analyses. Urine samples and urinalysis, done locally.
- Full chemistry panel (sodium, potassium, calcium, alkaline phosphatase, blood urea nitrogen, uric acid, lactate dehydrogenase, creatinine, chloride, bicarbonate, glucose, total protein, albumin, total bilirubin, ALT, AST, phosphorous, and magnesium), done locally if clinically indicated. Calculate or measure creatinine clearance (CrCl). Screening results may be used for Cycle 1 Day 1 if obtained within 72 hours of Cycle 1 Day 1.
- GPC and serum chemistry obtained on Days 1, 5, 15, and 19 of Cycles 1 and 2, and on Days 3 and 8 of Cycle 1. Day 1 samples for laboratory analyses can be drawn within 72 hours prior to dosing on Day 1 for all subsequent cycles after Cycle 1 only if clinically indicated.
- k Complete blood count (CBC) with differential, done locally, and includes the following: Hemoglobin, hematocrit, white blood cell (WBC) count with complete manual or automated differential (total neutrophils, lymphocytes, monocytes, eosinophils, basophils; reported as absolute counts), red blood cell (RBC) count, and platelet count. Screening results may be used for Cycle 1 Day 1 if obtained within 72 hours of Cycle 1 Day 1.



Supplemental Clinical Study Report: 20130411


> Onvx Therapeutics Oprozomib ER Tablets


#### APPENDIX A1 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE ESCALATION 5/14 SCHEDULE (CONT'D)

- Coagulation tests, done locally if clinically indicated, and includes the following: Prothrombin time, activated partial thromboplastin time, and international normalized ratio.
- m Screening pregnancy testing, done locally, for females of childbearing potential (FCBP) must have a sensitivity of at least 50 mIU/mL with TWO medically supervised tests performed before pomalidomide dosing starts. One test must be obtained within 10-14 days and one test within 24 hours prior to the start of pomalidomide on Cycle 1 Day 1. A medically supervised, serum pregnancy test will be done weekly during Cycle 1 (Days 1, 8, 15, and 22). Starting with Cycle 2, serum pregnancy tests will be done within 24 hours prior to each cycle of pomalidomide dosing in FCBP only. Pregnancy tests will be repeated on Day 15 of Cycle 2 and beyond if menses are irregular (i.e., not within ± 7 days of a 28-day cycle) or menses are not present in FCBP.
- Results for SPEP, UPEP, and SFLC, obtained locally, during Screening must be available before starting study drug treatment. When the subject is on study drug, the disease response assessments will be performed at the end of each cycle (Day 22–28 or prior to dosing on Day 1 of the next cycle) for the first 18 months (Cycles 1–18), then every 8 weeks thereafter (starting with Cycle 20). If the subject comes off study for reasons other than progressive disease, then disease response assessments will be performed every 4 weeks through 18 months on study, and then every 8 weeks thereafter. Obtain blood for SPEP (please refer to Section 11.3 for collection times for SPEP Immunofixation, UPEP and UPEP Immunofixation with 24-hr urine, and sFLC) within 7 days prior to next Cycle study drug dosing. If a response assessment indicates PD, confirmation of PD may be obtained any time at or before the next scheduled assessment.
- Subjects are required to have a skeletal survey at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) and at End of Study Treatment/Early Discontinuation. This does not need to be repeated if previously done within 30 days of consent. If a skeletal survey was done more than 30 days before consent, it may be acceptable with the Sponsor's study medical monitor approval. Skeletal survey includes: Lateral radiograph of the skull, anteroposterior, and lateral views of the spine, and anteroposterior views of the pelvis, ribs, femora, and humeri. If present at Baseline, bone lesion(s) must be monitored throughout the study only as needed to document response according to the IMWG-URC and modified EBMT criteria or if clinically indicated. For subjects who did not progress during treatment with bone lesions present at Baseline, skeletal survey will no longer be required. During long-term follow-up, skeletal survey evaluation will also no longer be required.
- P Subjects are required to have a plasmacytoma evaluation if known or suspected clinically at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) and at End of Study Treatment. This does not need to be repeated if previously done within 30 days of consent. If the assessment was done more than 30 days before consent, it may be acceptable with the Sponsor's study medical monitor approval. If present at Baseline, plasmacytoma evaluation is to be repeated during treatment only to document response according to the IMWG-URC and modified EBMT criteria or if clinically indicated. If clinically indicated due to history of extramedullary disease, the same technique (may include ultrasound, CT scan, MRI, PET, or other standard-of-care method) must be employed for each measurement. For subjects with plasmacytoma at Baseline and did not progress during treatment, plasmacytoma will **no longer be required**. During long-term follow-up, plasmacytoma evaluation will also no longer be required.
- <sup>q</sup> Bone marrow aspirate or biopsy is required at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) to quantitate percent myeloma cell involvement. Obtain bone marrow aspirate sample for fluorescence in situ hybridization (FISH) studies. A portion of the sample may be used for optional genomic biomarker analysis, for all patients who consent. If Baseline bone marrow aspirate or biopsy were previously obtained and included cytogenetics and FISH (with results available) within 45 days prior to Cycle 1 Day 1 dosing, collection does not need to be repeated unless the patient consents to the optional biomarker genomic samples, which include collection of additional bone marrow aspirate(s). Repeat bone marrow aspirate when appropriate to confirm achievement of stringent complete response (sCR) or complete response (CR) within 30 days (+ 5 days) of confirmation assessment. Bone marrow aspirate will also be collected at disease progression if clinically indicated (may be collected at End of Study Treatment/Early Discontinuation due to PD; it will no longer be required during Long-term Follow-up) for subjects who consent to optional genomic biomarker analysis.
- Optional genomic biomarker samples- blood and saliva: For subjects who consent to participate, blood and saliva samples (in addition to a portion of the bone marrow aspirate obtained for FISH analysis; no new sample is required, as applicable) will be collected at Baseline (within 45 days prior to Cycle 1 Day 1 dosing).
- Sampling times are indicated in Section 11.4 of the protocol, and volumes are provided in the Laboratory Manual.
- Oprozomib treatment will be administered on Days 1-5 and 15-19 during 28-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason. On days on which oprozomib and dexamethasone are administered concurrently (i.e., on Days 1, 2, 15, and 16 of each cycle), dexamethasone should be taken at least 30 minutes prior to oprozomib. Oprozomib should be taken with food. On the PK collection days, dosing of oprozomib in relation to the meal intake (within 2 hours before and 1 hour after dose) will be recorded.
- <sup>u</sup> Subjects will receive 20 mg of dexamethasone on Days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day treatment cycle.
- V Pomalidomide will be administered Days 1–21 of each 28-day cycle up to Cycle 24. Pomalidomide should be taken in the fasted state (i.e., 2 hours before or after a meal).



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


#### APPENDIX A1 SCHEDULE OF STUDY ASSESSMENTS - PHASE 1B DOSE ESCALATION 5/14 SCHEDULE (CONT'D)



w Record all AEs from time of consent through 30 days after the last dose of study drug or before start of subsequent anticancer treatment (whichever occurs first). Start to record concomitant medications from 30 days prior to Day 1 until 30 days after the last dose of study drug. If there is any change in the subject's concomitant medications during the study, it must be recorded on the

x All patients will be followed for survival status by telephone contact or other method approximately every 3 months (± 1 week), or as needed, until study closure.

**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


#### APPENDIX A2 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE ESCALATION 2/7 SCHEDULE

| | Screening | Baseline | | | | Cyc | cle 1 | | | | | Cy | cle 2 | | Cyc | le 3 + | End of Study | Long- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Day<br>-28 to -1 | (Pre-<br>C1D1<br>dose) | Day<br>1 | Day<br>2 | Day 3-7 | Day<br>8 | Day<br>9–14 | Day<br>15 | Day<br>16-21 | Day 22-28 | Day<br>1 | Day 2-14 | Day<br>15 | Day 22-28 | Day<br>1 | Day 22-28 | Treatment/<br>Early<br>Discon.a | term<br>Follow-<br>up |
| Written Informed<br>Consent | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | | | | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | | | | |
| Previous Treatment<br>History | X | | | | | | | | | | | | | | | | | |
| Physical Examination <sup>b</sup> | X | | X | | | | | | | | X | | | | X | | X | |
| Height | X | | | | | | | | | | | | | | | | | |
| Weight | X | | X | | | | | | | | X | | | | X | | X | |
| Neurological Assessment<br>(BPNS and NCI-CTCAE<br>Grading) <sup>e</sup> | X | | | | | | | | | | X | | | | X | | х | |
| Vital Signs <sup>d,e,f</sup> | X | | X | X | | X | X | X | X | X | X | X | X | | X | | X | |
| 12-lead ECGg (Local) | X | | X | | | | | | | | X | | | | X | | X | |
| Urinalysis <sup>h</sup> | X | | | | | | | | | | | | | | | | X | |
| Serum Chemistryi,j | X | | X | X | | X | X | X | X | | X | X | X | | X | | X | |
| CBC with Diff and<br>Platelets <sup>j,k</sup> | X | | X | Х | | X | X | X | Х | | X | X | Х | | X | | X | |
| Coagulation Tests <sup>1</sup> | X | | | | | | | | | | | | | | | | | |
| Pregnancy Test <sup>m</sup> | X | | X | | | X | | X | | X | X | | X | | X | | X | |
| SPEP/UPEP/ Serum FLC<br>Immunofixation <sup>n</sup> | X | X<br>(Day -7<br>to 1) | | | | | | X<br>sFLC<br>only | | | х | | | | Х | | X | |

Footnotes are defined on next page





**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


Onyx Therapeutics Oprozomib ER Tablets


#### APPENDIX A2 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE ESCALATION 2/7 SCHEDULE (CONT'D)

| | Screening | Baseline | | | | Cyc | ele 1 | | | | | Cyc | le 2 | | Cyc | le 3 + | | Long- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Day -28 to -1 | (Pre-<br>C1D1<br>dose) | Day<br>1 | Day<br>2 | Day 3-7 | Day<br>8 | Day<br>9-14 | Day<br>15 | Day<br>16-21 | Day 22-28 | Day<br>1 | Day 2-14 | Day<br>15 | Day 22-28 | Day<br>1 | Day 22-28 | End of Study<br>Treatment/<br>Early Discon. <sup>a</sup> | term<br>Follow-<br>up |
| β2 Microglobulin | X | | | | | | | | | | | | | | | | | |
| Skeletal Survey <sup>o</sup> | | X | | | | | | | | | | | | | | | X | |
| Plasmacytoma<br>Evaluation <sup>p</sup> | | X | | | | | | | | | | | | | | | Х | |
| Bone Marrow Aspirate<br>and FISH Analyses <sup>q,</sup> | | X | | | | | | | | | | | | | | | Х | |
| Optional – Genomic<br>Biomarker Assessment:<br>Blood <sup>r</sup> | | Х | | | | | | | | | | | | | | | | |
| Optional - Genomic<br>Biomarker Assessment:<br>Saliva <sup>r</sup> | | Х | | | | | | | | | | | | | | | | |
| Blood for PKs | | | X | X | | | | | | | X | | | | | | | |
| Blood for PDn Assays | | | X | X | | | | | | | X | | | | | | | |
| Oprozomib Dosing <sup>t</sup> | | | X | X | | X | X | X | X | X | X | X | X | X | X | X | | |
| Dexamethasone Dosing <sup>u</sup> | | | X | X | | X | X | X | X | X | X | X | X | X | X | X | | |
| Pomalidomide Dosing <sup>v</sup> | | | X | X | X | X | X | X | X | | X | X | X | | X | | | |
| AEs and Concomitant<br>Medications <sup>w</sup> | | | | | | | | | ' | | | | | ' | | | <b></b> | |
| Telephone or other<br>contact for disease and<br>survival status <sup>x</sup> | | | | | | | | | | | | | | | | | | X |

Footnotes are defined on next page





Supplemental Clinical Study Report: 20130411


AE = adverse event; BPNS = Brief Peripheral Neuropathy Screen; C = Cycle; CBC = complete blood count; D = Day; s; Discon. = discontinuation; EBMT = European Group for Blood and Marrow Transplantation; ECG = electrocardiogram; FISH = fluorescence in situ hybridization; FLC = free light chain; IMWG-URC = International Myeloma Working Group-Uniform Response Criteria; NCI-CTCAE = National Cancer Institute - Common Terminology Criteria for Adverse Event; PDn = pharmacodynamic(s); PK = pharmacokinetic(s); SFLC = serum free light chain; SPEP = serum protein electrophoresis; UPEP = urine protein electrophoresis.

- <sup>a</sup> All End of Study Treatment/Early Discontinuation Assessments must be performed within 30 days following the subject's last administration of study drug and prior to initiation of any other treatment, whichever comes first.
- b Complete physical examinations will be performed during Screening and at the End of Study Treatment/Early Discontinuation visits. All other physical examinations will be limited physical examinations only if clinically indicated. A complete physical examination will include examination of the skin, head and neck, chest (heart and lungs), abdomen, extremities, and a brief neurological examination including an assessment for peripheral neuropathy. Rectal and pelvic examinations are optional. Eastern Cooperative Oncology Group (ECOG) performance status (assessed only at the time of the Screening and End of Study Treatment/Early Discontinuation physical examination) will be conducted. A limited physical examination will include an examination of the chest (heart and lungs) and abdomen, with additional examinations as clinically indicated or directed by AEs. Screening Physicals may be used for Cycle 1 Day 1 if done within 7 days prior to Day 1. Physical exams for additional cycles can be conducted within 3 days of Day 1 of the next cycle prior to dosing.
- <sup>c</sup> Neurological assessments (BPNS and if applicable record AEs with CTCAE grading) will be performed at Screening and on Day 1 of every cycle starting from Cycle 2 **if clinically indicated** and at the End of Study Treatment/Early Discontinuation (See Appendix M).
- d Vital signs: On Cycle 1 Days 1, 2, 8, 9, 15, 16, 22, and 23. On days when oprozomib is administered measure vitals within 1 hour prior to oprozomib dose and approximately 1 hour after each oprozomib dose. Include measurement of orthostatic blood pressure, temperature, respiration rate, and pulse on every study visit, including Screening and End of Study Treatment/Early Discontinuation. Subject should lie down for 5 minutes and then have blood pressure and pulse measured consistently in either arm. This should be followed by having the subject stand and repeating the blood pressure and pulse at 1 and 3 minutes. A drop of 20 mmHg systolic, 10 mmHg diastolic or lightheadedness/dizziness between supine and standing blood pressures would indicate orthostatic hypotension. Usually an increase in pulse of 10 beats/min is associated but not required. Subject's dosage and use of antihypertensive agents in the setting of orthostatic hypotension should be evaluated and reassessed on an ongoing basis while on study. Fluid intake should be assessed to confirm the subject is acting in accordance with protocol requirements. Re-education should occur if subject is not adhering to protocol requirements. Fluid status should be repleted to normal levels. If protocol requirements for oral intake of fluids are being met, additional measures should be taken to increase volume status, and ongoing monitoring is warranted and can be managed per investigator discretion. For time points where PK and vital signs are to be done together, vital signs should be obtained first as the act of phlebotomy may impact vital sign measurement results.
- e At the investigator's medical discretion, vital signs monitoring may be extended beyond the time periods specified above (d).
- f For Cycle 2, if clinically indicated, vital signs are required within approximately 1 hour prior to oprozomib administration on Days 1, 2, and 15. For Cycles 3 and higher, if clinically indicated, vital signs are required within approximately 1 hour prior to oprozomib administration on Day 1.
- g Perform ECG approximately within 1 hour before (predose) and approximately 1 hour after (postdose) administration of oprozomib for Cycles 1, 2, 3, 4, 6, 8, 12, 18, 24, and then every 6 months solely if clinically indicated, until progression or unacceptable toxicity. Perform standard ECG assessment at Screening and End of Study Treatment/Early Discontinuation visit.
- h Subjects with urine positive for protein (> than trace) will need to collect a 24-hour urine sample for creatinine and protein analyses. Urine samples and urinalysis, done locally,
- <sup>i</sup> Full chemistry panel (sodium, potassium, calcium, alkaline phosphatase, blood urea nitrogen, uric acid, lactate dehydrogenase, creatinine, chloride, bicarbonate, glucose, total protein, albumin, total bilirubin, ALT, AST, phosphorous, and magnesium), done locally **if clinically indicated**. Calculate or measure creatinine clearance (CrCl). Screening results may be used for Cycle 1 Day 1 if obtained within 72 hours of Cycle 1 Day 1.
- j CBC and serum chemistry obtained Days 1, 2, and 15 of Cycles 1 and 2, and on Days 8, 9, and 16 of Cycle 1. Day 1 samples for laboratory analyses can be drawn within 72 hours prior to dosing on Day 1 for all subsequent cycles after Cycle 1 only if clinically indicated.
- k Complete blood count (CBC) with differential, done locally, and includes the following: Hemoglobin, hematocrit, white blood cell (WBC) count with complete manual or automated differential (total neutrophils, lymphocytes, monocytes, eosinophils, basophils; reported as absolute counts), red blood cell (RBC) count, and platelet count. Screening results may be used for Cycle 1 Day 1 if obtained within 72 hours of Cycle 1 Day 1.
- 1 Coagulation tests, done locally if clinically indicated, and includes the following: Prothrombin time, activated partial thromboplastin time, and international normalized ratio.



age 110


Product: Oprozomib

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019 Pag


- m Screening pregnancy testing, done locally, for females of childbearing potential (FCBP) must have a sensitivity of at least 50 mIU/mL with TWO medically supervised tests performed before pomalidomide dosing starts. One test must be obtained within 10–14 days and one test within 24 hours prior to the start of pomalidomide on Cycle 1 Day 1. A medically supervised, serum pregnancy test will be done weekly during Cycle 1 (Days 1, 8, 15, and 22). Starting with Cycle 2, serum pregnancy tests will be done within 24 hours prior to each cycle of pomalidomide dosing in FCBP only. Pregnancy tests will be repeated on Day 15 of Cycle 2 and beyond if menses are irregular (i.e., not within ± 7 days of a 28-day cycle) or menses are not present in FCBP.
- n Results for SPEP, UPEP, and SFLC, obtained locally, during Screening must be available before starting study drug treatment. When the subject is on study drug, the disease response assessments will be performed at the end of each cycle (Day 22–28 or prior to dosing on Day 1 of the next cycle) for the first 18 months (Cycles 1–18), then every 8 weeks thereafter (starting with Cycle 20). If the subject comes off study for reasons other than progressive disease, then disease response assessments will be performed every 4 weeks through 18 months on study, and then every 8 weeks thereafter. Obtain blood for SPEP (please refer to Section 11.3 for collection times for SPEP Immunofixation, UPEP and UPEP Immunofixation with 24-hr urine, and sFLC) within 7 days prior to next Cycle study drug dosing. If a response assessment indicates PD, confirmation of PD may be obtained any time at or before the next scheduled assessment.
- Subjects are required to have a skeletal survey at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) and at End of Study Treatment/Early Discontinuation. This does not need to be repeated if previously done within 30 days of consent. If a skeletal survey was done more than 30 days before consent, it may be acceptable with the Sponsor's study medical monitor approval. Skeletal survey includes: Lateral radiograph of the skull, anteroposterior and lateral views of the spine, and anteroposterior views of the pelvis, ribs, femora, and humeri. If present at Baseline, bone lesion (s) must be monitored throughout the study only as needed to document response according to the IMWG-URC and modified EBMT criteria or if clinically indicated. For subjects who did not progress during treatment with bone lesions present at Baseline, skeletal survey will no longer be required. During long-term follow-up, skeletal survey evaluation will also no longer be required.
- P Subjects are required to have a plasmacytoma evaluation if known or suspected clinically at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) and at End of Study Treatment/Early Discontinuation. This does not need to be repeated if previously done within 30 days of consent. If the assessment was done more than 30 days before consent, it may be acceptable with the Sponsor's study medical monitor approval. If present at Baseline, plasmacytoma evaluation is to be repeated during treatment only to document response according to the IMWG-URC and modified EBMT criteria or if clinically indicated. If clinically indicated due to history of extramedullary disease, the same technique (may include ultrasound, CT scan, MRI, PET, or other standard-of-care method) must be employed for each measurement. For subjects with plasmacytoma at Baseline and did not progress during treatment, plasmacytoma will no longer be required. During long-term follow-up, plasmacytoma evaluation will also no longer be required.
- <sup>q</sup> Bone marrow aspirate or biopsy is required at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) to quantitate percent myeloma cell involvement. Obtain bone marrow aspirate sample for fluorescence in situ hybridization (FISH) studies. A portion of the sample may be used for optional genomic biomarker analysis, for all patients who consent. If Baseline bone marrow aspirate or biopsy were previously obtained and included cytogenetics and FISH (with results available) within 45 days prior to Cycle 1 Day 1 dosing, collection does not need to be repeated unless the patient consents to the optional biomarker genomic samples, which include collection of additional bone marrow aspirate(s). Repeat bone marrow aspirate when appropriate to confirm achievement of stringent complete response (sCR) or complete response (CR) within 30 days (+ 5 days) of confirmation assessment. Bone marrow aspirate will also be collected at disease progression if clinically indicated (may be collected at End of Study Treatment/Early Discontinuation due to PD; it will no longer be required during Long-term Follow-up) for subjects who consent to optional genomic biomarker analysis.
- Optional genomic biomarker samples- blood and saliva: For subjects who consent to participate, blood and saliva samples (in addition to a portion of the bone marrow aspirate obtained for FISH analysis; no new sample is required, as applicable) will be collected at Baseline (within 45 days prior to Cycle 1 Day 1 dosing)
- s Sampling times are indicated in Section 11.4 of the protocol, and volumes are provided in the Laboratory Manual.
- Oprozomib treatment will be administered on Days 1, 2, 8, 9, 15, 16, 22, and 23 during 28-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason. On days on which oprozomib and dexamethasone are administered concurrently (i.e., on Days 1, 2, 8, 9, 15, 16, 22, 23 of each cycle), dexamethasone should be taken at least 30 minutes prior to oprozomib. Oprozomib should be taken with food. On the PK collection days, dosing of oprozomib in relation to the meal intake (within 2 hours before and 1 hour after dose) will be recorded.
- <sup>u</sup> Subjects will receive 20 mg of dexamethasone on Days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day treatment cycle.
- Pomalidomide will be administered Days 1-21 of each 28-day cycle up to Cycle 24. Pomalidomide should be taken in the fasted state (i.e., 2 hours before or after a meal).


Approved



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019




w Record all AEs from time of consent through 30 days after the last dose of study drug or before start of subsequent anticancer treatment (whichever occurs first). Start to record concomitant medications from 30 days prior to Day 1 until 30 days after the last dose of study drug. If there is any change in the subject's concomitant medications during the study, it must be recorded on

x All patients will be followed for survival status by telephone contact or other method approximately every 3 months (± 1 week), or as needed, until study closure.

**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


#### APPENDIX B1 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE EXPANSION 5/14 SCHEDULE

| | Screening | Baseline | | | | | Су | cle 1 | | | | | | | Cycle | 2 | | Cyc | le 3 + | End of | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Day<br>-28 to -1 | (Pre-<br>C1D1<br>dose) | Day<br>1 | Day<br>2 | Day 3-4 | Day<br>5 | Day 6-7 | Day<br>8 | Day<br>9–14 | | Day<br>16-21 | Day 22-28 | Day<br>1 | Day 2-14 | Day<br>15 | Day<br>16-21 | Day 22-28 | Day<br>1 | Day<br>22-28 | Study<br>Treatment/<br>Early<br>Discon.a | Long-<br>term<br>Follow-<br>up |
| Written Informed<br>Consent | X | | | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | | | | | | | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | | | | | | | |
| Previous Treatment<br>History | X | | | | | | | | | | | | | | | | | | | | |
| Physical Examination <sup>b</sup> | X | | X | | | | | | | | | | X | | | | | X | | X | |
| Height | X | | | | | | | | | | | | | | | | | | | | |
| Weight | X | | X | | | | | | | | | | X | | | | | X | | X | |
| Neurological<br>Assessment<br>(BPNS and<br>NCI-CTCAE Grading) <sup>c</sup> | х | | | | | | | | | | | | Х | | | | | Х | | X | |
| Patient Questionnaires <sup>d</sup> :<br>BPI-SF<br>EORTC QLQ-C30<br>EORTC QLQ-MY20<br>FACT/GOG-Ntx4<br>EQ-5D-5L | | | Х | | | | | | | | | | X | | | | | X | | X | |
| Vital Signs <sup>e,f</sup> | X | | X | X | X | X | | X | | X | X | | X | X | X | X | | X | | X | |
| 12-lead ECGg (Local) | X | | X | | | | | | | | | | X | | | | | X | | X | |
| Urinalysis <sup>h</sup> | X | | | | | | | | | | | | | | | | | | | X | |
| Serum Chemistry <sup>i,j</sup> | X | | X | | X | X | | X | | X | X | | X | X | X | X | | X | | X | |
| CBC with Diff and<br>Platelets <sup>j,k</sup> | X | | X | | X | X | | X | | X | X | | X | Х | X | X | | X | | X | |
| Coagulation Tests <sup>1</sup> | X | | | | | | | | | | | | | | | | | | | | |
| Pregnancy Test <sup>m</sup> | X | | X | | | | | X | | X | | X | X | | X | | | X | | X | |

Footnotes are defined on next page



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| APPENDIX | X B1 S0 | CHEDU | JLE ( | OF ST | <b>TUDY</b> | ASS | SESSI | MEN' | TS – | PHAS | SE 11 | B DOS | EE | <b>XPAN</b> | SIO | N 5/1 | 4 SCF | IED | ULE ( | CONT'D | ) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Baseline | | | | | Су | cle 1 | | | | | | | Cycle | 2 | | Cyc | le 3 + | | |
| Visit | Day<br>-28 to -1 | (Pre-<br>C1D1<br>dose) | Day<br>1 | Day<br>2 | Day<br>3-4 | Day<br>5 | Day 6-7 | Day<br>8 | Day<br>9–14 | Day<br>15 | Day<br>16–21 | Day 22-28 | Day<br>1 | Day<br>2–14 | Day<br>15 | Day<br>16–21 | Day<br>22–28 | Day<br>1 | Day<br>22-28 | End of<br>Study<br>Treatment/<br>Early<br>Discon. <sup>a</sup> | Long-<br>term<br>Follow-<br>up |
| SPEP/UPEP/Serum<br>FLC Immunofixation <sup>n</sup> | X | X<br>(Day -7<br>to 1) | | | | | | | | X<br>sFLC<br>only | | | X | | | | | X | | X | |
| β2 Microglobulin | X | | | | | | | | | | | | | | | | | | | | |
| Skeletal Survey <sup>o</sup> | | X | | | | | | | | | | | | | | | | | | X | |
| Plasmacytoma<br>Evaluation <sup>p</sup> | | X | | | | | | | | | | | | | | | | | | X | |
| Bone Marrow Aspirate<br>and FISH Analyses <sup>4,</sup> | | X | | | | | | | | | | | | | | | | | | X | |
| Optional – Genomic<br>Biomarker Assessment:<br>Blood <sup>r</sup> | | х | | | | | | | | | | | | | | | | | | | |
| Optional – Genomic<br>Biomarker Assessment:<br>Saliva <sup>r</sup> | | Х | | | | | | | | | | | | | | | | | | | |
| Blood for PKs | | | X | X | | | | | | | | | X | | | | | | | | |
| Blood for PDn Assays | | | X | X | | | | | | | | | X | | | | | | | | |
| Oprozomib Dosing <sup>t</sup> | | | X | X | X | X | | | | X | X | | X | X | X | X | | X | | | |
| Dexamethasone Dosing <sup>u</sup> | | | X | X | | | | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Pomalidomide Dosing <sup>v</sup> | | | X | X | X | X | X | X | X | X | X | | X | X | X | X | | X | | | |
| AEs and Concomitant<br>Medications <sup>w</sup> | | | | | | | | | | | | | | | | | | | | <b>→</b> | |
| Telephone or other<br>contact for disease and<br>survival status <sup>x</sup> | | | | | | | | | | | | | | | | | | | | | X |
| Footnotes are defined | on next pag | ge | | • | | | | | | | | • | | | | | | | | | |



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019

Onvx Therapeutics Oprozomib ER Tablets Clinical Study Protocol No. OPZ007 

#### APPENDIX B1 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE EXPANSION 5/14 SCHEDULE (CONT'D)

AE = adverse event; BPI-SF = Brief Pain Inventory - Short Form; BPNS = Brief Peripheral Neuropathy Screen; C = Cycle; CBC = complete blood count; D = Day; Discon. = discontinuation; EBMT = European Group for Blood and Marrow Transplantation; ECG = electrocardiogram; EORTC = European Organization for Research and Treatment; EO-5D-5L = a new facility for the measurement of health-related quality of life: FACT/GOG-Ntx = Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity subscale questionnaire: FISH = fluorescence in situ hybridization; FLC = free light chain; IMWG-URC = International Myeloma Working Group-Uniform Response Criteria; NCI-CTCAE = National Cancer Institute -Common Terminology Criteria for Adverse Events; PDn = pharmacodynamic(s); PK = pharmacokinetic(s); SFLC = serum free light chain; SPEP = serum protein electrophoresis; UPEP = urine protein electrophoresis.

- a All End of Study Treatment/Early Discontinuation Assessments must be performed within 30 days following the subject's last administration of study drug and prior to initiation of any other treatment, whichever comes first.
- b Complete physical examinations will be performed during Screening and at the End of Study Treatment/Early Discontinuation visits. All other physical examinations will be limited physical examinations only if clinically indicated. A complete physical examination will include examination of the skin, head and neck, chest (heart and lungs), abdomen, extremities, and a brief neurological examination including an assessment for peripheral neuropathy. Rectal and pelvic examinations are optional. Eastern Cooperative Oncology Group (ECOG) performance status (assessed only at the time of the Screening and End of Study Treatment/Early Discontinuation physical examination) will be conducted. A limited physical examination will include an examination of the chest (heart and lungs) and abdomen, with additional examinations as clinically indicated or directed by AEs. Screening Physicals may be used for Cycle 1 Day 1 if done within 7 days prior to Day 1. Physical exams for additional cycles can be conducted within 3 days of Day 1 of the next cycle prior to dosing.
- c Neurological assessments (BPNS and if applicable record AEs with CTCAE grading) will be performed at Screening and on Day 1 of every cycle starting from Cycle 2 if clinically indicated and at the End of Study Treatment/Early Discontinuation (See Appendix M).
- d BPI-SF, EORTC QLQ-C30, EORTC QLQ-MY20, FACT/GOG-Ntx4, and EQ-5D-5L to be collected at on Day 1 of every cycle through End of Study Treatment/Early Discontinuation visit. These patient-reported outcome instruments should be administered prior to administration of any study drug.
- e Vital signs: On Cycle 1 Days 1-5, 8, 15, and 19. On days when oprozomib is administered measure vitals within 1 hour prior to oprozomib dose and approximately 1 hour after each oprozomib dose. Include measurement of orthostatic blood pressure, pulse, respiration rate, and temperature on every study visit, including Screening and End of Study Treatment/Early Discontinuation. Subject should lie down for 5 minutes and then have blood pressure and pulse measured consistently in either arm. This should be followed by having the subject stand and repeating the blood pressure and pulse at 1 and 3 minutes. A drop of 20 mmHg systolic, 10 mmHg diastolic, or lightheadedness/dizziness between supine and standing blood pressures would indicate orthostatic hypotension. Usually an increase in pulse of 10 beats/min is associated but not required. Subject's dosage and use of antihypertensive agents in the setting of orthostatic hypotension should be evaluated and reassessed on an ongoing basis while on study. Fluid intake should be assessed to confirm the subject is acting in accordance with protocol requirements Re-education should occur if subject is not adhering to protocol requirements. Fluid status should be repleted to normal levels. If protocol requirements for oral intake of fluids are already being met, additional measures should be taken to increase volume status, and ongoing monitoring is warranted and can be managed per investigator discretion. At the investigator's medical discretion, vital sign monitoring may be extended beyond the time periods specified above. For time points where PK and vital signs are to be done together, vital signs should be obtained first as the act of phlebotomy may impact vital sign measurement results.
- For Cycles 2, if clinically indicated, vital signs are required within approximately 1 hour prior to oprozomib administration on Days 1, 5, 15, and 19. For Cycles 3 and higher, if clinically indicated, vital signs are required within approximately 1 hour prior to oprozomib administration on Day 1.
- g Perform ECG approximately within 1 hour before (predose) and approximately 1 hour after (postdose) administration of oprozomib for Cycles 1, 2, 3, 4, 6, 8, 12, 18, 24 and then every 6 months solely if clinically indicated, until progression or unacceptable toxicity. Perform standard ECG assessment at Screening and End of Study Treatment/Early Discontinuation visit.
- h Subjects with urine positive for protein (> than trace) will need to collect a 24-hour urine sample for creatinine and protein analyses. Urine samples and urinalysis, done locally.
- Full chemistry panel (sodium, potassium, calcium, alkaline phosphatase, blood urea nitrogen, uric acid, lactate dehydrogenase, creatinine, chloride, bicarbonate, glucose, total protein, albumin, total bilirubin, ALT, AST, phosphorous, and magnesium), done locally if clinically indicated. Calculate or measure creatinine clearance (CrCl). Screening results may be used for Cycle 1 Day 1 if obtained within 72 hours of Cycle 1 Day 1.



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


#### APPENDIX B1 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE EXPANSION 5/14 SCHEDULE (CONT'D)

- GBC and serum chemistry obtained Days 1, 5, 15, and 19 of Cycles 1 and 2, and on Days 3 and 8 of Cycle 1. Day 1 samples for laboratory analyses can be drawn within 72 hours prior to dosing on Day 1 for all subsequent cycles after Cycle 1 only if clinically indicated.
- k Complete blood count (CBC) with differential, done locally, and includes the following: Hemoglobin, hematocrit, white blood cell (WBC) count with complete manual or automated differential (total neutrophils, lymphocytes, monocytes, eosinophils, basophils; reported as absolute counts), red blood cell (RBC) count, and platelet count. Screening results may be used for Cycle 1 Day 1 if obtained within 72 hours of Cycle 1 Day 1.
- 1 Coagulation tests, done locally if clinically indicated, and includes the following: Prothrombin time, activated partial thromboplastin time, and international normalized ratio.
- m Screening pregnancy testing, done locally for females of childbearing potential (FCBP) must have a sensitivity of at least 50 mIU/mL with TWO medically supervised tests performed before pomalidomide dosing starts. One test must be obtained within 10-14 days and one test within 24 hours prior to the start of pomalidomide on Cycle 1 Day 1. A medically supervised, serum pregnancy test will be done weekly during Cycle 1 (Days 1, 8, 15, and 22). Starting with Cycle 2, serum pregnancy tests will be done within 24 hours prior to each cycle of pomalidomide dosing in FCBP only. Pregnancy tests will be repeated on Day 15 of Cycle 2 and beyond if menses are irregular (i.e., not within ± 7 days of a 28-day cycle) or menses are not present in FCBP.
- n Results for SPEP, UPEP, and SFLC, obtained locally, during Screening must be available before starting study drug treatment. When the subject is on study drug, the disease response assessments will be performed at the end of each cycle (Day 22–28 or prior to dosing on Day 1 of the next cycle) for the first 18 months (Cycles 1–18), then every 8 weeks thereafter (starting with Cycle 20). If the subject comes off study for reasons other than progressive disease, then disease response assessments will be performed every 4 weeks through 18 months on study, and then every 8 weeks thereafter. Obtain blood for SPEP (please refer to Section 11.3 for collection times for SPEP Immunofixation, UPEP and UPEP Immunofixation with 24-hr urine, and sFLC) within 7 days prior to next Cycle study drug dosing. If a response assessment indicates PD, confirmation of PD may be obtained any time at or before the next scheduled assessment.
- o Subjects are required to have a skeletal survey at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) and at End of Study Treatment/Early Discontinuation. This does not need to be repeated if previously done within 30 days of consent. If a skeletal survey was done more than 30 days before consent, it may be acceptable with the Sponsor's study medical monitor approval. Skeletal survey includes: Lateral radiograph of the skull, anteroposterior, and lateral views of the spine, and anteroposterior views of the pelvis, ribs, femora, and humeri. If present at Baseline, bone lesion (s) must be monitored throughout the study only as needed to document response according to the IMWG-URC and modified EBMT criteria or if clinically indicated. For subjects who did not progress during treatment with bone lesions present at Baseline, skeletal survey will **no longer be required**. During long-term follow-up, skeletal survey evaluation will also no longer be required.
- P Subjects are required to have a plasmacytoma evaluation if known or suspected clinically at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) and at End of Study Treatment. This does not need to be repeated if previously done within 30 days of consent. If the assessment was done more than 30 days before consent, it may be acceptable with the Sponsor's study medical monitor approval. If present at Baseline, plasmacytoma evaluation is to be repeated during treatment only to document response according to the IMWG-URC and modified EBMT criteria or if clinically indicated. If clinically indicated due to history of extramedullary disease, the same technique (may include ultrasound, CT scan, MRI, PET, or other standard-of-care method) must be employed for each measurement. For subjects with plasmacytoma at Baseline and did not progress during treatment, plasmacytoma will **no longer be required**. During long-term follow-up, plasmacytoma evaluation will also no longer be required.
- <sup>q</sup> Bone marrow aspirate or biopsy is required at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) to quantitate percent myeloma cell involvement. Obtain bone marrow aspirate sample for fluorescence in situ hybridization (FISH) studies. A portion of the sample may be used for optional genomic biomarker analysis, for all patients who consent. If Baseline bone marrow aspirate or biopsy were previously obtained and included cytogenetics and FISH (with results available) within 45 days prior to Cycle 1 Day 1 dosing, collection does not need to be repeated unless the patient consents to the optional biomarker genomic samples, which include collection of additional bone marrow aspirate(s). Repeat bone marrow aspirate when appropriate to confirm achievement of stringent complete response (sCR) or complete response (CR) within 30 days (+ 5 days) of confirmation assessment. Bone marrow aspirate will also be collected at disease progression if clinically indicated (may be collected at End of Study Treatment/Early Discontinuation due to PD; it will no longer be required during Long-term Follow-up) for subjects who consent to optional genomic biomarker analysis.
- Optional genomic biomarker samples- blood and saliva: For subjects who consent to participate, blood and saliva samples (in addition to a portion of the bone marrow aspirate obtained for FISH analysis; no new sample is required, as applicable) will be collected at Baseline (within 45 days prior to Cycle 1 Day 1 dosing).
- Sampling times are indicated in Section 11.4 of the protocol, and volumes are provided in the Laboratory Manual.

| _ | 'O | TEL | DI | 28.17 | CT A |
|---|----|-----|----|-------|------|



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


#### APPENDIX B1 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE EXPANSION 5/14 SCHEDULE (CONT'D)

- Oprozomib treatment will be administered on Days 1-5 and 15-19 during 28-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason. On days on which oprozomib and dexamethasone are administered concurrently (i.e., on Days 1, 2, 15, and 16 of each cycle), dexamethasone should be taken at least 30 minutes prior to oprozomib. Oprozomib should be taken with food. On the PK collection days, dosing of oprozomib in relation to the meal intake (within 2 hours before and 1 hour after dose) will be recorded.
- <sup>u</sup> Subjects will receive 20 mg of dexamethasone on Days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day treatment cycle.
- v Pomalidomide will be administered Days 1–21 of each 28-day cycle up to Cycle 24. Pomalidomide should be taken in the fasted state (i.e., 2 hours before or after a meal).
- w Record all AEs from time of consent through 30 days after the last dose of study drug or before start of subsequent anticancer treatment (whichever occurs first). Start to record concomitant medications from 30 days prior to Day 1 until 30 days after the last dose of study drug. If there is any change in the subject's concomitant medications during the study, it must be recorded on
- x All patients will be followed for survival status by telephone contact or other method approximately every 3 months (± 1 week), or as needed, until study closure.



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


#### APPENDIX B2 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE EXPANSION 2/7 SCHEDULE

| | Screening | Baseline | | | | Cyc | le 1 | | | | | Cyc | le 2 | | Cyc | le 3 + | End of Study | Long- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Day<br>-28 to -1 | (Pre-<br>C1D1<br>dose) | Day<br>1 | Day<br>2 | Day 3-7 | Day<br>8 | Day<br>9–14 | Day<br>15 | Day<br>16-21 | Day<br>22-28 | Day<br>1 | Day 2-14 | Day<br>15 | Day 22-28 | Day<br>1 | Day 22-28 | Treatment/<br>Early<br>Discon.a | term<br>Follow-<br>up |
| Written Informed<br>Consent | X | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | | | | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | | | | |
| Previous Treatment<br>History | X | | | | | | | | | | | | | | | | | |
| Physical Examination <sup>b</sup> | X | | X | | | | | | | | X | | | | X | | X | |
| Height | X | | | | | | | | | | | | | | | | | |
| Weight | X | | X | | | | | | | | X | | | | X | | X | |
| Neurological<br>Assessment<br>(BPNS and<br>NCI-CTCAE Grading) <sup>c</sup> | х | | | | | | | | | | X | | | | Х | | X | |
| Patient Questionnaires <sup>d</sup> :<br>BPI-SF<br>EORTC QLQ-C30<br>EORTC QLQ-MY20<br>FACT-COG-Ntx4<br>EQ-5D-5L | | | X | | | | | | | | х | | | | Х | | х | |
| Vital Signs <sup>e,f</sup> | X | | X | X | | X | X | X | X | X | X | X | X | | X | | X | |
| 12-lead ECGg (Local) | X | | X | | | | | | | | X | | | | X | | X | |
| Urinalysis <sup>h</sup> | X | | | | | | | | | | | | | | | | X | |
| Serum Chemistry <sup>i,j</sup> | X | | X | X | | X | X | X | X | | X | X | X | | X | | X | |
| CBC with Diff and<br>Platelets <sup>j,k</sup> | X | | X | X | | X | X | X | X | | X | X | X | | Х | | X | |
| Coagulation Tests <sup>1</sup> | X | | | | | | | | | | | | | | | | | |
| Pregnancy Test <sup>m</sup> | X | | X | | | X | | X | | X | X | | X | | X | | X | |

Footnotes are defined on the next page





**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


#### APPENDIX B2 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE EXPANSION 2/7 SCHEDULE (CONT'D)

| | Screening | Baseline | | | | Cyc | cle 1 | | | | | Cyc | cle 2 | | Cyc | le 3 + | End of Study | Long- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | Day<br>-28 to -1 | (Pre-<br>C1D1<br>dose) | Day<br>1 | Day<br>2 | Day 3-7 | Day<br>8 | Day<br>9–14 | Day<br>15 | Day<br>16-21 | Day 22-28 | Day<br>1 | Day 2- | Day<br>15 | Day 22-28 | Day 1 | Day 22-28 | Treatment/ Early Discon.a | term<br>Follow-<br>up |
| SPEP/UPEP/ Serum<br>FLC Immunofixation <sup>n</sup> | X | X<br>(Day -7<br>to 1) | | | | | | X<br>sFLC<br>only | | | Х | | | | х | | Х | |
| β2 Microglobulin | X | | | | | | | | | | | | | | | | | |
| Skeletal Survey <sup>o</sup> | | X | | | | | | | | | | | | | | | X | |
| Plasmacytoma<br>Evaluation <sup>p</sup> | | X | | | | | | | | | | | | | | | X | |
| Bone Marrow Aspirate<br>and FISH Analyses <sup>q,</sup> | | Х | | | | | | | | | | | | | | | X | |
| Optional – Genomic<br>Biomarker Assessment:<br>Blood <sup>r</sup> | | X | | | | | | | | | | | | | | | | |
| Optional – Genomic<br>Biomarker Assessment:<br>Saliva <sup>r</sup> | | X | | | | | | | | | | | | | | | | |
| Blood for PKs | | | X | X | | | | | | | X | | | | | | | |
| Blood for PDn Assays | | | X | X | | | | | | | X | | | | | | | |
| Oprozomib Dosing <sup>t</sup> | | | X | X | | X | X | X | X | X | X | X | X | X | X | X | | |
| Dexamethasone<br>Dosing <sup>u</sup> | | | X | X | | X | X | X | X | X | X | X | X | X | X | X | | |
| Pomalidomide Dosing <sup>v</sup> | | | X | X | X | X | X | X | X | | X | X | X | | X | | | |
| AEs and Concomitant<br>Medications <sup>w</sup> | | | | | | | | | | | | | | | | | <del></del> | |
| Telephone or other contact for disease and survival status <sup>x</sup> | | | | | | | | | | | | | | | | | | X |

Footnotes are defined on next page





Supplemental Clinical Study Report: 20130411

Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets

#### APPENDIX B2 SCHEDULE OF STUDY ASSESSMENTS - PHASE 1B DOSE EXPANSION 2/7 SCHEDULE (CONT'D)

AE = adverse event; BPI-SF = Brief Pain Inventory – Short Form; BPNS = Brief Peripheral Neuropathy Screen; C = Cycle; CBC = complete blood count; D = Day; Discon. = discontinuation; EBMT = European Group for Blood and Marrow Transplantation; ECG = electrocardiogram; EORTC = European Organization for Research and Treatment; EQ-5D-5L = a new facility for the measurement of health-related quality of life; FACT/GOG-Ntx = Functional Assessment of Cancer Therapy/Gynecologic Oncology Group Neurotoxicity subscale questionnaire; FISH = fluorescence in situ hybridization; FLC = free light chain; IMWG-URC = International Myeloma Working Group-Uniform Response Criteria; NCI-CTCAE = National Cancer Institute – Common Terminology Criteria for Adverse Events; PDn = pharmacodynamic(s); PK = pharmacokinetic(s); SFLC = serum free light chain; SPEP = serum protein electrophoresis; UPEP = urine protein electrophoresis.

- <sup>a</sup> All End of Study Treatment/Early Discontinuation Assessments must be performed within 30 days following the subject's last administration of study drug and prior to initiation of any other treatment, whichever comes first.
- Complete physical examinations will be performed during Screening and at the End of Study Treatment/Early Discontinuation visits. All other physical examinations will be limited physical examinations only if clinically indicated. A complete physical examination will include examination of the skin, head and neck, chest (heart and lungs), and abdomen, extremities, and a brief neurological examination including an assessment for peripheral neuropathy. Rectal and pelvic examinations are optional. Eastern Cooperative Oncology Group (ECOG) performance status (assessed only at the time of the Screening and End of Study Treatment/Early Discontinuation physical examination) will be conducted. A limited physical examination will include an examination of the chest (heart and lungs) and abdomen, with additional examinations as clinically indicated or directed by AEs. Screening Physicals may be used for Cycle 1 Day 1 if done within 7 days prior to Day 1. Physical exams for additional examinations as of Day 1 of the next cycle prior to dosing.
- c Neurological assessments (BPNS and if applicable record AEs with CTCAE grading) will be performed at Screening and on Day 1 of every cycle starting from Cycle 2 if clinically indicated and at the End of Study Treatment/Early Discontinuation (See Appendix M).
- d BPI-SF, EORTC QLQ-C30, EORTC QLQ-MY20, FACT/GOG-Ntx4, and EQ-5D-5L to be collected on Day 1 of every cycle through End of Study Treatment/Early Discontinuation visit. These patient-reported outcome instruments should be administered prior to administration of any study drug.
- <sup>c</sup> Vital signs: On Cycle 1 Days 1, 2, 8, 9, 15, 16, 22, and 23. On days when oprozomib is administered measure vitals within 1 hour prior to oprozomib dose and approximately 1 hour after each oprozomib dose. Include measurement of orthostatic blood pressure, pulse, respiration rate, and temperature on every study visit, including Screening and End of Study Treatment/Early Discontinuation. Subject should lie down for 5 minutes and then have blood pressure and pulse measured consistently in either arm. This should be followed by having the subject stand and repeating the blood pressure and pulse at 1 and 3 minutes. A drop of 20 mmHg systolic, 10 mmHg diastolic, or lightheadedness/dizziness between supine and standing blood pressure would indicate orthostatic hypotension. Usually an increase in pulse of 10 beats/min is associated but not required. Subject's dosage and use of antihypertensive agents in the setting of orthostatic hypotension should be evaluated and reassessed on an ongoing basis while on study. Fluid intake should be assessed to confirm the subject is acting in accordance with protocol requirements. Re-education should occur if subject is not adhering to protocol requirements. Fluid status should be repleted to normal levels. If protocol requirements for oral intake of fluids are already being met, additional measures should be taken to increase volume status and ongoing monitoring is warranted and can be managed per investigator discrection. At the investigator's medical discretion, vital sign monitoring may be extended beyond the time periods specified above. For time points where PK and vital signs are to be done together, vital signs should be obtained first as the act of phlebotomy may impact vital sign measurement results.
- f For Cycle 2, if clinically indicated, vital signs are required within approximately 1 hour prior to oprozomib administration on Days 1, 2, and 15. For Cycles 3 and higher, if clinically indicated, vital signs are required within approximately 1 hour prior to oprozomib administration on Day 1.
- g Perform ECG approximately within 1 hour before (predose) and approximately 1 hour after (postdose) administration of oprozomib for Cycles 1, 2, 3, 4, 6, 8, 12, 18, 24 and then every 6 months solely if clinically indicated, until progression or unacceptable toxicity. Perform standard ECG assessment at Screening and End of Study Treatment/Early Discontinuation visit.
- h Subjects with urine positive for protein (> than trace) will need to collect a 24-hour urine sample for creatinine and protein analyses. Urine samples and urinalysis, done locally.
- Full chemistry panel (sodium, potassium, calcium, alkaline phosphatase, blood urea nitrogen, uric acid, lactate dehydrogenase, creatinine, chloride, bicarbonate, glucose, total protein, albumin, total bilirubin, ALT, AST, phosphorous, and magnesium), done locally, **if clinically indicated**. Calculate or measure creatinine clearance (CrCl). Screening results may be used for Cycle 1 Day 1 if obtained within 72 hours of Cycle 1 Day 1.

| | | | | | | _ |
|-----|-----|-----|---|----|----|---|
| - ( | 'ON | IFI | D | EN | TΙ | А |





**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


#### APPENDIX B2 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE EXPANSION 2/7 SCHEDULE (CONT'D)

- CBC and serum chemistry obtained Days 1, 2, and 15 of Cycles 1 and 2, and on Days 8, 9, and 16 of Cycle 1. Day 1 samples for laboratory analyses can be drawn within 72 hours prior to dosing on Day 1 for all subsequent cycles after Cycle 1 only if clinically indicated.
- k Complete blood count (CBC) with differential, done locally, and includes the following: Hemoglobin, hematocrit, white blood cell (WBC) count with complete manual or automated differential (total neutrophils, lymphocytes, monocytes, eosinophils, basophils; reported as absolute counts), red blood cell (RBC) count, and platelet count. Screening results may be used for Cycle 1 Day 1 if obtained within 72 hours of Cycle 1 Day 1.
- 1 Coagulation tests, done locally if clinically indicated, and includes the following: Prothrombin time, activated partial thromboplastin time, and international normalized ratio.
- m Screening pregnancy testing, done locally, for females of childbearing potential (FCBP) must have a sensitivity of at least 50 mIU/mL with TWO medically supervised tests performed before pomalidomide dosing starts. One test must be obtained within 10-14 days and one test within 24 hours prior to the start of pomalidomide on Cycle 1 Day 1. A medically supervised, serum pregnancy test will be done weekly during Cycle 1 (Days 1, 8, 15, and 22). Starting with Cycle 2, serum pregnancy tests will be done within 24 hours prior to each cycle of pomalidomide dosing in FCBP only. Pregnancy tests will be repeated on Day 15 of Cycle 2 and beyond if menses are irregular (i.e., not within ± 7 days of a 28-day cycle) or menses are not present in FCBP.
- Results for SPEP, UPEP, and SFLC, obtained locally, during Screening must be available before starting study drug treatment. When the subject is on study drug, the disease response assessments will be performed at the end of each cycle (Day 22–28 or prior to dosing on Day 1 of the next cycle) for the first 18 months (Cycles 1–18), then every 8 weeks thereafter (starting with Cycle 20). If the subject comes off study for reasons other than progressive disease, then disease response assessments will be performed every 4 weeks through 18 months on study, and then every 8 weeks thereafter. Obtain blood for SPEP (please refer to Section 11.3 for collection times for SPEP Immunofixation, UPEP and UPEP Immunofixation with 24-hr urine, and sFLC) within 7 days prior to next Cycle study drug dosing. If a response assessment indicates PD, confirmation of PD may be obtained any time at or before the next scheduled assessment.
- o Subjects are required to have a skeletal survey at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) and at End of Study Treatment/Early Discontinuation. This does not need to be repeated if previously done within 30 days of consent. If a skeletal survey was done more than 30 days before consent, it may be acceptable with the Sponsor's study medical monitor approval. Skeletal survey includes: Lateral radiograph of the skull, anteroposterior, and lateral views of the spine, and anteroposterior views of the pelvis, ribs, femora, and humeri. If present at Baseline, bone lesion (s) must be monitored throughout the study only as needed to document response according to the IMWG URC and modified EBMT criteria or if clinically indicated. For subjects who did not progress during treatment with bone lesions present at Baseline, skeletal survey will no longer be required. During long-term follow-up, skeletal survey evaluation will also no longer be required.
- P Subjects are required to have a plasmacytoma evaluation if known or suspected clinically at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) and at End of Study Treatment/Early Discontinuation. This does not need to be repeated if previously done within 30 days of consent. If the assessment was done more than 30 days before consent, it may be acceptable with the Sponsor's study medical monitor approval. If present at Baseline, plasmacytoma evaluation is to be repeated during treatment only to document response according to the IMWG-URC and modified EBMT criteria or if clinically indicated. If clinically indicated due to history of extramedullary disease, the same technique (may include ultrasound, CT scan, MRI, PET, or other standard of care method) must be employed for each measurement. For subjects with plasmacytoma at Baseline and did not progress during treatment, plasmacytoma will no longer be required. During long-term follow-up, plasmacytoma evaluation will also no longer be required.
- <sup>q</sup> Bone marrow aspirate or biopsy is required at Baseline (within 45 days prior to Cycle 1 Day 1 dosing) to quantitate percent myeloma cell involvement. Obtain bone marrow aspirate sample for fluorescence in situ hybridization (FISH) studies. A portion of the sample may be used for optional genomic biomarker analysis, for all patients who consent. If Baseline bone marrow aspirate or biopsy were previously obtained and included cytogenetics and FISH (with results available) within 45 days prior to Cycle 1 Day 1 dosing, collection does not need to be repeated unless the patient consents to the optional biomarker genomic samples, which include collection of additional bone marrow aspirate(s). Repeat bone marrow aspirate when appropriate to confirm achievement of stringent complete response (sCR) or complete response (cR) within 30 days (+ 5 days) of confirmation assessment. Bone marrow aspirate will also be collected at disease progression if clinically indicated (may be collected at End of Study Treatment/Early Discontinuation due to PD; it will no longer be required during Long-term Follow-up) for subjects who consent to optional genomic biomarker analysis.
- Optional genomic biomarker samples- blood and saliva: For subjects who consent to participate, blood and saliva samples (in addition to a portion of the bone marrow aspirate obtained for FISH analysis; no new sample is required, as applicable) will be collected at Baseline (within 45 days prior to Cycle 1 Day 1 dosing).
- s Sampling times are indicated in Section 11.4 of the protocol, and volumes are provided in the Laboratory Manual.

| | ~~ | - T | | _ | _ | | _ | |
|-----|----|-----|----|----|---|----------|---|---|
| - 1 | CC | | нι | I) | ы | <b>V</b> | ш | Δ |





**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


#### APPENDIX B2 SCHEDULE OF STUDY ASSESSMENTS – PHASE 1B DOSE EXPANSION 2/7 SCHEDULE (CONT'D)

- Oprozomib treatment will be administered on Days 1, 2, 8, 9, 15, 16, 22, and 23 during 28-day cycles until disease progression, unacceptable toxicity, or study treatment discontinuation for any reason. On days on which oprozomib and dexamethasone are administered concurrently (i.e., on Days 1, 2, 8, 9, 15, 16, 22, 23 of each cycle), dexamethasone should be taken at least 30 minutes prior to oprozomib. Oprozomib should be taken with food. On the PK collection days, dosing of oprozomib in relation to the meal intake (within 2 hours before and 1 hour after dose) will be recorded.
- <sup>u</sup> Subjects will receive 20 mg of dexamethasone on Days 1, 2, 8, 9, 15, 16, 22, and 23 of each 28-day treatment cycle.
- V Pomalidomide will be administered Days 1-21 of each 28-day cycle up to Cycle 24. Pomalidomide should be taken in the fasted state (i.e., 2 hours before or after a meal).
- w Record all AEs from time of consent through 30 days after the last dose of study drug or before start of subsequent anticancer treatment (whichever occurs first). Start to record concomitant medications from 30 days prior to Day 1 until 30 days after the last dose of study drug. If there is any change in the subject's concomitant medications during the study, it must be recorded on
- x All patients will be followed for survival status by telephone contact or other method approximately every 3 months (± 1 week), or as needed, until study closure.



Date: 30 July 2019

Approved

Onyx Therapeutics Oprozomib ER Tablets


#### APPENDIX C RESPONSE CRITERIA FOR MULTIPLE MYELOMA

Table D1 Summary of International Myeloma Working Group-Uniform Response Criteria (IMWG-URC)

| Response<br>Subcategory <sup>a</sup> | Response Criteria |
|---|---|
| sCR <sup>b</sup> | <ul> <li>Negative immunofixation on the serum and urine and</li> <li>Disappearance of any soft tissue plasmacytomas and</li> <li>&lt; 5% plasma cells in bone marrow and</li> <li>Normal SFLC ratio and</li> <li>Absence of clonal cells in bone marrow<sup>c</sup></li> </ul> |
| CR <sup>b</sup> | <ul> <li>Negative immunofixation on the serum and urine and</li> <li>Disappearance of any soft tissue plasmacytomas and</li> <li>&lt; 5% plasma cells in bone marrow</li> </ul> |
| VGPR <sup>b, d</sup> | Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-component with urine M-component < 100 mg per 24 hours If the serum and urine M-protein are not measurable, a decrease of > 90% in the difference between the involved and uninvolved sFLC levels is required in place of the M-protein criteria |
| PR <sup>b, d</sup> | <ul> <li>≥ 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥ 90% or to &lt; 200 mg per 24 hours</li> <li>If the serum and urine M-protein are not measurable, a decrease ≥ 50% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria.</li> <li>If present at baseline, a ≥ 50% reduction in the size of soft tissue plasmacytomas is also required<sup>d, e</sup></li> </ul> |
| Stable | Not meeting criteria for CR, VGPR, PR, or PD |
| PDc | <ul> <li>Any one or more of the following increase of ≥ 25% from lowest response value in:</li> <li>Serum M-component (absolute increase must be ≥ 0.5 g/dL) and/or</li> <li>Urine M-component (absolute increase must be ≥ 200 mg per 24 hours) and/or</li> <li>Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase must be &gt; 10 mg/dL)</li> </ul> |
| | <ul> <li>Only in patients without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow plasma cell percentage (absolute percentage must be ≥ 10%)</li> <li>Bone marrow plasma cell percentages (absolute % must be ≥ 10%)</li> <li>Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in size of existing bone lesions or soft tissue plasmacytomas<sup>f, g, h</sup></li> <li>Development of hypercalcemia (corrected serum calcium &gt; 11.5 mg/dL or 2.65 mmol/L) attributed solely to the plasma cell proliferative disorder</li> </ul> |

Footnotes are defined on next page



Supplemental Clinical Study Report: 20130411


Table D1 Summary of International Myeloma Working Group-Uniform Response Criteria (IMWG-URC) (cont'd)

| Response | |
|--------------------------|-------------------|
| Subcategory <sup>a</sup> | Response Criteria |

Sources: Blade 1998; Durie 2006; Rajkumar 2011.

CR = complete response; sCR = stringent complete response; FLC = free light chain; PD = progressive disease; PR = partial response; SFLC = serum free light chain; VGPR = very good partial response.

- <sup>a</sup> Subjects with measurable disease in both serum (SPEP) and urine (UPEP) at study entry are required to meet response criteria in both UPEP and SPEP in order to qualify for a PR or better. Conversely, it should be noted that criteria for progressive disease only needs to be met, and confirmed, in one parameter.
- b All response categories (CR, sCR, VGPR, PR) require two consecutive assessments made at any time before the institution of any new therapy, as well as no known evidence of progressive or new bone lesions if radiographic studies were performed. Radiographic studies are not required to satisfy these response requirements. Bone marrow assessments are not required to be confirmed by repeat testing.
- c Presence/absence of clonal cells is based on the κ/λ ratio. An abnormal κ/λ ratio by immunohistochemistry and/or immunofluorescence requires a minimum of 100 plasma cells for analysis. An abnormal ratio reflecting presence of an abnormal clone is κ/λ of > 4:1 or < 1:2.</p>
- d Response criteria for all categories and subcategories of response except CR and VGPR are applicable only to patients that have "measurable" disease defined by at least one of SPEP ≥ 1.0 g/dL) or UPEP ≥ 200 mg per 24 hours; except for assessment of sCR, CR, or VGPR, patients with measurable disease restricted to SPEP will need to be followed only by SPEP. Correspondingly, patients with measurable disease restricted to UPEP will need to be followed only by UPEP.
- <sup>c</sup> Determination of PD based on based on M-protein, hypercalcemia, or FLC while on study requires two consecutive assessments made at any time before classification of progressive disease and/or the institution of new therapy. Serum M-component increases of ≥ 1 g/dL are sufficient to define progression if starting M-component is ≥ 5 g/dL.
- f Plasmacytomas: A definite increase in the size is defined as a ≥ 50% increase as measured serially by the sum of the products of the cross-diameters of the measurable lesion. A plasmacytoma is considered measurable if the longest diameter is at least 1 cm and the product of the cross diameters is at least 1 cm². Plasmacytomas of lesser size will be considered nonmeasurable.
- g The requirement for bi-directional measurements will only be applied to plasmacytomas.
- h The plasmacytoma specifications for PD are based on the sponsor's interpretation of the IMWG-URC and practical considerations for study execution.



Date: 30 July 2019


Table D2 Definition of Minimal Response per EBMT Criteria

| Minimal Response | |
|---|---|
| Response<br>Subcategory | Response Criteria |
| MR <sup>a</sup> | ≥ 25 but < 49% reduction in serum M-protein and a 50–89% reduction in 24-hour urinary M-protein, which still exceeds 200 mg per 24 h |
| | If the serum and urine M-protein are not measurable, a decrease of 25%–49% in the difference between involved and uninvolved FLC levels is required in place of the M-protein criteria. |
| | For patients with nonsecretory myeloma only, 25–49% reduction in plasma cells in a bone marrow aspirate and on trephine biopsy, if biopsy is performed |
| | 25–49% reduction in the size of soft tissue plasmacytomas (by radiography or clinical examination) |

Sources: Bladé 1998; Kyle 2009.

EBMT = European Group for Blood and Marrow Transplantation; FLC = free light chain; MR = minimal response.

Approved




<sup>&</sup>lt;sup>a</sup> The response category MR requires 2 consecutive assessments made at any time before the institution of any new therapy, as well as no known evidence of progressive or new bone lesions if radiographic studies were performed. Radiographic studies are not required to satisfy these response requirements. Bone marrow assessments are not required to be confirmed by repeat testing.

Supplemental Clinical Study Report: 20130411


## APPENDIX D EUROPEAN ORGANIZATION FOR RESEARCH AND TREATMENT OF CANCER (EORTC) CORE MODULE (QLQ-C30) AND EORTC MULTIPLE MYELOMA MODULE (QLQ-MY20)

Subjects should be instructed to fill out the EORTC QLC-C30 (Version 3) and EORTC QLC-MY20 questionnaires to the best of their abilities. The study staff will be responsible for confirming that the subject has completed the questionnaires.

Citations for the EORTC QLQ-C30 and the EORTC QLQ-MY20 are provided in the Reference List (Aaronson 1993; Fayers 2001; Cocks 2007).

Approved



Supplemental Clinical Study Report: 20130411


# APPENDIX E NEUROTOXICITY SUBSCALE OF THE GYNECOLOGIC ONCOLOGY GROUP'S FUNCTIONAL ASSESSMENT OF CANCER THERAPY (FACT/GOG-NTX4 [VERSION 4])

Subjects with neurotoxicities should be instructed to fill out the FACT/GOG-Ntx4 (Version 4) to the best of their abilities. The study staff will be responsible for confirming that the subject has completed the questionnaire.

Approved



**Supplemental Clinical Study Report: 20130411** 


### APPENDIX F EQ-5D-5L (V.2)

Subjects should be instructed to fill out the EQ-5D-5L (v.2) questionnaire to the best of their abilities. The study staff will be responsible for confirming that the subject has completed the questionnaire.

Approved



Supplemental Clinical Study Report: 20130411


#### EASTERN COOPERATIVE ONCOLOGY GROUP (ECOG) APPENDIX G PERFORMANCE SCALE

| Grade | Description |
|---|---|
| 0 | Normal activity, fully active, able to carry on all predisease performance without restriction. |
| 1 | Symptoms, but fully ambulatory, restricted in physically strenuous but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than $50\%$ of waking hours. |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | Completely disabled. Cannot carry on any self care. Totally confined to bed or chair. |
| 5 | Death |

Source: Oken 1982

Eastern Cooperative Oncology Group, Robert Comis M.D., Group Chair

Approved



Supplemental Clinical Study Report: 20130411


#### APPENDIX H DRUG-DRUG INTERACTION POTENTIAL OF OPROZOMIB AND POMALIDOMIDE

#### **Oprozomib**

| Alfentanil | Diergotamine | Quinidine |
|-------------------------|--------------|--------------|
| Astemizole <sup>a</sup> | Ergotamine | Sirolimus |
| Cisapride <sup>a</sup> | Fentanyl | Tacrolimus |
| Cyclosporine | Pimozide | Terfenadinea |

<sup>&</sup>lt;sup>a</sup> Not available in the United States.

Because oprozomib is a P-gp substrate, use of P-gp inhibitors and inducers (see table below) should be carefully monitored and such drugs should be substituted for others if necessary.

#### **Pomalidomide**

In accordance with the Pomalidomide Prescribing Information, use of the following concomitant medications is to be carefully monitored and these drugs should be substituted for others if necessary.

#### Drugs That May Increase Pomalidomide Plasma Concentrations

CYP3A, CYP1A2, or P-gp inhibitors: Co-administration of POMALYST with drugs that are strong inhibitors of CYP1A2, CYP3A (e.g., ketoconazole) or P-gp could increase exposure and should be avoided.

#### Drugs That May Decrease Pomalidomide Plasma Concentrations

CYP3A, CYP1A2, or P-gp inducers: Co-administration of POMALYST with drugs that are strong inducers of CYP1A2, CYP3A (e.g., rifampin) or P-gp could decrease exposure and should be avoided.

#### **Smoking**

Cigarette smoking may reduce pomalidomide exposure due to CYP1A2 induction. Subjects should be advised that smoking may reduce the efficacy of pomalidomide.





Supplemental Clinical Study Report: 20130411


The tables below provide lists of the inhibitors and inducers of concern.

| CYP 3A inhibitor | CYP1A2 inhibitor | |
|---|---|---|
| Strong: | Strong: | P-gp inhibitor |
| boceprevir | ciprofloxacin | amiodarone |
| clarithromycin | enoxacin | azithromycin |
| conivaptan | fluvoxamine | captopril |
| grapefruit juice | | carvedilol |
| indinavir | | clarithromycin |
| itraconazole | | conivaptan |
| ketoconazole | | cyclosporine |
| lopinavir/ritonavir | | diltiazem |
| mibefradil | | dronedarone |
| nefazodone | | erythromycin |
| nelfinavir | | felodipine |
| posaconazole | | itraconazole |
| ritonavir | | ketoconazole |
| saquinavir | | lopinavir and ritonavir |
| telaprevir, telithromycin, | | quercetin |
| voriconazole | | quinidine, ranolazine, ticagrelor, verapamil |

| CYP 3A inducer | | |
|-----------------|----------------|----------------------|
| Strong: | CYP1A2 inducer | P-gp inducer |
| avasimibe | | avasimibe |
| carbamazepine | | carbamazepine |
| phenytoin | | phenytoin |
| rifampin | | rifampin |
| St. John's wort | | St John's wort |
| | | tipranavir/ritonavir |



Supplemental Clinical Study Report: 20130411


### APPENDIX I POMALIDOMIDE RISKS OF FETAL EXPOSURE, PREGNANCY TESTING GUIDELINES, AND ACCEPTABLE BIRTH CONTROL METHODS

#### **Risks Associated with Pregnancy**

Pomalidomide was found to be teratogenic in a developmental study in rabbits.

Pomalidomide is an analogue of thalidomide. Thalidomide is a known human teratogen that causes severe life-threatening human birth defects. If pomalidomide is taken during pregnancy, it may cause birth defects or death to an unborn baby.

#### Criteria for Females of Childbearing Potential (FCBP)

This protocol defines a female of childbearing potential as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

#### Counseling

For an FCBP, pomalidomide is contraindicated unless all of the following are met (i.e., FCBP must be counseled concerning the following risks and requirements prior to the start of pomalidomide study therapy):

- She understands the potential teratogenic risk to the unborn child
- She understands the need for effective contraception, without interruption, 28 days before starting study treatment, throughout the entire duration of study treatment, dose interruption, and 28 days after the End of Study Treatment
- She should be capable of complying with effective contraceptive measures
- She is informed and understands the potential consequences of pregnancy and the need to notify her study doctor immediately if there is a risk of pregnancy
- She understands the need to commence the study treatment as soon as pomalidomide is dispensed following a negative pregnancy test
- She understands the need and accepts to undergo pregnancy testing based on the frequency outlined in this protocol
- She acknowledges that she understands the hazards and necessary precautions associated with the use of pomalidomide





Supplemental Clinical Study Report: 20130411


#### The Investigator must ensure that females of childbearing potential:

• Comply with the conditions for pregnancy risk minimization, including confirmation that she has an adequate level of understanding

• Acknowledge the aforementioned requirements

For a female NOT of childbearing potential, pomalidomide is contraindicated unless the following are met (i.e., all females NOT of childbearing potential must be counseled concerning the following risks and requirements prior to the start of pomalidomide study therapy):

• She acknowledges that she understands the hazards and necessary precautions associated with the use of pomalidomide

The effect of pomalidomide on spermatogenesis is not known and has not been studied.

Therefore, male subjects taking pomalidomide must meet the following conditions (i.e., all males must be counseled concerning the following risks and requirements prior to the start of pomalidomide study therapy):

- Understand the potential teratogenic risk if engaged in sexual activity with a woman of childbearing potential
- Understand the need for the use of a condom, even if he has had a vasectomy, if engaged in sexual activity with a female of childbearing potential.

#### Contraception

Females of childbearing potential enrolled in this protocol must agree to use 2 reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 28 days after study treatment discontinuation.

The 2 methods of reliable contraception must include 1 highly effective method and 1 additional effective (barrier) method. An FCBP must be referred to a qualified provider of contraceptive methods if needed.

Approved



Date: 30 July 2019


Onyx Therapeutics Oprozomib ER Tablets

The following are examples of highly effective and additional effective methods of contraception:

- Highly effective methods:
  - o Intrauterine device (IUD)
  - o Hormonal (birth control pills, injections, implants)
  - o Tubal ligation
  - Partner's vasectomy
- Additional effective methods:
  - o Male condom
  - Diaphragm
  - o Cervical cap

Because of the increased risk of venous thromboembolism in patients with multiple myeloma taking pomalidomide and dexamethasone, combined oral contraceptive pills are not recommended. If a subject is currently using combined oral contraception the subject should switch to another one of the effective methods listed above. The risk of venous thromboembolism continues for 4–6 weeks after discontinuing combined oral contraception.

The efficacy of contraceptive steroids may be reduced during co-treatment with dexamethasone.

Implants and levonorgestrel-releasing intrauterine systems are associated with an increased risk of infection at the time of insertion and irregular vaginal bleeding. Prophylactic antibiotics should be considered, particularly in subjects with neutropenia.

#### **Pregnancy testing**

Medically supervised pregnancy tests with a minimum sensitivity of 50 mIU/mL must be performed for females of childbearing potential, including females of childbearing potential who commit to complete abstinence, as outlined below.

Approved



Supplemental Clinical Study Report: 20130411


#### Before starting study drug

#### Female Subjects

Females of childbearing potential must have 2 negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to starting pomalidomide. The first pregnancy test must be performed within 10-14 days prior to the start of pomalidomide and the second pregnancy test must be performed within 24 hours prior to the start of pomalidomide. The subject may not receive study drug until the investigator has verified that the results of these pregnancy tests are negative.

#### Male Subjects

Must practice complete abstinence or agree to use a condom during sexual contact with FCBP while participating in the study, during dose interruptions, and for at least 90 days following study drug discontinuation, even if he has undergone a successful vasectomy.

#### During study participation and for 28 days following study drug discontinuation

#### Female Subjects

- Females of childbearing potential with regular or no menstrual cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while on study, at study discontinuation, and at Day 28 following study drug discontinuation. If menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days and then every 14 days while on study, at study discontinuation, and at Days 14 and 28 following study drug discontinuation.
- At each visit, the investigator must confirm with the FCBP that she is continuing to use 2 reliable methods of birth control.
- Counseling about pregnancy precautions and the potential risks of fetal exposure must be conducted at a minimum of every 28 days.
- If pregnancy or a positive pregnancy test does occur in a study subject, pomalidomide must be immediately discontinued.
- Pregnancy testing and counseling must be performed if a subject misses her period or if her pregnancy test or her menstrual bleeding is abnormal. Study drug treatment must be discontinued during this evaluation.
- Females must agree to abstain from breastfeeding during study participation and for at least 28 days after study drug discontinuation.

Approved



Supplemental Clinical Study Report: 20130411


#### Male Subjects

- Counseling about the requirement for condom use during sexual contact with FCBP and the potential risks of fetal exposure must be conducted at a minimum of every 28 days.
- If pregnancy or a positive pregnancy test does occur in the partner of a male study subject during study participation, the investigator must be notified immediately.

#### **Additional precautions**

- Subjects should be instructed never to give this medicinal product to another person and to return any unused capsules to the investigator at the End-of-Treatment.
- Subjects should not donate blood during therapy and for at least 28 days following discontinuation of pomalidomide.
- Male subjects should not donate semen or sperm during therapy or for at least 90 days following discontinuation of pomalidomide.
- Only enough pomalidomide for 1 cycle of therapy may be dispensed with each cycle of therapy.

Approved




Supplemental Clinical Study Report: 20130411


#### POMALIDOMIDE EDUCATION AND COUNSELLING APPENDIX J **GUIDANCE DOCUMENT**

| Prot | tocol Number: OPZ007 |
|---|---|
| Patio | ent Name (Print): DOB:/(mm/dd/yyyy) |
| Fem | <u>rale</u> |
| If fe | male, check one: |
| | FCBP (female of childbearing potential): Sexually mature female who: 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months) |
| | NOT FCBP |
| To be completed prior to each dispensing of pomalidomide | |

#### Do Not Dispense pomalidomide if:

- The patient is pregnant.
- No pregnancy tests were conducted for a FCBP.
- The patient states she did not use TWO reliable methods of birth control (unless practicing complete abstinence of heterosexual intercourse) [at least 28 days prior while taking pomalidomide, during dose interruption, and 28 days after discontinuation of pomalidomide].

#### **FCBP**

- 1. I verified that the required pregnancy tests performed are negative.
- 2. I counseled FCBP regarding the following:
- Potential fetal harm: If pomalidomide is taken during pregnancy, it may cause birth defects or death to any unborn baby. Females are advised to avoid pregnancy while taking pomalidomide. The teratogenic potential of pomalidomide in humans cannot be ruled out. Females of childbearing potential must agree not to become pregnant while taking pomalidomide.






- Using TWO reliable methods of birth control at the same time or complete abstinence from heterosexual intercourse [at least 28 days prior, while taking pomalidomide, during dose interruption, and 28 days after discontinuation of pomalidomide].
- Continuation of TWO reliable methods of birth control or complete abstinence if therapy is interrupted.
- That even if she has amenorrhea she must comply with advice on contraception.
- Use of one highly effective method and one additional method of birth control AT THE SAME TIME. The following are examples of highly effective and additional effective methods of contraception:
  - Highly effective methods:
    - Intrauterine device (IUD)
    - Hormonal (birth control pills, injections, implants)
    - **Tubal ligation**
    - Partner's vasectomy
  - Additional effective methods:
    - Male condom
    - Diaphragm
    - Cervical cap
- Pregnancy tests before and during treatment, even if the patient agrees not to have reproductive heterosexual intercourse. Two pregnancy tests will be performed prior to receiving study drug, one within 10-14 days and the second within 24 hours of the start of pomalidomide.
- Frequency of pregnancy tests to be done:
  - o Every week during the first 28 days of this study and a pregnancy test every 28 days during the patient's participation in this study if menstrual cycles are regular or every 14 days if cycles are irregular.
  - If the patient missed a period or has unusual menstrual bleeding.
  - When the patient is discontinued from the study and at Day 28 after study drug discontinuation if menstrual cycles are regular. If menstrual cycles are irregular, pregnancy tests will be done at discontinuation from the study and at Days 14 and 28 after study drug discontinuation.
- Stop taking pomalidomide immediately in the event of becoming pregnant and to call their study doctor as soon as possible.
- NEVER share pomalidomide with anyone else.



Supplemental Clinical Study Report: 20130411


- Do not donate blood while taking pomalidomide and for 28 days after stopping pomalidomide.
- Do not breastfeed a baby while participating in this study and for at least 28 days after study drug discontinuation.
- Do not break, chew, or open pomalidomide capsules.
- Return unused pomalidomide to the investigator.
- 3. Provide Pomalidomide Information Sheet to the patient.

## <u>Female not of childbearing potential (natural menopause for at least 24 consecutive months, a hysterectomy, or bilateral oophorectomy):</u>

- 1. I counseled the female NOT of childbearing potential regarding the following:
- Potential fetal harm (Refer to item #2 in FCBP).
- NEVER share pomalidomide with anyone else.
- Do not donate blood while taking pomalidomide and for 28 days after stopping pomalidomide.
- Do not break, chew, or open pomalidomide capsules.
- Return used pomalidomide capsules to the investigator.
- 2. Provide Pomalidomide Information Sheet to the patient.

## Male

- 1. I counseled the Male patient regarding the following:
- Potential fetal harm (Refer to item #2 in FCBP).
- To engage in complete abstinence or use a condom when engaging in sexual intercourse (including those who have had a vasectomy) with a FCBP, while taking pomalidomide, during dose interruptions, and for 28 days after stopping pomalidomide.
- Males should notify their study doctor when their female partner becomes pregnant and
  female partners of males taking pomalidomide should be advised to call their healthcare
  provider immediately if they get pregnant.
- NEVER share pomalidomide with anyone else.
- Do not donate blood while taking pomalidomide and for 28 days after stopping pomalidomide.
- Do not donate semen or sperm while taking pomalidomide and for 90 days after stopping pomalidomide.
- Do not break, chew, or open pomalidomide capsules.


Approved



patient records.

Supplemental Clinical Study Report: 20130411


| Clinical Sti | ady Proto | ocol No. OPZ<br>Page 146 of |
|--------------|-----------|-----------------------------|
| t. | | |
| _ | | |
| Date | / | / |
| _ Date | / | / |
| | <b>t.</b> | <b>t.</b> |

Approved



Supplemental Clinical Study Report: 20130411


# APPENDIX K POMALIDOMIDE INFORMATION SHEET FOR PATIENTS ENROLLED IN CLINICAL RESEARCH STUDIES

Please read this Pomalidomide Information Sheet before you start taking pomalidomide and each time you get a new supply, since there may be new information. This Pomalidomide Information Sheet does not take the place of an informed consent to participate in clinical research or talking to your study doctor or healthcare provider about your medical condition or your treatment.

## What is the most important information I should know about pomalidomide?

Pomalidomide may cause birth defects (deformed babies) or death of an unborn baby.

Pomalidomide is similar to the medicine thalidomide. It is known that thalidomide causes life-threatening birth defects. Pomalidomide has not been tested in pregnant women but may also cause birth defects. Pomalidomide was found to cause birth defects when tested in pregnant rabbits.

If you are a female who is able to become pregnant:

- Do not take pomalidomide if you are pregnant or plan to become pregnant
  - o For 28days before starting pomalidomide
  - While taking pomalidomide
  - o During dose interruptions of pomalidomide
  - o For 28 days after stopping pomalidomide
- Stop taking pomalidomide if you become pregnant during pomalidomide treatment
- Do not breastfeed while taking pomalidomide
- You must have pregnancy testing done at the following times:
  - o Within 10–14 days and again 24 hours prior to the first dose of pomalidomide
  - Weekly for the first 28 days
  - Every 28 days after the first month or every 14 days if you have irregular menstrual periods
  - o If you miss your period or have unusual menstrual bleeding





Supplemental Clinical Study Report: 20130411


- 28 days after the last dose of pomalidomide (14 and 28 days after the last dose if menstrual periods are irregular)
- You must either not have any sexual relations with a man or use 2 reliable, separate forms of effective birth control at the same time:
  - o For 28 days before starting pomalidomide
  - While taking pomalidomide
  - During dose interruptions of pomalidomide and for 28 days after stopping pomalidomide
  - The study doctor will be able to advise you where to get additional advice on contraception.
  - If you suspect you are pregnant at any time during the study, you must stop
    pomalidomide immediately and immediately inform your study doctor.
    The study doctor will report all cases of pregnancy to Celgene Corporation
    and to Onyx Therapeutics.

If you are a female not of childbearing potential:

In order to ensure that an unborn baby is not exposed to pomalidomide, your study doctor will confirm that you are not able to become pregnant.

If you are a male:

The effect of pomalidomide on sperm development is not known and has not been studied. The risk to the fetus in females of childbearing potential whose male partner is receiving pomalidomide is unknown at this time.

- Male patients (including those who have had a vasectomy) must either not have any
  sexual relations with a female who can become pregnant or a pregnant female or must
  use a condom during sexual intercourse with a pregnant female or a female that can
  become pregnant:
  - o While you are taking pomalidomide
  - During dose interruptions of pomalidomide
  - o For 90 days after you stop taking pomalidomide
- Male patients should not donate sperm or semen while taking pomalidomide and for 90 days after stopping pomalidomide.
- If you suspect that your partner is pregnant any time during the study, you must immediately inform your study doctor. The study doctor will report all cases of pregnancy to Celgene Corporation and to Onyx Therapeutics.





Supplemental Clinical Study Report: 20130411


## Pomalidomide restrictions in sharing pomalidomide and donating blood:

- Do not share pomalidomide with other people. It must be kept out of the reach of children and should never be given to any other person.
- Do not give blood while you take pomalidomide and for 28 days after stopping pomalidomide.
- Do not break, chew, or open pomalidomide capsules.
- You will be supplied with no more than 1 cycle of pomalidomide
- Return unused pomalidomide capsules to your study doctor.

Additional information is provided in the informed consent form and you can ask your study doctor for more information.

Approved





#### APPENDIX L ACTG BRIEF PERIPHERAL NEUROPATHY SCREENING TOOL

Source: NIAID Adult AIDS Clinical Trials Group

## 1. Elicit Subjective Symptoms

Ask the patient to rate the severity of each symptom listed in Question 1 on a scale of 01 (mild) to 10 (most severe) for right and left feet and legs. Enter the score for each symptom in the columns marked R (right lower limb) and L (left lower limb). If a symptom has been present in the past, but not since the last visit, enter "00 - Currently Absent." If the symptom has never been present, enter "11 - Always Been Normal."

| Always Been Normal | $\mathbf{Mild} \longleftarrow \mathbf{Severe}$ | | |
|---|---|---|---|
| 11 | 11 00 01 02 03 04 05 06 07 | 09 | 10 |
| Symptoms | | | L |
| a. Pain, aching, or burning | a. Pain, aching, or burning in feet, legs | | |
| b. "Pins and needles" in feet, legs | | | |
| c. Numbness (lack of feeling | ng) in feet, legs | | |

# Approved

### 2. Grade Subjective Symptoms

Use the single highest severity score from Question 1 above to obtain a subjective sensory neuropathy score. If all severity scores are "00" or "11," the subjective sensory neuropathy score will equal "0."



Supplemental Clinical Study Report: 20130411


## APPENDIX M ACTG BRIEF PERIPHERAL NEUROPATHY SCREENING TOOL (CONT'D)

Subjective Sensory Neuropathy Score (based on highest severity rating)

01-03 = grade of 1

04-06 = grade of 2

07-10 = grade of 3

11 or 00 = grade of 0

| R | L |
|---|---|

## 3. Evaluate Perception of Vibration

Compress the ends of a 128-Hz tuning fork just hard enough that the sides touch. Place the vibrating tuning fork on a bony prominence on the patient's wrist or hand to be sure that he/she can recognize the vibration or "buzzing" quality of the tuning fork. Again, compress the ends of the tuning fork just hard enough that the sides touch. Immediately place the vibrating tuning fork gently but firmly on the top of the distal interphalangeal (DIP) joint of one great toe and begin counting the seconds. Instruct the patient to tell you when the "buzzing" stops. Repeat for the other great toe.

### Vibration perception

a. Great toe DIP joint perception of vibration in seconds

b. Vibration perception score

0 = felt > 10 seconds (normal)

1 = felt 6-10 seconds (mild loss)

2 = felt < 5 seconds (moderate loss)

3 = not felt (severe loss)

8 = unable to or did not assess

| R | L |
|---|---|





Supplemental Clinical Study Report: 20130411


# APPENDIX M ACTG BRIEF PERIPHERAL NEUROPATHY SCREENING TOOL (CONT'D)

## 4. Evaluate Deep Tendon Reflexes

With the patient seated, the examiner uses one hand to press upward on the ball of the foot, dorsiflexing the patient's ankle to 90 degrees. Using a reflex hammer, the examiner then strikes the Achilles tendon. The tendon reflex is felt by the examiner's hand as a plantar flexion of the foot, appearing after a slight delay from the time the Achilles tendon is struck. Use reinforcement by having the patient clench his/her fist before classifying the reflex as absent.

#### **Ankle Reflexes Score**

0 = absent

1 = hypoactive

2 = normal deep tendon reflexes

3 = hyperactive

4 = clonus

8 = unable to or did not assess

| L |
|---|

From Peripheral Neuropathy

**Primary Care of Veterans with HIV** 

Office of Clinical Public Health Programs

Veterans Health Administration, 2009

Approved



Supplemental Clinical Study Report: 20130411


## APPENDIX M SAMPLE BRIEF PAIN INVENTORY – SHORT FORM (BPI-SF)

Source: Cleeland 2006. Date: Study ID: Hospital: **Brief Pain Inventory (Short Form)** 1. Throughout our lives, most of us have had pain from time to time (such as minor headaches, sprains, and toothaches). Have you had pain other than these everyday kinds of pain today? □No 2. On the diagram, shade in the areas where you feel pain. Put an X on the area that hurts the most. 3. Please rate your pain by marking the box beside the number that be describes your pain at its worst in the last 24 hours. □ 1 □ 2 □ 3 8 🗌 □9 □ 0 □ 10 Pain As Bad As You Can Imagine 4. Please rate your pain by marking the box peside the number that best describes your pain at its least in the last 24 hours. □ 1 □ 2 □ 3 **4** 8 9 5 □6 **7** Pain As Bad As You Can Imagine 5. Please rate your pain by marking the box beside the number that best describes your pain on the average. □ 0 □ 1 □ 2 □ 3 □ 4 □ 5 □ 6 □ 7 10 Pain As Bad As You Can Imagine □8 □9 6. Please rate your pain by marking the box beside the number that tells how much pain you have right □ 0 
 □1
 □2
 □3
 □4
 □5
 □6
 □7
 □8
 □9
 No Pain Pain As Bad As Copyright 1991 Charles S. Cleeland, PhD Pain Research Group Page 1 of 2 All rights reserved



Product: Oprozomib Supplemental Clinical Study Report: 20130411


| Date | e: | | | | | Study ID: | | | _ | |
|---|---|---|---|---|---|---|---|---|---|---|
| Hos | spital: | | | _ | | | | | | |
| 7. <b>W</b> hat | t treatı | ments or m | edication | ns are you | ı receivin | g for you | r pain? | | | |
| | $\dagger \dagger$ | | | | | | | | | |
| mark<br>0%<br>□ | | 24 hours, hox below th | | | • | | | | | ved.<br>100%<br>□ |
| No<br>Relief | ш | | | | | | Ш | | | Complete<br>Relief |
| A. Gen | | | □3 | <b>□</b> 4 | □ 5 | □6 | <b>□</b> 7 | □8 | □9 | ☐ 10 |
| Does No<br>Interfere<br>B. Moo | | 1 □2 | ∏3 | □4 | ∏5 | □6 | | . □8 | ∏9 | Comple<br>Interfere |
| Does No Interference C. Wal | ot —<br>∍ | | | | | | | | | Compl |
| 0<br>Does No | ot - | _ | 3 | | □5 | □6 | 7 | □8 | □9 | ☐ 10<br>Compl<br>Interfe |
| D. Nor | mal W | ork (includ | e hoth w | vork oatsi | de the ho | me and l | ousewo | rk) | | |
| 0<br>Does No<br>Interfere | | 1 | <b>\</b> | □4 | □ 5 | □6 | <b>□</b> 7 | □8 | □9 | ☐ 10<br>Comple<br>Interfer |
| | | with other | · ·_ | _ | _ | _ | _ | _ | _ | _ |
| ☐ 0<br>Does No<br>Interfere | | 1 | □3 | <b>□</b> 4 | □ 5 | □6 | <b>□</b> 7 | □8 | □9 | ☐ 10<br>Comple<br>Interfer |
| F. Slee | · | . – | | | | | | | | |
| 0 Does No | | | □3 | □ 4 | □ 5 | □6 | <b>□</b> 7 | □8 | □9 | 10<br>Comple<br>Interfer |
| G. Enjo | oymen<br> | | □3 | □4 | □5 | □6 | □7 | <b>□</b> 8 | □9 | □ 10 |
| Does No | | . Ц | | _ → | | | | _ u | | Complete |




#### EXAMPLE ELECTRONIC SERIOUS ADVERSE EVENT APPENDIX N **CONTINGENCY REPORT FORM**

| AMGEN | . El | lectronic | Seri | ous Ad | vers | e E | ven | t Co | on | ting | end | у Г | Rep | ort Fo | rm |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study # 201304 <sup>a</sup><br>Oprozomib | 11 | | | | For i | Rest | ricte | d U | se | | | | | | |
| Оргодонны | | | | | | | | | _ | | | | | | |
| Reason for reporting | | | | | | | | | | | | | | | |
| The Clinical Trial Da | | | | | | | | | | | | | | | |
| ☐ Is not available du | | _ | ny site | | | | | | | | | | | | |
| ☐ Is not yet available | for this stu | udy | | | | | | | | | | | | | |
| ☐ Has been closed for | or this stud | y | | | | | | | | | | | | | |
| | | on by COM p | orior to | providing | g to si | tes: | SELE | CT O | )R 1 | YPE | IN A | FAX | (#>> | | |
| 1. SITE INFORMATION Site Number | | Investig | ator | | | _ | | | | | Cour | ntrv | | | |
| | | - | | | | | | | | | | • | | | |
| F | Reporter | | Pho | one Number | | | | | | Fax Num | ber | | | | |
| | | | ( | ) | | | | | | ( | ) | | | | |
| 2. SUBJECT INFORMA Subject ID Number | | Age at event on: | sat | | | Sex | | | Race | | H | annlin | ahla ne | ovide End of | Shudu |
| | - | Age at event on | 361 | | | 1 | De Dr | м | nava | = | | ate | aute, pri | ovide End of | Siady |
| | | | | | | | | ** | | | | | | | |
| If this is a follow-up to an e | | | tem (eg | , Rave), prov | ide the | advers | e event | term: | _ | | | | | | _ |
| and start date: Day 3. SERIOUS ADVERSE | | Year | | | | | | | | | | | | | |
| Provide the date the Invest | | e aware of this in | nformatio | on: Day | Month | Ye | ar | | | | | | | | |
| Serious Adverse Event diagno<br>If diagnosis is unknown, enter: | | | | | Check<br>only if | č | ifserious<br>enter | le the | | Rak<br>easonable | ionehip<br>nossih | | theFuen | Outcome<br>t of Event | Check only |
| and provide diagnosis, when ke | | | | Date Ended | event | serions? | Serious | | n | nay have b<br>ngen devi | een ca | used by | | -Resolved | related to<br>study |
| up report<br>List one event per line. If event | is fatal, enter the | | <sup>2</sup> 1 | Date Elided | before<br>first dose | t se | Criteria<br>code | 1 0 | an Ai | ngen dem | IP? | 10 00111 | mater an | -Fatal | |
| cause of eeath. Entry of "death"<br>as this is an outco | | e, | | | of IP | event | (see<br>codes | | | | | | | -Unknown | eg, biops |
| da inio la di Outco | me. | Day Month | Year Day | Month Year | | <u>00</u> | below) | 4Pid<br>No-∕ | evice><br>Yes• | ◆Piderice No-/ Yes | | | ◆Pidevio<br>No-1 Ye | | |
| | | | | | | □Yes<br>□No | | П | | | | | | | |
| | | | | | | □Yes | | H | $\dashv$ | | | | _ | | +- |
| | | | | | | □No | | Ш | _ | | | | _ | | |
| | | | | | | □Yes<br>□No | | | | | | | | | |
| Serious 01 Fatal<br>Criteria: 02 immediately | life-threatening | | | onged hospitaliz<br>Ignificant disabi | | pacity | | | | | | | | irth defect<br>ant serious e | vent |
| 4. Was subject hospita | | | | | | | nt? □N | 4o 🗆 | Yes | | | | | | |
| | Date Admi | itted | | T | | | | | Da | te Disc | harge | d | | | |
| D | ay Month | Year | | | | | | D | ay | Mont | h | Year | | | |
| 5. Was IP/drug under s | study admii | nistered/taker | n prior t | to this even | ıt? □N | n ПУ | es If ve | s nle | 956 | comple | te all | of Se | ction 5 | | |
| or trad it raining attack to | raay aanin | | | | Prior to | o, or at | time of E | vent | | | A | ction 1 | Taken | | |
| | | Date of Initial [ | Dose | Date of D | )ose | Do | 98 F | Route | F | requenc | | ith Pro | | | |
| | | | | | | | | | | | Adi | ministe | red | Lot # and | Serial # |
| | | | | | | | | | | | dis | continu | | | |
| IP/Amgen Device: | | Day Month | Year [ | Day Month | Year | + | - | | + | | 03 | Withh | eld | Lot# | |
| | | | | | | | | | | | | | | ☐ Unknown | |
| | | | | | | | | | | | | | | Serial # | |
| Oprozomib 🗆 ынde | ed 🗆 open label | | | | | | | | | | | | | Unknown | sle / |
| | | | | | | | | | Τ | | | | | Lot# | |
| | | | | | | | | | | | | | | Serial # | |
| | | | | | | | | | | | | | | Unevailed | ole / |
| Oprozomib 🗆 blinde | ed □ open label | | | | | | | | | | | | | Unknown | |






Supplemental Clinical Study Report: 20130411


| AMGEN<br>Study # 20130411 | Electronic Serious Adverse Event Contingency Report Form |
|---|---|
| Oprozomib | For Restricted Use |

| | | | | Site N | umber | | | | | Su | bject II | ) Num | ber | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| . CONC | OMITANT M | IEDICATION | | | | | | | | | | | | es, p | olease | complete: | | | |
| Med | dication Name | e(s) | Dey 8 | Start Da | | Dey | Stop | Date<br>th Y | | | uspect<br>Yæ√ | Con<br>No. | tinuing<br>Yæ√ | | Dose | Route | Freq. | Treat | ment Me<br>Yee |
| | | | | | | | | | Τ, | | 100 | | 1 | | | | | 1.2 | 1 |
| | | | | | | | | | + | $\dashv$ | | | | | | | | <del> </del> | + |
| | | | | | | | | | + | | | | | | | | | | $\vdash$ |
| | | | | | | | | | 4 | _ | | | | | | | | | <u> </u> |
| . RELE | VANT MEDI | CAL HIST | ORY | (inclu | ide da | tes, | allei | rgies | and | l any | relev | ant p | rior th | eraj | oy) | | | | |
| DELE | VANT LABO | DATORY | 7.1/4.1.1 | IIE¢ / | inalu | do ha | nodi | no 14 | alua | al A | Dala | | abazat | | -12 | | a Maria ale | | ! |
| , KLLL | Test | MATORI | VAL | JE3 ( | morac | re va | Sen | ne v | aiuea | <i>3)</i> ~ | ly rese | vanu | abolati | луч | alues: | 100016 | s II yes, pi | ease ou | mpiete |
| | Unit | | | _ | | | + | | | | - | | | $\dashv$ | | | | | |
| Date<br>Dev Mo | onth Year | | | _ | | | ╄ | | | | 1 | | | 4 | | | | | |
| 207 80 | 700 | | | | | | | | | | | | | | | | | | |
| | | | | | | | ╄ | | | | _ | | | $\dashv$ | | | | | |
| . OTHE | R RELEVAN | NT TESTS | (diag | nosti | cs an | d pro | oceo | lures | ;) | | Any C | ther F | Relevan | t test | ts? [ | □ No □ Ye | s If yes, ple | ease co | mplete |
| | ate<br>onth Year | | | Add | itional | Test | s | | _ | | | | | Res | ults | | | Unit | s |
| July 101 | 1001 | | | | | | | | | | Π | | | | | | | | |
| | | | | | | | | | | | + | | | | | | - | | |
| | | | | | | | | | | | _ | | | | | | $\perp$ | | |
| | | | | | | | | | | | I | | | | | | - 1 | | |


Approved

FORM-056006

Version 7.0 Effective Date: 1 February 2016



Supplemental Clinical Study Report: 20130411


| AMGEN<br>Study # 20130411 | Electronic Serious Adverse Event Contingency Report Form |
|---|---|
| Oprozomib | For Restricted Use |

| | Sit | e Numb | er | | | | Subje | ct ID N | lumb | er | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | Π | | | | |
| <ol> <li>CASE DESCRIPTION (Provide event in section 3, where relations)</li> </ol> | de <i>nai</i><br>nip=Y | rrative<br>es, ple | detail:<br>ase pro | s of | evei<br>e rati | nts list<br>onale. | ed in | secti | on 3 | ) P | rovide | add | itional pages if ne | ecessary. For each |
| Signature of Investigator or Designee - | | | | | | | | Title | 1 | | | | | Date |
| I confirm by signing this report that the infi<br>causality assessments, is being provided to<br>a Qualified Medical Person authorized by t | Amge | n by the | investige | ator f | for thi | eriousne<br>is study, | ss and<br>or by | | | | | | | |
| | | | | | | | | | | | | | | • |


Approved

FORM-056006

Version 7.0 Effective Date: 1 February 2016




## APPENDIX O EXAMPLE AMGEN PREGNANCY NOTIFICATION WORKSHEET

## **AMGEN** Pregnancy Notification Worksheet

Fax Completed Form to the Country-respective Safety Fax Line

| | SELECT O | OR TYPE IN A FAX# | • | l | |
|---|---|---|---|---|---|
| 1. Case Administrative Inf | | | | | |
| Protocol/Study Number: 2013041 | 1 | | | | |
| Study Design: Interventional | Observational | (If Observational: | Prospective | Retrospective) | |
| 2. Contact Information | | | | | |
| Investigator Name | | | | Site # | |
| Phone () | Fax ( | ) | | Email | |
| Institution | | | | | |
| Address | | | | | |
| 3. Subject Information | | | | | |
| Subject ID # | Subject Gen | der: Female | Male Su | bject DOB: mm/ dd// yyy | у |
| 4. Amgen Product Exposu | ire | | | | |
| Amgen Product | Dose at time of conception | Frequency | Route | Start Date | |
| Oih | conception | | | | |
| Oprozomib | | | | mml/ddl/yyyy | |
| Was the Amgen product (or st | | | - | | |
| If yes, provide product (or | | | <u></u> /yyyy | | |
| Did the subject withdraw from | the study? 🗌 Yes | No | | | |
| 5. Pregnancy Information | | | | | |
| Pregnant female's LMP mm | ▼ / dd ▼ / | yyyy Un | known | | |
| Estimated date of delivery mm | ▼ / dd ▼ / | yyyy Un | known N | 1/4 | |
| If N/A, date of termination (act | ual or planned) mm | ▼ /dd ▼ | / 5000 | | |
| Has the pregnant female already d | | | | - | |
| If yes, provide date of deliver | | | | | |
| Was the infant healthy? Yes | | | | | |
| If any Adverse Event was experien | iced by the infant, pr | ovide brief details: | | | |
| Form Completed by: | | | | | |
| Print Name: | | Tit | le: | | |
| Signature: | | Dat | te: | | |
| Effective Date: March 27, 2011 | | | | | 4 -64 |


Approved


# APPENDIX P EXAMPLE AMGEN LACTATION NOTIFICATION WORKSHEET

## AMGEN Lactation Notification Worksheet

| Fax Completed Form to the C | Fax Completed Form to the Country-respective Safety Fax Line SELECT OR TYPE IN A FAX# enter fax number | | | |
|---|---|---|---|---|
| 1. Case Administrative Info | ormation | | | |
| Protocol/Study Number: 2013041 | | | | |
| Study Design: Interventional | | (If Observational: | Prospective | Retrospective) |
| 2. Contact Information | | | | |
| Investigator Name | | | | Site # |
| Phone () | Fax ( | ) | | Email |
| Institution | | | | |
| Address | | | | |
| 3. Subject Information | | | | |
| Subject ID # | Subject Date | of Birth: mm | / dd/ y | yyy |
| 4. Amgen Product Exposur | re | | | |
| Amgen Product | Dose at time of<br>breast feeding | Frequency | Route | Start Date |
| Oprozomib | | | | mm/dd/yyyyy |
| If yes, provide product (or some product of some product of some provide product of the subject withdraw from the subject withdraw from the subject withdraw from the subject of the subje | ion ie the infant with pu //dd //yyyy | No mped breast milk whi | le actively tak | ting an Amgen product? ☐ Yes ☐ No |
| Form Completed by: Print Name: | | | | |
| | | Titl | | |
| Signature: | | Dai | · - | |
| | | | *************************************** | |
| Effective Date: 03 April 2012, version 2 | | | | Page 1 of 1 |


Approved


#### APPENDIX O SUMMARY OF CHANGES IN STUDY OPZ007 AMENDMENT 2.0

Study OPZ007 was amended to include the following:

- 1. Revised inclusion and exclusion criteria to allow subjects with prior carfilzomib exposure to be considered for inclusion in the study, if carfilzomib was not withdrawn due to toxicity.
- 2. Revised exclusion criteria to allow subjects with prior pomalidomide exposure to be considered for inclusion in the dose-escalation portion of the study, if pomalidomide was neither dose-reduced nor withdrawn due to toxicity.
- 3. Revised alkylator language to specify that only subjects who have been treated with adequate alkylator therapy are eligible to be considered for inclusion in the Phase 1b dose-escalation portion and Phase 3 portion of the study.
- 4. An exclusion criterion for previous GI bleed was added, proton-pump inhibitors were changed from recommended to required, and additional text has been added to the dose modification table for nonhematologic toxicities and guidance to investigators because of toxicities observed in Study 2011-001.
- 5. The planned number of study sites for Part 1 of the study was increased from 20 to 35 sites, and the number of sites planned for the Dose-Escalation versus Dose-Expansion portions were clarified (15 and 20 sites, respectively).
- 6. The health-related quality of life measurement by Brief Pain Inventory Short Form was added as an exploratory objective and endpoint for the dose-expansion portion of the study, and as a secondary objective and endpoint for the Phase 3 portion of the study.
- 7. The text for secondary and exploratory objectives for Part 2 (randomized Phase 3) portion of the study) was revised for accuracy and consistency within the protocol.
- 8. The text "at sponsor discretion" was added for Part 1 (Phase 1b dose-escalation and dose-expansion portions of the study) for flexibility if MTD cannot be achieved with 4 mg of pomalidomide.
- 9. The ">" sign before Grade 3 fatigue in the Dose-Limiting Toxicities sections was removed as there is no > Grade 3 fatigue per NCI-CTCAE.
- 10. The carfilzomib status stratification factors were revised to "carfilzomib naïve/sensitive versus carfilzomib-refractory" to reflect allowed enrollment of carfilzomib-refractory patients to the study.
- 11. The sample size justification text was revised for clarity.
- 12. The 8 hour postdose PK sample timepoint was removed, and a 3 hour postdose PK sample timepoint was added to further characterize the PK profile for oprozomib.
- 13. Genomic measurements language was revised for clarity.




- 14. Endpoints language was revised for accuracy and consistency within the protocol.
- 15. The efficacy and safety analyses sections were revised for clarity.
- 16. The clinical background information for Study 2009-003 and Study 2011-001 were updated per the most recent information.
- 17. Updated clinical background information was added for Study 2012-001 and OPZ003 for consistency with other oprozomib protocols.
- 18. Text that allows for the potential use of blister packs in Phase 3 of the study was added to the Study Drug Accountability section.
- 19. The text "or fosaprepitant" was added for consistency with other oprozomib protocols to allow IV administration of this antiemetic if needed.
- 20. Additional guidance for subjects who may experience orthostatic hypotension was added.
- 21. A new subsection "11.5 Patient-Reported Outcomes Assessments" was added in the Study Procedures section to further clarify these assessments in the dose-expansion and Phase 3 portions of the study.
- 22. The term "on study" and additional text was added for clarity on the long-term follow-up based on disease progression status.
- 23. Subgroups of interest were revised for clarity, including potential inclusion of subjects with prior carfilzomib exposure in the study.
- 24. For Appendices A1, A2, B1, B2, C1, and C2, "X"s in the Schedule of Assessment tables were removed and added, and the text of footnotes was revised for clarity and consistency with the protocol body text.
- 25. Definition of "Baseline" (within 45 days prior to Cycle 1 Day 1 dosing) versus Screening (Days -1 to -28 prior to Cycle 1 Day 1 dosing) was added, and skeletal survey, plasmacytoma evaluation, bone marrow aspirate and FISH analyses, and optional genomic biomarker assessments on blood and saliva in Appendices A1, A2, B1, B2, C1, and C2 were moved from Screening to Baseline to provide clarity on the use of the tests. Screening tests are mandated to confirm eligibility, whereas baseline tests are used for disease assessments after patient enrollment.
- 26. The ACTG Brief Peripheral Neuropathy Screening Tool was added as Appendix M.
- 27. The Brief Pain Inventory Short Form was added as Appendix N.

In addition, administrative updates, editorial changes, and style and formatting revisions have been made to improve clarity and consistency throughout the document. Changes noted in specific sections were also made in the protocol synopsis and elsewhere in the document, as applicable. Significant changes are presented in the table below. Detailed changed text is displayed for **first major** occurrence only. All affected sections are noted in the "Section(s)"



Supplemental Clinical Study Report: 20130411


column. Text that has been deleted is presented in strikethrough format. Added text is presented in bold format.

Superseded




**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Pag

Onyx Therapeutics Oprozomib Tablets Clinical Study Protocol No. OPZ007 

| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Cover Page<br>Signature Page<br>Protocol<br>Acceptance Page | - | Added: Amendment 2 and 08 July 2014 | Updated for new amendment |
| Confidentiality and approval statements | This document is signed with electronic signatures at Onyx Therapeutics, Inc. (a wholly owned subsidiary of Onyx Pharmaceuticals, Inc.). | This document is signed with electronic signatures at Onyx Therapeutics, Inc. (a wholly owned subsidiary of Onyx Pharmaceuticals Inc., an Amgen subsidiary). | Updated confidentiality and<br>approval statements where<br>Onyx Therapeutics and<br>Onyx Pharmaceuticals are<br>listed to be consistent with<br>current company name and<br>study sponsorship |
| Global: In all sections listing "Inc." | | Deleted: Inc. | Removed all references to<br>"Inc." to be consistent with<br>current company name and<br>study sponsorship |
| Global: Oprozomib<br>tablets (where<br>applicable) | - | Added: ER | In instances where this was<br>missing, it was clarified that<br>Oprozomib ER Tablets will<br>be used |
| Global: Oprozomib<br>and dexamethasone<br>dosing regimens | Days 1–2, 8–9, 15–16, and 22–23 | Days 1, 2, 8, 9, 15, 16, 22, and 23 | Oprozomib and<br>dexamethasone dosing<br>regimens were made<br>consistent throughout the<br>protocol |
| Global: In all<br>instances of "End of<br>Study" and "End of<br>Treatment" | "End of Study" or "End of Treatment" | End of Study Treatment | Corrected for accuracy and consistency throughout the protocol, and to distinguish between "End of Study" and "End of Study Treatment" |
| Global: In instances where the timing of disease response | Treatment cycles will last 28 days. Disease response assessments will be performed at the end of every 4-week cycle for the first 18 months on study, and at | Treatment cycles will last 28 days. Disease response assessments will be performed at the end of every 4-week cycle for the first 18 months on study, and at | Added text for clarity |




Superseded

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Page

Onyx Therapeutics Oprozomib Tablets

| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| assessments are described | the end of every other cycle (every 8 weeks) thereafter. | the end of every other cycle (every 8 weeks) thereafter, beginning with Month 20. | |
| Global: In instances<br>of "first dose"<br>(where applicable) | "first dose" | "first dose of study drug" or "first dose of study treatment" | Added "of study drug" or<br>"of study treatment" for<br>clarity |
| Synopsis: Study<br>objectives<br>Section 4.1 Part 1:<br>Phase 1b<br>Dose-Escalation and<br>Expansion Portions<br>of the Study (by<br>Schedule) | Part 1: Phase 1b Dose Escalation and Expansion Portions of the Study | Part 1: Phase 1b Dose-Escalation and <b>Dose</b> -Expansion Portions of the Study (by schedule) | Added text to clarify that<br>each individual schedule<br>will be assessed<br>independently for Part 1 of<br>the study |
| Synopsis: Study<br>Objectives | Part 1: Phase 1b Dose Escalation and Expansion<br>Portions of the Study<br>Exploratory Objectives | Part 1: Phase 1b Dose Escalation and Dose-Expansion Portions of the Study Exploratory Objectives | Added Brief Pain Inventory – Short Form as a HRQoL exploratory objective in the |
| Section 4.1.3<br>Exploratory<br>Objectives | To evaluate quality of life (in the dose expansion phase only) on the basis of patient-reported outcomes tools listed below: Global health scale as measured by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Module (QLQ-C30) questionnaire Health status assessed by the European Quality of Life descriptive system EQ-5D-5L (EuroQol EQ-5D-5L) Disease symptoms subscale as measured by EORTC Multiple Myeloma Module (QLQ-MY20) questionnaire Neurotoxicity symptoms as measured by the Functional Assessment of Cancer Therapy Scale / Gynecological Oncology Group – Neurotoxicity (FACT/GOG-Ntx4 [(Version 4]) for patients with neurotoxicity score | To evaluate quality of life (in the dose-expansion phase portion only) on the basis of patient-reported outcomes (PRO) using the tools listed below: Bone pain and the impact of bone pain measured with the Brief Pain Inventory Short Form (BPI-SF) Health-related quality of life (HRQoL) measured by the global health seale status/QoL scale as measured by of the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Core Module (QLQ-C30) questionnaire Health status assessed by the European Quality of Life descriptive system—EQ-5D-5L (EuroQol EQ-5D-5L) Disease symptoms subscale as measured by the disease symptoms subscale of the EORTC Multiple Myeloma Module | dose-expansion portion of<br>the study |





| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | (QLQ-MY20) questionnaire Neurotoxicity symptoms as measured by the neurotoxicity subscale of the Functional Assessment of Cancer Therapy Seale / Gynecological Oncology Group – Neurotoxicity (FACT/GOG-Ntx4 [(Version 4]) for patients with neurotoxicity score questionnaire | |
| Synopsis: | Part 2: Randomized Phase 3 Portion of the Study | Part 2: Randomized Phase 3 Portion of the Study | Removed and added text for |
| Secondary<br>objectives | To compare the following between subjects treated with OPomd and those treated with Pomd: | To compare the following between subjects treated with OPomd and those treated with Pomd: | accuracy of secondary<br>objectives for Part 2 of the<br>study |
| Section 4.2.2<br>Secondary<br>Objectives | Improvement in renal function over time, as defined by an increase in glomerular filtration rate (GFR) of at least 10 mL/min over baseline Improvement in hemoglobin over time, as defined by an increase of at least 2 g/dL over baseline Population–based PK parameters of oprozomib in the OPomd regimen Safety and tolerability Health-related quality of life (HRQoL) QLQ-30 global health status score measured by EORTC QLQ-C30 Disease symptoms as measured by the disease symptoms subscale of EORTC QLQ-MY20 Health status as assessed with EuroQol EQ-5D-5L | Incidence of improvement in renal function over time, as defined by an increase in glomerular filtration rate (GFR) of at least 10 mL/min over baseline at least once after the start of treatment Incidence of improvement in hemoglobin over time, as defined by an increase of at least 2 g/dL over baseline at least once after the start of treatment Population-based PK parameters of oprozomib in the OPomd regimen Safety and tolerability Bone pain and the impact of bone pain measured with the BPI-SF Health-related quality of life (HRQoL) QLQ-30 global health status score measured by the global health status/QoL scale of the EORTC QLQ-C30 Disease symptoms as measured by the disease symptoms subscale of EORTC QLQ-MY20 Neurotoxicity symptoms as measured by the neurotoxicity subscale of the FACT/GOG- | |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | Ntx4 (Version 4) Health status as assessed with EuroQol EQ-5D-5L To evaluate population-based PK parameters of oprozomib in the OPomd regimen | |
| Synopsis: Study objectives Section 4.2.3 Exploratory Objectives | Part 2: Randomized Phase 3 Portion of the Study Exploratory Objectives To compare the following between subjects treated with OPomd and those treated with Pomd: • PFS and ORR as determined by the investigator • Duration of response (DOR), defined as the time from the first evidence of confirmed PR or better to disease progression or death due to any cause as determined by the investigator according to the IMWG-URC and modified EBMT criteria • Clinical benefit rate (CBR) as determined by the investigator according to the modified EBMT criteria • Duration of clinical benefit (DOCB), defined as the time from first evidence of ≥ MR as determined by ORCA and the investigator according to the modified EBMT criteria • Genomic biomarkers that may correlate with antitumor activity and resistance following treatment with proteasome inhibitors • The incidence of neuropathy events (defined as Grade 2 or higher peripheral neuropathy incidence) • The number of neuropathy events (defined as Grade 2 or higher peripheral neuropathy incidence, and neurotoxicity symptoms scores assessed by FACT/GOG-Ntx4 [Version 4]) • Health status assessed with subscale scores of | Part 2: Randomized Phase 3 Portion of the Study Exploratory Objectives To compare the following between subjects treated with OPomd and those treated with Pomd: • PFS and ORR as determined by the investigator according to the IMWG-URC • Duration of response (DOR), defined as the time from the first evidence of confirmed PR or better to disease progression or death due to any cause as determined by the investigator according to the IMWG-URC-and modified EBMT criteria • Clinical benefit rate (CBR) as determined by the investigator according to the IMWG-URC and the modified EBMT criteria • Duration of clinical benefit (DOCB), defined as the time from first evidence of ≥ MR or better to disease progression or death due to any cause, as determined by ORCA and the investigator according to the IMWG-URC and the modified EBMT criteria • Genomic biomarkers that may be correlated with antitumor activity and resistance following treatment with proteasome inhibitors • The incidence of neuropathy events (defined as Grade 2 or higher peripheral neuropathy incidence, and neurotoxicity symptoms scores assessed by | Revised text for corrections and for consistency within the protocol |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | EORTC QLQ-C30 (excluding global health status scale) and EORTC QLQ-MY20 (excluding disease symptom subscale) | FACT/GOG-Ntx4 [Version 4]) Health status HRQoL assessed with subscale scores of EORTC QLQ-C30 (excluding global health status scale) and EORTC QLQ-MY20 (excluding disease symptom subscale) | |
| Synopsis: Study<br>design<br>Synopsis: Study<br>population<br>Section 5 Study<br>design | This study will include subjects with primary refractory or relapsed and refractory multiple myeloma, i.e., those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy including bortezomib and lenalidomide or thalidomide and adequate alkylator therapy. | This study will include subjects with primary refractory or relapsed and refractory multiple myeloma, i.e., those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy (including bortezomib and lenalidomide and/or thalidomide, and in the dose-expansion and Phase 3 portions of the study only, been treated with adequate alkylator therapy). | Revised alkylator language<br>to specify that only subjects<br>who have been treated with<br>adequate alkylator therapy<br>are eligible to be considered<br>for inclusion in the Phase<br>1b dose-escalation portion<br>and Phase 3 portion of the<br>study |
| Synopsis: Study design | Part 1: Phase 1b Dose Escalation and Expansion Portions of the Study If the starting dose of oprozomib cannot be safely administered with the labeled pomalidomide dose, then up to 2 possible alternative paths for oprozomib with lower pomalidomide doses will be explored. (See tables below for primary and alternative dose-escalation paths.) Dose escalation will continue until ≥ 2 DLTs occur in a cohort, which will be declared the maximal administered dose for that dose level of pomalidomide (if more than 1 dose level is explored). The prior cohort will be expanded to at least 6 subjects if not previously done to establish that dose as the MTD. There may be more than 1 MTD for oprozomib if more than 1 dose level of pomalidomide is studied. The MTD of oprozomib associated with each dose level of pomalidomide assessed will be the dose level where < 2 DLTs in 6 subjects are observed. There will be no planned maximum dose of oprozomib | Part 1: Phase 1b Dose-Escalation and <b>Dose</b> -Expansion Portions of the Study If the starting dose of oprozomib cannot be safely administered with the labeled pomalidomide dose, or at sponsor discretion, after the MTD with 4 mg of pomalidomide is determined, then up to 2 possible alternative paths for oprozomib with lower pomalidomide doses will be explored. (See tables below for primary and alternative dose-escalation paths.) Dose escalation will continue until sponsor discretion, the maximum planned dose of pomalidomide is reached, or ≥ 2 DLTs occur in a cohort, whoever occurs firstwhich will be declared the maximal administered dose for that dose level of pomalidomide (if more than 1 dose level is explored). The prior cohort will be expanded to at least 6 subjects if not previously done to establish that dose as the MTD. There may be more than 1 MTD for oprozomib if more than 1 dose level of pomalidomide is studied. | Added text for flexibility if MTD cannot be achieved with 4 mg of pomalidomide |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | to be studied as it is being added to the FDA approved regimen of pomalidomide/dexamethasone. The starting dose of oprozomib for the 5/14 schedule is 150 mg, 3 dose levels below the established 5/14 single-agent MTD of 240 mg | The MTD of oprozomib associated with each dose level of pomalidomide assessed will be the dose level where < 2 DLTs in 6 subjects are observed. There will be is no planned maximum dose of oprozomib to be studied as it is being added to the FDA approved regimen of pomalidomide/dexamethasone, however, this could be imposed at any time during the course of the study, based on sponsor discretion. The starting dose of oprozomib for the 5/14 schedule is 150 mg, 3 dose levels below the established 5/14 single-agent MTD of 240 mg. | |
| Synopsis: Study<br>design<br>Section 5.1.1 Dose<br>Escalation Schema<br>for the 5/14<br>Oprozomib Dosing<br>Schedule | The starting dose for the 5/14 schedule will be 150 mg of oprozomib and 4 mg of pomalidomide. The 5/14 primary and alternate paths are summarized below. 5/14 Schedule Study Dose-Escalation Paths* Pom(mg) | The starting dose for the 5/14 schedule will be 150 mg of oprozomib and 4 mg of pomalidomide. The 5/14 primary and alternate paths are summarized below; these are examples, and are not inclusive of all possible dose-escalation paths. 5/14 Schedule Primary Study Dose-Escalation Paths*a Pem (mg) Daby 21/28d Days 1.2 8.9, 3 15, 16, 22, 23 2 150 mg 180 mg 210 mg OPZ (mg) 5/14 schedule 5/14 = Dosing on Days 1-5 and 15-19; Dex = dexamethasone; OPZ = oprozomib; Pom = pomalidomide. * There is no predefined maximum dose level of oprozomib being studied. | Added text to clarify that the dose-escalation paths are examples, and not inclusive of all possible dose-escalation paths. Revised in schema "Dex 20 mg Days 1, 2, 8, 9" for consistency with the rest of the protocol |
| Synopsis Study | Table 3 Primary Dose-Escalation Path for Oprozomib | Table 3 Primary Dose-Escalation Path for Oprozomib | Revised titles and notes for |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Page


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Design Section 5.1.1 Dose Escalation Schema for the 5/14 Oprozomib Dosing Schedule Section 5.1.2 Dose Escalation Schema for the 2/7 Oprozomib Dosing Schedule | and Pomalidomide on 5/14 Schedule in Phase 1b Note: This is an example of the primary dose-escalation cohort and dose-escalation will continue in 30 mg increments of oprozomib until the MTD is identified. Table 6 Primary Dose-Escalation Path for Oprozomib and Pomalidomide on the 2/7 Schedule in Phase 1b Note: This is an example of the primary dose-escalation cohort and dose-escalation will continue in 30 mg increments of oprozomib until the MTD is identified. | and Pomalidomide on 5/14 Schedule with Pomalidomide 4 mg in Phase 1b Note: This is an example of the primary dose-escalation cohort and dose-escalation will continue in 30-mg increments of oprozomib at sponsor discretion or until the MTD is identified. Table 6 Primary Dose-Escalation Path for Oprozomib and Pomalidomide on the 2/7 Schedule with Pomalidomide 4 mg in Phase 1b Note: This is an example of the primary dose-escalation cohort and dose-escalation will continue in 30-mg increments of oprozomib at sponsor discretion or until the MTD is identified. | Table 3 and Table 6 for clarity. |
| Synopsis: Study design Section 5.1.1 Dose Escalation Schema for the 5/14 Oprozomib Dosing Schedule Section 5.1.2 Dose Escalation Schema for the 2/7 Oprozomib Dosing Schedule | Table 4 Alternative Dose-Escalation Path 1 for Oprozomib andPomalidomide on 5/14 Schedule in Phase 1b if Cohort 1a Exceeds the MTD Table 5 Alternative Dose-Escalation Path 2 for Oprozomib and Pomalidomide in Phase 1b if Cohort 1b Exceeds the MTD Table 7 Alternative Dose-Escalation Path 1 for Oprozomib and Pomalidomide on 2/7 Schedule in Phase 1b if Cohort 101a Exceeds the MTD Table 8 Alternative Dose-Escalation Path 2 for Oprozomib and Pomalidomide on 2/7 Schedule in Phase 1b if Cohort 101b Exceeds the MTD | Table 4 Alternative Dose-Escalation Path 1 for Oprozomib and Pomalidomide on 5/14 Schedule with Pomalidomide in Phase 1b if Cohort 1a Exceeds the MTD, or at Sponsor Discretion Table 5 Alternative Dose-Escalation Path 2 for Oprozomib and Pomalidomide on 5/14 Schedule with Pomalidomide in Phase 1b if Cohort 1b Exceeds the MTD, or at Sponsor Discretion Table 7 Alternative Dose-Escalation Path 1 for Oprozomib and Pomalidomide on 2/7 Schedule with Pomalidomide in Phase 1b if Cohort 101a Exceeds the MTD or at Sponsor Discretion Table 8 Alternative Dose-Escalation Path 2 for | Added "or at Sponsor<br>Discretion" to Table 4,<br>Table 5, Table 7, and Table<br>8 titles match earlier added<br>text, and revised titles for<br>clarity |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | Oprozomib and Pomalidomide on 2/7 Schedule with Pomalidomide in Phase 1b if Cohort 101b Exceeds the MTD or at Sponsor Discretion | |
| Synopsis: Study<br>design<br>Section 5.1.2 Dose<br>Escalation Schema<br>for the 2/7<br>Oprozomib Dosing<br>Schedule | The starting doses for the 2/7 oprozomib dosing schedule will be 210 mg of oprozomib and 4 mg of pomalidomide. The 2/7 primary and alternate paths are summarized below. 2/7 Schedule Study Dose-Escalation Paths 2/7 Schedule Study Dose-Escalation Paths 2/7 Schedule Study Dose-Escalation Paths 2/7 Schedule Study Dose-Escalation Paths 2/8 Dose 20 mg 2/9 Dally 21/28d | The starting doses for the 2/7 oprozomib dosing schedule will be 210 mg of oprozomib and 4 mg of pomalidomide. The 2/7 primary and alternate paths are summarized below; these are examples, and are not inclusive of all possible dose-escalation paths. 2/7 Schedule Primary Study Dose-Escalation Paths <sup>a</sup> Pom (mg) Daly, 21/23d Dev 20 mg Days 1, 2, 8, 9, 15, 16, 22, 23 2 101b> 201c> 301c 210 mg 240 mg 270 mg OPZ (mg) 2/7 schedule 2/7 = Dosing on Days 1, 2, 8, 9, 15, 16, 22, and 23; Dex = dexamethasone; OPZ = oprozomib; Pom = pomalidomide. a There is no predefined maximum dose level of oprozomib being studied. | Added text to clarify that the dose-escalation paths are examples, and not inclusive of all possible dose-escalation paths. Revised in schema "Dex 20 mg Days 1, 2, 8, 9" for consistency with the rest of the protocol. Added note below figure for consistency with the figure of 5/14 Schedule Study Dose-Escalation Paths. |
| Synopsis: Study<br>design | At the sponsor's discretion, once the MTD for oprozomib is reached on 1 or both schedules, additional dose escalation with oprozomib may continue with lower doses of pomalidomide down to the 2 mg dose level. The sponsor, with input from the Cohort Safety Review Committee ([CSRC] consisting of investigators, sponsor's medical monitor, and sponsor's Drug Safety representative), will determine which single dose combination to use for the dose expansion (i.e., the RP3D) portion of the study. The | At the sponsor's discretion, once the MTD for oprozomib is reached on 1 or both schedules, or if the initial cohort exceeds the MTD, additional dose escalation with oprozomib may continue with lower doses of pomalidomide down to the 2-mg dose level. The sponsor, with input from the Cohort Safety Review Committee ([CSRC] consisting of investigators, sponsor's medical monitor, and sponsor's drug safety representative, will determine which single dose combination dose and schedule of oprozomib in combination with Pomd to use for the dose-expansion | Revised text for consistency within the protocol |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | RP3D may differ from the MTD, but will not be higher than the MTD, and will be selected based upon the assessment of the safety, tolerability, PK, PDn, preliminary activity, and other variables to be observed across multiple cycles of combination therapy. | (i.e., the RP3D) portion of the study. The sponsor has the option of expanding 1 or both schedules in order to establish the RP3D and schedule. The RP3D may differ from the MTD, but will not be higher than the MTD, and will be selected based upon the assessment of the safety, tolerability, PK, PDn, preliminary activity, and other variables to be observed across multiple cycles of combination therapy. | |
| Synopsis: Study<br>Design<br>Section 10.5<br>Definition of<br>Dose-Limiting<br>Toxicity | Dose-Limiting Toxicities o > Grade 3 fatigue lasting < 14 days is not considered a DLT | Dose-Limiting Toxicities ○ > Grade 3 fatigue lasting < 14 days is not considered a DLT | Removed ">" sign for<br>accuracy as there is no<br>> Grade 3 fatigue per<br>NCI-CTCAE |
| Synopsis: Study<br>Design<br>Section 5.1.4<br>Subject<br>Replacement | In the Phase 1b portion of the study, subjects must meet the following criteria to be considered evaluable for MTD determination during the 4-week DLT evaluation period unless a study drug-related DLT occurs before the subject receives all planned doses of oprozomib for both the 5/14 and 2/7 dosing schedules: | In the Phase 1b portion of the study, subjects must meet the following criteria to be considered evaluable for MTD determination during the 4-week DLT evaluation period unless a study drug-related DLT occurs before the subject receives all planned doses of oprozomib for both the 5/14 and 2/7 dosing schedules: | Deleted text for clarity |
| Synopsis: Study<br>Design<br>Section 5.1.5 Dose<br>Expansion<br>Section 5.2 Part 2:<br>Randomized Phase<br>3 Portion of the<br>Study | Dose Expansion The criteria for selecting the RP3D for 1 or both schedules of oprozomib at the sponsor's discretion will include assessment of the safety, tolerability, and preliminary activity observed across multiple cycles of therapy. In addition, both PK and PDn assessments to demonstrate adequate exposure and proteasome inhibition will be a key factor. Therefore, the RP3D may differ from the MTD. Once the MTD(s) has been determined and the RP3D has been selected, a minimum of 20 additional subjects for 1 or both schedules of oprozomib at the sponsor's discretion will be enrolled in the dose-expansion portion of Part 1 in order to continue the evaluation of the safety and | Dose Expansion The criteria for selecting the RP3D for 1 or both schedules of oprozomib at the sponsor's discretion will include assessment of the safety, tolerability, and preliminary activity observed across multiple cycles of therapy. In addition, both PK and PDn assessments to demonstrate adequate exposure and proteasome inhibition will be a key factor. Therefore, the RP3D may differ from the MTD. Once the MTD(s) has been determined and the RP3D recommended dose for the expansion phase has been selected, a minimum of 20 additional subjects for 1 or both schedules of oprozomib at the sponsor's discretion will be enrolled in the dose-expansion portion of Part 1 in order to | Revised text for clarity |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | efficacy of the regimen as a prelude to initiation of the Phase 3 portion of the study. The safety of subjects in the Dose Expansion will be monitored on an ongoing basis by the CSRC during bimonthly calls. Enrollment to the Phase 3 portion will not commence until the CSRC has evaluated all available safety information from a minimum of 10 subjects who have completed ≥ 2 cycles of therapy at the R3PD and enrollment of the remaining 10 subjects in Dose Expansion has occurred in 1 or both schedules if both were opened. | continue the evaluation of the safety and efficacy of the regimen as a prelude to initiation of the Phase 3 portion of the study. The safety of subjects in the Dose Expansion will be monitored on an ongoing basis by the CSRC during bimonthly regularly scheduled calls. Enrollment to the Phase 3 portion will not commence until the CSRC has evaluated all available safety information from a minimum of 10 subjects who have completed ≥ 2 cycles of therapy at the R3PD and enrollment of the remaining 10 subjects in Dose Expansion has occurred in 1 or both schedules if both were opened. This information will inform the selection of a RP3D and schedule by the sponsor and CSRC. | |
| Synopsis: Study design Section 5.4.1 Randomization Section 14.5.2.2 Part 2 Randomized Phase 3 Portion of the Study | Part 2: Randomized Phase 3 Portion of the Study Randomization After screening and eligibility determination, eligible subjects will be randomized in a 2:1 ratio to receive a regimen consisting of OPomd or Pomd plus oprozomib placebo, respectively. Central randomization will be implemented in this part of the study through the use of an interactive voice response system / interactive web response system (IVRS/IWRS). Eligible subjects will be stratified by: • Age: <75 years versus ≥ 75 years • Number of prior therapies: 2 versus 3 or more • Carfilzomib status: Carfilzomib naïve versus carfilzomib sensitive Within each stratum, treatment assignment will be made using a random permuted blocked randomization scheme. | Part 2: Randomized Phase 3 Portion of the Study Randomization After screening and eligibility determination, eligible subjects will be randomized in a 2:1 ratio to receive a regimen consisting of OPomd or Pomd plus oprozomib placebo, respectively. Central randomization will be implemented in this part of the study through the use of an Interactive Voice Response System / Interactive Web Response System (IVRS/IWRS). Eligible subjects will be stratified by: ■ Age: <75 years versus ≥75 years ■ Number of prior therapies: 2 versus 3 or more ■ Carfilzomib status: Carfilzomib-naïve/sensitive versus carfilzomib-refractory sensitive. Carfilzomib-sensitive multiple myeloma patients are defined as having had previously achieved a PR or greater with therapy that includes carfilzomib (or carfilzomib monotherapy), and did not experience PD until more than 60 days after their last dose of carfilzomib. Carfilzomib-refractory | Correction made to remove "oprozomib" before "placebo" Revised carfilzomib status stratification factors to reflect potential inclusion of subjects with prior carfilzomib exposure in the study |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | multiple mycloma is defined as disease that is nonresponsive while on primary or salvage therapy that includes carfilzomib, or that progresses on or within 60 days of last therapy. Within each stratum, treatment assignment will be made using a-random permuted blocked randomization scheme. | |
| Synopsis: Number<br>of investigational<br>sites<br>Section 5 Study<br>Design | Up to 20 study sites will participate in Part 1 of the study (Phase 1b Dose-Escalation and Dose-Expansion portion of the study). Approximately 70 sites will participate in Part 2 of the study (Phase 3 portion of the study). | Approximately Up to 35 20 study sites will participate in Part 1 of the study (15 sites for the Phase 1b dose-escalation and 20 sites for the dose-expansion portions of the study). An additional 35 sites, for a total of approximately 70 sites will participate in Part 2 of the study (Phase 3 portion of the study). | Increased the planned<br>number of study sites for<br>Part 1 of the study, and<br>clarified how many sites are<br>planned for the<br>Dose-Escalation versus<br>Dose-Expansion portions |
| Synopsis: Planned<br>number of subjects<br>Section 14.7<br>Determination of<br>Sample Size | Part 1: Phase 1b (Dose Escalation and Expansion Portions of the Study) A total enrollment of approximately 82 subjects is planned for Part 1 of the study. During the Phase 1b Dose Escalation portion of Part 1, up to 21 subjects will be enrolled for each schedule. Part 2: Randomized Phase 3 Portion of the Study During Part 2, the planned enrollment is approximately 270 subjects. Therefore, a total enrollment of approximately 352 subjects is planned. | Part 1: Phase 1b (Dose-Escalation and Dose-Expansion Portions of the Study) A total enrollment of up to approximately 82 subjects is planned for Part 1 of the study. During the Phase 1b dose-escalation portion of Part 1, approximately 21 subjects will be enrolled for each schedule. Part 2: Randomized Phase 3 Portion of the Study During Part 2, the planned enrollment is approximately 270 subjects. Therefore, a the total planned enrollment of will be approximately 352 subjects is planned. | Revised text for flexibility<br>and for clarity |
| Synopsis: Sample size justification | Part 2: Randomized Phase 3 Portion of the Study The estimated sample size for the Phase 3 portion of the study is based on comparison of PFS (death or disease progression events) distributions for subjects treated with Pomd plus placebo versus those treated with OPomd based on the log-rank test statistic. It is assumed that the risk of a PFS event for subjects | Part 2: Randomized Phase 3 Portion of the Study For the Phase 3 portion of the study, 157 PFS events are required to detect a 45.7% reduction in the risk of PFS (HR=0.543) with 95% power and a 1-sided significance level of 0.025. Enrollment of 270 subjects (2:1 OPomd versus Pomd, respectively) is consistent with reaching the required 157 events | Revised text for clarity |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Pag


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | randomized to OPomd will be 45.7% lower than for subjects randomized to Pomd. Therefore, the target hazard ratio (HR) is 0.543. The statistical hypothesis being tested is as follows: $H_0\colon \text{PFS (Pomd)} = \text{PFS (OPomd)} \\ H_a\colon \text{PFS (Pomd)} < \text{PFS(OPomd)} \\ \text{For a 1-sided } \alpha = 0.025 \text{ level of significance and 95\% power, 157 PFS events are required.} \\ \dots$ | in approximately 14 months, assuming an enrollment rate of approximately 22 subjects per month, a drop-out rate of 5% at 18 months, and a median PFS of 3.8 and 7 months for Pomd and OPomd, respectively. The estimated sample size for the Phase 3 portion of the study is based on comparison of PFS (death or disease progression events) distributions for subjects treated with Pomd plus placebo versus those treated with OPomd based on the log-rank test statistic. It is assumed that the risk of a PFS event for subjects randomized to OPomd will be 45.7% lower than for subjects randomized to Pomd. Therefore, the target hazard ratio (HR) is 0.543. The statistical hypothesis being tested is as follows: H <sub>u</sub> : PFS (Pomd) = PFS (OPomd) H <sub>n</sub> : PFS (Pomd) < PFS(OPomd) For a 1-sided α = 0.025 level of significance and 95% power, 157 PFS events are required. | |
| Synopsis: Study<br>population | The study population will consist of subjects with primary refractory or relapsed and refractory, symptomatic multiple myeloma that have been treated with at least 2 prior lines of therapy including lenalidomide and bortezomib or thalidomide and been treated with adequate alkylator therapy, who have progressed on or within 60 days of their last therapy, and who are considered to be appropriate for this clinical study by their treating physicians. | The study population will consist of subjects with primary refractory or relapsed and refractory, symptomatic multiple mycloma that had been treated with, i.e., those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy (including lenalidomide and bortezomib and lenalidomide and/or thalidomide, and in the dose-expansion and Phase 3 portions of the study only, been treated with adequate alkylator), and who have progressed on or within 60 days of their last therapy; and who are considered to be appropriate for this clinical study by their treating physicians. | Revised text for consistency within the protocol |
| Synopsis: Inclusion<br>Criteria<br>Section 6.1<br>Inclusion Criteria | Multiple myeloma that is primary refractory or relapsed and refractory after at least 2 lines of standard therapy for multiple myeloma including: a. ≥ 2 consecutive cycles of both bortezomib | Multiple myeloma that is primary refractory, of relapsed and refractory, or intolerant after at least 2 lines of standard therapy for multiple myeloma including: | Revised alkylator language<br>to specify that only subjects<br>who have been treated with<br>adequate alkylator therapy |




Superseded


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | and lenalidomide or thalidomide (alone or in combination) i. Patients who received bortezomib as their last therapy who were not refractory but developed bortezomib intolerance, as defined by the development of Grade 2 peripheral neuropathy with pain or ≥ Grade 3 peripheral neuropathy after ≥ 2 consecutive cycles, are eligible b. Adequate alkylator therapy defined as: i. High-dose melphalan or other alkylating agent as conditioning for autologous or allogeneic stem cell transplant (SCT), or ii. ≥ 6 cycles of induction therapy, or iii. Progressive disease after ≥ 2 cycles | a. ≥ 2 consecutive cycles of both bortezomib and lenalidomide or thalidomide (alone or in combination) i. Patients who received bortezomib as their last therapy who were not refractory but developed bortezomib intolerance, as defined by the development of Grade 2 peripheral neuropathy with pain or ≥ Grade 3 peripheral neuropathy after ≥ 2 consecutive cycles, are eligible b. In the dose-expansion and Phase 3 portions of the study only: In addition to the above, treatment with adequate alkylator therapy defined as: i. High-dose melphalan or other alkylating agent as conditioning for autologous or allogeneic stem cell transplant (SCT), or ii. ≥ 6 cycles of induction therapy, or iii. Progressive disease after ≥ 2 cycles | are eligible to be considered for inclusion in the Phase 1b dose-escalation portion and Phase 3 portion of the study Moved definition of bortezomib intolerance from Inclusion Criterion 1 to Inclusion Criterion 3 for clarity |
| Synopsis: Inclusion<br>Criteria<br>Section 6.1<br>Inclusion Criteria | Measurable disease as indicated by 1 or more of the following: d. Serum M-protein ≥ 500 mg/dL e. Urine M-protein ≥ 200 mg/24 h f. For subjects without measurable M-protein by serum protein electrophoresis (SPEP) or urine protein electrophoresis (UPEP), involved free light chain (FLC) concentration ≥ 10 mg/dL provided serum free light chain (SFLC) ratio is abnormal | 2. Measurable disease as indicated by 1 or more of the following: a. Serum M-protein ≥ 500 mg/dL b. Urine M-protein ≥ 200 mg/24 h c. Only for subjects without measurable M-protein by serum protein electrophoresis (SPEP) er and urine protein electrophoresis (UPEP), involved free light chain (FLC) concentration ≥ 10 mg/dL provided serum free light chain (SFLC) ratio is abnormal | Added "only" and added "and" for clarity |
| Synopsis: Inclusion<br>Criteria<br>Section 6.1<br>Inclusion Criteria | Disease progression on or within 60 days of completion of the last therapy as long as the last treatment was not carfilzomib. | 3. Disease progression on or within 60 days of completion of the last therapy, or intolerance to bortezomib if received as their last therapy as long as the last treatment was not carfilzomib. a. Patients who received bortezomib as their last therapy who were not refractory but | Revised to allow subjects<br>with prior carfilzomib<br>exposure to be considered<br>for inclusion in the study<br>Moved definition of |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | developed bortezomib intolerance, as defined<br>by the development of Grade 2 peripheral<br>neuropathy with pain or ≥ Grade 3<br>peripheral neuropathy after ≥ 2 consecutive<br>cycles, are eligible | bortezomib intolerance<br>from Inclusion Criterion 1<br>to Inclusion Criterion 3 for<br>clarity |
| Synopsis: Inclusion<br>Criteria<br>Section 6.1<br>Inclusion Criteria | 4. Prior carfilzomib is not required but is allowed if a subject had at least 2 cycles of carfilzomib alone or in combination with a dose of at least 20/27 mg/m² as long as the subject: a. Had at least a PR to prior carfilzomib therapy b. Was not removed from carfilzomib therapy due to toxicity c. Was not removed from carfilzomib therapy for progressive disease nor experienced progressive disease within 6 months of any prior carfilzomib therapy. | 4. Prior carfilzomib is not required but is allowed if a subject was not removed from carfilzomib therapy due to toxicity, unless approved by the Onyx study medical monitor had at least 2 eycles of carfilzomib alone or in combination with a dose of at least 20/27 mg/m² as long as the subject: a. Had at least a PR to prior carfilzomib therapy b. Was not removed from carfilzomib therapy due to toxicity c. Was not removed from carfilzomib therapy for progressive disease nor experienced progressive disease within 6 months of any prior carfilzomib therapy. | Revised to allow subjects<br>with prior carfilzomib<br>exposure to be considered<br>for inclusion in the study, if<br>carfilzomib was not<br>withdrawn due to toxicity |
| Synopsis:<br>Exclusion Criteria<br>Section 6.2<br>Exclusion Criteria | 7. Prior treatment of any duration with pomalidomide | 7. Prior treatment of any duration with pomalidomide exposure a. For the dose-escalation portion of the study: Subjects requiring pomalidomide dose reduction or removal due to toxicity b. For the dose-expansion portion and Part 2 of the study: Prior pomalidomide treatment of any duration | Revised to allow subjects with prior pomalidomide exposure to be considered for inclusion in the dose-escalation portion of the study, if pomalidomide was neither dose-reduced nor withdrawn due to toxicity |
| Synopsis:<br>Exclusion Criteria<br>Section 6.2<br>Exclusion Criteria | 11. Primary refractory or relapsed and refractory to carfilzomib alone or in combination with at least 2 cycles at a dose of at least 20/27 mg/m <sup>2</sup> | 11. Primary refractory or relapsed and refractory to earfilzomib alone or in combination with at least 2 eyeles at a dose of at least 20/27 mg/m <sup>2</sup> | Revised to allow subjects<br>with prior carfilzomib<br>exposure to be considered<br>for inclusion in the study;<br>subsequent Exclusion<br>Criteria were renumbered<br>accordingly |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Synopsis:<br>Exclusion Criteria<br>Section 6.2<br>Exclusion Criteria | _ | 14. History of previous clinically significant GI bleed in the 6 months prior to first dose of study drug | Added an Exclusion<br>Criterion for previous GI<br>bleed to potentially reduce<br>the risk for GI hemorrhage;<br>subsequent Exclusion<br>Criteria were renumbered<br>accordingly |
| Synopsis: Criteria<br>for evaluation:<br>Other<br>Section 11.4.1.1.<br>Phase 1b Dose<br>Escalation and<br>Expansion<br>Section 14.5.5<br>Pharmacokinetic<br>Analyses | Pharmacokinetics In the Phase 1b Dose Escalation and Expansion portions of the study, blood samples will be collected from all subjects for determination of plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 4, 6, and 8 hours postdose) and 1 predose time point on Day 2 of Cycle 1 for both schedules. In the Phase 3 portion of the study, PK samples will be collected from all randomized subjects at Cycle 1 Day 1 and Cycle 3 Day 1 and will be analyzed for oprozomib concentrations. | Pharmacokinetics In the Phase 1b dose-escalation and dose-expansion portions of the study, blood samples will be collected from all subjects for determination of plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 3, 2, 4, and 6, and 8 hours postdose) and 1 predose time point on Day 2 of Cycle 1 for both schedules. In the Phase 3 portion of the study, PK samples will be collected from all randomized subjects at Cycle 1 Day 1 and Cycle 3 Day 1 and will be analyzed for oprozomib concentrations in OPomd subjects. | Removed 8 hour postdose<br>PK sample timepoint and<br>added 3 hour postdose PK<br>sample timepoint to further<br>characterize the PK profile<br>for oprozomib |
| Synopsis: Criteria<br>for evaluation:<br>Other<br>Section 11.4.3<br>Genomic<br>Measurements | Genomics Analysis of genomic biomarkers that may predict response and resistance following treatment with proteasome inhibitors will be conducted for all subjects from all phases of the study who consent to optional genomic biomarker analysis. These analyses will be performed on Screening bone marrow aspirate (a portion of the bone marrow aspirate sample obtained at Screening will be used, no additional sample is required), blood, and saliva. Additional bone marrow samples for biomarkers may be collected at the time of progression or at the End of Treatment visit from all subjects who consent. | Genomics Analysis of genomic biomarkers that may predict response and resistance following treatment with proteasome inhibitors will be conducted for all subjects receiving oprozomib from all phases of the study who consent to optional genomic biomarker analysis. These analyses will be performed on-Sereening a bone marrow aspirate-(obtained at Baseline (within 45 days prior to Cycle 1 Day 1 dosing, only after all other eligibility criteria have been met (a portion of the bone marrow aspirate obtained at Sereening Baseline will be used; no additional sample is required), as well as a sample of blood; and saliva, also collected at Baseline. Bone marrow aspirate or | Revised text for clarity;<br>definition of "Baseline"<br>added |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Pag


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | biopsy collection does not need to be repeated if previously completed within 45 days prior to Cycle 1 Day 1 dosing, and for Phase 3 only, if it was processed at the central laboratory. Additional bone marrow samples for biomarkers may be collected at the time of disease progression or at the (End of Study Treatment visit due to progressive disease [PD], or Long-term Follow-up) from all subjects who consent. | |
| Synopsis:<br>Statistical methods<br>and analyses<br>Section 14.1 Study<br>Endpoints | Endpoints Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study Primary Endpoints-Part 1 Nature of DLTs | | Revised for accuracy and consistency within the protocol |
| ~4 | <ul> <li>Nature and severity of AEs Adverse events and select laboratory abnormalities graded according to<br/>NCI-CTCAE, v-Version 4.03</li> </ul> | | |
| | Changes from baseline in Vital signs and select clinical laboratory results during and following study drug administration | | |
| | Secondary Endpoints-Part 1 | | |
| | <ul> <li>Overall response rate of OPomd defined as the pro<br/>VGPR, or PR as determined by investigator and d</li> </ul> | oportion of subjects with best response of sCR, CR,<br>lefined by according to the IMWG-URC | |
| | Clinical benefit rate of OPomd, defined as the pro-<br>better as determined by investigator according to the control of the pro-<br>better as determined by investigator according to the pro- | portion of subjects with overall best response of MR or the IMWG-URC and modified EBMT criteria | |
| | <ul> <li>Pharmacokinetics parameters, including maximum<br/>concentration (T<sub>max</sub>), area under the plasma conce<br/>(AUC<sub>0-τ</sub>), and area under the plasma concentration<br/>noncompartmental methods</li> </ul> | | |
| | Exploratory Endpoints-Part 1 | | |
| | Pharmacodynamic biomarkers that may be correlated treatment with proteasome inhibitors | ated with antitumor activity and resistance following | |
| | Genomic biomarkers that may be correlated with a | antitumor activity | |
| | Change over time in bone pain and the impact of lonly) | bone pain measured with the BPI-SF (Dose Expansion | |
| | Change over time in the global health-scale status | s/QoL scale of the EORTC QLQ-C30 (Dose Expansion | |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | only) | | |
| | Change over time in health status assessed by EuroQol EQ-5D-5L (Dose Expansion only) | | |
| | Change over time in the disease symptoms subscale of the EORTC QLQ-MY20 (Dose Expansion only) | | |
| | Change over time in neurotoxicity symptoms measured by the FACT/GOG-Ntx4 score (Version 4) (Dose Expansion only) | | |
| | Part 2: Randomized Phase 3 Portion of the Study | | |
| | Primary Endpoint-Part 2 | | |
| | <ul> <li>Progression-free survival, defined as time from rated determined by ORCA according to the IMWG-and according to the IMWG-URC and modified E</li> </ul> | | |
| | Secondary Endpoints-Part 2 | | |
| | Overall survival, defined as time from randomizat | ion to death due to any cause | |
| | Overall response, defined as an overall the best re<br>ORCA and defined by according to the IMWG-U | sponse of sCR, CR, VGPR, or PR as determined by JRC | |
| | <ul> <li>Clinical benefit, defined as an overall- the best resaccording to the IMWG-URC and modified EBM'</li> </ul> | | |
| | Duration of response, defined as the time from the<br>progression as determined by ORCA according to<br>determined by ORCA | first evidence of confirmed PR or better to disease the IMWG-URC or death due to any cause as | |
| | <ul> <li>Improvement in renal function over time, as define</li> </ul> | ed by an increase in GFR of at least 10 mL/min | |
| | Improvement in hemoglobin over time, as defined | by an increase of at least 2 g/dL | |
| | Duration of response, defined as the time from the progression or death due to any cause as determine | first evidence of confirmed PR or better to disease ed by ORCA | |
| | Population based PK parameters including, but no<br>be determined from OPomd subjects | ot limited to, area under the curve (AUC) and C <sub>max</sub> , will | |
| | Adverse events and <b>select</b> laboratory abnormalities time | s graded according to NCI-CTCAE, <b>v Version</b> 4.03 over | |
| | Vital signs and select clinical laboratory results du | aring and following study drug administration over time | |
| | Change over time in bone pain and the impact of bone. | one pain measured with the BPI-SF | |
| | Change over time in the global health seale status | <b>/QoL scale</b> of the EORTC QLQ-C30 | |



| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | Change over time in the disease symptoms subscale of the E | | |
| | Change over time in health status assessed by EuroQol EQ- | | |
| | Population-based PK parameters including, but not lim<br>concentration-time curve (AUC) and C <sub>max</sub> , will be deter | | |
| | Exploratory Endpoints-Part 2 | | |
| | Progression-free survival and ORR-overall response, as det IMWG-URC | termined by the investigator according to the | |
| | <ul> <li>Duration of response, defined as the time from the first evid<br/>progression as determined by the investigator according<br/>as determined by the investigator according to the IMWG-U</li> </ul> | to the IMWG-URC or death due to any cause | |
| | Clinical benefit rate as determined by the investigator accor<br>EBMT criteria | ding to the IMWG-URC and modified | |
| | Duration of clinical benefit (DOCB), defined as the time fro<br>progression or death due to any cause, as determined by C<br>IMWG-URC and modified EBMT criteria | | |
| | Genomic biomarkers that may be correlated with antitumor<br>with proteasome inhibitors | | |
| | Neuropathy events (defined as Grade 2 or higher peripheral | neuropathy incidence) | |
| | Change in the neurotoxicity symptoms as measured by FAC | CT/GOG-Ntx4 score (Version 4) | |
| | Change over time in all domains of the EORTC QLQ-C30 QLQ-MY20 (excluding the global health scale and disease section). | | |
| Synopsis: | Efficacy Analyses | | Revised text for clarity |
| Statistical methods | Part 1: Phase 1b Dose Escalation and <b>Dose</b> -Expansion Portions of | f the Study | |
| and analyses | Response assessment data, PFS, Progression-free survival and duration of response will be listed for all subjects by dose level and schedule. Overall response rate and clinical benefit rate will be estimated for all subjects treated at the RP3D along with the associated 95% exact binomial confidence intervals (CIs). | | |
| | Part 2: Randomized Phase 3 Portion of the Study | | |
| | Median PFS will be estimated for each treatment arm using Kaplar interval (CI) for the median PFS will be constructed using the met of PFS and other efficacy endpoints will be based on the ITT p randomized. The primary inferential comparison for PFS between | hod of Brookmeyer (1982) primary analysis opulation, defined as all subjects | |
| | stratified log-rank test using stratified by the randomization strati | | |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | 2 treatment arms HR will be estimated using a stratified stratification factors. Duration of follow-up for PFS will including medians, will be summarized descriptively group. Overall survival will be analyzed using the san DOCB will be summarized for each treatment group | | |
| | Statistical methods for analyses of OS will be identical t<br>will also be used for estimating median DOR. no forma<br>responders constitute a nonrandom subset of the ITT pop | l inferential comparisons of DOR will be made, as pulation. | |
| | Point estimates and 95% exact <b>binomial</b> CIs will be calc<br>Inferential comparison between treatment groups for thi<br>Cochran-Mantel Haenszel chi-square test, stratified by the | | |
| | Inferential testing of the primary efficacy endpoint and s CBR, improvement in renal function, improvement i scale, and change over time in QLQ-C30 total scale) accordance with a closed testing procedure. | | |
| | Safety Analyses Part 1: Phase 1b Dose Escalation and Dose-Expansion 1 | | |
| | For the Phase 1b portion of the study, safety will be asse<br>laboratory test results, ECGs, vital signs, and oprozomib<br>data collected will be listed by study site, cohort, subject | | |
| Section 3.1<br>Introduction | - | This is a Phase 1b/Phase 3 clinical trial of the oral proteasome inhibitor, oprozomib, in subjects with primary refractory or relapsed and refractory multiple myeloma. See Section 5 for a complete description of the study design. The protocol has been amended with changes to the study design as new data became available from other ongoing oprozomib studies, and based on review of safety results from these studies. A summary of changes for each amendment is included in the appendix of each version of the protocol. The main purposes for each amendment are summarized below. | Added text in a new subsection "Introduction" to provide a top level summary of the amendments thus far. All subsequent headings in this section were renumbered accordingly |
| [ | | Amendment 1: | |




Product: Oprozomib Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | 1. Added an alternative oprozomib dosing schedule consisting of 2 consecutive days every 7 days (2/7), as preliminary data suggest that a 2/7 schedule has single-agent activity, and may be better tolerated than the existing schedule of 5 consecutive days every 14 days (5/14 schedule). | |
| | | <ol><li>Clarified that plasmapheresis is not<br/>permitted at any time during the study.</li></ol> | |
| | | 3. The starting dose of oprozomib was changed from 210 mg to 150 mg to provide increased margin of safety for subjects participating in this study. This dose (150 mg) is 3 dose levels below the single-agent MTD and was selected due to the overlapping toxicities of oprozomib with pomalidomide. | |
| | | <ol> <li>Additional dose modification text was<br/>added to the dose modification table for<br/>nonhematologic toxicities and guidance to<br/>investigators to mitigate Grade 4<br/>gastrointestinal (GI) hemorrhage.</li> </ol> | |
| | | Amendment 2: | |
| | | <ol> <li>To allow subjects with prior carfilzomib<br/>exposure to be considered for inclusion in<br/>the study, if carfilzomib was not withdrawn<br/>due to toxicity.</li> </ol> | |
| | | <ol> <li>To allow subjects with prior pomalidomide<br/>exposure to be considered for inclusion in<br/>the dose-escalation portion of the study, if<br/>pomalidomide was neither dose-reduced<br/>nor withdrawn due to toxicity.</li> </ol> | |
| | | <ol> <li>To specify that only subjects who have been<br/>treated with adequate alkylator therapy are<br/>eligible to be considered for inclusion in the<br/>Phase 1b dose-escalation portion and Phase</li> </ol> | |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | 3 portion of the study. 4. Additional safety guidance regarding Grade 3 or 4 GI hemorrhage (see Section 10.4.2.1.2), mandatory proton-pump inhibitors (see Section 10.6.1.5), and the addition of an exclusion criterion for patients with prior clinically significant bleed in the 6 months prior to first dose of study treatment, because of toxicities observed in Study 2011-001. 5. Revisions in synopsis, statistical sections, objectives, and endpoints for accuracy, clarity, and consistency within the protocol. | |
| Section 3.2 Multiple<br>Myeloma<br>Background | Median OS from diagnosis was reported at 3 years for high-risk patients, 4 to 5 years for intermediate-risk patients, and 8 to 20 years for standard-risk patients (Mikhael 2013). | Median OS from diagnosis was reported at 3 years for high-risk patients, 4 to 5 years for intermediate-risk patients, and 8 to 10 20 years for standard-risk patients (Mikhael 2013). | Corrected text |
| Section 3.4<br>Oprozomib<br>Background | Oprozomib is a tripeptide epoxyketone proteasome inhibitor and structural analogue of carfilzomib (Kyprolis) that primarily targets the chymotrypsin-like activity of the 20S proteasome. Carfilzomib is a tetrapeptide epoxyketone proteasome inhibitor approved in the US for the treatment of relapsed and refractory multiple myeloma. Similar to carfilzomib, oprozomib is a potent, selective, and irreversible inhibitor of the CT-L activity of the constitutive proteasome (the form of proteasome found in most cell types) and the immunoproteasome (the form of proteasome found in many hematopoietic cells) (Zhou 2009). In addition, when measured against a broad panel of proteases containing metallo-, aspartyl, cysteine, and serine proteases, oprozomib demonstrated minimal reactivity against nonproteasomal proteases. | Oprozomib (formerly ONX 0912) is a tripeptide epoxyketone proteasome inhibitor and structural analogue of carfilzomib (Kyprolis) that primarily targets the CT-L ehymotrypsin-like activity of the 20S proteasome. Carfilzomib received accelerated approval in the US for the treatment of patients with multiple myeloma who have received at least 2 prior therapies, including bortezomib and an immunomodulatory agent, and have demonstrated disease progression on or within 60 days of completion of the last therapy (Kyprolis Prescribing Information [Onyx Pharmaceuticals, 2012]). Carfilzomib is a tetrapeptide epoxyketone proteasome inhibitor approved in the US for the treatment of relapsed and refractory multiple myeloma. Similar to carfilzomib, oprozomib is a potent, selective, and irreversible inhibitor of the CT-L activity of the constitutive proteasome (the form of proteasome found in most cell types) and the immunoproteasome (the | Updated text to provide missing information on carfilzomib label, and for consistency with other oprozomib protocols. |



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Page


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | form of proteasome found in many hematopoietic cells) (Zhou 2009). In addition, when measured against a broad panel of proteases containing metallo-, aspartyl, cysteine, and serine proteases, oprozomib demonstrated minimal reactivity against nonproteasomal proteases. | |
| Section 3.4.2<br>Relevant Clinical<br>Background | (SD) was observed in 6 subjects (30%) in the once da daily dosing group. Safety The majority of adverse events (AEs) were Grade 1 a cumulative toxicities. The most common AEs were in preclinical animal studies with oprozomib. Dose-limication of the maximum tolerated dose (MTD) for the once daily toxicities for the split daily x5 days dosing group in S 180 mg and Grade 5 upper GI hemorrhage and Grade dosing is 180 mg. The first-in-human clinical trial (2009-003) of oprozomis subject visit in November 2012 in 44 subjects with adva 19 March 2013. This was an open-label, Phase I study a Capsules orally, once daily, on a 5 consecutive day, bim 14 days. The primary objectives of the study were to eve dose (MTD) of oprozomib in this patient population. Sa were collected at various time points during Cycles I and Amendment 4, oprozomib was administered as a split degastrointestinal (GI) toxicity and to support additional dedosing. Differences in PDn and tolerability between fas for subjects enrolled under Protocol Amendment 4. Efficacy Powder in Capsule | subject achieved an objective response. Stable disease ily dosing group and 4 subjects (23.5%) in the split and 2, manageable, and there were no apparent in the GI system organ class. This was consistent with iting toxicities for the once daily dose group in Study 1 Grade 3 hypophosphatemia in the 180 mg cohort. By x5 days dose group is 150 mg. Dose-limiting tudy 2009-003 included Grade 3 hypophosphatemia at le 3 hallucinations at 210 mg. The MTD for the split be was initiated in May 2010 and completed the last need solid tumors; the database was closed in which subjects initially received Oprozomib in onthly treatment schedule, with cycles repeated every aluate the safety, tolerability, and maximum tolerated in mples for pharmacokinetics (PK) and PDn evaluations d 2. For subjects enrolled under 2009-003 Protocol use (doses administered 4 to 6 hours apart) to mitigate use escalation after reaching the MTD with single daily ted (Cycle 1) and fed (Cycle 2) states were also explored | Updated clinical background information for Study 2009-003 per most recent information |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | the first 4 treatment cycles, and either had at least 1 post-due to progressive disease (PD) prior to the first schedule achieved a partial response (PR). Stable disease (SD) wa the once-daily dosing group and 4 subjects (23.5%) in the progression was 43 days for the once daily group and 57 (CBR; best response > minimal response [MR]) was 28.6 twice-daily dosing group. | as the best response achieved by 6 subjects (28.6%) in<br>e twice daily dosing group. The median time to<br>days for the twice-daily group. The clinical benefit rate | |
| | <u>Safety</u> | | |
| | Once-Daily Group Powder in Capsule | | |
| | All 25 subjects who received a once-daily dose of Oproze All subjects are off study; reasons for study discontinuati consent (3 subjects, 12.0%), adverse event (AE)/toxicity 12.0%). The latter category includes subject decision in | on included PD (18 subjects, 72.0%), withdrawal of (1 subject, 4.0%), and "Other" reasons (3 subjects, | |
| | One subject in the 180-mg cohort experienced a dose-lim dehydration and a second subject in the same dose cohort prompting the expansion of the 150-mg cohort to 7 subjection was determined to be 150 mg. | t experienced a DLT of Grade 3 hypophosphatemia, | |
| | Twenty-four subjects (96.0%) experienced at least 1 treat ≥ 25% of subjects included nausea (23 subjects, 92.0%), 56.0%), diarrhea (13 subjects, 52.0%), decreased appetite and anemia (7 subjects each, 28.0%). | vomiting (20 subjects, 80.0%), fatigue (14 subjects, | |
| | The majority of treatment-emergent AEs were GI and Groceurring in more than 1 subject were Grade 3 dehydratic hyponatremia, and hypophosphatemia (2 subjects each, 8 treatment-emergent AE of hyperuricemia that resolved al subjects (28.0%) experienced at least 1 treatment-emerge SAEs in the once-daily dosing group. Grade 3 dehydratic experienced by more than 1 subject. | on (3 subjects, 12.0%) and Grade 3 vomiting,<br>1.0%). One subject (4.0%) experienced a Grade 4<br>fter 13 days; no action was taken with study drug. Seven<br>tent serious AE (SAE). There were no Grade 4 or Grade 5 | |
| | Twice Daily Group Powder in Capsule | | |
| | The safety population comprised all 19 enrolled subjects All subjects are off study; reasons for study discontinuati subjects, 15.8%), symptomatic deterioration (1 subject, 5 including subject decision/preference (3 subjects) and lace | on included PD (11 subjects, 57.9%), AE/toxicity (3 .3%), and "Other" reasons (4 subjects, 21.1%), the latter | |
| | One subject in the 180-mg cohort experienced a DLT of the 180-mg cohort to 7 subjects (1 subject did not complete the 180-mg cohort to 7 subjects (1 subject did not complete the 180-mg cohort to 7 subjects (1 subject did not complete the 180-mg cohort experienced a DLT of the 180-mg cohort to 7 subjects (1 subject did not complete the 180-mg cohort experienced a DLT of the 180-mg cohort experienced a DLT of the 180-mg cohort to 7 subjects (1 subject did not complete the 180-mg cohort experienced a DLT of the 180-mg cohort to 7 subjects (1 subject did not complete the 180-mg cohort experienced a DLT of the 180-mg cohort experienced a D | Grade 3 hypophosphatemia, prompting the expansion of ete Cycle 1 for reasons other than DLT and was therefore | |




| Section(s) | Changed from | m | | Changed to | Rationale |
|---|---|---|---|---|---|
| | replaced). No additional DLTs w<br>cohort (120 mg, 90 mg), including<br>hallucinations. The MTD for the | | | | |
| | | subjects, 94.7%); nause | a (17 subjects, 89.5 | The most frequent AEs seen in ≥ 25% (3%); diarrhea (14 subjects, 73.7%); rexia, dysguesia, and anemia (5 | , de |
| | decreased were the only ≥ Grade: Grade 3 anemia, and 2 subjects (1 | 3 AEs occurring in more 0.5%) experienced Graceurred in the twice daily addy drug due to a GI bloom to the two security of the control of the | than 1 subject. For<br>le 3 lymphocyte co-<br>dosing group. On | mia, fatigue, and lymphocyte count<br>our subjects (21.1%) experienced<br>unt decreased and Grade 3 fatigue,<br>e subject in the 210-mg cohort died | |
| Section 3.4.2<br>Relevant Clinical<br>Background | 3.3.2.2. Study 2011-001: Hemate Efficacy As of 21 January 2014, the Phase evaluable subjects with hematol Oprozomib Tablets with daily day weekly (2/7) schedule in Phasubjects with Waldenström made in Table 1 and Table 2, respecti Table 1 Phase 1 Response Rates | Updated clinical background information for Study 2011-001 per most recent information | | | |
| | Formulation/Schedule (n) | Dose Range (mg) | ORR | Clinical Benefit Rate | |
| | PIC 5/14 (10) | 120-210 | 40% | 50% | |
| | Tablets 5/14 (18) | 150-270 | 27.8% | 38.9% | |
| I | <b>Tablets 2/7 (15)</b> | 150-330 | 20.0% | 46.7% | |
| | ORR = overall response rate; PIC = powder in capsule. Table 2 Phase 1 Response Rates for Subjects with Waldenström macroglobulinemia, by Schedule and Formulation | | | | |
| | Formulation/Schedule | (n) Dose Range (m | g) ORR <sup>a</sup> | Major Response <sup>b</sup> | |




| Section(s) | Changed from | m | | Changed to | Rationale |
|---|---|---|---|---|---|
| | Tablets 5/14 (11) | 150-270 | 63.6% | 54.5% | |
| | <b>Tablets 2/7 (7)</b> | 150-330 | 42.9% | 14.3% | |
| | MR = minimal response <sup>a</sup> ORR is defined as ≥ M <sup>b</sup> Major response is defi The Phase 2 portion of Study 20 Oprozomib Tablets on the 5/14 s 1 subject was off study prior to a Safety In the Phase 1 portion of the stu • Thirty-two (32) subjects have schedule observed at the mass | IR. ined as ≥ PR. i11-001 is ongoing. E schedule with once da any disease response dy (as of 21 January, e been enrolled on th | ight (8) response-ev-<br>illy dosing in Phase<br>assessment.<br>2014):<br>e 5/14 schedule. Do | aluable subjects have rece<br>2; 7 subjects had SD, and<br>se-limiting toxicities for th | ne 5/14 |
| | (TLS) and Grade 3 vomiting Phase 2 portion for the 5/14; high rate of discontinuations reduced. The Phase 2 portio 150 mg as the initial dose lev • Twenty-nine (29) subjects ha schedule observed at the MA MTD was defined as 300 mg 240 mg as the initial dose lev | schedule. Due to toxicobserved at this doson of the study will real, with an increase to the been enrolled on the LD of 330 mg were Grant With the opening of | cities, including fata<br>e level, the dose und<br>open using a step-up<br>o 180 mg in Cycle 2.<br>the 2/7 schedule. Do<br>rade 3 diarrhea and<br>f Amendment 6, a st | al GI bleeding in 2 subject<br>er evaluation in Phase 2 h<br>o dose approach starting v<br>se-limiting toxicities for th<br>Grade 4 thrombocytopen<br>ep-up dosing regimen usi | s, and a as been with the 2/7 ia. The |
| | for the 2/7 schedule. In the Phase 2 portion of the stu | dy (as of 21 January | 2014)• | | |
| | A total of 13 subjects have be | • • | * | | |
| | No subjects have been enroll | | | | |
| | Nineteen (19) subjects experience<br>related SAEs comprised 4 GI even dehydration), 2 hematological even 1 general event (fatigue/dehthese are expected events based. There were also 2 Grade 5 GI hematological events based. | ents (diarrhea, nause<br>vents (anemia and ne<br>ydration/nausea; eve<br>on the Oprozomib IE | a/vomiting, fatigue/<br>utropenia), 2 cases onts could be counted<br>to (Version 6). There | dehydration/nausea, and of TLS, 1 infection (pneum d in more than 1 category) were 2 cases of renal fails | nonia),<br>). All of |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | The second clinical trial (2011-001) was initiated in Sept This is an ongoing, open-label, Phase 1b/2, multicenter's March 2013. The primary objectives for the Phase 1b es of oprozomib in this patient population. Differences in a fasted and fed state are also being explored. The study worally, twice daily (doses separated by 4 to 6 hours), on eyele) treatment schedule. For subjects enrolled under 2 Oprozomib Tablets, once daily, either on a 5 consecutive schedule (Days 1, 2, 8, and 9 of a 14-day cycle). Under earfilzomib-refraetory multiple myeloma (n = 20) will be the efficacy and safety of oprozomib in this patient popul myeloma will be treated using the 5 consecutive day, bir | tudy of oprozomib with 37 subjects treated as of calation are to evaluate the safety, tolerability, and MTD prozomib tolerability and PDn in subjects treated in a ras initiated with Oprozomib in Capsules administered in 5 consecutive day, bimonthly (Days 1 to 5 of a 14-day 011-001 Protocol Amendment 2, subjects received aday, bimonthly schedule or a 2 consecutive day, weekly Protocol Amendment 3, a cohort of subjects with a enrolled in the Phase 2 portion of the study to evaluate lation. Subjects with carfilzomib-refractory multiple | |
| | Twice Daily × 5 Bimonthly Powder in Capsule | | |
| | As of 25 March 2013, 13 subjects have received Oprozoschedule with split daily dosing. Twelve subjects are exfrom the study. Among the subjects with multiple mycle their best response. In addition, 1 subject on study with response. | aluable for response assessment and 1 has withdrawn<br>oma, 3 had a PR, 2 had a MR, 4 had SD, and 2 had PD as | |
| | Once Daily × 5 Bimonthly Powder in Capsule | | |
| | Thirteen multiple myeloma and 5 Waldenström macrogl-<br>bimonthly schedule were included in the response evalua<br>(multiple myeloma) and 80.0% (WM). In subjects with-<br>response (VGPR), 2 (210 mg/d) had a PR, 6 (150–240 m<br>evaluable for response. In WM subjects, 4 (150–210 mg | ttion. The clinical benefit rates (CBR) were 23.1% multiple myeloma, 1 (150 mg/d) had a very good partial g/d) had SD, 1 (150 mg/d) had PD, and 3 were not | |
| | Safety | , , , | |
| | Twice Daily × 5 Bimonthly Powder in Capsule | | |
| | As of 25 March 2013, 13 subjects (5 males, 8 females) whave received Oprozomib in Capsules on a 5 consecutive 13 subjects received at least 1 dose of study drug and we up to 210 mg/day. At study entry, 11 subjects had relaps At least 1 treatment-emergent AE has been recorded in a | day, bimonthly schedule with twice-daily dosing. All re evaluable for safety. No DLTs were observed at doses ed multiple myeloma and 2 subjects had CLL. | |
| | of subjects were nausea (11 subjects), diarrhea (9 subject subjects), thrombocytopenia (4 subjects), and decreased | | |
| | Seven subjects had at least 1 treatment-emergent Grade | 11 | |






| Section(s) | Ch | anged from | Change | d to | Rationale |
|---|---|---|---|---|---|
| | and nausea (2 subjects<br>neutropenia, pneumoni<br>emergent Grade 4 AE ( | or Adverse Events (NCI-CTCAE), Veeach), and thrombocytopenia, abdomia, back pain, and vomiting (1 subject (thrombocytopenia in all 3 subjects). One death due to PD occurred, 71 decemble of the control | inal pain, fatigue, Herpes zo<br>each). Three subjects had a<br>No Grade 5 AEs were repor | ster ophthalmic,<br>t least 1 treatment-<br>ted within 30 days of the | |
| | cohort), Herpes zoster The pneumonia resolve after 2 days and require days and required dose | ophthalmic (1 subject in the 120-mg c<br>ed after 2 days without oprozomib dose<br>ed the subject's oprozomib dose to be<br>reduction and concomitant mediation | ped at least 1 treatment-emergent SAE, including pneumonia (1 subject in the 120-mg phthalmic (1 subject in the 120-mg cohort), and nausea (1 subject in the 150-mg cohort). I after 2 days without oprozomib dose modification. The Herpes zoster event resolved 1 the subject's oprozomib dose to be held or delayed. The nausea event resolved after 2 | | |
| | | thly Tablet and Once Daily × 2 Table<br>edian treatment duration was 11.3 eye | | | |
| | schedule and once dail<br>once daily × 5 bimonth<br>dose of 240 mg/day. T | y × 2 weekly schedule, respectively. Ly schedule: renal failure on a dose of the most common Grade 1–2 adverse verse Events in > 25% of Subjects | | | |
| | | Grade 1-2 Adverse Events | Number of Subjects | | |
| | | Nausea | 28 | | |
| | | Diarrhea | 20 | | |
| | | Fatigue | 20 | | |
| | | Vomiting | 14 | | |
| | | Constipation | 11 | | |
| | The most common Gra | de 3-4 AEs (≥ 2 subjects) are summar | rized in Table 2. | | |
| | Table 2 Grade 3-4 Ad | Table 2 Grade 3-4 Adverse Events (≥ 2 Subjects) | | | |
| | | Grade 1-2 Adverse Events | Number of Subjects | | |
| | | Diarrhea | 9 | | |
| | | Anemia | 4 | | |
| | | Nausea | 4 | | |
| | | Neutropenia | 4 | | |




| Section(s) | Cha | nged from | Change | d to | Rationale |
|---|---|---|---|---|---|
| | | Hypophosphatemia | 3 | | |
| | | Thrombocytopenia | 3 | | |
| | | Vomiting | 3 | | |
| | | Dehydration | 2 | | |
| | | Fatigue | 2 | | |
| | Further details are provide | led in the Oprozomib IB. | | - | |
| Section 3.4.2<br>Relevant Clinical<br>Background | | | 3.2.3 Study 2012-001: Oprovith Dexamethasone in Multificacy For the 2012-001 Phase 1b/2 014, 5 response-evaluable refractory multiple myeloma Dprozomib Tablets on a 5 commonthly (5/14) schedule with ombination with dexamethate and 4 subjects had SD at as of 31 March 2014, 8 response received Oprozomib Tarally, once daily, on Days 1, yele (2/7) in combination with dexamethasone; 1 subject has unconfirmed), 2 subjects has provided and 4 subjects had SD at a subject has and 4 subjects had SD at a subject has and 4 subjects had SD at a subject | study, as of 31 March elapsed and/or a subjects received onsecutive day ith daily dosing in asone; 1 subject had a their best response. Onse-evaluable subjects ablets administered and a their best response med), 1 subject had a partial response med), 1 subject had a sa the best response. dy assessing safety and their ombination with enrolling in the Phase exts have been enrolled med (n = 5) to 210 mg ule, and 4 subjects | Added updated clinical background information for Study 2012-001 for consistency with other oprozomib protocols. |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Pag


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | experienced DLTs at the 210 mg dose, including 1 subject with a subarachnoid hemorrhage (SAH), 1 subject with Grade 3 transaminitis, and 1 subject with Grade 4 thrombocytopenia. In addition, 1 subject had 3 SAEs (esophagitis, urinary tract infection, and pneumonia). Data suggest that the 180-mg dose level will be the tolerable dose in combination with dexamethasone. This dose level exceeds the starting dose for the combination of oprozomib, pomalidomide, and dexamethasone (OPomd). • As of May 2014, 13 subjects have been enrolled and treated at doses of 180 mg (n = 3), 210 mg (n = 3), 240 mg (n = 3), to 270 mg (n = 4) on the 2/7 schedule, and 7 subjects remain on study. One DLT of Grade 4 thrombocytopenia has been observed. Dose escalation is ongoing at the 300-mg dose level, suggesting that doses lower than 300 mg in combination with dexamethasone are tolerable. Current doses explored in this schedule exceed the starting dose for the combination of OPomd. | |
| | | As of 31 March 31 2014, ten (10) subjects experienced serious adverse events (SAEs) across both schedules. The 3 treatment-related SAEs were 1 subject with a SAH, hypertension, and headache, 1 subject with thrombocytopenia, pneumonia, and sepsis, and 1 subject with delirium. Thrombocytopenia and infection were expected events based on the Oprozomib IB (Version 6), but the SAH, hypertension, headache, and delirum were not. | |
| Section 3.4.2<br>Relevant Clinical<br>Background | _ | 3.3.2.4 Study OPZ003: Oprozomib in Combination with Lenalidomide and Dexamethasone in Multiple Myeloma <u>Efficacy</u> | Added updated clinical<br>background information for<br>Study OPZ003 for<br>consistency with other |




Superseded


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | No efficacy data are available at this time. Safety The OPZ003 Phase 1b/2 study, assessing oprozomib in combination with lenalidomide and dexamethasone, is currently enrolling in the Phase 1b portion of the study in newly diagnosed subjects with multiple myeloma. As of 21 January 2014, 3 subjects have been enrolled. Two (2) subjects remain on study. One subject, a very remain on study. One subject, a very remain of the subject discontinued treatment, and the SAE resolved. Subsequently, the subject experienced a second event of syncope. The dose level in this study has since been de-escalated to 180 mg and syncope has been identified as an event of interest for oprozomib. | oprozomib protocols. |
| Section 3.5.3<br>Pomalidomide | but far greater antiproliferative and immunomodula 2007; Payvandi 2004). Pomalidomide has also been statement of relativity (ADCC) (Bartlett 2007). Pomalidomide received accelerated approval in the Factory and the European Commission has granted approval for for the treatment of relapsed and refractory multiple and have demonstrated disease progression on the la approval for patients with multiple myeloma with 2 plenalidomide and who are refractory to their last the dose of pomalidomide is 4 mg given 21 days of a 28-d Approval was based on Study MM002, a randomized with low-dose therapeutic dexamethasone (POM + L The overall response rate (ORR) was 34%, with a multiple myeloma state of the state o | s an IMiD that displays similar antiangiogenic activity tory activity compared with the parent drug (Bartlett shown to stimulate antibody-dependent cytotoxic EU in August 2013 and in the US in February 2013. pomalidomide in combination with dexamethasone, emyeloma who received at least two prior therapies st drug taken and the US FDA granted accelerated prior therapies including both bortezomib and rapy or progressed within 60 days. The approved lay cycle until progressive disease (PD). In Phase 2 comparison of pomalidomide in combination to Dex.) to pomalidomide alone (Jagannath 2012), edian PFS of 4.6 months and median OS of | Reorganized sections for clarity and to reduce redundancy |






| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | (10%), and urinary tract infection (9%). Grade 3 or years and in 35% of subjects aged > 65 years. Febrile age group (2%). Overall, 78% of subjects who develor granulocyte-colony stimulating factor (G-CSF) durin peripheral neuropathy (PN) reported, although Grad POM + LoDex. Deep vein thrombosis (DVT) occurre provide an efficacious option with a manageable toxic and refractory multiple myeloma. | | |
| | The approved dose of pomalidomide is 4 mg given 21 da | ays of a 28-day cycle until PD. | |
| | The MM003 study assessed relapsed and/or refractory su treated with bortezomib and lenalidomide or thalidomide A regimen of pomalidomide and dexamethasone was con | bjects with multiple myeloma who had been previously and progressed on or within 60 days of the last therapy. | |
| | Subjects were randomized 2:1 to receive 28-day cycles of pomalidomide 4 mg on Days 1–21 + dexamethasone 40 mg (20 mg for subjects more than 75 years old) weekly or dexamethasone 40 mg (20 mg for subjects more than 75 years old) on Days1–4, 9–12, and 17–20. Treatment continued until PD or unacceptable toxicity. The primary endpoint was PFS. Secondary endpoints included OS, <del>overall response rate (</del> ORR (≥ PR), and safety. Analyses were based on intent to treat. A total of 455 subjects were randomized to pomalidomide + low-dose dexamethasone (n = 302) or high-dose dexamethasone (n = 153). The median number of prior therapies was 5 (range: 1–17). Seventy-two percent (72%) of subjects were refractory to lenalidomide and bortezomib. Median follow-up was 4 months. Pomalidomide + low-dose dexamethasone significantly extended median PFS (3.6 versus 1.8 months, hazard ratio [HR] = 0.45, p < 0.001) and OS (not reached versus 7.8 months, HR = 0.53, p < 0.001) compared with high-dose dexamethasone. The OS benefit was observed despite 29% of high-dose dexamethasone subjects receiving pomalidomide after PD (Jagannath 2012). With updated data, the ORR was 21% for pomalidomide + low-dose dexamethasone versus 3% for high-dose dexamethasone (p < 0.001) and 24% versus 3% for subjects randomized ≥ 6 months after enrollment (p < 0.001). Median OS overall survival was 12.7 months for pomalidomide and 8.1 months for high-dose dexamethasone; HR = 0.74 (p = 0.28). The most frequent Grade 3/4 AEs for pomalidomide + low-dose dexamethasone versus high-dose dexamethasone were neutropenia (42% versus 15%), anemia (27% versus 29%), and infection (24% versus 23%). Discontinuation due to AEs was infrequent (7% versus 6%) (San Miguel 2013). | | |
| Section 3.5 Dose | 3.5.1 Oprozomib | 3.5.1 Oprozomib | Text was rearranged and |
| Rationale | Early development of oprozomib focused on the 5 consecutive day bimonthly (either once or twice daily) (5/14) and 2 consecutive days weekly (2/7) schedules, | Early development of oprozomib focused on the 5 consecutive day bimonthly (either once or twice daily) (5/14) and 2 consecutive days weekly (2/7) schedules, | revised for clarity |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | both on 14-day treatment cycles. The maximum administered dose for Oprozomib Tablets administered once daily on a 5 consecutive day bimonthly schedule has been reached with a total daily dose of up to 270 mg in subjects with hematologic malignancies, with 1 DLT of TLS and one Grade 3 vomiting out of 6 subjects. At the 240 mg dose, 6 subjects were dosed with 1 DLT of TLS, therefore 240 mg was the declared as the MTD. The starting dose of 150 mg of oprozomib will be added to the FDA approved regimen of pomalidomide/dexamethasone, 3 dose levels below the MTD in the 5/14 schedule in the single-agent study. The starting dose for the 2/7 schedule will be 210 mg, 3 dose levels below the single agent MTD of 300 mg. One DLT of grade 3 orthostatic hypotension was reported in this cohort. The maximum administered dose was reached with a total daily dose of 330 mg with 1 DLT of Grade 3 diarrhea and 1 DLT of Grade 4 thrombocytopenia. The most significant AEs noted are GI toxicities. This study will assess both schedules in Part 1 of the study, as oprozomib has demonstrated preliminary activity in subjects with hematologic malignancies on both schedules. (Kaufman 2013). | both on 14-day treatment cycles. The maximum administered dose MAD for Oprozomib Tablets administered dose MAD for Oprozomib Tablets administered once daily on a 5 consecutive day bimonthly schedule has been reached with a total daily dose of up to 270 mg in subjects with hematologic malignancies, with 1 dose-limiting toxicity (DLT) of TLS and 1 one Grade 3 vomiting out of 6 subjects. At the 240-mg dose, 6 subjects were dosed with 1 DLT of TLS, therefore 240 mg was the declared as the MTD. For the 5/14 schedule, the starting dose of 150 mg of oprozomib will be added to the Food and Drug Administration (FDA)-approved regimen of pomalidomide/dexamethasone, 3 dose levels below the MTD in the single-agent study in the 5/14 schedule in the single-agent study. The starting dose for the 2/7 schedule will be 210 mg, 3 dose levels below the single agent MTD of 300 mg. One DLT of grade 3 orthostatic hypotension was reported in this cohort. The maximum administered dose was reached with a total daily dose of 330 mg with 1 DLT of Grade 3 diarrhea and 1 DLT of Grade 4 thrombocytopenia. For the 2/7 schedule, the MAD was reached with a total daily dose of 330 mg with 1 DLT of Grade 3 diarrhea and 1 DLT of Grade 4 thrombocytopenia. One DLT of Grade 3 orthostatic hypotension was reported in the 300-mg cohort, therefore 300 mg was declared the MTD. The starting dose for the 2/7 schedule will be 210 mg, 3 dose levels below the single agent MTD of 300 mg. The most significant AEs noted are GI toxicities. This study will assess both schedules in Part 1 of the study, as oprozomib has demonstrated preliminary activity in subjects with hematologic malignancies on both schedules (Kaufman 2013). | |
| Section 3.5 Dose<br>Rationale | Dexamethasone will be administered in this study based on data from the SUMMIT trial (Richardson | Dexamethasone will be administered in this study based on data from the SUMMIT trial (Richardson | Deleted text that is now redundant with newly |






| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | 2003) and an expanded access trial (Mikhael 2009), in which dexamethasone was shown to have improved efficacy when administered with proteasome inhibitors. Preclinical studies also suggest the potential therapeutic advantage of dexamethasone combined with carfilzomib (Kuhn 2007) and bortezomib (Hideshima 2001) in multiple myeloma. In earlier clinical studies, dexamethasone was shown to mitigate AEs temporally associated with single-agent oprozomib. | 2003) and an expanded access trial (Mikhael 2009), in which dexamethasone was shown to have improved efficacy when administered with proteasome inhibitors. Preclinical studies also suggest the potential therapeutic advantage of dexamethasone combined with carfilzomib (Kuhn 2007) and bortezomib (Hideshima 2001) in multiple myeloma. In earlier elinical studies, dexamethasone was shown to mitigate AEs temporally associated with single-agent oprozomib. | added clinical background<br>information for Study<br>2012-001 |
| Section 3.6 Study Rationale | Carfilzomib (Kyprolis) is an irreversible inhibitor of the epoxyketone class (proteasome) that is selective and structurally distinct from bortezomib (O'Connor 2009). Proteasome inhibition by bortezomib is slowly reversible. Consequently, proteasome inhibition is more sustained with carfilzomib than with bortezomib (Demo 2007; Suzuki 2011). In comparison to bortezomib, carfilzomib exhibits equal potency, but greater selectivity for the CT-L activity of the proteasome. In cell culture, carfilzomib is more cytotoxic than bortezomib following brief treatments that mimic the in vivo PK of both molecules (Demo 2007) Data collected in these 2 trials suggested that the 2 consecutive day weekly schedule was better tolerated and demonstrated clinically meaningful response rates. Subsequent Phase 2 and Phase 3 carfilzomib studies have utilized this dose and schedule and have provided data indicating both tolerability and efficacy in advanced stage, heavily pretreated multiple myeloma subjects. | Carfilzomib (Kyprolis) is an irreversible inhibitor of the epoxyketone class (proteasome) that received accelerated approval in the US for the treatment of patients with multiple myeloma who have received at least 2 prior therapies, including bortezomib and an immunomodulatory agent, and have demonstrated disease progression on or within 60 days of completion of the last therapy (Kyprolis Prescribing Information [Onyx Pharmaceuticals 2012]). Carfilzomib is selective and structurally distinct from bortezomib (O'Connor 2009). Proteasome inhibition by bortezomib is slowly reversible. Consequently, proteasome inhibition is more sustained with carfilzomib than with bortezomib (Demo 2007; Suzuki 2011). In comparison to bortezomib, carfilzomib exhibits equal potency, but greater selectivity for the CT-L activity of the proteasome. In cell culture, carfilzomib is more cytotoxic than bortezomib following brief treatments that mimic the in vivo PK of both molecules (Demo 2007). Data collected in these 2 trials suggested that the 2 consecutive day weekly schedule was better tolerated and demonstrated clinically meaningful response rates. | Added text for clarity |



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Page


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | Subsequent Phase 2 and Phase 3 carfilzomib studies have utilized this dose and schedule and have provided data indicating both tolerability and efficacy in advanced stage, heavily pretreated multiple myeloma subjects. Both schedules will be assessed with oprozomib to determine which schedule provides an advantage in tolerability and efficacy. | |
| Section 5 Study<br>Design | During Part 2 of the study, subjects will be randomized to oprozomib or placebo (subjects in the Pomd arm) at the RP3D and schedule determined during Part 1 of the study. Up to 20 study sites will participate in Part 1 of the study (Phase 1b Dose Escalation and Expansion portions of the study). Approximately 70 sites will participate in Part 2 of the study (Phase 3 portion of the study). | During Part 2 of the study, subjects will be randomized to oprozomib in combination with pomalidomide and dexamethasone (OPomd) or placebo (subjects in the Pomd arm) at the RP3D and schedule determined during Part 1 of the study or placebo in combination with pomalidomide and dexamethasone (Pomd). Approximately 35 study sites will participate in Part 1 of the study (15 sites for the Phase 1b dose-escalation and 20 additional sites for the dose-expansion portions of the study). An additional 35 sites, for a total of approximately 70 sites will participate in Part 2 of the study (Phase 3 portion of the study). | Revised text for clarity. |
| Section 5 Study<br>Design | Moved from: 5.1.2 Dose-Escalation Schema for the 2/7 Oprozomib Dosing Schedule Treatment cycles for both parts of the study will last 28 days. Disease assessments will be performed every 4 weeks for subjects in both arms for 18 months. Further disease assessments will be conducted every 8 weeks after this period. Details of the study assessments required for this study are provided in Appendices A1 and A2. | Moved to: (End of) 5 Study Design Treatment cycles are 28 days in duration. Two (2) oprozomib dosing schedules will be assessed during dose-escalation. Subjects will receive oprozomib once daily either on Days 1–5 and 15–19, referred to hereafter as the 5/14 schedule, or an alternate schedule of once daily on Days 1, 2, 8, 9, 15, 16, 22, and 23, referred to hereafter as the 2/7 schedule. Pomalidomide will be given on Days 1–21 and dexamethasone will be given on Days 1, 2, 8, 9, 15, 16, 22, and 23 of every 28-day cycle. | Revised text for clarity and moved text to the appropriate location in the protocol |
| Section 5.1 Part 1:<br>Phase 1b Dose-<br>Escalation and<br><b>Dose-</b> Expansion | The safety of subjects in the Dose Expansion will be monitored on an ongoing basis by the CSRC during bimonthly calls. Enrollment to the Phase 3 portion will | The safety of subjects in the Dose Expansion will be monitored on an ongoing basis by the CSRC during bimonthly calls. Enrollment to the Phase 3 portion will | Deleted text as it is<br>redundant with the text in<br>the following section (5.2<br>Part 2: Randomized Phase |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Portions of the<br>Study | not commence until the CSRC has evaluated all available safety information from a minimum of 10 subjects who have completed ≥ 2 cycles of therapy at the RP3D and enrollment of the remaining 10 subjects in Dose Expansion has occurred in 1 or both schedules if both were opened. | not commence until the CSRC has evaluated all available safety information from a minimum of 10 subjects who have completed $\geq$ 2 cycles of therapy at the RP3D and enrollment of the remaining 10 subjects in Dose Expansion has occurred in 1 or both schedules if both were opened. | 3 Postion of the Study) |
| Section 5.1.3<br>Dose-Limiting<br>Toxicities | Deleted text from Section 5.1.4 Subject Replacement and Subjects in both dosing schedules will be evaluated for I the 28-day period of Cycle 1 combination therapy. Intra once that dose has been determined and after a discussion study medical monitor. The decision to escalate to the nother study will be based on an assessment of study drug-reconsists of investigators, the Onyx medical monitor, at the cohort under review will be discussed and assessed decide on the most appropriate course of action regards Study drug is defined as the combination of oprozod drug-related is defined as a reasonable likelihood of clinidechallenge improvement and that the AE was not likely disease, concomitant medication, or study/nonstudy procoprovided in Section 10.5. | DLTs according to the NCI-CTCAE, version 4.03 during subject dose escalation to the RP3D may be permitted in has occurred between the treating physician and Onyx ext higher dose of oprozomib in the Phase 1b portion of elated DLTs during Cycle 1 by the CSRC. The CSRC and Onyx Drug Safety representative. Each subject in d. Once all data have been presented, the CSRC will reding dose escalation based on guidance in Section 5.1. alidomide, and dexamethasone. Study ical causality based on time of event, biology, explained by the subject's clinical state, underlying | Reorganized text so that it is in the appropriate location in the protocol. Added definition of "study drug" |
| Section 5.2<br>Randomized Phase<br>3 (Part 2) Portion of<br>the Study | Part 2 will consist of a placebo-controlled, double-blind RP3D component. | Part 2 will consist of a placebo-controlled, double-blind RP3D randomized Phase 3 component. | Corrected text |
| Section 5.3<br>Estimated Study<br>Duration and Study<br>Closure | The total study duration is expected to be approximately 32-33 months. • The Phase 1b portion of the study will take approximately 7–8 months to complete. • Approximately 5 months will be required to enroll and evaluate response status of subjects in the dose expansion portion of the study. • Approximately 13 additional months will be required to enroll subjects in the Phase 3 portion of the study. | The total study duration is expected to be approximately 32–33 months. • The Phase 1b portion of the study will take approximately 7–8 months to complete • Approximately 5 months will be required to enroll and evaluate response status of subjects in the dose-expansion portion of the study • Approximately 13 additional months will be required to enroll subjects in the Phase 3 portion of the study | Deleted redundant text |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Page


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | Assuming an enrollment rate of 22 subjects per month, it is estimated that the final analysis of PFS will occur approximately 17 months after the first subject is enrolled in the Phase 3 portion of the study. Distriction of the Study Colored to the Study Colored | Assuming an enrollment rate of 22 subjects per month, it is estimated that the final analysis of PFS will occur approximately 17 months after the first subject is enrolled in the Phase 3 portion of the study | |
| | Prior to initiating the Phase 3 portion of the study, an assessment of the safety and efficacy data from a minimum of 10 subjects treated during the expansion portion of the study and the enrollment of the remaining 10 subjects in the expansion cohort will be completed in 1 or both schedules if each will be opened per the sponsor's discretion. | Prior to initiating the Phase 3 portion of the study, an assessment of the safety and efficacy data from a minimum of 10 subjects treated during the expansion portion of the study and the enrollment of the remaining 10 subjects in the expansion cohort will be completed in 1 or both schedules if each will be opened per the sponsor's discretion. | |
| Section 5.4.2<br>Blinding | For Phase 3 only, an independent, external Data<br>Monitoring Committee (DMC) will monitor the<br>conduct of the study and undertake periodic unblinded<br>assessments of safety data to optimize the safety of<br>study subjects and ensure integrity of the study. | For Phase 3 only, an independent, external Data Monitoring Committee (DMC) will monitor the conduct of the study and undertake periodic unblinded assessments of safety data to <b>protect</b> optimize the safety of study subjects and ensure integrity of the study. | Revised text for accuracy. |
| Section 9.4 Study<br>Drug Accountability | Onyx (or designee) and the investigator will maintain records of each shipment of investigational product (IP). Upon receipt of IP, the designated recipient at the study site will inspect the shipment, verify the number and condition of the vials, and prepare an inventory or drug accountability record. The records will document shipment dates, method of shipment, batch numbers, product presentation, quantity of bottles contained in the shipment, and dispensation to individual subjects using the subject identification number. | Onyx (or designee) and the investigator will maintain records of each shipment of investigational product (IP). Upon receipt of IP, the designated recipient at the study site will inspect the shipment, verify the number and condition of the <b>bottles or blister packs vials</b> , and prepare an inventory or drug accountability record. The records will document shipment dates, method of shipment, batch numbers, product presentation, quantity of bottles <b>or blister packs</b> contained in the shipment, and dispensation to individual subjects using the subject identification number. | Corrected text and added<br>text to allow for the<br>potential use of blister<br>packs in Phase 3 of the<br>study |
| Section 10.1<br>Oprozomib<br>Treatment<br>Administration | It is recommended that oprozomib not be taken on an empty stomach. Subjects will be instructed to take the oprozomib doses after eating with approximately 8 ounces of water. | It is recommended that oprozomib not be taken on an empty stomach. Subjects will be instructed to take the oprozomib doses after eating with approximately 8 ounces of water. On the PK collection days, dosing of oprozomib in relation to the meal intake (within 2 hours before and 1 hour after dose) will be | Added text for consistency with other oprozomib protocols |




Superseded


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | recorded. | |
| Section 10.3 Dose<br>Modification<br>Guidelines | This section provides dose reduction and other modification guidelines for oprozomib, pomalidomide, and dexamethasone to manage possible toxicity. Administration of oprozomib or pomalidomide will be discontinued in the event of a treatment-related toxicity that, in the opinion of the investigator, warrants permanent discontinuation. Monotherapy with dexamethasone is not allowed in the | This section provides dose reduction and other modification guidelines for oprozomib, pomalidomide, and dexamethasone to manage possible toxicity. Administration of oprozomib or pomalidomide will be discontinued in the event of a treatment-related toxicity that, in the opinion of the investigator, warrants permanent discontinuation. Monotherapy with dexamethasone is not allowed in the | Added text for clarity |
| | Phase 1b Dose-Escalation and Expansion portions of the study. In the event that oprozomib or pomalidomide is permanently discontinued in Phase 3 only, dexamethasone may be continued. | Phase 1b dose-escalation and dose-expansion portions of the study. In the event that oprozomib or pomalidomide is permanently discontinued in Phase 3 only, dexamethasone may be continued. | |
| Section 10.4.1 Dose<br>Reductions | Modifications of the dose of oprozomib/placebo will occur in up to three 30-mg decrements down to a minimum of 150 mg. Additional reductions will be managed by schedule change. | Modifications of the dose of oprozomib/placebo will occur in up to three 30-mg decrements down to a minimum dose of 150 mg. Additional reductions will be managed by schedule change. | Corrected text and rearranged text for clarity |
| | Treatment guidelines for specific hematologic toxicities are outlined in Section 10.4.2.1.1 and nonhematologic toxicities in Section 10.4.2.1.2. In addition to dose reductions, administration of oprozomib, and pomalidomide may be temporarily interrupted for a maximum of 4 weeks in the event of a treatment-related toxicity. | Treatment guidelines for specific hematologic toxicities are outlined in Section 10.4.2.1.1 and nonhematologic toxicities in Section 10.4.2.1.2. In addition to dose reductions, administration of oprozomib, and pomalidomide, and dexamethasone may be temporarily interrupted for a maximum of 4 weeks in the event of a treatment-related toxicity. | |
| | If dexamethasone dosing is permanently stopped due to toxicity in accordance with the dose modification guidelines described in Table 15, the subject should stay on oprozomib and/or pomalidomide, depending on the arm to which they are randomized, and continue to follow protocol required therapy, procedures, and assessments. In the event oprozomib or pomalidomide is permanently discontinued in Phase 3 only, | If dexamethasone dosing is permanently stopped due to toxicity in accordance with the dose modification guidelines described in Table 15, the subject should stay on oprozomib and/or pomalidomide, depending on the arm to which they are randomized, and continue to follow protocol required therapy, procedures, and assessments. Subjects may continue to take antiemetic doses of dexamethasone (4 mg) on days | |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | dexamethasone may be continued. Subjects may continue to take antiemetic doses of dexamethasone (4 mg) on days of oprozomib dosing at the investigator's discretion. | of oprozomib dosing, if tolerated, at the investigator's discretion. In the event oprozomib or pomalidomide is permanently discontinued in Phase 3 only, dexamethasone may be continued. Subjects may continue to take antiemetic doses of dexamethasone (4 mg) on days of oprozomib dosing at the investigator's discretion. | |
| Section 10.4.2.1.1<br>Hematologic<br>Toxicities | Additional guidance regarding hematologic toxicities and dosing actions is as follows: • To initiate a new cycle of pomalidomide, the neutrophil count must be at least 500 per mcL and the platelet count must be at least 50,000 per mcL. If toxicities occur after dose reductions to 1 mg, then discontinue pomalidomide. • Non-treatment-related events: If the toxicity resolves to ≤ Grade 1 or baseline and the toxicity is not treatment-related, oprozomib may be restarted at the same dose level. • If required by continued or recurrent toxicity, a second or third dose reduction may be permitted after discussion with the Onyx study medical monitor. No more than 3 dose reductions down to a minimum of 150 mg will be permitted for an individual subject on study and additional reductions will be managed by schedule change. If toxicity continues, oprozomib should be discontinued. | Additional guidance regarding hematologic toxicities and dosing actions is as follows: • To initiate a new cycle of pomalidomide, the neutrophil count must be at least 500 per mcL and the platelet count must be at least 50,000 per mcL. If toxicities <b>continue to</b> occur after dose reductions to <b>down</b> 1 mg, then discontinue pomalidomide. • Non-treatment-related events: If the toxicity resolves to ≤ Grade 1 or baseline and the toxicity is not treatment-related, oprozomib may be restarted at the same dose level • If required by continued or recurrent toxicity, a second or third dose reduction <b>of oprozomib</b> may be permitted after discussion with the Onyx study medical monitor. No more than 3 dose reductions down to a minimum of 150 mg will be permitted for an individual subject on study and additional reductions will be managed by schedule change. If toxicity continues, oprozomib should be discontinued. | Added text for clarity |
| Section 10.4.2.1.2<br>Nonhematologic<br>Toxicities – Table<br>14 | Symptom: Grade 4 GI Hemorrhage | Added the following to the table: Symptom: Grade 1 or 2 GI hemorrhage Findings: Assessed as oprozomib-related Oprozomib Dosing Action: • DELAY until Grade 0 • DECREASE one dose level for Grade 2 Pomalidomide Dosing Action: Full dose at | Additional text has been added to the dose modification table for nonhematologic toxicities and guidance to investigators to potentially reduce the risk for GI hemorrhage |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | physician discretion | |
| Section 10.4.2.1.2 | Additional guidance regarding nonhematologic | Changed to: Symptom: Grade <b>3 or</b> 4 GI Hemorrhage Additional guidance regarding nonhematologic | Added text for clarity and |
| Nonhematologic<br>Toxicities | <ul> <li>toxicities and dosing actions is as follows:</li> <li>Nontreatment-related events: If the toxicity resolves to ≤ Grade 1 or baseline and the toxicity is not treatment-related, oprozomib may be restarted at the same dose level.</li> </ul> | toxicities and dosing actions is as follows: Nontreatment-related events: If the toxicity resolves to ≤ Grade 1 or baseline and the toxicity is not treatment-related, oprozomib may be restarted at the same dose level | to reflect change in dose<br>modification guidelines for<br>GI hemorrhage |
| | If the subject tolerates the reduced dose for 1 cycle,<br>the subject's dose may be re-escalated to the dose<br>being taken prior to the dose reduction. | If the subject tolerates the reduced dose for 1 cycle,<br>the subject's dose may be re-escalated to the dose<br>being taken prior to the dose reduction | |
| | If required by continued or recurrent toxicity, a second or third dose reduction may be permitted after discussion with the Onyx study medical monitor. No more than 3 dose reductions down to a minimum of 150 mg will be permitted for an individual subject on study and additional reductions will be managed by schedule change. If toxicity continues, oprozomib should be discontinued. | If required by continued or recurrent toxicity, a second or third dose reduction of oprozomib may be permitted after discussion with the Onyx study medical monitor. No more than 3 dose reductions down to a minimum of 150 mg will be permitted for an individual subject on study and additional reductions will be managed by schedule change. If toxicity continues, oprozomib should be discontinued. | |
| | Subjects who develop Grade 4 GI hemorrhage<br>should not be rechallenged with oprozomib. Oprozomib should be permanently discontinued. | Subjects who develop Grade 3 or 4 GI hemorrhage<br>should not be rechallenged with oprozomib. Oprozomib should be permanently discontinued. Endoscopy should be strongly considered for any<br>subject with GI hemorrhage. | |
| Section 10.6.1.2<br>Antinausea and<br>Antiemetics | It is strongly recommended that subjects be premedicated with a 5-HT <sub>3</sub> inhibitor, such as ondansetron or granisetron, prior to administration of the first dose of oprozomib each day and throughout the day as needed to prevent nausea and vomiting. If nausea/vomiting at any grade persists, aprepitant is recommended if needed. Additional antiemetics may | It is strongly recommended that subjects be premedicated with a 5-HT <sub>3</sub> inhibitor, such as ondansetron or granisetron, prior to administration of the first dose of oprozomib each day and throughout the day as needed to prevent nausea and vomiting. If nausea/vomiting at any grade persists, aprepitant or fosaprepitant is recommended. Additional | Added "or fosaprepitant"<br>for consistency with other<br>oprozomib protocols to<br>allow IV administration of<br>this antiemetic if needed |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | be used if needed per investigator discretion. | antiemetics may be used per investigator discretion. | |
| Section 10.6.1.5<br>Acid-related<br>Medications | Lansoprazole or another oral proton-pump inhibitor is recommended for the duration of treatment to prevent peptic disease or other GI disorders. | Lansoprazole or another oral proton-pump inhibitor is recommended required (unless subject has intolerance or hypersensitivity) for the duration of treatment to prevent peptic disease or other GI toxicities. | Revised text for consistency<br>with other oprozomib<br>protocols and to potentially<br>reduce the risk for GI<br>hemorrhage |
| Section 10.6.1.7<br>Tumor Lysis<br>Syndrome | Tumor Lysis Syndrome Laboratory Abnormalities Subjects with laboratory abnormalities prior to dosing that are consistent with lysis of tumor cells (e.g., as defined by increases in at least 3 of the following 4 categories: [1] a 2-fold increase of lactate dehydrogenase above the ULN; [2] increases in serum creatinine, uric acid, or phosphorus > 50% over baseline; [3] potassium > 30% above the ULN; or [4] calcium decreases from baseline of > 20% in the absence of concomitant bisphosphonate therapy) (Sezer 2006) should not receive the scheduled dose prior to institution of the aforementioned preventive measures. | Tumor Lysis Syndrome Laboratory Abnormalities Subjects with laboratory abnormalities prior to dosing that are consistent with lysis of tumor cells (e.g., as defined by abnormalities increases in at least 3 of the following 4 categories: [1] a 2-fold increase of lactate dehydrogenase above the ULN; [2] increases in serum creatinine, uric acid, or phosphorus > 50% over baseline; [3] potassium > 30% above the ULN; or [4] calcium decreases from baseline of > 20% in the absence of concomitant bisphosphonate therapy) (Sezer 2006). Subjects should must not receive the scheduled dose prior to institution of the aforementioned preventive measures. | Revised as corrections and for consistency with other oprozomib protocols |
| Section 10.6.1.8<br>Orthostatic<br>Hypotension | | 10.6.1.8 Orthostatic Hypotension Orthostatic hypotension has been reported in subjects taking oprozomib. The following guidelines should be employed in the management of subjects exhibiting orthostatic hypotension. An etiology should be sought for the orthostatic hypotension to determine its cause is neurogenic, non-neurogenic or iatrogenic. Dose modifications should be taken in accordance with Table 13 and Table 14. • For those subjects with orthostatic hypotension who are taking antihypertensives, the subject's dosage and use of antihypertensive agents should be evaluated and reassessed on an ongoing basis while on study • Fluid intake should be assessed to confirm the | Added additional guidance for subjects who may experience orthostatic hypotension. |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | subject is getting appropriate hydration in accordance with protocol requirements of 6–8 eight ounce glasses of fluids in the 24–48 hours prior to dosing and on every day of oprozomib dosing • Fluid status should be repleted to normal levels in subjects with orthostatic hypotension | |
| | | If protocol requirements for oral intake of fluids are already being met, additional measures should be taken to increase blood pressure per investigator discretion, such as increased oral intake, florinef or midodrine, others depending on the etiology. Holding the dose and dose reduction upon resolution may be a consideration. | |
| | | Ongoing monitoring of fluid status is warranted<br>and should be managed per investigator<br>discretion | |
| | | • In addition, vital signs monitoring may be extended beyond the time periods specified in the Schedules of Assessments (Appendices A1, A2, B1, B2, C1, and C2) | |
| Section 10.6.2<br>Optional and<br>Allowed<br>Concomitant<br>Medications | Additional antiemetics that are not required may be used as well as antidiarrheal agents as necessary | Additional antiemetics that are not required may be used as well as antidiarrheal agents, and/or laxatives as necessary | Removed extraneous text,<br>and added "and/or<br>laxatives" for consistency<br>with other oprozomib<br>protocols |
| Section 10.6.3<br>Excluded<br>Concomitant<br>Medications | Other antimyeloma agents are not permitted prior to the subject developing confirmed progressive disease. | Other antimyeloma <b>or investigational</b> agents are not permitted prior to the subject developing confirmed progressive disease. | Added text for clarity |
| Section 11.1.1 Vital<br>Signs | Vital signs will include measurement of orthostatic blood pressure, pulse rate, and temperature. Subjects should lie down for 5 minutes and then have blood | All vital signs assessments will include measurement of orthostatic blood pressure, pulse rate, respiration rate, and temperature. Subjects should lie down for | Revised text for consistency with other oprozomib protocols |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | pressure and pulse measured. This should be followed by having the subject stand and the blood pressure and pulse should be repeated at 1 and 3 minutes. Any drop of 20 mmHg systolic, 10 mmHg diastolic or lightheadedness/dizziness between supine and standing blood pressures would indicate orthostatic hypotension. Usually an increase in pulse of 10 beats/min is associated with but not required for identification of orthostatic hypotension. Subject's dosage and use of antihypertensive agents in the setting of orthostatic hypotension should be evaluated and reassessed on an ongoing basis while on study. Fluid intake should be assessed to confirm the subject is acting in accordance with protocol requirements. Reeducation should occur if subject is not adhering to protocol requirements. Fluid status should be repleted to normal levels. If protocol requirements for oral intake of fluids are already being met, additional measure should be taken to increase volume status per investigator discretion. Ongoing monitoring of fluid status is warranted and should also be managed per investigator discretion. In addition, vital signs monitoring may be extended beyond the time periods specified in the Schedules of Assessments (Appendices A1, A2, B1, B2, C1, and C2) as needed. | 5 minutes and then have blood pressure and pulse measured consistently in either arm. Following the supine blood pressure/pulse reading, This should be followed by having the subject should stand and the blood pressure and pulse should be repeated after at 1 and 3 minutes. Any drop of 20 mmHg systolic, 10 mmHg diastolic or lightheadedness/dizziness between supine and standing blood pressures would indicate orthostatic hypotension. Usually an increase in pulse of 10 beats/min is associated with but not required for identification of orthostatic hypotension. For time points where PK and vital signs are to be done together, vital signs should be obtained first as the act of phlebotomy may impact vital sign measurement results. Subject's dosage and use of antihypertensive agents in the setting of orthostatic hypotension should be evaluated and reassessed on an ongoing basis while on study. Fluid intake should be assessed to confirm the subject is acting in accordance with protocol requirements. Re-education should occur if subject is not adhering to protocol requirements. Fluid status should be repleted to normal levels. If protocol requirements for oral intake of fluids are already being met, additional measure should be taken to increase volume status per investigator discretion. Ongoing monitoring of fluid status is warranted and should also be managed per investigator discretion. In addition, vital signs monitoring may be extended beyond the time periods specified in the Schedules of Assessments (Appendices A1, A2, B1, B2, C1, and C2) as needed. | |
| Section 11.3<br>Disease Response<br>Assessments | Disease response and progression assessments include: Serum protein electrophoresis (SPEP) Urine protein electrophoresis (UPEP) Serum immunofixation, serum free light chain | Disease response and progression assessments include: Serum protein electrophoresis (SPEP) Urine protein electrophoresis (UPEP) Serum immunofixation, serum free light chain | Separated bullet points for<br>clarity; revised text to<br>reflect updated Schedules<br>of Assessment |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | (SFLC) | (SFLC) | |
| | Urine immunofixation | Urine immunofixation | |
| | Serum calcium, bone marrow sample as<br>clinically indicated to confirm CR | <ul> <li>Serum calcium, bone marrow sample as<br/>elinically indicated to confirm CR</li> </ul> | |
| | Radiographic assessments including<br>plasmacytoma evaluation if baseline<br>assessments were positive and as clinically<br>indicated per the response criteria | Bone marrow sample as clinically indicated to confirm CR Radiographic assessments including plasmacytoma evaluation if baseline | |
| | <ul> <li>Skeletal survey if baseline assessments were<br/>positive and as clinically indicated per the<br/>response criteria</li> </ul> | assessments were positive and as clinically indicated per the response criteria | |
| | Serum protein electrophoresis and immunofixation assessments will be conducted according to the | <ul> <li>Skeletal survey if baseline assessments were<br/>positive and as clinically indicated per the<br/>response criteria</li> </ul> | |
| | schedule outlined in Appendices A1, A2, B1, B2, C1, and C2, Schedule of Assessments. Immunofixation will only be required after Screening and End of Study Treatment, if results of the previous SPEP are zero/undetectable. | Serum protein electrophoresis and immunofixation assessments will be conducted according to the schedule outlined in Appendices A1, A2, B1, B2, C1, and C2, Schedule of Assessments. Immunofixation will only be required after Screening, Baseline (Day -7 | |
| | Urine protein electrophoresis and immunofixation will be performed on a 24-hour urine specimen collected | to 1), and End of Study Treatment, if results of the previous SPEP are zero/undetectable. | |
| | from all subjects during the Screening period and at the End of Study Treatment visit. The UPEP with 24-hour urine collection will be conducted according to the schedule outlined in Appendices A1, A2, B1, B2, C1, | Urine protein electrophoresis and immunofixation will be performed on a 24-hour urine specimen collected from all subjects during the Screening period, <b>Baseline</b> | |
| | and C2, Schedule of Assessments, and is required: 1) only if Screening UPEP was ≥ 200 mg/24 hours, and 2) to confirm a disease response or disease | (Day -7 to 1), and at the End of Study Treatment visit. The UPEP with 24-hour urine collection will be conducted according to the schedule outlined in Appendices A1, A2, B1, B2, C1, and C2, Schedule of | |
| | progression. If the Screening UPEP was negative, spot<br>urine is required at each time point. If positive for<br>paraprotein, a 24-hour urine collection with UPEP | Assessments, and is required: 1) only if Screening Baseline UPEP was ≥ 200 mg/24 hours, and 2) to | |
| | must be done at the next assessment and at each subsequent assessment unless the UPEP shows an absence of paraprotein. | confirm a disease response or disease progression. If<br>the Screening-Baseline UPEP was negative, spot urine<br>is required at each time point. If positive for<br>paraprotein, a 24-hour urine collection with UPEP must | |
| | Serum free light chain assay and kappa:lambda $(K/\lambda)$ ratio will be conducted according to the schedule | be done at the next assessment and at each subsequent assessment unless the UPEP shows an absence of | |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | outlined in the Schedule of Assessments, Appendices A1, A2, B1, B2, C1, and C2. Only in subjects without measurable serum and urine M-protein levels (serum M-protein < 0.5 g/dL or urine M-protein < 200 mg/24 hours) at Screening will SFLC assays be used to determine eligibility and response. In subjects with measurable SPEP and/or UPEP, SFLC may be used in conjunction with those assessments to determine response per disease response criteria but only SPEP and/or UPEP will be used to determine eligibility. | paraprotein. Serum free light chain assay and kappa:lambda (K/λ) ratio will be conducted according to the schedule outlined in the Schedule of Assessments, Appendices A1, A2, B1, B2, C1, and C2. Only in subjects without measurable serum and urine M-protein levels (serum M-protein < 0.5 g/dL or urine M-protein < 200 mg/24 hours) at Screening Baseline will SFLC assays be used to determine eligibility and response. In subjects with measurable SPEP and/or UPEP, SFLC may be used in conjunction with those assessments to determine response per disease response criteria but only SPEP and/or UPEP will be used to determine eligibility. | |
| Section 11.3 Disease Response Assessments | All response categories (CR, sCR, VGPR, PR, MR, PD) require 2 consecutive assessments made at any time before the institution of any new therapy, as well as no known evidence of progressive or new bone lesions. All subjects will be followed until disease progression (confirmed by 2 consecutive measurements that are also verified by the Onyx medical monitor prior to treatment discontinuation), unacceptable toxicity, or withdrawal of consent, whichever occurs first. Disease progression will be determined using the IMWG-URC (Appendices A1, A2, B1, B2, C1, and C2). Serum M component increases of ≥ 1.0 g/dL are sufficient to define progression if the starting component is ≥ 0.5 g/dL according to these criteria. However, it is understood from these criteria that a single measurement is adequate in cases of clear increased bone marrow plasma cell percentage, development of new or worsened bone lesions from a skeletal survey, or development of new or worsened soft tissue plasmacytomas. | All response categories (CR, sCR, VGPR, PR, MR, PD) require 2 consecutive assessments made at any time before the institution of any new therapy, as well as no known evidence of progressive or new bone lesions. All subjects will be followed until disease progression (confirmed by 2 consecutive measurements that are also verified by the Onyx medical monitor prior to treatment discontinuation), unacceptable toxicity, or withdrawal of consent, whichever occurs first. Disease progression will be determined and confirmed with the medical monitor by two consecutive assessments using the IMWG-URC (Appendices A1, A2, B1, B2, C1, and C2). Serum M component increases of ≥ 1.0 g/dL are sufficient to define progression if the starting component is ≥ 0.5 g/dL according to these criteria. However, it is understood from these criteria that a single measurement is adequate in cases of clear increased bone marrow plasma cell percentage, development of new or worsened bone lesions from a skeletal survey, or development of new or worsened soft tissue | Revised text for clarification of the requirements for the assessment of disease disease progression |



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Pag


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | plasmacytomas. | |
| Section 11.4.3<br>Genomic<br>Measurements | Whole genome sequencing (WGS), whole exome sequencing (WES), and/or whole transcriptome sequencing will be conducted on isolated tumor (CD138 <sup>+</sup> ) cells from bone marrow samples taken at Screening and disease progression. In addition, WGS or WES will be performed on a normal tissue sample (e.g., saliva, CD3 <sup>+</sup> T-cells, or isolated PBMCs) in order to determine the presence of somatic mutations in tumor cell samples. Data will be analyzed to examine specific hypotheses about whether drug response is related to alterations in genes regulated by or involved in activation of nuclear factor kappa light chain enhancer of activated B cell (NF-kB) transcription factors as well as genes involved in immunoglobulin production and plasma cell protein homeostasis. These data will also be used to derive new hypotheses about mechanisms of drug response, resistance, and safety. | Whole genome sequencing (WGS), whole exome sequencing (WES), and/or whole transcriptome sequencing, and/or other methods of nucleic acid quantification, will be conducted on isolated tumor (CD138°) cells from bone marrow samples taken at Screening and disease progression. In addition, WGS or WES will be performed on a normal tissue sample (e.g., saliva or peripheral blood, CD3° T-cells, or isolated PBMCs) in order to determine the presence of somatic mutations in tumor cell samples. Data will be analyzed to examine specific hypotheses about whether drug response is related to alterations in genes regulated by or involved in activation of nuclear factor kappa light chain enhancer of activated B cell (NF-kB) transcription factors as well as genes involved in immunoglobulin production and plasma cell protein homeostasis. Immunoglobulin levels in tumor cells will be quantified by enzyme-linked immunosorbent assay (ELISA) and/or other protein quantification methods. These data will also be used to derive new hypotheses about mechanisms of drug response, resistance, and safety. | Added text for clarity and consistency with other oprozomib protocols |
| Section 11.5 Quality | - | Added subsection: | Added subsection to further |
| of Life Assessments | | 11.5 Patient-Reported Outcomes Assessments | clarify the quality of life assessments to be |
| | | Beginning with Cycle 1, HRQoL/PRO assessments are to be completed at the beginning of every cycle prior to drug administration through End of Study Treatment/Early Discontinuation visit during the dose-expansion portion of the trial, and at the beginning of every cycle prior to drug administration through End of Study Treatment/Early Discontinuation visit and then every 12 weeks during the long-term follow-up in the Phase 3 portion of the study. The HRQoL/PRO | performed in the<br>dose-expansion and Phase 3<br>portions of the study |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | assessments include: BPI-SF (see Appendix N for a sample Brief Pain Inventory – Short Form) | |
| | | EORTC QLQ-C30 (Appendix E) EORTC QLQ MV20 (Appendix E) | |
| | | EORTC QLQ-MY20 (Appendix E) Neurotoxicity subscale of the FACT/GOG-Ntx4 (Appendix F) | |
| | | • EQ-5D-5L (Appendix G) | |
| Section 12 Study<br>and Study<br>Treatment<br>Discontinuation | An individual subject who discontinues study treatment for PD is considered to have completed the study after the safety follow-up visit | An individual subject who discontinues study treatment for PD will be followed for OS in long-term follow-up is considered to have completed the study after the safety follow-up visit. | Revised text for clarity |
| Section 12.1 Study<br>Treatment<br>Discontinuation | Subjects who discontinue from study treatment will be monitored for AEs for 30 days after the last dose of oprozomib or before the start of subsequent anticancer treatment (whichever occurs first). Treatment discontinuation due to progression should be recorded on the Treatment/Discontinuation eCRF as "Disease Progression." Onyx Therapeutics, or designee must be notified within 24 hours if a subject is withdrawn from treatment for any reason (i.e., disease progression, toxicity, etc.). Disease progression must be confirmed by the medical monitor before any subject is discontinued from study treatment. | Subjects who discontinue from study treatment will be monitored for AEs for 30 days after the last dose of oprozomib or immediately before the start of subsequent anticancer treatment (whichever occurs first). Treatment discontinuation due to progression should be recorded on the Study Drug Completion Treatment/Discontinuation eCRF as "Disease Progression." Onyx Therapeutics, or designee must be notified within 24 hours if a subject is withdrawn from treatment for any reason (i.e., disease progression, toxicity, etc.). Disease progression with 2 consecutive disease assessments must be confirmed by the medical monitor before any subject is discontinued from study treatment. | Corrected text and revised text for clarification of the requirements for the duration of AE collection |
| Section 12.2 Study<br>Discontinuation | The sponsor, Onyx Therapeutics, Inc., may elect to discontinue the study at any time. Each subject will be followed until death or study closure. The reason for | The sponsor, Onyx Therapeutics, Inc., may elect to discontinue the study at any time. Each subject will be followed until death or study closure. The reason for | Deleted text as it was in the inappropritate location in the protocol |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | discontinuation from the study will be documented on the eCRF. | discontinuation from the study will be documented on the eCRF. | |
| Section 12 Study and Study Treatment Discontinuation Section 12.3 Long- Term Follow-up | Long-Term Follow-up After completion of the post treatment visit, subjects will be followed for disease and survival status by telephone contact or other method every 3 months in addition to disease assessments. Long-term follow-up will continue until the subject has withdrawn consent for further participation, is lost to follow-up, has died, or the sponsor makes a decision to close the study. For any subject who is lost to follow-up, the study site will attempt to ascertain survival information via public database search. Informed consent to obtain these data will be obtained from subjects at the time of enrollment. | Long-Term Follow-up After completion of the post treatment End of Study Treatment visit, subjects will be followed for disease progression, OS, and quality of life (QOL). and survival status by telephone contact or other method every 3 months in addition to disease assessments. Subjects will be followed based on their disease progression status at End of Study Treatment. Progression and Overall Survival • For subjects who have not progressed at end of study treatment, disease response assessments will be performed every 4 weeks through 18 months on study, and then every 8 weeks thereafter, beginning with Month 20, until progression or initiation of next therapy • Subjects who progressed at end of study treatment or long-term follow-up will be followed for survival status approximately every 3 months, or as needed Quality of Life For Phase 3 only, in long-term follow-up, QOL questionnaires will be collected from subjects (regardless of disease status) every 12 weeks. Long-term follow-up will continue until the subject has withdrawn consent for further participation, is lost to follow-up, has died, or the sponsor makes a decision to close the study. For any subject who is lost to follow- up, the study site will attempt to ascertain survival information via public database search. Informed consent to obtain these data will be obtained from subjects at the time of enrollment. | Added "on study" and additional text for clarity on the long-term follow-up based on disease progression status |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 12.4 Study<br>Termination | Onyx has the right to terminate this study or a study site from participating in a study at any time. | Onyx has the right to terminate this study, <b>either schedule</b> , or a study site from participating in a study at any time | Added text to provide flexibility in terminating either schedule |
| Section 14.2<br>Analysis of the<br>Conduct of the<br>Study | Enrollment, subject disposition, study treatment administration, and discontinuation from the study will be summarized. Eligibility exceptions and major protocol deviations will be summarized. | Enrollment, subject disposition, study treatment administration, and discontinuation from the study will be summarized. Eligibility exceptions and major important protocol deviations will be summarized. | Revised to match ICH E3<br>Guidance |
| Section 14.3 Data<br>Monitoring<br>Committee | | terim analyses are planned for the PFS primary endpoint. | Revised text for clarity |
| | An interim analysis of OS,—the key secondary endpoint Details of the monitoring plan for OS are described in | | |
| | Overall survival may also be evaluated without penalty by risk during the course of the study. Details of the monite the objective of this evaluation is not to declare OS of analyses of OS, alpha level will not be adjusted for the | | |
| | An independent DMC will be convened for this the Pha capacity to the sponsor with respect to safeguarding the efficacy (OS secondary only) data, and for monitoring the of the study, the DMC may also formulate recommendat of subjects, management of subjects, improving adherent management and quality control. | | |
| | The DMC will meet to review safety data on a periodic between the initial meeting should occur within 3 months. The initial meeting should occur within 3 months Phase 3 part portion of the study. Unplanned safety review sponsor or the DMC Chair if additional review of safety and the part of th | | |
| | The membership criteria and other details of the DMC w | rill be described in the DMC Charter. | |
| Section 14.4<br>Analysis of<br>Treatment Group<br>Comparability | Descriptive statistics will be used to summarize baseline subject characteristics, treatment administration, efficacy, and safety outcomes. Summaries of discrete data will include number of subjects and incidence as a frequency and as a percentage. Summaries of continuous data will include | Descriptive statistics will be used to summarize baseline subject characteristics, treatment administration, efficacy, and safety outcomes. Summaries of discrete data will include number of subjects and incidence as a frequency and as a percentage. Summaries of continuous data will include | Corrected text |



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | mean, standard deviation, median, minimum, maximum, and sample size. | mean, standard deviation, median, minimum, maximum, and sample size. | |
| Section 14.4.1<br>Treatment Exposure<br>and Medication<br>Compliance | The average relative dose intensity for each treatment group will be calculated by summarizing the average relative dose intensity for individual subjects. These results will be provided to determine the presence of any major differences between the treatment groups for the planned versus actual dose and schedule of pomalidomide and dexamethasone administered. For each subject, a compliance measure will be calculated based on the information provided in the CRFs. Compliance will be defined as the percentage of the actual number of days with treatment intake over the expected number of days with treatment intake. Summary statistics will be provided on percent compliance by treatment group. | The average relative dose intensity for each treatment group will be calculated by summarizing the average relative dose intensity for individual subjects. These The results for pomalidomide and dexamethasone will be provided to determine the presence of any major differences between the treatment groups for the planned versus actual dose and schedule of pomalidomide and dexamethasone administered these two (2) study medications. For each subject, a compliance measure will be calculated based on the information provided in the CRFs. Compliance will be defined as the percentage of the actual number of days with treatment intake over the expected number of days with treatment intake. Summary statistics will be provided on percent compliance by treatment group. | Revised text for clarity and as corrections |
| Section 14.5.1.1<br>Safety Population | All subjects receiving any amount of study treatment (oprozomib, pomalidomide, or dexamethasone) will be included in safety analyses. | All subjects receiving any amount of study treatment (oprozomib, <b>placebo</b> , pomalidomide, or dexamethasone) will be included in safety analyses. | Corrected text by adding "placebo" |
| Section 14.5.2<br>Efficacy Analyses | | | Revised for clarity and as corrections |




| Section(s) | | Changed from | Changed | Changed to |
|---|---|---|---|---|
| | ana trea Prin The to the IMV algorians of the prin For | ess otherwise noted, all primary and secondalyzed according to the ITT analysis principal truent assigned at randomization. Mary Efficacy Analysis Primary efficacy endpoint for the Phase 3 pare earlier of disease progression or death duw WG-URC (Appendix D). Response and disease progression or death duw WG-URC (Appendix D). Response and disease doutcomes. The PFS outcomes assessed mary analysis of PFS. Purposes of calculating PFS, the start date for duration of PFS will be right-censored according to the property of the proposed according to the primary analysis of PFS. | e (Section 14.5.1), i.e., subjects will be grant or to find the study is PFS, defined as the set of any cause. Disease progression will be asse progression will be determined using tors. The primary analysis of PFS will be d by the investigators will serve as a support of PD is the date at which progression is f | time from randomization to determined using the a validated computer based on ORCA-pritive analysis of the first observed. |
| | | le 18 Date of Progression or Censoring for I | - | |
| | | Situation | Date of Progression or Censoring | Outcome |
| | | No baseline disease assessments | Date of randomization | Censored |
| | | No postbaseline disease assessments and alive | Date of randomization + 1 day | Censored |
| | | New anticancer treatment started before documentation of PD or death | Date of last disease assessment prior to start of a new anticancer treatment | Censored |
| | | Death or PD immediately after more<br>than 1 consecutively missed disease<br>assessment visit | Date of last disease assessment visit without documentation of PD that is before the first missed visit | Censored |
| | | Alive and without PD documentation | Date of last disease assessment | Censored |
| | | Death or PD between planned disease assessments | Date of death or first disease assessment showing PD, whichever occurs first | Progressed |
| | | Death before first disease assessment | Date of death | Progressed |
| | | PD = progressive disease. | | <u> </u> |
| | The | primary analysis of PFS will be conducted | after approximately when 157 PFS events | s have occurred. |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | The hypothesis to be tested is as given below: | | |
| | H <sub>u</sub> : PFS (Pomd) | = PFS (OPomd) | |
| | H <sub>a</sub> : PFS (Pomd) | < PFS (OPomd) | |
| | The primary inferential comparison between treatment gratest at an overall 0.025 (1-sided) significance level using a | | |
| | • Age: < 75 years versus ≥ 75 years | | |
| | <ul> <li>Number of prior therapies: 2 versus 3 or more</li> </ul> | | |
| | Carfilzomib status: carfilzomib-naïve/sensitive | versus carfilzomib-sensitive refractory | |
| | The hazard ratio between the 2 treatment arms will be est model. | imated using a stratified Cox proportional hazards | |
| | The distribution of PFS times, including medians, will be method. Median PFS will be estimated for each treatmen Kaplan-Meier estimates. The 95% CIs for median and of method of Brookmeyer and Crowley (1982). Duration o Kaplan-Meier method of Schemper (1996). | t group from the 50th percentile of the corresponding ther quartiles of PFS will be constructed using the | |
| | Secondary Efficacy Analyses | | |
| | At the time of the primary PFS analysis, the first of 2 inte endpoint of OS will also be conducted. Overall survival it to any cause. Subjects who are alive or lost to follow-up as of the data analysis cutoff date will be right the subject's last known date alive of last contact or data. Determination of the required number of events and timin randomized to treatment with Pomd plus placebo versus tupon the following assumptions: | s defined as the time from randomization to death due censored. The censoring date will be determined from analysis cutoff date, whichever event occurs first. | |
| | The risk of death in subjects randomized to OPomd is 32% the target hazard ratio is 0.68 | | |
| | The hypothesis test of interest is: | | |
| | H <sub>o</sub> : OS (Pomd) | = OS (OPomd) | |
| | H <sub>a</sub> : OS (Pomd) | < OS (OPomd) | |
| | Inference will be made using the log-rank testing procedu | re. | |
| | <ul> <li>1-sided 0.025 level of significance</li> </ul> | | |
| | • 75% power | | |
| | • 1 interim and 1 final analysis (30%, 100%) | | |




| | Changed from | | | Changed to | |
|---|---|---|---|---|---|
| • mOS (Pe | omd) = 16 months | and mOS (OPomd) | = 23.5 months | | |
| <ul> <li>Duration</li> </ul> | of OS is exponent | ially distributed | | | |
| • 10% Los | st to Follow-Up at ( | 60 months | | | |
| total of 211 death<br>for OPomd versu<br>exponential distr<br>Pomd arms, resp<br>study of pomalide | s will provide 75% s Pomd ( <del>16 vs. 23.5</del> ribution, 23.5 mon pectively. The assumide/dexamethasc | power to detect a 25 months HR = 0.6 ths versus 16 mortimed median OS of one (Jagannath 201 | 32% decrease in the state of th | | ne OPomd and<br>ed on a Phase 2<br>ssuming 10% lost |
| anticipated to occ<br>total number of d<br>of OS will be per<br>include an upper<br>Demets alpha spe<br>interim analysis o | eur approximately 1<br>eath events is expect<br>formed using an O'<br>boundary for benef | 4 months after the cted at the time of the Brien-Fleming ground to constructed using roach will be used to the projected in | first subject is ran-<br>the primary PFS at<br>our sequential mon<br>g a false-positive e<br>to adjust the O'Br<br>iformation time. | domized. Approximalysis. The interimitoring plan. The m | and final analysis<br>nonitoring plan will<br>Table 19). The Lan- |
| Information<br>Fraction | Death Events | Study Month | Boundary<br>(Reject H <sub>o</sub> ) | 1-Sided<br>Significance<br>Level | Alpha Spent |
| 30% | 63 | 14 | 3.929 | 0.000042 | 0.000 |
| | | _ | | | |




| Section(s) | Changed from Changed to | Rationale |
|---|---|---|
| | at the 1-sided 0.025 level of significance, then testing of the aforementioned secondary endpoints w a sequential step-down manner. The nominal level of significance at interim analysis will be as presim Table 19, consistent with the monitoring plan for the key secondary endpoint of OS. Testing of selected secondary efficacy endpoints will continue, provided the null hypothesis for each tested endpoint is rejected. Otherwise, no further testing will be done. The sequential order in which efficacy endpoints will be tested is as follows: | ch previously |
| | PFS | |
| | • OS | |
| | • ORR | |
| | • CBR | |
| | Time to Improvement in renal function | |
| | Time to Improvement in hemoglobin | |
| | Change from baseline over time in QLQ-C30 global health scale | |
| | Change from baseline over time in QLQ-MY20 disease symptoms subscale | |
| | Overall response rate will be estimated based on the proportion of subjects in each treatment group sCR, CR, VGPR, or PR as their best response across the entire treatment duration. The inferential of between treatment groups for this endpoint will be made using the Cochran-Mantel Haenszel chi-sq stratified by the randomization stratification factors. Approximate 95% CIs will be calculated by the for the true ORR. An estimate of the common odds ratio for the odds of overall response will be promeasure of the relative treatment effect. The odds ratio (and 95% CI) will be estimated using the Mantel-Haenszel method. The Pomd plus placebo arm group will serve as the reference treatment calculation of the odds ratio. Homogeneity of the odds ratio across randomization strata will be exasting frame level of 0.05 by the Breslow-Day test. | comparison quare test, eatment group rovided as a group in the |
| | Clinical benefit rate (CBR) will be estimated based on the proportion of subjects in each group who CR, VGPR, PR, or MR and will be analyzed in the same manner as described previously for ORR. | achieve sCR, |
| | Improvement in renal function is defined as an increase in glomerular filtration rate (GFR) of at least $\geq 10 \text{ mL/min}$ . | <del>st</del> |
| | Improvement in hemoglobin is defined as an increase of $\geq 2g/dL$ . | |
| | Inferences for time to Incidence of improvement in renal function and improvement in hemoglobic those for the other time to event outcomes of PFS and OS, be analyzed in the same manner as depreviously for ORR. | |
| | The Kaplan-Meier methodology Duration of response and DOCB will also be used for estimating DOR. be summarized for each treatment group by Kaplan-Meier method; however no formal | |


Product: Oprozomib Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | comparisons of DOR will be made, as responders constit | ute a nonrandom subset of the ITT population | |
| Section 14.5.3<br>Safety Analyses | The safety population will be used in all safety analyses of presented separately for Part 1 and Part 2 of the study. Part 1: Phase 1b Dose Escalation and Dose-Expansion P | • • | Revised for clarity and as corrections |
| | cohorts. Safety will be assessed through summaries of D | For the Phase 1b portion of the study, safety data will be summarized for each cohort and for the pooled cohorts. Safety will be assessed through summaries of DLTs, AEs, changes in laboratory test results, ECGs, vital signs, and oprozomib, pomalidomide, and dexamethasone exposure. All AE data collected will be listed by study site, cohort, subject number, and cycle day. | |
| | Part 2: Randomized Phase 3 Portion of the Study For the Phase 3 portion of the study, safety data will be s received. | e Phase 3 portion of the study, safety data will be summarized grouped according to treatment actually | |
| | For both Part 1 and Part 2 of the study, safety analyses will include all AEs occurring on or after treatment on Cycle 1 Day 1. Summaries of AEs will include number and percentage of subjects experiencing 1 or more AEs, relationship to study drug, and severity. Treatment-emergent AEs are defined as AEs that start on or after the first day study treatment is administered and within 30 days of the last administration of study treatment or befor start of subsequent anticancer treatment (whichever occurs first). Treatment-emergent AEs Adverse events-wi be summarized by the number and percentage of subjects who experienced the event, according to system organ class and preferred term. A subject experiencing multiple instances of the same AE will be counted once within each system organ class and similarly counted once within each preferred term. These conventions will be appropriately modified to calculate AE incidence rates separately for each cycle that study therapy is administered. Adverse event incidence rates may also be calculated based on other measures of subject exposure (e.g., total number of treatment cycles administered). Adverse events will also be summarized by NCI-CTCAE Version 4.03 severity grade and by relationship to each study drug. For AEs not adequately addressed by NCI-CTCAE version 4.03, the severity grading described in Table 17 may be used. Additional summaries may also be provided for SAEs and events resulting in the permanent discontinuation of therapy. All AEs will be | | |
| | Incidence, severity, and duration of specific signs and syneurotoxicities will be assessed. The appropriate terms is performed to provide a subject incidence of those with the | n these categories will be codified and analyses<br>be relevant events. | |
| | Laboratory parameters will be summarized using descrip select laboratory parameters relative to baseline, chang significant abnormalities. The changes in hematology, cl summarized descriptively for each scheduled and unsche calculated relative to the values collected at baseline and The incidence of Grade 3 and 4 hematological toxicities | ges from baseline, and data listings of clinically hemistry, and other laboratory values will be duled protocol assessment time point. Changes will be on the first day of each cycle of treatment. | |



Product: Oprozomib Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | will be provided by treatment cycle and across all treatm RBC) and/or growth factor support will be summarized Similar analyses will be done for selected chemistry test listings of all laboratory data collected during the study limits will be identified in the subject listings and will in Vital sign results (systolic and diastolic blood pressure, p summarized descriptively for each scheduled and unsche relative to the assessments at baseline and on the first day | reported in the Concomitant Medications section. s (including liver and renal function tests). Subject will be presented. Laboratory values outside normal clude flags for high and low values. bulse, respiration, and temperature) and ECGs will be reduled protocol time point. Changes will be calculated | |
| Section 14.5.4<br>Subgroup Analyses<br>and Effects of<br>Baseline Factors | To determine whether the treatment effect is consistent a (or odds ratio) for treatment group (with 95% CI) will be efficacy endpoints and plotted within each of the followi sample size in the subgroups of interest: | provided for the primary and selected secondary | Revised text for clarity,<br>including the potential<br>inclusion of subjects with<br>prior carfilzomib exposure |
| | Refractory status: primary refractory versus rel | apsed, and refractory versus bortezomib intolerant | in the study |
| | • Number of prior therapies: 2 versus 3 or more ( | (stratification factor) | |
| | • Age (< 75 years versus ≥ 75 years) (stratificatio | n factor) | |
| | Prior carfilzomib (naïve/sensitive versus sensiti | ve refractory) (stratification factor) | |
| | Refractory status: Primary refractory versus r<br>bortezomib-intolerant | elapsed-refractory, <del>and refractory</del> versus | |
| | Refractory to lenalidomide | | |
| | Refractory to bortezomib (refractory to lenalid) | lomide and bortezomib) | |
| | Double refractory | | |
| | | ard-risk group. The high-risk group consists of the 17p. The standard-risk group consists of all other | |
| | <ul> <li>No prior transplant versus prior transplant</li> </ul> | | |
| | <ul> <li>Bone marrow infiltration by plasma cells ≤ 50%</li> </ul> | versus > 50% at baseline | |
| | • Renal function ≤ 60 mL/min versus > 60 mL/m | in at baseline | |
| | • Age (< 65 years versus ≥ 65 years) | | |
| | • Race (Caucasian versus all others) | | |
| | <ul> <li>Sex (male versus female)</li> </ul> | | |
| | Study center | | |



Product: Oprozomib Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 14.7<br>Determination of<br>Sample Size | The CSRC will review the data and provide guidance in selection of the RP3D. Therefore the RP3D may differ from the MTD. | The CSRC will review the data and provide guidance in selection of the RP3D. Therefore the RP3D may differ from the MTD, <b>but will not be higher than the MTD.</b> | Added text for clarity and for consistency within the protocol |
| Section 14.7 | Part 2: Randomized Phase 3 Portion of the Study | | Revised text for clarity |
| Determination of Sample Size | The estimated sample size For the Phase 3 portion of the disease progression events) distributions for subjects tree OPomd based upon the log-rank test statistic. It is assum will be 45.7% lower than for subjects randomized to Pon order to have 95% power with 157 PFS events are requ (HR = 0.543) with 95% power and a 1-sided $\alpha$ = 0.025 difference in PFS risk versus a 45.7% reduction in risk b Enrollment of 270 subjects (2:1 OPomd versus Pomd, re events in approximately 14 months, assuming an enrollm drop-out rate at 18 months, and a median PFS of 3.8 and Therefore, a the total planned enrollment of will be app. | ted with Pomd plus placebo versus those treated with ned that the PFS risk for subjects randomized to OPomd and. Therefore, the target HR of interest is 0.543. In ired to detect a 45.7% reduction in the risk of PFS level of significance level of 0.025. for testing no etween the 2 treatments, 157 PFS events are required spectively) is consistent with reaching the required 157 tent rate of approximately 22 subjects per month, a 5% 7 months for Pomd and OPomd, respectively. | |
| Section 16<br>References | _ | Cleeland CS. The measurement of pain from metastatic bone disease: capturing the patient's experience. Clin Cancer Res. 2006;12(20 Pt 2):6236s–42s. Oken MM, Creech RH, Tormey DC, et al. Toxicity and Response Criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982;5(6):649–55. Onyx Pharmaceuticals. Kyprolis (carfilzomib) for Injection full prescribing information. 2012. | Added references |
| Appendix A1, A2,<br>B1, B2, C1, and C2 | Appendices updated per body of protocol. See updated appendices for further details. | | Removed and added "X"s in the Schedule of Assessment tables and revised text of footnotes for clarity and consistency with the protocol body text |
| Appendix D | Response Criteria for Multiple Myeloma | | Revised text for minor corrections |




**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Appendix M | _ | Added: Appendix M ACTG Brief Peripheral Neuropathy Screening Tool | Added ACTG Brief<br>Peripheral Neuropathy<br>Screening Tool as<br>Appendix M |
| Appendix N | _ | Added: Appendix N Sample Brief Pain Inventory – Short Form | Added Sample Brief Pain<br>Inventory – Short Form as<br>Appendix N |



Supplemental Clinical Study Report: 20130411


**Document Title:** 

protocol-OPZ007-a2.docx

**Workflow Number:** 

14118445

UserName:

Title: Senior Vice President, Development

Date: Tuesday, 08 July 2014, 07:31 PM Pacific Daylight Time

Meaning: I have reviewed and approved this document.

Superseded

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


#### APPENDIX Q **SUMMARY OF CHANGES IN STUDY OPZ007 AMENDMENT 3.0**

Study OPZ007 was amended to include the following:

- The Phase 3 portion of the study was never executed; therefore, all text pertaining to the Phase 3 portion of the study was removed.
- Study visits are less frequent with data collection (eg, labs) being pared down to instances of clinical need or adverse event reporting for subjects on active treatment. This amendment is based on the completion of the primary analysis of the study and abbreviated clinical study report.

In addition, administrative updates, editorial changes, and style and formatting revisions have been made to improve clarity and consistency throughout the document. Changes noted in specific sections were also made in the protocol synopsis and elsewhere in the document, as applicable. Significant changes are presented in the table below. Detailed changed text is displayed for first major occurrence only. All affected sections are noted in the "Section(s)" column. Text that has been deleted is presented in strikethrough format. Added text is presented in bold format.

Approved




**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Global | Phase 1b/3 | Phase 1b/3 | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Global | International Conference on Harmonisation (ICH) | International Council for Harmonisation (ICH) | Change in regulatory body name |
| Global | Onyx Drug Safety | Amgen Global Patient Safety | New<br>sponsor<br>protocol<br>standard<br>operating<br>procedure<br>(SOP) |
| Global | Onyx | Sponsor | New<br>sponsor<br>protocol<br>SOP |
| Title page | New text added | NCT Number: NCT01999335 | New<br>protocol<br>SOP |
| Title page | Onyx Therapeutics<br>249 East Grand Ave.<br>South San Francisco, CA 94080 | Onyx Therapeutics, Inc. One Amgen Center Drive Thousand Oaks, CA 91320, USA Phone: (805) 447-1000 | Change in<br>sponsor title<br>and contact<br>information |





Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Title page | Study Medical Monitor: MD 249 East Grand Avenue Phone: Email: | Study Medical Monitor: MD Medical Director, Early Development 1120 Veterans Blvd South San Francisco, CA 94080 USA Phone: Email: | Change in responsibilit ies |
| Title page | New text added | Amendment 3.0: 07 March 2018 | New<br>amendment<br>identifiers |
| [Protocol<br>Approval<br>Signature Page] | Protocol Approval Signature Page | [page removed] | New<br>sponsor<br>protocol<br>SOP |
| Protocol<br>Acceptance<br>Page | Issue/Date: OPZ007 (08 July 2014) | Issue/Date: OPZ007 (07 March 2018) | New<br>amendment<br>identifiers |
| Synopsis<br>(Study<br>objectives) | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study (by Schedule) | Part 1: Phase 1b Dose Escalation and Dose Expansion Portions of the Study (by Schedule) | Study is no longer divided into 2 parts |




**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


# Synopsis (Study objectives)

Section 4.2 (Part 2: Randomized Phase 3 Portion of the Study) -Whole Section deleted

Part 2: Randomized Phase 3 Portion of the Study

Phase 3 objectives involve comparison of key outcome measures for subjects with primary refractory or relapsed and refractory multiple myeloma who are randomized to either oprozomib or placebo, in combination with pomalidomide and dexamethasone, hereafter denoted by OPomd or Pomd, respectively.

## Primary Objective

• To compare progression free survival (PFS), as determined by Onyx Response Computational Assessment (ORCA) according to the IMWG-URC. between subjects treated with OPomd and those treated with Pomd

## Secondary Objectives

- To compare the following between subjects treated with OPomd and those treated with Pomd:
  - o Overall survival (OS)
  - o Overall response rate (ORR), the clinical benefit rate (CBR), and duration of response (DOR) as determined by ORCA according to the IMWG-URC and modified EBMT criteria
  - o Incidence of improvement in renal function, as defined by an increase in glomerular filtration rate (GFR) of at least 10 mL/min over baseline at least once after the start of treatment
  - o Incidence of improvement in hemoglobin, as defined by an increase of at least 2 g/dL over baseline at least once after the start of treatment
  - o Safety and tolerability
  - o Bone pain and the impact of bone pain measured with the BPI-SF
  - o Health-related quality of life (HRQoL) measured by the global health status/QoL scale of the EORTC QLQ-C30

Part 2: Randomized Phase 3 Portion of the Study

Phase 3 objectives involve comparison of key outcome measures for subjects with primary refractory or relapsed and refractory multiple myeloma who are randomized to either oprozomib or placebo, in combination with pomalidomide and dexamethasone, hereafter denoted by OPomd or Pomd, respectively.

## Primary Objective

• To compare progression free survival (PFS), as determined by Onyx Response Computational Assessment (ORCA) according to the IMWG-URC, between subjects treated with OPomd and those treated with Pomd

# Secondary Objectives

- To compare the following between subjects treated with OPomd and those treated with Pomd:
  - o Overall survival (OS)
  - o Overall response rate (ORR), the clinical benefit rate (CBR), and duration of response (DOR) as determined by ORCA according to the IMWG-URC and modified EBMT criteria
  - o Incidence of improvement in renal function, as defined by an increase in glomerular filtration rate (GFR) of at least 10 mL/min over baseline at least once after the start of treatment
  - o Incidence of improvement in hemoglobin, as defined by an increase of at least 2 g/dL over baseline at least once after the start of treatment
  - o Safety and tolerability
  - o Bone pain and the impact of bone pain measured with the BPI-SF
  - o Health-related quality of life (HRQoL) measured by the global health status/QoL scale of the EORTC OLO-C30

Removed Phase 3 text to reflect what data was collected for the study



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Page

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | o Disease symptoms as measured by the disease<br>symptoms subscale of EORTC QLQ-MY20 | o Disease symptoms as measured by the disease symptoms subscale of EORTC QLQ-MY20 | |
| | <ul> <li>Neurotoxicity symptoms as measured by the<br/>neurotoxicity subscale of the FACT/GOG-Ntx4<br/>(Version 4)</li> </ul> | <ul> <li>Neurotoxicity symptoms as measured by the<br/>neurotoxicity subscale of the FACT/GOG-Ntx4<br/>(Version 4)</li> </ul> | |
| | o Health status assessed with EQ-5D-5L | o Health status assessed with EQ-5D-5L | |
| | <ul> <li>To evaluate population-based PK parameters of<br/>oprozomib in the OPomd regimen.</li> </ul> | <ul> <li>To evaluate population based PK parameters of<br/>oprozomib in the OPomd regimen.</li> </ul> | |
| | Exploratory Objectives | Exploratory Objectives | |
| | To compare the following between subjects treated with OPomd and those treated with Pomd: | To compare the following between subjects treated with OPomd and those treated with Pomd: | |
| | <ul> <li>PFS and ORR as determined by the investigator<br/>according to the IMWG-URC</li> </ul> | <ul> <li>PFS and ORR as determined by the investigator<br/>according to the IMWG-URC</li> </ul> | |
| | Duration of response (DOR), defined as the time from<br>the first evidence of confirmed PR or better to disease<br>progression or death due to any cause as determined<br>by the investigator according to the IMWG-URC | Duration of response (DOR), defined as the time from<br>the first evidence of confirmed PR or better to disease<br>progression or death due to any cause as determined<br>by the investigator according to the IMWG-URC | |
| | <ul> <li>Clinical benefit rate (CBR) as determined by the<br/>investigator according to the IMWG-URC and<br/>modified EBMT criteria</li> </ul> | Clinical benefit rate (CBR) as determined by the investigator according to the IMWG-URC and modified EBMT-criteria | |
| | Duration of clinical benefit (DOCB), defined as the time from first evidence of MR or better to disease progression or death due to any cause, as determined by ORCA and the investigator according to the IMWG-URC and modified EBMT criteria | Duration of clinical benefit (DOCB), defined as the time from first evidence of MR or better to disease progression or death due to any cause, as determined by ORCA and the investigator according to the IMWG-URC and modified EBMT-criteria | |
| | <ul> <li>Genomic biomarkers that may correlate with<br/>antitumor activity and resistance following treatment<br/>with proteasome inhibitors</li> </ul> | Genomic biomarkers that may correlate with<br>antitumor activity and resistance following treatment<br>with proteasome inhibitors | |
| | <ul> <li>The incidence of neuropathy (events are defined as<br/>Grade 2 or higher peripheral neuropathy)</li> </ul> | The incidence of neuropathy (events are defined as<br>Grade 2 or higher peripheral neuropathy) | |
| | <ul> <li>HRQoL assessed with subscale scores of EORTC<br/>QLQ-C30 (excluding global health status scale) and<br/>EORTC QLQ-MY20 (excluding disease symptom<br/>subscale)</li> </ul> | HRQoL assessed with subscale scores of EORTC QLQ-C30 (excluding global health status scale) and EORTC QLQ-MY20 (excluding disease symptom subscale) | |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Synopsis<br>(Study design) | There are 2 parts to this study. Part 1 includes an open-label, Phase 1b, dose-escalation and dose-expansion portion (equivalent to a small Phase 2), during which the RP3D will be identified. | This study includes an open-label, Phase 1b, dose-escalation and dose-expansion portion (equivalent to a small Phase 2), during which the RP3D will be identified. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Study design) | During the Phase 1b portion of the study, subjects will receive Oprozomib extended release (ER) Tablets according to their assigned dose cohort. | During this study, subjects will receive Oprozomib extended release (ER) Tablets according to their assigned dose cohort. | Study is no longer divided into 2 Parts. |
| Synopsis<br>(Study design) | Part 2 will consist of a placebo-controlled, double-blind, randomized Phase 3 component, where subjects will be randomized to receive the RP3D of oprozomib or placebo administered orally in combination with pomalidomide and dexamethasone in 28-day cycles until disease progression or unacceptable toxicity. | Part 2 will consist of a placebo-controlled, double-blind, randomized Phase 3 component, where subjects will be randomized to receive the RP3D of oprozomib or placebo administered orally in combination with pomalidomide and dexamethasone in 28-day cycles until disease progression or unacceptable toxicity. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Study design)<br>Section 5<br>(Study Design) | This study will include subjects with primary refractory or relapsed and refractory multiple myeloma, i.e., those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy (including bortezomib and lenalidomide and/or thalidomide, and in the dose-expansion and Phase 3 portions of the study only, been treated with adequate alkylator therapy). | This study will include subjects with primary refractory or relapsed and refractory multiple myeloma, i.e., those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy (including bortezomib and lenalidomide and/or thalidomide, and in the dose-expansion and Phase 3 portions of the study only, been treated with adequate alkylator therapy). | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Synopsis<br>(Study design) | All study subjects (i.e., Part 1 and Part 2) will receive oprozomib once daily (or placebo in the case of Phase 3 subjects in the Pomd arm) either on Days 1–5 and 15–19, referred to hereafter as the 5/14 schedule, or an alternate schedule of once daily on Days 1, 2, 8, 9, 15, 16, 22, and 23, referred to hereafter as the 2/7 schedule. | All study subjects (i.e., Part 1 and Part 2) will receive oprozomib once daily (or placebo in the case of Phase 3 subjects in the Pomd arm) either on Days 1–5 and 15–19, referred to hereafter as the 5/14 schedule, or an alternate schedule of once daily on Days 1, 2, 8, 9, 15, 16, 22, and 23, referred to hereafter as the 2/7 schedule. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Study design) | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study | Part 1: Phase 1b Dose Escalation and Dose Expansion Portions of the Study | Study no longer divided into 2 parts. |
| Synopsis<br>(Study design) | In Part 1 of the study, the safety, MTD, PK/PDn, and RP3D of oprozomib when given in combination with pomalidomide and dexamethasone will be assessed using a standard 3+3 dose-escalation design. | The safety, MTD, PK/PDn, and RP3D of oprozomib when given in combination with pomalidomide and dexamethasone will be assessed using a standard 3+3 dose-escalation design. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Study design) | Part 1: Phase 1b Dose Escalation and Dose Expansion Portions of the Study In Part 1 of the study, the safety, MTD, PK/PDn, and RP3D of oprozomib when given in combination with pomalidomide and dexamethasone will be assessed using a standard 3+3 dose-escalation design. For each of the 2 schedules being studied, groups of 3 to 6 subjects will be enrolled into dose-escalation cohorts. As long as fewer than 33% of subjects experience a dose limiting toxicity (DLT) in a given cohort, escalation will continue by 30 mg increments of oprozomib onto the next designated cohort(s). A minimum of 6 subjects must be treated at the MTD to establish the dose as the MTD. If the starting dose of oprozomib cannot be safely administered with the labeled pomalidomide dose, or at sponsor discretion, then up to | Part 1: Phase 1b Dose Escalation and Dose Expansion Portions of the Study In Part 1 of the study, the safety, MTD, PK/PDn, and RP3D of oprozomib when given in combination with pomalidomide and dexamethasone will be assessed using a standard 3+3 dose escalation design. For each of the 2 schedules being studied, groups of 3 to 6 subjects will be enrolled into dose-escalation cohorts. As long as fewer than 33% of subjects experience a dose limiting toxicity (DLT) in a given cohort, escalation will continue by 30 mg increments of oprozomib onto the next designated cohort(s). A minimum of 6 subjects must be treated at the MTD to establish the dose as the MTD. If the starting dose of oprozomib cannot be safely administered with the labeled pomalidomide dose, or at sponsor discretion, then up to 2 | Removed<br>duplicated<br>text |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | 2 possible alternative paths for oprozomib with lower pomalidomide doses will be explored. (See tables below for primary and alternative dose escalation paths.) Dose escalation will continue until sponsor discretion, the maximum planned dose of pomalidomide is reached, or $\geq 2$ DLTs occur in a cohort, whichever occurs first. The prior cohort will be expanded to at least 6 subjects if not previously done to establish that dose as the MTD. There may be more than 1 MTD for oprozomib if more than 1 dose level of pomalidomide is studied. The MTD of oprozomib associated with each dose level of pomalidomide assessed will be the dose level where $\leq 2$ DLTs in 6 subjects are observed. | possible alternative paths for oprozomib with lower pomalidomide doses will be explored. (See tables below for primary and alternative dose escalation paths.) Dose escalation will continue until sponsor discretion, the maximum planned dose of pomalidomide is reached, or ≥ 2 DLTs occur in a cohort, whichever occurs first. The prior cohort will be expanded to at least 6 subjects if not previously done to establish that dose as the MTD. There may be more than 1 MTD for oprozomib if more than 1 dose level of pomalidomide is studied. The MTD of oprozomib associated with each dose level of pomalidomide assessed will be the dose level where < 2 DLTs in 6 subjects are observed. | |
| | There is no planned maximum dose of oprozomib to be studied as it is being added to the FDA approved regimen of pomalidomide/dexamethasone, however, this could be imposed at any time during the course of the study, based on Sponsor discretion. The starting dose of oprozomib for the 5/14 schedule is 150 mg, 3 dose levels below the established 5/14 single agent MTD of 240 mg. The starting dose of oprozomib for the 2/7 schedule is 210 mg, 3 dose levels below the established 2/7 single-agent MTD of 300 mg. Following dose escalation, the sponsor has the option of expanding 1 or both schedules in order to establish the RP3D and schedule. | There is no planned maximum dose of oprozomib to be studied as it is being added to the FDA approved regimen of pomalidomide/dexamethasone, however, this could be imposed at any time during the course of the study, based on Sponsor discretion. The starting dose of oprozomib for the 5/14 schedule is 150 mg, 3 dose levels below the established 5/14 single agent MTD of 240 mg. The starting dose of oprozomib for the 2/7 schedule is 210 mg, 3 dose levels below the established 2/7 single-agent MTD of 300 mg. Following dose escalation, the sponsor has the option of expanding 1 or both schedules in order to establish the RP3D and schedule. | |
| Synopsis<br>(Study design) | During the Phase 1b portion of the study, assessment of DLTs will occur during the 28-day period of Cycle 1 combination therapy. | During this study, assessment of DLTs will occur during the 28-day period of Cycle 1 combination therapy. | Study is no longer divided into 2 parts |
| Synopsis<br>(Study design) | In the Phase 1b portion of the study, subjects must meet the following criteria to be considered evaluable for MTD determination during the 4-week DLT evaluation period unless a DLT occurs before the subject receives all planned doses of oprozomib for both the 5/14 and 2/7 dosing schedules: | Subjects must meet the following criteria to be considered evaluable for MTD determination during the 4-week DLT evaluation period unless a DLT occurs before the subject receives all planned doses of oprozomib for both the 5/14 and 2/7 dosing schedules: | Study no<br>longer<br>divided into<br>2 parts |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Synopsis<br>(Study design) | Once the MTD(s) has been determined and the recommended dose for the expansion phase has been selected, a minimum of 20 additional subjects for 1 or both schedules of oprozomib at the sponsor's discretion will be enrolled in the dose-expansion portion of Part 1 in order to continue the evaluation of the safety and efficacy of the regimen as a prelude to initiation of the Phase 3 portion of the study. | Once the MTD(s) has been determined and the recommended dose for the expansion phase has been selected, a minimum of 20 additional subjects for 1 or both schedules of oprozomib at the sponsor's discretion will be enrolled in the dose-expansion portion of the study in order to continue the evaluation of the safety and efficacy of the regimen. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Study design) | Enrollment to the Phase 3 portion will not commence until the CSRC has evaluated all available safety information from a minimum of 10 subjects who have completed ≥ 2 cycles of therapy and enrollment of the remaining 10 subjects in Dose Expansion has occurred in 1 or both schedules if both were opened. | Enrollment to the Phase 3 portion will not commence until the CSRC has evaluated all available safety information from a minimum of 10 subjects who have completed ≥2 cycles of therapy and enrollment of the remaining 10 subjects in Dose Expansion has occurred in 1 or both schedules if both were opened. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Study design) | Part 2: Randomized Phase 3 Portion of the Study Randomization After screening and eligibility determination, eligible subjects will be randomized in a 2:1 ratio to receive a regimen consisting of OPomd or Pomd plus placebo, respectively. Central randomization will be implemented in this part of the study through the use of an Interactive Voice Response System / Interactive Web Response System (IVRS/IWRS). Eligible subjects will be stratified by: • Age: <75 years versus ≥ 75 years | Part 2: Randomized Phase 3 Portion of the Study Randomization After screening and eligibility determination, eligible subjects will be randomized in a 2:1 ratio to receive a regimen consisting of OPomd or Pomd plus placebo, respectively. Central randomization will be implemented in this part of the study through the use of an Interactive Voice Response System / Interactive Web Response System (IVRS/IWRS). Eligible subjects will be stratified by: | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| | Number of prior therapies: 2 versus 3 or more Carfilzomib status: Carfilzomib-naïve/sensitive versus carfilzomib-refractory. Carfilzomib-sensitive multiple myeloma patients are defined as having had previously achieved a PR or greater with therapy that includes carfilzomib (or carfilzomib monotherapy), and did not experience PD until more than 60 days after their last dose of carfilzomib. Carfilzomib-refractory multiple myeloma is defined as | Number of prior therapies: 2 versus 3 or more Carfilzomib status: Carfilzomib naïve/sensitive versus carfilzomib refractory. Carfilzomib sensitive multiple myeloma patients are defined as having had previously achieved a PR or greater with therapy that includes carfilzomib (or carfilzomib monotherapy), and did not experience PD until more than 60 days after their last dose of carfilzomib. Carfilzomib-refractory multiple myeloma is defined as | |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | disease that is nonresponsive while on primary or<br>salvage therapy that includes carfilzomib, or that<br>progresses on or within 60 days of last therapy. | disease that is nonresponsive while on primary or<br>salvage therapy that includes carfilzomib, or that<br>progresses on or within 60 days of last therapy. | |
| | Within each stratum, treatment assignment will be made using a permuted block randomization scheme. | Within each stratum, treatment assignment will be made using a permuted block randomization scheme. | |
| | Randomized treatment is to commence on the day of randomization (Day 1), if possible, but not more than 5 calendar days after randomization. Treatment initiation beyond 5 days after randomization must be approved by the Onyx study medical monitor or designee. | Randomized treatment is to commence on the day of randomization (Day 1), if possible, but not more than 5-calendar days after randomization. Treatment initiation beyond 5-days after randomization must be approved by the Onyx study medical monitor or designee. | |
| Synopsis<br>(Number of<br>investigational<br>sites)<br>Section 5<br>(Study Design) | Approximately 35 study sites will participate in Part 1 of the study (15 sites for the Phase 1b dose-escalation and 20 additional sites for the dose-expansion portions of the study). An additional 35 sites, for a total of approximately 70 sites, will participate in Part 2 of the study (Phase 3 portion of the study). | Approximately 35 study sites will participate in <b>this</b> study (15 sites for the dose-escalation and 20 additional sites for the dose-expansion portions of the study). | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Planned<br>number of<br>subjects) | Part 1: Phase 1b (Dose-Escalation and Dose-Expansion Portions of the Study) | Part 1: Phase 1b (Dose-Escalation and Dose-Expansion Portions of the Study) | Study is<br>longer<br>divided into<br>2 parts |
| Synopsis<br>(Planned<br>number of<br>subjects) | A total enrollment of approximately 82 subjects is planned for Part 1 of the study. During the Phase 1b Dose-Escalation portion of Part 1, approximately 21 subjects will be enrolled for each schedule. | A total enrollment of approximately 82 subjects is planned for this study. During the Dose-Escalation portion, approximately 21 subjects will be enrolled for each schedule. | Study is no longer divided into 2 parts |
| Synopsis<br>(Planned<br>number of<br>subjects) | A minimum of 20 additional subjects are planned for enrollment for each schedule at the sponsor's discretion and treatment at the RP3D during the Phase 1b Dose-Expansion portion of Part 1 of the study. Part 2: Randomized Phase 3 Portion of the Study | A minimum of 20 additional subjects are planned for enrollment for each schedule at the sponsor's discretion and treatment at the RP3D during the <del>Phase 1b</del> Dose-Expansion portion of <del>Part 1 of</del> the study. Part 2: Randomized Phase 3 Portion of the Study | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected |
| | During Part 2, the planned enrollment is approximately 270 subjects. | During Part 2, the planned enrollment is approximately 270 subjects. | for the<br>study |



Approved

**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | Therefore, the total planned enrollment will be approximately 352 subjects. | Therefore, the total planned enrollment will be approximately 352 subjects. | |
| Synopsis<br>(Sample size<br>justification) | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study | Study is no longer divided into 2 parts |
| Synopsis<br>(Sample size<br>justification) | Part 2: Randomized Phase 3 Portion of the Study For the Phase 3 portion of the study, 157 PFS events are required to detect a 45.7% reduction in the risk of PFS (hazard ratio [HR] = 0.543) with 95% power and a 1-sided significance level of 0.025. Enrollment of 270 subjects (2:1 OPomd versus Pomd, respectively) is consistent with reaching the required 157 events in approximately 14 months, assuming an enrollment rate of approximately 22 subjects per month, a drop-out rate of 5% at 18 months, and a median PFS of 3.8 and 7 months for Pomd and OPomd, respectively. | Part 2: Randomized Phase 3 Portion of the Study For the Phase 3 portion of the study, 157 PFS events are required to detect a 45.7% reduction in the risk of PFS (hazard ratio [HR] = 0.543) with 95% power and a 1-sided significance level of 0.025. Enrollment of 270 subjects (2:1 OPomd versus Pomd, respectively) is consistent with reaching the required 157 events in approximately 14 months, assuming an enrollment rate of approximately 22-subjects per month, a drop-out rate of 5% at 18 months, and a median PFS of 3.8 and 7 months for Pomd and OPomd, respectively. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Study<br>population) | The study population will consist of subjects with primary refractory or relapsed and refractory, multiple myeloma, i.e., those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy (including bortezomib and lenalidomide and/or thalidomide, and in the dose-expansion and Phase 3 portions of the study only, been treated with adequate alkylator), and who are considered to be appropriate for this clinical study by their treating physicians. | The study population will consist of subjects with primary refractory or relapsed and refractory, multiple myeloma, i.e., those who have demonstrated disease progression on or within 60 days of their last therapy, and who have received at least 2 prior lines of therapy (including bortezomib and lenalidomide and/or thalidomide, and in the dose-expansion and Phase 3 portions of the study only, been treated with adequate alkylator), and who are considered to be appropriate for this clinical study by their treating physicians. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Reference<br>therapy dose,<br>and mode of<br>administration) | Placebo Oprozomib placebo tablet for Phase 3 | Placebo Oprozomib placebo tablet for Phase 3 | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



*spproved* 

**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


Onyx TherapeuticsClinical Study Protocol No. OPZ007Oprozomib ER TabletsPage 171 of 223

| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Synopsis<br>(Treatment<br>regimen[s]) | Oral oprozomib or placebo taken Days 1–5 and 15-19 or Days 1, 2, 8, 9, 15, 16, 22, and 23, pomalidomide taken on 21 of 28 days, and oral dexamethasone taken on Days 1, 2, 8, 9, 15, 16, 22, and 23 | Oral oprozomib or placebo-taken Days 1–5 and 15–19 or Days 1, 2, 8, 9, 15, 16, 22, and 23, pomalidomide taken on 21 of 28 days, and oral dexamethasone taken on Days 1, 2, 8, 9, 15, 16, 22, and 23 | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Inclusion<br>criteria)<br>Section 6.1<br>(Inclusion<br>Criteria) | b. In the dose-expansion and Phase 3 portions of the study only: In addition to the above, treatment with adequate alkylator therapy, defined as: | b. In the dose-expansion and Phase 3 portions of the study only: In addition to the above, treatment with adequate alkylator therapy, defined as: | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Exclusion<br>criteria:<br>Disease<br>Related)<br>Section 6.2<br>(Exclusion<br>Criteria) | b. For the Dose-Expansion portion and Part 2 of the study: Prior pomalidomide treatment of any duration | b. For the Dose-Expansion portion-and Part 2 of the study: Prior pomalidomide treatment of any duration | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Criteria for<br>evaluation –<br>Other | In the Phase 1b Dose-Escalation and Dose-Expansion portions of the study, blood samples will be collected from all subjects for determination of plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose) and 1 predose time point on Day 2 of Cycle 1 for both schedules. In the Phase 3 portion of the study, PK samples will be collected from all randomized subjects at Cycle 1 Day 1 and Cycle 3 Day 1 and will be analyzed for oprozomib concentrations in OPomd subjects. | In the Phase 1b-Dose-Escalation and Dose-Expansion portions of the study, blood samples will be collected from all subjects for determination of plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose) and 1 predose time point on Day 2 of Cycle 1 for both schedules. In the Phase 3 portion of the study, PK samples will be collected from all randomized subjects at Cycle 1 Day 1 and Cycle 3 Day 1 and will be analyzed for oprozomib concentrations in OPomd subjects. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Synopsis<br>(Criteria for<br>evaluation –<br>Other) | Blood samples for quantitation of proteasome inhibition by oprozomib will be collected from all subjects in the Phase 1b portion of the study. | Blood samples for quantitation of proteasome inhibition by oprozomib will be collected from all subjects in this study. | Study is no longer divided into 2 parts |
| Synopsis<br>(Criteria for<br>evaluation –<br>Other | Analysis of genomic biomarkers that may predict response and resistance following treatment with proteasome inhibitors will be conducted for all subjects receiving oprozomib from all phases of the study who consent to optional genomic biomarker analysis. | Analysis of genomic biomarkers that may predict response and resistance following treatment with proteasome inhibitors will be conducted for all subjects receiving oprozomib from all phases of the study who consent to optional genomic biomarker analysis. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Synopsis<br>(Criteria for<br>evaluation –<br>Other) | Bone marrow aspirate or biopsy collection does not need to be repeated if previously completed within 45 days prior to Cycle 1 Day 1 dosing, and for Phase 3 only, if it was processed at the central laboratory. Additional bone marrow samples for biomarkers may be collected at disease progression (End of Study Treatment due to progressive disease [PD] or Long-term Follow-up) from all subjects who consent. | Bone marrow aspirate or biopsy collection does not need to be repeated if previously completed within 45 days prior to Cycle 1 Day 1 dosing, and for Phase 3 only, if it was processed at the central laboratory. Additional bone marrow samples for biomarkers may be collected at disease progression (End of Study Treatment due to progressive disease [PD]-or Long term Follow-up) from all subjects who consent. | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |
| Synopsis<br>(Statistical<br>methods and<br>analyses –<br>Safety<br>Population and<br>Efficacy<br>Population) | Safety Population (All Subjects) For Part 1 (Phase 1b Dose Escalation and Expansion) and Part 2 (Randomized Phase 3 Portion) of the study, the safety population includes all subjects receiving any amount of study treatment (oprozomib, placebo, pomalidomide, or dexamethasone). Efficacy Population Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study For the Phase 1b Dose-Escalation and Expansion portions of the study, the efficacy population is equivalent to the safety population. | Safety Population (All Subjects) The safety population includes all subjects receiving any amount of study treatment (oprozomib, pomalidomide, or dexamethasone). Efficacy Population For this study, the efficacy population is equivalent to the safety population. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | Part 2: Randomized Phase 3 Portion of the Study For the Phase 3 portion of the study, the efficacy population will include all randomized subjects according to randomized treatment, consistent with the intent-to-treat (ITT) principle. | | |
| Synopsis<br>(Statistical<br>methods and<br>analyses –<br>Endpoints) | Endpoints Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study (by Schedule) | Endpoints Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study (by Schedule) | Study is no longer divided into 2 parts |
| Synopsis<br>(Statistical<br>methods and<br>analyses –<br>Primary,<br>Secondary, and<br>Exploratory<br>headings) | Primary Endpoints-Part 1 Secondary Endpoints-Part 1 Exploratory Endpoints-Part 1 | Primary Endpoints-Part 1 Secondary Endpoints-Part 1 Exploratory Endpoints-Part 1 | Study is no longer divided into 2 parts |
| Synopsis<br>(Statistical<br>methods and<br>analyses) | Part 2: Randomized Phase 3 Portion of the Study Primary Endpoint-Part 2 • Progression-free survival, defined as time from randomization to the earlier of disease progression | Part 2: Randomized Phase 3 Portion of the Study Primary Endpoint-Part 2 Progression-free survival, defined as time from randomization to the earlier of disease progression | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |




**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


determined by ORCA according to the IMWG-URC, or death due to any cause

## Secondary Endpoints-Part 2

- Overall survival, defined as time from randomization to death due to any cause
- Overall response, defined as the best response of sCR, CR, VGPR, or PR as determined by ORCA according to the IMWG-URC
- Clinical benefit, defined as the best response of MR or better, as determined by ORCA according to the the IMWG-URC and modified EBMT criteria
- Duration of response, defined as the time from the first evidence of confirmed PR or better to disease progression as determined by ORCA according to the IMWG-URC, or death due to any cause
- Improvement in renal function, as defined by an increase in GFR of at least 10 mL/min
- Improvement in hemoglobin, as defined by an increase of at least 2 g/dL
- Adverse events and laboratory abnormalities graded according to NCI-CTCAE, Version 4.03
- Vital signs and clinical laboratory results during and following study drug administration
- Change over time in bone pain and the impact of bone pain measured with the BPI-SF
- Change over time in the global health status/QoL scale of the EORTC QLQ-C30
- Change over time in the disease symptoms subscale of the EORTC OLO-MY20
- Change over time in neurotoxicity symptoms measured by the FACT/GOG-Ntx4 score (Version 4)
- Change over time in health status assessed by EQ-5D-5L

determined by ORCA according to the IMWG-URC, or death due to any cause

### Secondary Endpoints-Part 2

- Overall survival, defined as time from randomization to death due to any cause
- Overall response, defined as the best response of sCR, CR, VGPR, or PR as determined by ORCA according to the IMWG-URC
- Clinical benefit, defined as the best response of MR or better, as determined by ORCA according to the the IMWG-URC and modified EBMT criteria
- Duration of response, defined as the time from the first evidence of confirmed PR or better to disease progression as determined by ORCA according to the IMWG-URC, or death due to any cause
- Improvement in renal function, as defined by an increase in GFR of at least 10 mL/min
- Improvement in hemoglobin, as defined by an increase of at least 2 g/dL
- Adverse events and laboratory abnormalities graded according to NCI-CTCAE, Version 4.03
- · Vital signs and clinical laboratory results during and following study drug administration
- Change over time in bone pain and the impact of bone pain measured with the BPI-SF
- Change over time in the global health status/QoL scale of the EORTC OLO-C30
- Change over time in the disease symptoms subscale of the EORTC OLO-MY20
- Change over time in neurotoxicity symptoms measured by the FACT/GOG-Ntx4 score (Version 4)
- Change over time in health status assessed by EO-5D-5L



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Page

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | Population based PK parameters including, but not limited to, area under the plasma concentration-time curve (AUC) and C <sub>max</sub> , will be determined from OPomd subjects | Population based PK parameters including, but not limited to, area under the plasma concentration time curve (AUC) and C <sub>max</sub> , will be determined from OPomd subjects | |
| | Exploratory Endpoints-Part 2 | Exploratory Endpoints-Part 2 | |
| | <ul> <li>Progression-free survival and overall response as<br/>determined by the investigator according to the<br/>IMWG-URC</li> </ul> | Progression-free survival and overall response as<br>determined by the investigator according to the<br>IMWG-URC | |
| | Duration of response, defined as the time from the first evidence of confirmed PR or better to disease progression as determined by the investigator according to the IMWG-URC or death due to any cause | Duration of response, defined as the time from the first evidence of confirmed PR or better to disease progression as determined by the investigator according to the IMWG-URC or death due to any eause | |
| | <ul> <li>Clinical benefit as determined by the investigator<br/>according to the IMWG-URC and modified EBMT<br/>criteria</li> </ul> | <ul> <li>Clinical benefit as determined by the investigator<br/>according to the IMWG-URC and modified EBMT<br/>eriteria</li> </ul> | |
| | Duration of clinical benefit (DOCB), defined as the time from first evidence of MR or better to disease progression or death due to any cause, as determined by ORCA and the investigator according to the IMWG-URC and modified EBMT criteria | Duration of clinical benefit (DOCB), defined as the time from first evidence of MR or better to disease progression or death due to any cause, as determined by ORCA and the investigator according to the IMWG-URC and modified EBMT-criteria | |
| | <ul> <li>Genomic biomarkers that may be correlated with<br/>antitumor activity and resistance following treatment<br/>with proteasome inhibitors</li> </ul> | <ul> <li>Genomic biomarkers that may be correlated with<br/>antitumor activity and resistance following treatment<br/>with proteasome inhibitors</li> </ul> | |
| | <ul> <li>Neuropathy events (defined as Grade 2 or higher<br/>peripheral neuropathy)</li> </ul> | <ul> <li>Neuropathy events (defined as Grade 2 or higher<br/>peripheral neuropathy)</li> </ul> | |
| | <ul> <li>Change over time in all domains of the EORTC<br/>QLQ-C30 and EORTC</li> </ul> | Change over time in all domains of the EORTC QLQ-C30 and EORTC | |
| | QLQ-MY20 (excluding the global health scale and disease symptoms subscale, respectively) | QLQ-MY20 (excluding the global health scale and disease symptoms subscale, respectively) | |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Synopsis<br>(Statistical | Part 1: Phase 1b Dose-Escalation and Dose-Expansion<br>Portions of the Study | Part 1: Phase 1b Dose Escalation and Dose Expansion Portions of the Study | Removed<br>Phase 3 tex |
| methods and<br>analyses –<br>Efficacy<br>Analyses) | Progression-free survival and duration of response will be listed for all subjects by dose level and schedule. Overall response rate and clinical benefit rate will be estimated for all subjects treated at the RP3D along with the associated 95% exact binomial confidence intervals (CIs). | Progression-free survival and duration of response will be listed for all subjects by dose level and schedule. Overall response rate and clinical benefit rate will be estimated for all subjects treated at the RP3D along with the associated 95% exact binomial confidence intervals (CIs). | to reflect<br>what data<br>was<br>collected<br>for the |
| | Part 2: Randomized Phase 3 Portion of the Study | Part 2: Randomized Phase 3 Portion of the Study | study |
| | The primary analysis of PFS and other efficacy endpoints will be based on the ITT population, defined as all subjects randomized. The primary inferential comparison for PFS between treatment groups will use the log-rank test stratified by the randomization stratification factors. The HR will be estimated using a stratified Cox proportional hazards model. The distribution of PFS, including medians, will be summarized descriptively using the Kaplan-Meier method for each treatment group. Overall survival will be analyzed using the same method as for PFS. Duration of response and DOCB will be summarized for each treatment group by Kaplan-Meier method; however, no formal inferential comparisons will be made for these endpoints, as responders constitute a nonrandom subset of the ITT population. Point estimates and 95% exact binomial CIs will be calculated for the ORR and CBR for each treatment group. Inferential comparison between treatment groups for these endpoints will be made using the Cochran-Mantel Haenszel chi-square test, stratified by the randomization stratification factors. | The primary analysis of PFS and other efficacy endpoints will be based on the ITT population, defined as all subjects randomized. The primary inferential comparison for PFS between treatment groups will use the log-rank test stratified by the randomization stratification factors. The HR will be estimated using a stratified Cox proportional hazards model. The distribution of PFS, including medians, will be summarized descriptively using the Kaplan-Meier method for each treatment group. Overall survival will be analyzed using the same method as for PFS. Duration of response and DOCB will be summarized for each treatment group by Kaplan-Meier method; however, no formal inferential comparisons will be made for these endpoints, as responders constitute a nonrandom subset of the ITT population. Point estimates and 95% exact binomial CIs will be calculated for the ORR and CBR for each treatment group. Inferential comparison between treatment groups for these endpoints will be made using the Cochran-Mantel Haenszel chi-square test, stratified by the randomization stratification factors. | |
| | Inferential testing of the primary efficacy endpoint and selected secondary endpoints (OS, ORR, CBR, improvement in renal function, improvement in hemoglobin, change over time in QLQ-MY20 total scale, and change over time in QLQ-C30 total scale) will be performed against an overall 1-sided significance level of 0.025 in accordance with a closed testing procedure. | Inferential testing of the primary efficacy endpoint and selected secondary endpoints (OS, ORR, CBR, improvement in renal function, improvement in hemoglobin, change over time in QLQ-MY20 total scale, and change over time in QLQ-C30 total scale) will be performed against an overall 1-sided significance level of 0.025 in accordance with a closed testing procedure. | |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Synopsis<br>(Statistical<br>methods and<br>analyses –<br>Safety<br>Analyses) | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study For the Phase 1b portion of the study, safety will be assessed through summaries of DLTs, AEs, changes in laboratory test results, ECGs, vital signs, and oprozomib, pomalidomide, and dexamethasone exposure. All AE data collected will be listed by study site, cohort, subject number, and study day. | For this study, safety will be assessed through summaries of DLTs, AEs, changes in laboratory test results, ECGs, vital signs, and oprozomib, pomalidomide, and dexamethasone exposure. All AE data collected will be listed by study site, cohort, subject number, and study day. | Study is no<br>longer<br>divided into<br>2 parts |
| Synopsis<br>(Statistical<br>methods and<br>analyses –<br>Safety<br>Analyses) | Part 2: Randomized Phase 3 Portion of the Study For the Phase 3 portion of the study, safety data will be summarized according to treatment actually received. Safety analyses will be presented separately for Part 1 and Part 2 of the study and will include all AEs occurring on or after treatment on Cycle 1 Day 1 summarized by system organ class and preferred term using the Medical Dictionary for Regulatory Activities (current version of MedDRA), and NCI-CTCAE (Version 4.03) toxicity grade. In addition, all serious adverse events, including deaths, will be listed separately and summarized. Safety will be assessed through summaries of changes in laboratory results, ECGs, and vital signs. Extent of exposure to the study treatment will be summarized using descriptive statistics. | Part 2: Randomized Phase 3 Portion of the Study For the Phase 3 portion of the study, safety data will be summarized according to treatment actually received. Safety analyses will be presented separately for Part 1 and Part 2 of the study and will include all AEs occurring on or after treatment on Cycle 1 Day 1 summarized by system organ class and preferred term using the Medical Dictionary for Regulatory Activities (current version of MedDRA), and NCI-CTCAE (Version 4.03) toxicity grade. In addition, all serious adverse events, including deaths, will be listed separately and summarized. Safety will be assessed through summaries of changes in laboratory results, ECGs, and vital signs. Extent of exposure to the study treatment will be summarized using descriptive statistics. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 3.1<br>(Introduction) | This is a Phase 1b/Phase 3 clinical trial of the oral proteasome inhibitor, oprozomib, in subjects with primary refractory or relapsed and refractory multiple myeloma. | This is a Phase 1b/Phase 3 clinical trial of the oral proteasome inhibitor, oprozomib, in subjects with primary refractory or relapsed and refractory multiple myeloma. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 3.1<br>(Introduction) | New text added | Amendment 3: 1. Data collection for subjects on active treatment is being pared down due to both the completion of this study's analysis and its abbreviated clinical study report. | Update text<br>to reflect<br>the rationale<br>for<br>Amendment<br>3 |
| Section 3.5.1 (Oprozomib) | This study will assess both schedules in Part 1 of the study, as oprozomib has demonstrated preliminary activity in subjects with hematologic malignancies on both schedules (Kaufman 2013). | This study will assess both schedules in this study, as oprozomib has demonstrated preliminary activity in subjects with hematologic malignancies on both schedules (Kaufman, 2013). | Study is no longer divided into 2 parts |
| Section 4<br>(Study<br>Objectives) | 4.1 PART 1: PHASE 1B DOSE-ESCALATION AND DOSE-EXPANSION PORTIONS OF THE STUDY (BY SCHEDULE) | 4.1 PART 1: PHASE 1B DOSE ESCALATION AND DOSE-EXPANSION PORTIONS OF THE STUDY (BY SCHEDULE) | Study is no longer divided into 2 parts |



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


# Section 4.5 (Part 2: Randomization Phase 3 Portion of the Study)

### 4.5 PART 2: RANDOMIZED PHASE 3 PORTION OF THE STUDY

Phase 3 objectives involve comparison of key outcome measures for subjects with primary refractory or relapsed and refractory multiple myeloma who are randomized to either oprozomib or placebo in combination with pomalidomide and dexamethasone, hereafter denoted by OPomd or Pomd, respectively.

#### PRIMARY OBJECTIVE 4.5.1

To compare progression free survival (PFS), as determined by Onyx Response Computational Assessment (ORCA) according to the IMWG-URC, between subjects treated with OPomd and those treated with Pomd

#### 4.5.2 SECONDARY OBJECTIVES

- To compare the following between subjects treated with OPomd and those treated with Pomd:
  - o Overall survival (OS)
  - Overall response rate (ORR), the clinical benefit rate (CBR), and duration of response (DOR) as determined by ORCA according to the IMWG-URC and modified EBMT criteria
  - o Incidence of improvement in renal function, as defined by an increase in glomerular filtration rate (GFR) of at least 10 mL/min over baseline at least once after the start of treatment
  - o Incidence of improvement in hemoglobin as defined by an increase of at least 2 g/dL over baseline at least once after the start of treatment
  - Safety and tolerability

# PART 2: RANDOMIZED PHASE 3 PORTION OF THE STUDY

Phase 3 objectives involve comparison of key outcome measures for subjects with primary refractory or relapsed and refractory multiple myeloma who are randomized to either oprozomib or placebo in combination with pomalidomide and dexamethasone, hereafter denoted by OPomd or Pomd, respectively.

## 4.5.1 PRIMARY OBJECTIVE

 To compare progression free survival (PFS), as determined by Onyx Response Computational Assessment (ORCA) according to the IMWG-URC, between subjects treated with OPomd and those treated with Pomd

## 4.5.2 SECONDARY OBJECTIVES

- To compare the following between subjects treated with OPomd and those treated with Pomd:
  - Overall survival (OS)
  - Overall response rate (ORR), the clinical benefit rate (CBR), and duration of response (DOR) as determined by ORCA according to the IMWG-URC and modified EBMT criteria
  - o Incidence of improvement in renal function, as defined by an increase in glomerular filtration rate (GFR) of at least 10 mL/min over baseline at least once after the start of treatment
  - o Incidence of improvement in hemoglobin as defined by an increase of at least 2 g/dL over baseline at least once after the start of treatment
  - Safety and tolerability

Removed Phase 3 text to reflect what data was collected for the study



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | <ul> <li>Bone pain and the impact of bone pain measured<br/>with the BPI-SF</li> </ul> | Bone pain and the impact of bone pain measured with the BPI-SF | |
| | <ul> <li>Health-related quality of life (HRQoL)<br/>measured by the global health status/QoL scale<br/>of the EORTC QLQ-C30</li> </ul> | <ul> <li>Health-related quality of life (HRQoL) measured by the global health status/QoL scale of the EORTC QLQ-C30</li> </ul> | |
| | <ul> <li>Disease symptoms as measured by the disease<br/>symptoms subscale of EORTC QLQ-MY20</li> </ul> | <ul> <li>Disease symptoms as measured by the disease<br/>symptoms subscale of EORTC QLQ MY20</li> </ul> | |
| | <ul> <li>Neurotoxicity symptoms as measured by the<br/>neurotoxicity subscale of the FACT/GOG-Ntx4<br/>(Version 4)</li> </ul> | <ul> <li>Neurotoxicity symptoms as measured by the<br/>neurotoxicity subscale of the FACT/GOG-Ntx4<br/>(Version 4)</li> </ul> | |
| | o Health status assessed with EQ-5D-5L | → Health status assessed with EQ-5D-5L | ı |
| | To evaluate population-based PK parameters of oprozomib in the OPomd regimen A SOLUTION OF TRANSPORTED FOR THE PROPERTY OF THE PROPERTY | To evaluate population-based PK parameters of oprozonib in the OPomd regimen | |
| | 4.5.3 EXPLORATORY OBJECTIVES To compare the following between subjects treated with OPomd and those treated with Pomd: | 4.5.3 EXPLORATORY OBJECTIVES To compare the following between subjects treated with OPomd and those treated with Pomd: | |
| | <ul> <li>Progression-free survival (PFS) and ORR as<br/>determined by the investigator according to the<br/>IMWG-URC</li> </ul> | Progression-free survival (PFS) and ORR as<br>determined by the investigator according to the<br>IMWG-URC | |
| | Duration of response (DOR), defined as the time from<br>the first evidence of confirmed PR or better to disease<br>progression or death due to any cause as determined<br>by the investigator according to the IMWG-URC | Duration of response (DOR), defined as the time from<br>the first evidence of confirmed PR or better to disease<br>progression or death due to any cause as determined<br>by the investigator according to the IMWG-URC | |
| | <ul> <li>Clinical benefit rate (CBR) as determined by the<br/>investigator according to the IMWG-URC and<br/>modified EBMT criteria</li> </ul> | <ul> <li>Clinical benefit rate (CBR) as determined by the<br/>investigator according to the IMWG-URC and<br/>modified EBMT criteria</li> </ul> | 1 |
| | Duration of clinical benefit (DOCB), defined as the<br>time from first evidence of MR or better to disease<br>progression or death due to any cause, as determined | Duration of clinical benefit (DOCB), defined as the<br>time from first evidence of MR or better to disease<br>progression or death due to any cause, as determined | |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | by ORCA and the investigator according to the IMWG-URC and the modified EBMT criteria | by ORCA and the investigator according to the<br>IMWG-URC and the modified EBMT criteria | |
| | Genomic biomarkers that may correlate with<br>antitumor activity and resistance following treatment<br>with proteasome inhibitors | Genomic biomarkers that may correlate with<br>antitumor activity and resistance following treatment<br>with proteasome inhibitors | |
| | The incidence of neuropathy (events are defined as<br>Grade 2 or higher peripheral neuropathy) | <ul> <li>The incidence of neuropathy (events are defined as<br/>Grade 2 or higher peripheral neuropathy)</li> </ul> | |
| | HRQoL assessed with subscale scores of EORTC<br>QLQ-C30 (excluding global health status scale) and<br>EORTC QLQ-MY20 (excluding disease symptom<br>subscale) | <ul> <li>HRQoL assessed with subscale scores of EORTC<br/>QLQ-C30 (excluding global health status scale) and<br/>EORTC QLQ MY20 (excluding disease symptom<br/>subscale)</li> </ul> | |
| Section 5<br>(Study Design) | There are 2 parts to this study. Part 1 includes an open-label, Phase 1b, dose-escalation and dose-expansion portion (the equivalent of a small Phase 2) during which the RP3D will be identified. | This study includes an open-label, Phase 1b, dose-escalation and dose-expansion portion (the equivalent of a small Phase 2) during which the RP3D will be identified. | The study is<br>no longer<br>divided into<br>2 parts |
| Section 5<br>(Study Design) | During the Phase 1b portion of the study, subjects will receive Oprozomib ER Tablets according to their assigned dose cohort | During this study, subjects will receive Oprozomib ER<br>Tablets according to their assigned dose cohort | The study is no longer divided into 2 parts |
| Section 5<br>(Study Design) | Part 2 will consist of a placebo-controlled, double-blind, randomized Phase 3 component where subjects will be randomized to receive the RP3D of oprozomib or placebo administered orally in combination with pomalidomide and dexamethasone in 28-day cycles until disease progression or unacceptable toxicity. | Part 2 will consist of a placebo-controlled, double-blind, randomized Phase 3 component where subjects will be randomized to receive the RP3D of oprozomib or placebo administered orally in combination with pomalidomide and dexamethasone in 28-day cycles until disease progression or unacceptable toxicity. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |




| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 5<br>(Study Design) | During Part 2 of the study, subjects will be randomized to oprozomib in combination with pomalidomide and dexamethasone (OPomd) at the RP3D and schedule determined during Part 1 of the study or placebo in combination with pomalidomide and dexamethasone (Pomd). | During Part 2 of the study, subjects will be randomized to oprozomib in combination with pomalidomide and dexamethasone (OPomd) at the RP3D and schedule determined during Part 1 of the study or placebo in combination with pomalidomide and dexamethasone (Pomd). | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 5<br>(Study Design) | Treatment cycles for both parts of the study will last 28 days. | Treatment cycles for both parts of the study will last 28 days. | Redundant<br>text |
| Section 5<br>(Study Design) | Details of the study assessments required for both parts of this study are provided in Appendices A1, A2, B1, B2, C1, and C2. | Details of the study assessments required for this study are provided in Appendices A1, A2, B1, and B2. | Removed reference to Phase 3 part of study. |
| Section 5.1<br>(Dose-<br>escalation and<br>Dose-<br>expansion<br>Portions of the<br>Study) | 5.1 PART 1: PHASE 1B DOSE-ESCALATION AND DOSE-EXPANSION PORTIONS OF THE STUDY | 5.1 PART 1: PHASE 1B-DOSE-ESCALATION AND DOSE-EXPANSION PORTIONS OF THE STUDY | The study is<br>no longer<br>divided into<br>2 parts |
| Section 5.1<br>(Dose-<br>escalation and<br>Dose-<br>expansion<br>Portions of the<br>Study) | In Part 1 of the study, the safety, MTD, PK/PDn, and RP3D of oprozomib when given in combination with pomalidomide and dexamethasone will be assessed using a standard 3 + 3 dose-escalation design. | In <b>this</b> study, the safety, MTD, PK/PDn, and RP3D of oprozomib when given in combination with pomalidomide and dexamethasone will be assessed using a standard 3 + 3 dose-escalation design. | The study is<br>no longer<br>divided into<br>2 parts |

**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets





Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 5.1.1 Dose- escalations Schema for the 5/14 Oprozomi b Dosing Schedule | The primary and alternative pathways for dose escalation of oprozomib and pomalidomide in the Phase 1b portion of the study for the 5/14 schedule are summarized in Table 3 through Table 5; these are examples, and are not inclusive of all possible dose-escalation paths. | The primary and alternative pathways for dose escalation of oprozomib and pomalidomide in the Phase 1b portion of the study-for the 5/14 schedule are summarized in Table 3 through Table 5; these are examples, and are not inclusive of all possible dose-escalation paths. | The study is<br>no longer<br>divided into<br>2 parts |
| Section 5.1.3<br>(Dose-limiting<br>Toxicities) | The decision to escalate to the next higher dose of oprozomib in the Phase 1b portion of the study will be based on an assessment of study drug-related DLTs during Cycle 1 by the CSRC. | The decision to escalate to the next higher dose of oprozomib in this study will be based on an assessment of study drug-related DLTs during Cycle 1 by the CSRC. | The study is<br>no longer<br>divided into<br>2 parts |
| Section 5.1.4<br>(Subject<br>Replacement) | In the Phase 1b portion of the study, subjects must meet the following criteria to be considered evaluable for MTD determination during the 4-week DLT evaluation period unless a DLT occurs before the subject receives all planned doses of oprozomib for both the 5/14 and 2/7 dosing schedules: | Subjects must meet the following criteria to be considered evaluable for MTD determination during the 4-week DLT evaluation period unless a DLT occurs before the subject receives all planned doses of oprozomib for both the 5/14 and 2/7 dosing schedules: | The study is<br>no longer<br>divided into<br>2 parts |
| Section 5.1.5<br>(Dose<br>Expansion) | Once the MTD and the recommended dose for the expansion phase have been determined, a minimum of 20 additional subjects at 1 or both schedules of oprozomib at the sponsor's discretion will be enrolled in the dose-expansion portion of Part 1 in order to continue the evaluation of the safety and efficacy of the regimen as a prelude to initiation of the Phase 3 portion of the study. | Once the MTD and the recommended dose for the expansion phase have been determined, a minimum of 20 additional subjects at 1 or both schedules of oprozomib at the sponsor's discretion will be enrolled in the dose-expansion portion of the study in order to continue the evaluation of the safety and efficacy of the regimen. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 5.2<br>(Part 2:<br>Randomization<br>Phase 3 Portion<br>of the Study) | 5.2 PART 2: RANDOMIZED PHASE 3 PORTION OF THE STUDY Part 2 will consist of a placebo-controlled, double-blind randomized Phase 3 component. Enrollment to the Phase 3 portion will not commence until the CSRC has evaluated all available safety information from a minimum of 10 subjects who have completed ≥ 2 cycles of therapy and enrollment of the remaining 10 subjects in the dose expansion has occurred at 1 or both schedules per the sponsor's discretion. This information will inform the selection of a RP3D and schedule by the sponsor and CSRC. During Part 2, subjects will be randomized in a 2:1 to receive oprozomib or placebo administered orally in combination with pomalidomide and dexamethasone in 28-day cycles until disease progression or unacceptable toxicity. | 5.2 PART 2: RANDOMIZED PHASE 3 PORTION OF THE STUDY Part 2 will consist of a placebo-controlled, double blind randomized Phase 3 component. Enrollment to the Phase 3 portion will not commence until the CSRC has evaluated all available safety information from a minimum of 10 subjects who have completed > 2 cycles of therapy and enrollment of the remaining 10 subjects in the dose expansion has occurred at 1 or both schedules per the sponsor's discretion. This information will inform the selection of a RP3D and schedule by the sponsor and CSRC. During Part 2, subjects will be randomized in a 2:1 to receive oprozomib or placebo administered orally in combination with pomalidomide and dexamethasone in 28-day cycles until disease progression or unacceptable toxicity. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 5.2<br>(Estimated<br>Study Duration<br>and Study<br>Closure) –<br>previously<br>Section 5.3 in<br>Amendment 2 | The total study duration is expected to be approximately 32-33 months. | The total study duration is expected to be approximately 12-13 months. | Changed to<br>reflect<br>removal of<br>Part 2<br>(Phase 3) of<br>the study |
| Section 5.2<br>(Estimated<br>Study Duration<br>and Study<br>Closure) –<br>previously<br>Section 5.3 in<br>Amendment 2 | Approximately 13 additional months will be required to enroll subjects in the Phase 3 portion of the study Assuming an enrollment rate of 22 subjects per month, it is estimated that the final analysis of PFS will occur approximately 17 months after the first subject is enrolled in the Phase 3 portion of the study | Approximately 13 additional months will be required to enroll subjects in the Phase 3 portion of the study Assuming an enrollment rate of 22 subjects per month, it is estimated that the final analysis of PFS will occur approximately 17 months after the first subject is enrolled in the Phase 3 portion of the study | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 5.3 | 5.4.1 RANDOMIZATION | 5.4.1 RANDOMIZATION | |
| (Minimizing<br>Bias) –<br>previously<br>Section 5.4 in<br>Amendment 2 | After screening and eligibility determination, eligible subjects will be randomized in a 2:1 ratio to receive a regimen consisting of OPomd or Pomd plus placebo, respectively. Central randomization will be implemented in this part of the study through the use of an Interactive Voice Response System/Interactive Web Response System (IVRS/IWRS). | After screening and eligibility determination, eligible subjects will be randomized in a 2:1 ratio to receive a regimen consisting of OPomd or Pomd plus placebo, respectively. Central randomization will be implemented in this part of the study through the use of an Interactive Voice Response System/Interactive Web Response System (IVRS/IWRS). | |
| | Eligible subjects will be stratified by: | Eligible subjects will be stratified by: | |
| | • Age: < 75 years old versus ≥ 75 years old | <ul> <li>Age: &lt; 75 years old versus ≥ 75 years old</li> </ul> | |
| | • Number of prior therapies: 2 versus 3 or more | <ul> <li>Number of prior therapies: 2 versus 3 or more</li> </ul> | |
| | Carfilzomib status: Carfilzomib-naïve/sensitive versus carfilzomib-refractory. Carfilzomib-sensitive multiple myeloma patients are defined as having had previously achieved a PR or greater with therapy that includes carfilzomib (or carfilzomib monotherapy), and did not experience PD until more than 60 days after their last dose of carfilzomib. Carfilzomib-refractory multiple myeloma is defined as disease that is nonresponsive while on primary or salvage therapy that includes carfilzomib, or that progresses on or within 60 days of last therapy. Within each stratum, treatment assignment will be made using a permuted block randomization scheme. Treatment will begin on the day of randomization, if possible, but not more than 5 calendar days after randomization according to treatment group assignment. Treatment initiation beyond 5 days after randomization must be approved by the Onyx medical monitor or designee. | Carfilzomib status: Carfilzomib-naïve/sensitive versus carfilzomib-refractory. Carfilzomib-sensitive multiple myeloma patients are defined as having had previously achieved a PR or greater with therapy that includes carfilzomib (or carfilzomib monotherapy), and did not experience PD until more than 60 days after their last dose of carfilzomib. Carfilzomib-refractory multiple myeloma is defined as disease that is nonresponsive while on primary or salvage therapy that includes carfilzomib, or that progresses on or within 60 days of last therapy. Within each stratum, treatment assignment will be made using a permuted block randomization scheme. Treatment will begin on the day of randomization, if possible, but not more than 5 calendar days after randomization according to treatment group assignment. Treatment initiation beyond 5 days after randomization must be approved by the Onyx medical monitor or designee. | |
| Section 5.3.1<br>(Blinding) –<br>previously<br>Section 5.4.2 in<br>Amendment 2 | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study Both the Phase 1b dose-escalation and -expansion portions of Part 1 are open-label. | Both the dose-escalation and dose-expansion portions of <b>this study</b> are open-label. | The study<br>no longer is<br>divided into<br>2 parts |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 5.3.1<br>(Blinding) –<br>previously<br>Section 5.4.2 in<br>Amendment 2 | Part 2: Randomized Phase 3 Portion of the Study The second part of the study is a Phase 3, randomized, double-blind, placebo-controlled, multicenter clinical trial. In accordance with regulatory reporting requirements, Onyx will unblind the identity of the study medication for all unexpected SAEs that are considered by the investigator to be related to the study drug (oprozomib). Unblinding for other reasons except as noted above before final analysis of the primary efficacy endpoint is not permitted. Under no circumstances are subjects who enroll in this study permitted to be rerandomized to this study and enroll for a second course of treatment. The password-protected and/or encrypted electronic randomization list will be kept in a central repository by the sponsor's unblinding statistician. An open key to the code will not be available at the study site, to the sponsor's monitors, project statisticians, or the project team at Onyx. All other individuals directly involved in this study will remain blinded until the final analysis of the primary efficacy endpoint. For Phase 3 only, an independent, external Data Monitoring Committee (DMC) will monitor the conduct of the study and undertake periodic unblinded assessments of safety data to protect the safety of study subjects and ensure integrity of the study. | Part 2: Randomized Phase 3 Portion of the Study The second part of the study is a Phase 3, randomized, double-blind, placebo-controlled, multicenter clinical trial. In accordance with regulatory reporting requirements, Onyx will unblind the identity of the study medication for all unexpected SAEs that are considered by the investigator to be related to the study drug (oprozomib). Unblinding for other reasons except as noted above before final analysis of the primary efficacy endpoint is not permitted. Under no circumstances are subjects who enroll in this study permitted to be rerandomized to this study and enroll for a second course of treatment. The password-protected and/or encrypted electronic randomization list will be kept in a central repository by the sponsor's unblinding statistician. An open key to the code will not be available at the study site, to the sponsor's monitors, project statisticians, or the project team at Onyx. All other individuals directly involved in this study will remain blinded until the final analysis of the primary efficacy endpoint. For Phase 3 only, an independent, external Data Monitoring Committee (DMC) will monitor the conduct of the study and undertake periodic unblinded assessments of safety data to protect the safety of study subjects and ensure integrity of the study. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 9<br>(Study Drug) | New text added | No changes in drug product, dosage, or treatment-<br>regimen occurred in this protocol amendment from the<br>previous version. | Added text<br>to explain<br>no changes<br>to dose in<br>Amendment<br>3 |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 10.1<br>(Oprozomib<br>Treatment<br>Administration) | 10.1 OPROZOMIB AND PLACEBO TREATMENT ADMINISTRATION Oprozomib ER Tablets or placebo (for Phase 3 only) will be administered in single daily doses. | 10.1 OPROZOMIB AND PLACEBO-TREATMENT ADMINISTRATION Oprozomib ER Tablets or placebo (for Phase 3 only) will be administered in single daily doses. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 10.1<br>(Oprozomib<br>Treatment<br>Administration) | In the Phase 1b dose-escalation and dose-expansion portions of the study, subjects who permanently discontinue pomalidomide or oprozomib may continue on study. If both pomalidomide and oprozomib are permanently discontinued, study treatment will be discontinued but the subject will be followed until disease progression. In the Phase 3 portion of the study, subjects who permanently discontinue any or all components of study treatment for reasons other than progressive disease will continue the remaining study treatment, if any, and be followed for disease progression. | In the Phase 1b-dose-escalation and dose-expansion portions of the study, subjects who permanently discontinue pomalidomide or oprozomib may continue on study. If both pomalidomide and oprozomib are permanently discontinued, study treatment will be discontinued but the subject will be followed until disease progression. In the Phase 3 portion of the study, subjects who permanently discontinue any or all components of study treatment for reasons other than progressive disease will continue the remaining study treatment, if any, and be followed for disease progression. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 10.2<br>(Pomalidomide<br>Treatment<br>Administration) | The starting dose of pomalidomide for the Phase 1b portion of the study is 4 mg once daily, orally, on Days 1–21 of repeated 28-day cycles until disease progression. | The starting dose of pomalidomide for this study is 4 mg once daily, orally, on Days 1–21 of repeated 28-day cycles until disease progression. | The study is<br>no longer<br>divided into<br>2 parts |
| Section 10.4<br>(Dose<br>Modification<br>Guidelines) | Monotherapy with dexamethasone is not allowed in the Phase 1b dose-escalation and dose-expansion portions of the study. In the event that oprozomib or pomalidomide is permanently discontinued in Phase 3 only, dexamethasone may be continued. | Monotherapy with dexamethasone is not allowed in the Phase 1b dose-escalation and dose-expansion portions of the study.—In the event that oprozomib or pomalidomide is permanently discontinued in Phase 3 only, dexamethasone may be continued. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 10.4.1<br>(Dose<br>Reductions) | For the Phase 1b study, the initial cohort will start at an oprozomib dose level of 150 mg for the 5/14 schedule and 210 mg for the 2/7 schedule. | For this study, the initial cohort will start at an oprozomib dose level of 150 mg for the 5/14 schedule and 210 mg for the 2/7 schedule. | The study is no longer divided into 2 parts |




**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 10.4.1<br>(Dose<br>Reductions) | Modifications of the dose of oprozomib/placebo will occur in up to three 30-mg decrements down to a minimum dose of 150 mg. | Modifications of the dose of oprozomib/ <del>placebo</del> will occur in up to three 30-mg decrements down to a minimum dose of 150 mg. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 10.4.1<br>(Dose<br>Reductions) | For Parts 1 and 2 of the study, dose reduction levels for pomalidomide are provided in Table 11. | The dose reduction levels for pomalidomide are provided in Table 11. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 10.4.1<br>(Dose<br>Reductions) | In the event oprozomib or pomalidomide is permanently discontinued in Phase 3 only, dexamethasone may be continued. | In the event oprozomib or pomalidomide is permanently discontinued in Phase 3 only, dexamethasone may be continued. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 10.5<br>(Definition of<br>Dose-limiting<br>Toxicity) | During the Phase 1b portion of the study, assessment of DLTs will occur during the 28-day period of Cycle 1 combination therapy. | During this study, assessment of DLTs will occur during the 28-day period of Cycle 1 combination therapy. | The study is no longer divided into 2 parts. |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 11.3<br>(Disease<br>Response<br>Assessments) | The schedule of disease assessments for treated subjects is provided in Appendices A1, A2, B1, B2, C1, and C2. Disease response will be assessed by the investigator. Beginning with Cycle 1, assessments are to be completed at the end of every 4-week cycle for the first 18 months of study treatment, and then at the end of every other cycle (every 8 weeks), beginning with Month 20, for the remainder of study treatment and throughout long-term follow-up. | The schedule of disease assessments for treated subjects is provided in Appendices A1, A2, B1, and B2, C1, and C2. Disease response will be assessed by the investigator. Beginning with Cycle 1, assessments are to be completed at the end of every 4-week cycle for the first 18 months of study treatment, and then at the end of every other cycle (every 8 weeks), beginning with Month 20, for the remainder of study treatment and throughout long-term follow-up. | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |
| Section 11.4.1<br>(Pharmacokinet<br>ic<br>Measurements) | 11.4.1.1 PHASE 1B DOSE ESCALATION AND EXPANSION In the Phase 1b dose-escalation and dose-expansion portions of the study, blood samples will be collected from all subjects from both schedules to measure plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose) and 1 predose time point on Day 2 of Cycle 1. Estimates of oprozomib PK parameters will be determined when possible. 11.4.1.2 Phase 3 In the Phase 3 portion of the study, samples will be collected from all subjects enrolled in the OPomd and the Pomd + placebo treatment arms. The plasma samples will be randomly obtained from each sampling window below on Day 1 of Cycle 1 and Cycle 3. The first postdose sampling window in Cycle 1 and Cycle 3 will be between 1 to 2.5 hours and the second postdose sampling window will be between 2.75 to 5 hours. Plasma samples from the OPomd arm will be analyzed for oprozomib concentrations (note the difference between sample collection and sample analysis). Population PK parameter estimates and variability in these estimates will be determined using a population-based analysis method. | 11.4.1.1 PHASE 1B DOSE ESCALATION AND EXPANSION In the Phase 1b dose-escalation and dose-expansion portions of the study, blood samples will be collected from all subjects from both schedules to measure plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose) and 1 predose time point on Day 2 of Cycle 1. Estimates of oprozomib PK parameters will be determined when possible. 11.4.1.2 Phase 3 In the Phase 3 portion of the study, samples will be collected from all subjects enrolled in the OPomd and the Pomd + placebo treatment arms. The plasma samples will be randomly obtained from each sampling window below on Day 1 of Cycle 1 and Cycle 3. The first postdose sampling window in Cycle 1 and Cycle 3 will be between 1 to 2.5 hours and the second postdose sampling window will be between 2.75 to 5 hours. Plasma samples from the OPomd arm will be analyzed for oprozomib concentrations (note the difference between sample collection and sample analysis). Population PK parameter estimates and variability in these estimates will be determined using a population-based analysis method. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 11.4.2<br>(Pharmacodyna<br>mic<br>Measurements) | In the Phase 1b dose-escalation and dose-expansion portions of the study, blood samples for the quantitation of proteasome inhibition by oprozomib will be collected from all subjects for both schedules at 1 predose time point, up to 2 postdose time points (4 and 6 hours postdose) on Day 1 of Cycle 1 and Cycle 2, and 1 predose timepoint on Day 2 of Cycle 1. These timepoints are also specified in the Laboratory Manual. Blood samples for PDn analyses will not be collected in Phase 3. | In the Phase 1b-dose-escalation and dose-expansion portions of the study, blood samples for the quantitation of proteasome inhibition by oprozomib will be collected from all subjects for both schedules at 1 predose time point, up to 2 postdose time points (4 and 6 hours postdose) on Day 1 of Cycle 1 and Cycle 2, and 1 predose timepoint on Day 2 of Cycle 1. These timepoints are also specified in the Laboratory Manual. Blood samples for PDn analyses will not be collected in Phase 3. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 11.4.3<br>(Genomic<br>Measurements) | Analysis of genomic biomarkers that may predict for response and resistance following treatment with proteasome inhibitors will be conducted for all subjects from all phases of the study who consent to optional genomic biomarker analysis. | Analysis of genomic biomarkers that may predict for response and resistance following treatment with proteasome inhibitors will be conducted for all subjects in the study who consent to optional genomic biomarker analysis. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 11.4.3<br>(Genomic<br>Measurements) | Bone marrow aspirate or biopsy collection does not need to be repeated if previously completed within 45 days prior to Cycle 1 Day 1 dosing, and for Phase 3 only, if it was processed at the central laboratory. Additional bone marrow samples for biomarkers may be collected at disease progression (End of Study Treatment due to PD or Long-Term Follow-Up) from all subjects who consent. | Bone marrow aspirate or biopsy collection does not need to be repeated if previously completed within 45 days prior to Cycle 1 Day 1 dosing, and for Phase 3 only, if it was processed at the central laboratory. Additional bone marrow samples for biomarkers may be collected at disease progression (End of Study Treatment due to PD-or Long-Term Follow-Up) from all subjects who consent. | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |
| Section 11.5<br>(Patient-reported<br>Outcomes<br>Assessments | Beginning with Cycle 1, HRQoL/PRO assessments are to be completed at the beginning of every cycle prior to drug administration through End of Study Treatment/Early Discontinuation visit during the dose-expansion portion of the trial, and at the beginning of every cycle prior to drug administration through End of Study Treatment/Early Discontinuation visit and then every 12 weeks during the long-term follow-up in the Phase 3 portion of the study. | Beginning with Cycle 1, HRQoL/PRO assessments are to be completed at the beginning of every cycle prior to drug administration through End of Study Treatment/Early Discontinuation visit during the dose-expansion portion of the trial, and at the beginning of every cycle prior to drug administration through End of Study Treatment/Early Discontinuation visit and then every 12 weeks during the long-term follow-up in the Phase 3 portion of the study. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |


pproved

**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 12<br>(Study and<br>Study<br>Treatment<br>Discontinuation | New text added | Any subject who withdraws without PD will <b>no longer</b> be followed with long-term assessments every 4 weeks through 18 months on study, and then every 8 weeks thereafter, beginning with Month 20, until progression or initiation of next therapy <b>under Amendment 3</b> . | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |
| Section 12.1<br>(Study<br>Treatment<br>Discontinuation<br>) | For both parts of the study, subjects may withdraw from study treatment at any time. | For this study, subjects may withdraw from study treatment at any time. | Study is no<br>longer<br>divided into<br>2 parts |
| Section 12.1<br>(Study<br>Treatment<br>Discontinuation | Part 1 Phase 1b Dose Escalation and Expansion Only | Part 1 Phase 1b Dose Escalation and Expansion Only | Study is no longer divided into 2 parts |
| Section 12.3<br>(Long-term<br>Follow-up | After completion of the End of Study Treatment visit, subjects will be followed for disease progression, OS, and quality of life (QOL). | After completion of the End of Study Treatment visit, subjects will be followed for disease progression, OS, and quality of life (QOL). | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 12.3<br>(Long-term<br>Follow-up | For subjects who have not progressed at end of study treatment, disease response assessments will be performed every 4 weeks through 18 months on study, and then every 8 weeks thereafter, beginning with Month 20, until progression or initiation of next therapy | For subjects who have not progressed at end of study treatment, disease response assessments will no longer be performed every 4 weeks through 18 months on study, and then every 8 weeks thereafter, beginning with Month 20, until progression or initiation of next therapy under Amendment 3 | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |
| Section 12.3<br>(Long-term<br>Follow-up) | Quality of Life • For Phase 3 only, in long-term follow-up, QOL questionnaires will be collected from subjects (regardless of disease status) every 12 weeks. | Quality of Life • For Phase 3 only, in long-term follow-up, QOL questionnaires will be collected from subjects (regardless of disease status) every 12 weeks. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 12.4<br>(Study<br>Treatment) | The DMC recommends termination of the Phase 3 portion of the study | The DMC recommends termination of the Phase 3 portion of the study | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 13.5<br>(Serious<br>Adverse Event<br>Reporting and<br>Documentation<br>Requirements) | Onyx Drug Safety must be notified of the occurrence of any SAE within 24 hours of the investigator, designee, or site personnel's knowledge of the event. The SAE will be reported by completing and submitting the SAE report form through the EDC system. In the event that the EDC system is not available, paper SAE report forms may be used to report the SAE to Onyx Drug Safety. Please refer to the SAE Reporting Guidelines in the study reference manual. | Amgen Global Patient Safety must be notified of the occurrence of any SAE within 24 hours of the investigator, designee, or site personnel's knowledge of the event. The SAE will be reported by completing and submitting the SAE report form through the EDC system. In the event that the EDC system is not available, paper SAE report forms may be used to report the SAE to Amgen Global Patient Safety. Please refer to the SAE Reporting Guidelines below. | Update<br>safety<br>reporting<br>language<br>with latest<br>template. |
| | Follow-up reports must be submitted in a timely fashion as additional information becomes available. | The primary mechanism for reporting serious adverse events will be the electronic data capture system (EDC) via the Safety Report Form. If the EDC system is unavailable for more than 24 hours, then the site will report the information to Amgen using an electronic Serious Adverse Contingency Report Form (see Appendix N) within 24 hours of the investigator's knowledge of the event. The site will enter the serious adverse event data into the electronic system as soon as it becomes available. | |
| | | After the study is completed at a given site, the EDC system will be taken off line to prevent the entry of new data or changes to existing data. | |
| | | If a site receives a report of a new serious adverse event from a study subject or receives updated data on a previously reported serious adverse event after the EDC has been taken off line, then the site can report this information on a paper Serious Adverse Event Report Form (see Appendix N). | |
| | | If a subject is permanently withdrawn from protocol-<br>required therapies because of a serious adverse event,<br>this information must be submitted to Amgen. | |
| | | New or updated information will be recorded in the originally completed Event CRF. | |
| | | The investigator will submit any updated serious adverse event data to Amgen Global Patient Safety within 24 hours of receipt of the information. | |



Supplemental Clinical Study Report: 20130411


> Onvx Therapeutics Oprozomib ER Tablets


Update

pregnancy

reporting

language

with latest template.

### Section 13.6 (Pregnancy Reporting)

Pregnancy occurring in a female subject, or in a male subject's partner, while enrolled in this clinical trial through 30 days after the subject's last dose of study drug, although not considered an SAE, must be reported to Onyx Drug Safety on a Pregnancy Reporting Form within 24 hours of the investigator, designee, or site personnel learning of the event. If the subject is pregnant, all study treatment must be discontinued immediately and the pregnancy must be reported to the investigator and sponsor within 24 hours.

In the event of a pregnancy in the partner of a male subject, the pregnant partner will be asked to complete an authorization form prior to the collection of any pregnancy data. If such authorization is provided by the partner, the investigator will follow the pregnancy of the male subject's partner until completion or termination of the pregnancy.

Any abnormal maternal, fetal, or neonatal outcomes must be reported to Onyx Drug Safety as a follow-up on the Pregnancy Reporting Form within the same time parameters as stated above for report of a pregnancy. If the outcome of the pregnancy meets an SAE criterion (e.g., spontaneous abortion, stillbirth, neonatal death, or fetal or neonatal congenital anomaly), the investigator will report the SAE through the EDC system.

A fetus exposed to study drug by a parent (female subject or male subject's partner) will be followed until a minimum of 12 weeks after birth. Follow-up may be extended at the discretion of the Onyx study medical monitor. All findings inclusive of SAEs will be reported to Onvx Drug Safety within 24 hours of the investigator, designee, or site personnel learning of the event. Subject to the parents' continuing authorization, SAEs that may occur in these infants will be reported to Onyx Drug Safety.

Pregnancy occurring in a female subject, or in a male subject's partner, while enrolled in this clinical trial through 30 days after the subject's last dose of study drug, although not considered an SAE, must be reported to **Amgen Global** Patient Safety on an Amgen Pregnancy Notification Worksheet (Appendix O) within 24 hours of the investigator, designee, or site personnel learning of the event. If the subject is pregnant, all study treatment must be discontinued immediately and the pregnancy must be reported to the investigator and sponsor within 24 hours. To report a pregnancy to Amgen Global Patient Safety. please refer to the pregnancy reporting guidelines below. **Collection of Pregnancy Information** 

Female Subjects Who Become Pregnant

- Investigator will collect pregnancy information on any female subject who becomes pregnant while taking protocol-required therapies through 30 days after stopping oprozomib.
- Information will be recorded on the Pregnancy Notification Worksheet (Appendix O). The worksheet must be submitted to Amgen Global Patient Safety within 24 hours of learning of a subject's pregnancy. Note: Sites are not required to provide any information on the Pregnancy Notification Worksheet that violates the country or regions local privacy laws.
- After obtaining the female subject's signed authorization for release of pregnancy and infant health information, the investigator will collect pregnancy and infant health information and complete the pregnancy questionnaire for any female subject who becomes pregnant while taking protocol-required therapies through 30 days after stopping oprozomib. This information will be forwarded to Amgen Global Patient Safety. Generally, infant follow-up will be conducted up to 12 months after the birth of the child (if applicable).



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019

| Onyx Therapeutics | Clinical Study Protocol No. OPZ007 |
|----------------------|------------------------------------|
| Oprozomib ER Tablets | |

- Any termination of pregnancy will be reported to Amgen Global Patient Safety, regardless of fetal status (presence or absence of anomalies) or indication for procedure.
- While pregnancy itself is not considered to be an adverse event or serious adverse event, any pregnancy complication or report of a congenital anomaly or developmental delay, fetal death, or suspected adverse reactions in the neonate will be reported as an adverse event or serious adverse event. Note that an elective termination with no information on fetal congenital malformation or maternal complication is generally not considered an adverse event, but still must be reported to Amgen as a pregnancy exposure case.
- If the outcome of the pregnancy meets a criterion for immediate classification as a serious adverse event (eg, female subject experiences a spontaneous abortion, stillbirth, or neonatal death or there is a fetal or neonatal congenital anomaly) the investigator will report the event as a serious adverse
- Any serious adverse event occurring as a result of a post-study pregnancy which is considered reasonably related to the study treatment by the investigator will be reported to Amgen Global Patient Safety as described in Section 13.5. While the investigator is not obligated to actively seek this information in former study subjects, he or she may learn of a serious adverse event through spontaneous reporting.
- Any female subject who becomes pregnant while participating will discontinue study treatment.

Male Subjects With Partners Who Become Pregnant or Were Pregnant at the Time of Enrollment

In the event a male subject fathers a child during treatment, and for an additional 90 days after





**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

| zomib ER Tablets | P |
|---|---|
| | discontinuing protocol-required therapies, the information will be recorded on the Pregnancy Notification Worksheet (Appendix O). The worksheet must be submitted to Amgen Global Patient Safety within 24 hours of the site's awareness of the pregnancy. Note: Sites are not required to provide any information on the Pregnancy Notification Worksheet that violates the country or regions local privacy laws. |
| | <ul> <li>The investigator will attempt to obtain a signed<br/>authorization for release of pregnancy and infant<br/>health information directly from the pregnant<br/>female partner to obtain additional pregnancy<br/>information.</li> </ul> |
| | <ul> <li>After obtaining the female partner's signed<br/>authorization for release of pregnancy and infant<br/>health information, the investigator will collect<br/>pregnancy outcome and infant health information on<br/>the pregnant partner and her baby and complete the<br/>pregnancy questionnaires. This information will be<br/>forwarded to Amgen Global Patient Safety.</li> </ul> |
| | <ul> <li>Generally, infant follow-up will be conducted up to<br/>12 months after the birth of the child (if applicable).</li> </ul> |
| | <ul> <li>Any termination of the pregnancy will be reported to<br/>Amgen Global Patient Safety regardless of fetal<br/>status (presence or absence of anomalies) or<br/>indication for procedure.</li> </ul> |
| | Collection of Lactation Information |
| | <ul> <li>Investigator will collect lactation information on any<br/>female subject who breastfeeds while taking<br/>protocol-required therapies through 30 days after<br/>stopping oprozomib.</li> </ul> |
| | Information will be recorded on the Lactation |


Notification Worksheet (Appendix P) and submitted to Amgen Global Patient Safety within 24 hours of

the investigator's knowledge of event.





**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | Study treatment will be discontinued if female subject breastfeeds during the study as described in exclusion criterion 22. With the female subjects signed authorization for release of mother and infant health information, the investigator will collect mother and infant health information and complete the lactation questionnaire on any female subject who breastfeeds while taking protocol-required therapies through 30 days after discontinuing protocol-required therapies. | |
| Section 14.1<br>(Study<br>Endpoints) | 14.1.1 PART 1: PHASE 1B DOSE ESCALATION AND DOSE EXPANSION PORTIONS OF THE STUDY (BY SCHEDULE) | 14.1.1 PART 1: PHASE 1B DOSE ESCALATION AND DOSE EXPANSION PORTIONS OF THE STUDY (BY SCHEDULE) | The study is no longer divided into 2 parts |
| Section 14.1.1<br>(Primary<br>Endpoints) –<br>previously<br>Section 14.1.1.<br>1 in<br>Amendment 2 | 14.1.1 PRIMARY ENDPOINTS-PART 1 | 14.1.1 PRIMARY ENDPOINTS-PART 1 | The study is<br>longer<br>divided into<br>2 parts |
| Section 14.1.2<br>(Secondary<br>Endpoints) –<br>previously<br>Section 14.1.1.<br>2 in<br>Amendment 2 | 14.1.2 SECONDARY ENDPOINTS-PART 1 | 14.1.2 SECONDARY ENDPOINTS-PART 1 | The study is<br>no longer<br>divided into<br>2 parts |
| Section 14.1.3<br>(Exploratory<br>Endpoints) –<br>previously<br>Section 14.1.1.<br>3 in<br>Amendment 2 | 14.1.3 EXPLORATORY ENDPOINTS-PART 1 | 14.1.3 EXPLORATORY ENDPOINTS-PART 1 | The study is<br>no longer<br>divided into<br>2 parts |





**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


# Section 14.1.2 (Part 2: Randomized Phase 3 Portion of the Study)

### 14.1.2 PART 2: RANDOMIZED PHASE 3 PORTION OF THE STUDY

#### 14.1.2.1 Primary Endpoint-Part 2

 Progression-free survival, defined as time from randomization to the earlier of disease progression determined by ORCA according to the IMWG-URC, or death due to any cause.

#### 14.1.2.2 Secondary Endpoints-Part 2

- Overall survival defined as time from randomization to death due to any cause
- Overall response, defined as the best response of sCR, CR, VGPR, or PR as determined by ORCA according to the IMWG-URC
- Clinical benefit, defined as the best response of MR or better, as determined by ORCA according to the IMWG-URC and modified EBMT criteria
- Duration of response, defined as the time from the first evidence of confirmed PR or better to disease progression, as determined by ORCA according to the IMWG-URC, or death due to any cause
- Improvement in renal function, as defined by an increase in GFR of at least 10 mL/min
- Improvement in hemoglobin, as defined by an increase of at least 2 g/dL
- Adverse events and laboratory abnormalities graded according to NCI-CTCAE, Version 4.03
- Vital signs and clinical laboratory results during and following study drug administration
- Bone pain and the impact of bone pain measured with the BPI-SF
- Change over time in the global health status/QoL scale of the EORTC QLQ-C30
- Change over time in the disease symptoms subscale of the EORTC OLO-MY20

### 14.1.2 PART 2: RANDOMIZED PHASE 3 PORTION OF THE STUDY

### 14.1.2.1 Primary Endpoint-Part 2

• Progression-free survival, defined as time from randomization to the earlier of disease progression determined by ORCA according to the IMWG-URC, or death due to any cause.

#### 14.1.2.2 Secondary Endpoints-Part 2

- Overall survival defined as time from randomization to death due to any cause
- Overall response, defined as the best response of sCR, CR, VGPR, or PR as determined by ORCA according to the IMWG-URC
- Clinical benefit, defined as the best response of MR or better, as determined by ORCA according to the IMWG-URC and modified EBMT criteria
- Duration of response, defined as the time from the first evidence of confirmed PR or better to disease progression, as determined by ORCA according to the IMWG-URC, or death due to any cause
- Improvement in renal function, as defined by an increase in GFR of at least 10 mL/min
- Improvement in hemoglobin, as defined by an increase of at least 2 g/dL
- Adverse events and laboratory abnormalities graded according to NCI-CTCAE, Version 4.03
- · Vital signs and clinical laboratory results during and following study drug administration
- Bone pain and the impact of bone pain measured with the BPI-SF
- Change over time in the global health status/OoL scale of the EORTC OLO-C30
- Change over time in the disease symptoms subscale of the EORTC OLO-MY20

Removed Phase 3 text to reflect what data was collected for the study



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Date: 30 July 2019 Page:

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | Change over time in neurotoxicity symptoms<br>measured by the FACT/GOG-Ntx4 score (Version 4) | Change over time in neurotoxicity symptoms<br>measured by the FACT/GOG-Ntx4 score (Version 4) | |
| | Change over time in health status assessed by<br>EQ-5D-5L | Change over time in health status assessed by<br>EQ-5D-5L | |
| | <ul> <li>Population based PK parameters including, but not<br/>limited to, area under the plasma concentration time<br/>curve (AUC) and C<sub>max</sub>, determined for OPomd<br/>subjects</li> </ul> | Population based PK parameters including, but not<br>limited to, area under the plasma concentration time<br>curve (AUC) and C <sub>max</sub> , determined for OPomd<br>subjects | |
| | 14.1.2.3 Exploratory Endpoints-Part 2 | 14.1.2.3 Exploratory Endpoints-Part 2 | |
| | Progression-free survival and overall response, as<br>determined by the investigator according to the<br>IMWG-URC | Progression-free survival and overall response, as<br>determined by the investigator according to the<br>IMWG-URC | |
| | Duration of response, defined as the time from the<br>first evidence of confirmed PR or better to disease<br>progression as determined by the investigator<br>according to the IMWG-URC or death due to any<br>cause | Duration of response, defined as the time from the first evidence of confirmed PR or better to disease progression as determined by the investigator according to the IMWG-URC or death due to any cause | |
| | <ul> <li>Clinical benefit as determined by the investigator<br/>according to the IMWG-URC and modified EBMT<br/>criteria</li> </ul> | Clinical benefit as determined by the investigator<br>according to the IMWG-URC and modified EBMT<br>criteria | |
| | Duration of clinical benefit (DOCB), defined as the time from first evidence of MR or better to disease progression or death due to any cause, as determined by ORCA and the investigator according to the IMWG-URC and modified EBMT criteria | Duration of clinical benefit (DOCB), defined as the time from first evidence of MR or better to disease progression or death due to any cause, as determined by ORCA and the investigator according to the IMWG-URC and modified EBMT criteria | |
| | <ul> <li>Genomic biomarkers that may be correlated with<br/>antitumor activity and resistance following treatment<br/>with proteasome inhibitors</li> </ul> | Genomic biomarkers that may be correlated with<br>antitumor activity and resistance following treatment<br>with proteasome inhibitors | |
| | <ul> <li>Neuropathy events (defined as Grade 2 or higher<br/>peripheral neuropathy)</li> </ul> | Neuropathy events (defined as Grade 2 or higher<br>peripheral neuropathy) | |
| | <ul> <li>Change over time in all domains of the EORTC<br/>QLQ-C30 and EORTC QLQ-MY20 (excluding the<br/>global health scale and disease symptoms subscale,<br/>respectively)</li> </ul> | Change over time in all domains of the EORTC QLQ C30 and EORTC QLQ MY20 (excluding the global health scale and disease symptoms subscale, respectively) | |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 14.3<br>(Data<br>Monitoring | In Part 1 of the study, safety will be monitored by a CSRC for both the Phase 1b dose-escalation and dose-expansion portions of the study. | In this study, safety will be monitored by a CSRC for both the dose-escalation and dose-expansion portions of the study. | Removed<br>Phase 3 tex<br>to reflect |
| Committee) | In the Phase 3 portion of the study, no formal efficacy interim analyses are planned for the PFS primary endpoint. An interim analysis of OS, the key secondary endpoint, is planned at the time of primary analysis of PFS. Details of the efficacy monitoring plan for OS are described in Section 14.5.2.2. | | what data<br>was<br>collected<br>for the<br>study |
| | Overall survival may be evaluated by the DMC in their ongoing safety review during the course of the study. As the objective of this evaluation is not to declare OS efficacy before the planned efficacy interim and final analyses of OS, alpha level will not be adjusted for these reviews. | | |
| | An independent DMC will be convened for the Phase 3 portion of the study and will act in an advisory capacity to the sponsor with respect to safeguarding the interests of study subjects, assessing interim safety and efficacy (OS | | |
| | secondary only) data, and for monitoring the overall conduct<br>of the study. To enhance the integrity of the study, the DMC<br>may also formulate recommendations relating to the<br>selection, recruitment, and retention of subjects, | | |
| | management of subjects, improving adherence to protocol treatment, and the procedures for data management and quality control. | | |
| | The DMC will meet to review safety data on a periodic basis, but no less frequently than approximately every 6 months. The initial meeting should occur within 3 months after approximately 30 subjects are enrolled in the Phase 3 portion of the study. Unplanned safety review meetings of the DMC may be called at any time by the sponsor or the DMC Chair if additional review of safety data is warranted. | | |
| | The membership criteria and other details of the DMC will be described in the DMC Charter. | | |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section<br>14.5.1.1 (Safety<br>Population) | All subjects receiving any amount of study treatment (oprozomib, placebo, pomalidomide, or dexamethasone) will be included in safety analyses. In the Phase 3 portion of the study, subjects will be included in the treatment group corresponding to the actual treatment received. | All subjects receiving any amount of study treatment (oprozomib, <del>placebo, pomalidomide, or dexamethasone) will be included in safety analyses. In the Phase 3 portion of the study, subjects will be included in the treatment group corresponding to the actual treatment received.</del> | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section<br>14.5.1.2<br>(Efficacy<br>Population) | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study For Part 1 of the study, the efficacy population is equivalent to the safety population. Part 2: Randomized Phase 3 Portion of the Study For the Phase 3 portion of the study, the efficacy population will include all randomized subjects as randomized, i.e., according to the intent to treat (ITT) principle. | For this study, the efficacy population is equivalent to the safety population. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 14.5.2<br>(Efficacy<br>Analyses) | All efficacy analyses will be presented separately for Part 1 and Part 2 of the study. 14.5.2.1 Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study | All efficacy analyses will be presented separately for Part 1 and Part 2 of the study. 14.5.2.1 Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


> Removed Phase 3 text

to reflect

what data

collected

for the

study

was

# Section 14.5.2 (Efficacy Analyses)

14.5.2.2 Part 2: Randomized Phase 3 Portion of the Study Unless otherwise noted, all primary and secondary efficacy analyses will include all randomized subjects analyzed according to the ITT principle (Section 14.5.1), i.e., subjects will be analyzed by the treatment assigned at randomization. Primary Efficacy Analysis

The primary efficacy endpoint for the Phase 3 portion of the study is PFS, defined as the time from randomization to the earlier of disease progression or death due to any cause. Disease progression will be determined using the IMWG-URC (Appendix D). Response and disease progression will be determined using a validated computer algorithm (ORCA) as well as by local investigators. The primary analysis of PFS will be based on ORCA-assessed outcomes. The PFS outcomes assessed by the investigators will serve as a supportive analysis of the primary analysis of

For purposes of calculating PFS, the start date for PD is the date at which progression is first observed. The duration of PFS will be right censored according to the conventions described in Table 18.

Table 18Date of Progression or Censoring for Progression free Survival

14.5.2.2 Part 2: Randomized Phase 3 Portion of the Study Unless otherwise noted, all primary and secondary efficacy analyses will include all randomized subjects analyzed according to the ITT principle (Section 14.5.1), i.e., subjects will be analyzed by the treatment assigned at randomization. Primary Efficacy Analysis

The primary efficacy endpoint for the Phase 3 portion of the study is PFS, defined as the time from randomization to the earlier of disease progression or death due to any cause. Disease progression will be determined using the IMWG-URC (Appendix D). Response and disease progression will be determined using a validated computer algorithm (ORCA) as well as by local investigators. The primary analysis of PFS will be based on ORCA-assessed outcomes. The PFS outcomes assessed by the investigators will serve as a supportive analysis of the primary analysis of

For purposes of calculating PFS, the start date for PD is the date at which progression is first observed. The duration of PFS will be right censored according to the conventions described in Table 18.

Table 18Date of Progression or Censoring for Progression free Survival

| iice Suivivai | | | iicc Suivivai | | |
|---|---|---|---|---|---|
| Situation | Date of Progression or Censoring | Outcome | Situation | Date of Progression or Censoring | Outcome |
| No baseline disease assessments | Date of randomization | Censored | No baseline disease assessments | Date of randomization | Censored |
| No postbaseline<br>disease assessments<br>and alive | Date of<br>randomization + 1<br>day | Censored | No postbaseline disease assessments and alive | Date of randomization + 1 day | Censored |
| New anticancer<br>treatment started<br>before<br>documentation of<br>PD or death | Date of last disease<br>assessment prior to<br>start of a new<br>anticancer treatment | Censored | New anticancer<br>treatment started<br>before<br>documentation of<br>PD or death | Date of last disease<br>assessment prior to<br>start of a new<br>anticancer treatment | Censored |



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


| Death or PD<br>immediately after<br>more than<br>1 consecutively<br>missed disease<br>assessment visit | Date of last disease<br>assessment visit<br>without<br>documentation of<br>PD that is before the<br>first missed visit | Censored | Death or PD<br>immediately after<br>more than 1<br>consecutively<br>missed disease<br>assessment visit | Date of last disease<br>assessment visit<br>without<br>documentation of<br>PD that is before the<br>first missed visit | Censored |
|---|---|---|---|---|---|
| Alive and without PD documentation | Date of last disease assessment | Censored | Alive and without PD documentation | Date of last disease assessment | Censored |
| Death or PD<br>between planned<br>disease assessments | Date of death or<br>first disease<br>assessment showing<br>PD, whichever<br>occurs first | Progressed | Death or PD<br>between planned<br>disease assessments | Date of death or<br>first disease<br>assessment showing<br>PD, whichever<br>occurs first | Progressed |
| Death before first disease assessment | Date of death | Progressed | Death before first<br>disease assessment | Date of death | Progressed |

PD = progressive disease.

The primary analysis of PFS will be conducted when 157 PFS events have occurred.

The primary inferential comparison between treatment groups for PFS will be based on the stratified log-rank test at an overall 0.025 (1-sided) significance level using randomization stratification factors as strata:

- Age: < 75 years versus  $\ge 75$  years
- Number of prior therapies: 2 versus 3 or more
- Carfilzomib status: carfilzomib naïve/sensitive versus carfilzomib-refractory. Carfilzomib-sensitive multiple myeloma patients are defined as having had previously achieved a PR or greater with therapy that includes carfilzomib (or carfilzomib monotherapy), and did not experience PD until more than 60 days after their last dose of carfilzomib. Carfilzomib-refractory multiple myeloma is defined as disease that is nonresponsive while on primary or

PD = progressive disease.

The primary analysis of PFS will be conducted when 157 PFS events have occurred.

The primary inferential comparison between treatment groups for PFS will be based on the stratified log-rank test at an overall 0.025 (1-sided) significance level using randomization stratification factors as strata:

- Age: < 75 years versus ≥ 75 years
- Number of prior therapies: 2 versus 3 or more
- Carfilzomib status: carfilzomib naïve/sensitive versus carfilzomib-refractory. Carfilzomib-sensitive multiple myeloma patients are defined as having had previously achieved a PR or greater with therapy that includes carfilzomib (or carfilzomib monotherapy), and did not experience PD until more than 60 days after their last dose of carfilzomib. Carfilzomib-refractory multiple myeloma is defined as

disease that is nonresponsive while on primary or



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


salvage therapy that includes carfilzomib, or that progresses on or within 60 days of last therapy.

The hazard ratio between the 2 treatment arms will be estimated using a stratified Cox proportional hazards model. The distribution of PFS, including medians, will be summarized descriptively using the Kaplan-Meier method for each treatment group. The 95% CIs for median and other quartiles of PFS will be constructed using the method of Brookmeyer and Crowley (1982). Duration of follow-up for PFS will be estimated by the reverse Kaplan-Meier method of Schemper (1996).

Secondary Efficacy Analyses

Overall survival is defined as the time from randomization to death due to any cause. Subjects who are alive or lost to follow-up as of the data analysis cutoff date will be right censored. The censoring date will be determined from the subject's last known date alive.

Final analysis of OS will be performed when 211 deaths have occurred. Two hundred and eleven (211) deaths will provide 75% power to detect a 32% decrease in the risk of OS for OPomd versus Pomd (HR = 0.68) at the 1-sided 0.025 level of significance. Under exponential distribution, 23.5 months versus 16 months is assumed for median OS for the OPomd and Pomd arms, respectively. The assumed median OS of 16 months for the Pomd group is based on a Phase 2 study of pomalidomide/dexamethasone (Jagannath 2012). Under these assumptions, and assuming 10% lost to follow-up for OS at 60 months, 211 deaths are expected to occur approximately 56 months after the study starts.

The interim analysis for OS will occur at the time of the primary analysis of PFS. The primary analysis of PFS is anticipated to occur approximately 14 months after the first subject is randomized. Approximately 30% of the total number of death events is expected at the time of the primary PFS analysis. The interim and final analysis of OS will be performed using an O'Brien-Fleming group

salvage therapy that includes carfilzomib, or that progresses on or within 60 days of last therapy.

The hazard ratio between the 2 treatment arms will be estimated using a stratified Cox proportional hazards model. The distribution of PFS, including medians, will be summarized descriptively using the Kaplan-Meier method for each treatment group. The 95% CIs for median and other quartiles of PFS will be constructed using the method of Brookmeyer and Crowley (1982). Duration of follow-up for PFS will be estimated by the reverse Kaplan-Meier method of Schemper (1996).

Secondary Efficacy Analyses

Overall survival is defined as the time from randomization to death due to any cause. Subjects who are alive or lost to follow-up as of the data analysis cutoff date will be right censored. The censoring date will be determined from the subject's last known date alive.

Final analysis of OS will be performed when 211 deaths have occurred. Two hundred and eleven (211) deaths will provide 75% power to detect a 32% decrease in the risk of OS for OPomd versus Pomd (HR = 0.68) at the 1-sided 0.025 level of significance. Under exponential distribution, 23.5 months versus 16 months is assumed for median OS for the OPomd and Pomd arms, respectively. The assumed median OS of 16 months for the Pomd group is based on a Phase 2 study of pomalidomide/dexamethasone (Jagannath 2012). Under these assumptions, and assuming 10% lost to follow-up for OS at 60 months, 211 deaths are expected to occur approximately 56 months after the study

The interim analysis for OS will occur at the time of the primary analysis of PFS. The primary analysis of PFS is anticipated to occur approximately 14 months after the first subject is randomized. Approximately 30% of the total number of death events is expected at the time of the primary PFS analysis. The interim and final analysis of OS will be performed using an O'Brien-Fleming group



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


sequential monitoring plan. The monitoring plan will include an upper boundary for benefit constructed using a false-positive error rate of 0.025 (Table 19). The Lan-Demets alpha spending function approach will be used to adjust the O'Brien-Fleming boundary if the actual interim analysis does not correspond to the projected information

Table 19O'Brien-Fleming Monitoring Boundary for Benefit

| ,,,, | | | | | |
|---|---|---|---|---|---|
| Informati<br>on<br>Fraction | Deat<br>h<br>Even<br>ts | Stud<br>y<br>Mont<br>h | Bounda<br>ry<br>(Reject<br>H <sub>o</sub> ) | 1-Sided<br>Significan<br>ce Level | Alph<br>a<br>Spen<br>t |
| 30% | 63 | 14 | 3.929 | 0.000042 | 0.00 |
| 100% | 211 | 56 | 1.96 | 0.025 | 0.02 |

Statistical analyses conducted for OS will be identical to those described for PFS. In addition to the key secondary

endpoint of OS, inferential testing will be conducted for

hemoglobin, change over time in QLQ-MY20 total scale,

ORR, CBR, improvement in renal function, improvement in

and change over time in QLQ-C30 total scale. Inferential testing of primary and selected secondary endpoints will be performed against an overall 1-sided significance level of 0.025 in accordance with a closed testing procedure (CTP). The CTP will be used to account for inflation of the overall type 1 error rate due to hypothesis testing of multiple endpoints.

The CTP will be structured as follows: If the null hypothesis for the primary efficacy endpoint of PFS is rejected at the 1-sided 0.025 level of significance, then testing of the aforementioned secondary endpoints will proceed in a sequential step down manner.

sequential monitoring plan. The monitoring plan will include an upper boundary for benefit constructed using a false-positive error rate of 0.025 (Table 19). The Lan-Demets alpha spending function approach will be used to adjust the O'Brien-Fleming boundary if the actual interim analysis does not correspond to the projected information

Table 19O'Brien-Fleming Monitoring Boundary for Benefit

| Informati<br>on<br>Fraction | Deat<br>h<br>Even<br>ts | Stud<br><del>y</del><br>Mont<br>h | Bounda<br>ry<br>(Reject<br>H <sub>e</sub> ) | 1-Sided<br>Significan<br>ce Level | Alph<br>a<br>Spen<br>t |
|---|---|---|---|---|---|
| 30% | 63 | 14 | 3.929 | 0.000042 | 0.00 |
| 100% | 211 | <del>56</del> | 1.96 | 0.025 | 0.02<br>5 |

Statistical analyses conducted for OS will be identical to those described for PFS. In addition to the key secondary endpoint of OS, inferential testing will be conducted for ORR, CBR, improvement in renal function, improvement in hemoglobin, change over time in OLO-MY20 total scale. and change over time in QLQ-C30 total scale.

Inferential testing of primary and selected secondary endpoints will be performed against an overall 1-sided significance level of 0.025 in accordance with a closed testing procedure (CTP). The CTP will be used to account for inflation of the overall type 1 error rate due to hypothesis testing of multiple endpoints.

The CTP will be structured as follows: If the null hypothesis for the primary efficacy endpoint of PFS is rejected at the 1-sided 0.025 level of significance, then testing of the aforementioned secondary endpoints will proceed in a sequential step down manner.



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


Testing of selected secondary efficacy endpoints will continue, provided the null hypothesis for each previously tested endpoint is rejected. Otherwise, no further testing will be done. The sequential order in which efficacy endpoints will be tested is as follows:

- PFS
- OS
- ORR
- CBR
- Improvement in renal function
- Improvement in hemoglobin
- Change over time in QLQ-C30 global health scale
- Change over time in QLQ-MY20 disease symptoms

Overall response rate will be estimated based on the proportion of subjects in each treatment group who achieve sCR, CR, VGPR, or PR as their best response across the entire treatment duration. The inferential comparison between treatment groups for this endpoint will be made using the Cochran-Mantel Haenszel chi-square test, stratified by the randomization stratification factors. Approximate 95% CIs will be calculated by treatment group for the true ORR. An estimate of the common odds ratio for overall response will be provided as a measure of the relative treatment effect. The odds ratio (and 95% CI) will be estimated using the Mantel-Haenszel method. The Pomd group will serve as the reference treatment group in the calculation of the odds ratio.

Clinical benefit rate will be estimated based on the proportion of subjects in each group who achieve sCR, CR, VGPR, PR, or MR, and will be analyzed in the same manner as described previously for ORR.

Improvement in renal function is defined as an increase in GFR of > 10 mL/min.

Testing of selected secondary efficacy endpoints will continue, provided the null hypothesis for each previously tested endpoint is rejected. Otherwise, no further testing will be done. The sequential order in which efficacy endpoints will be tested is as follows:

- PFS
- OS
- ORR
- CBR
- Improvement in renal function
- Improvement in hemoglobin
- Change over time in QLQ-C30 global health scale
- Change over time in OLO-MY20 disease symptoms

Overall response rate will be estimated based on the proportion of subjects in each treatment group who achieve sCR, CR, VGPR, or PR as their best response across the entire treatment duration. The inferential comparison between treatment groups for this endpoint will be made using the Cochran-Mantel Haenszel chi-square test, stratified by the randomization stratification factors. Approximate 95% CIs will be calculated by treatment group for the true ORR. An estimate of the common odds ratio for overall response will be provided as a measure of the relative treatment effect. The odds ratio (and 95% CI) will be estimated using the Mantel-Haenszel method. The Pomd group will serve as the reference treatment group in the calculation of the odds ratio.

Clinical benefit rate will be estimated based on the proportion of subjects in each group who achieve sCR, CR. VGPR, PR, or MR, and will be analyzed in the same manner as described previously for ORR.

Improvement in renal function is defined as an increase in GFR of > 10 mL/min.



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


Improvement in hemoglobin is defined as an increase of  $\geq 2 \text{ g/dL}$ .

Incidence of improvement in renal function and improvement in hemoglobin will be analyzed in the same manner as described previously for ORR.

Duration of response and DOCB will be summarized for each treatment group by Kaplan-Meier method; however, no formal inferential comparisons will be made for these endpoints, as responders constitute a nonrandom subset of the ITT population.

Quality of life will be assessed by the European Organization for Research and Treatment (EORTC) 30-item QLQ-C30 test and by the 20-item QLQ-MY20 module specifically designed to address the quality of life for those with multiple myeloma (Appendix E). The primary constructed scales from the QLC-C30 are:

- Global Health Status/QoL
- Physical Functioning, Role Functioning
- **Emotional Functioning**
- Cognitive Functioning
- Social Functioning

Nine additional scales can be derived: Fatigue, Nausea and Vomiting, Pain, Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrhea, and Financial Difficulties.

The QLQ-MY20 EORTC questionnaire was developed to assess the quality of life in cancer subjects with multiple myeloma. The QLQ-MY20 includes 20 items assessing disease symptoms, side effects of treatment, body image, and future perspective. There are 3 multi-item scales (Disease Symptoms Scale, Side Effects of Treatment Scale, and Future Perspective Scale) and 1 single-item scale (Body Image).

Scoring procedures are similar for both questionnaires and can be found in the EORTC QLQ-C30 Scoring Manual, Version 3. The analysis and reporting of all QOL data will be performed using the ITT population.

Improvement in hemoglobin is defined as an increase of  $\geq 2 \text{ g/dL}$ .

Incidence of improvement in renal function and improvement in hemoglobin will be analyzed in the same manner as described previously for ORR.

Duration of response and DOCB will be summarized for each treatment group by Kaplan-Meier method; however, no formal inferential comparisons will be made for these endpoints, as responders constitute a nonrandom subset of the ITT population.

Quality of life will be assessed by the European Organization for Research and Treatment (EORTC) 30-item QLQ-C30 test and by the 20-item QLQ-MY20 module specifically designed to address the quality of life for those with multiple myeloma (Appendix E). The primary constructed scales from the OLC-C30 are:

- Global Health Status/OoL
- Physical Functioning, Role Functioning
- Emotional Functioning
- Cognitive Functioning
- Social Functioning

Nine additional scales can be derived: Fatigue, Nausea and Vomiting, Pain, Dyspnoea, Insomnia, Appetite Loss, Constination, Diarrhea, and Financial Difficulties.

The OLO-MY20 EORTC questionnaire was developed to assess the quality of life in cancer subjects with multiple myeloma. The QLQ-MY20 includes 20 items assessing disease symptoms, side effects of treatment, body image. and future perspective. There are 3 multi-item scales (Disease Symptoms Scale, Side Effects of Treatment Scale, and Future Perspective Scale) and 1 single-item scale (Body

Scoring procedures are similar for both questionnaires and can be found in the EORTC OLO-C30 Scoring Manual, Version 3. The analysis and reporting of all QOL data will be performed using the ITT population.



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | Changes over time in QLQ-C30 global health status scores | Changes over time in QLQ-C30 global health status scores | |
| | will be compared between treatment groups using a | will be compared between treatment groups using a | |
| | restricted maximum likelihood-based linear mixed model for | restricted maximum likelihood-based linear mixed model for | |
| | repeated measures data under the missing at random | repeated measures data under the missing at random | |
| | assumption. Formal inferential testing will not be performed | assumption. Formal inferential testing will not be performed | |
| | for the QOL subscales of EORTC QLQ-C30 and | for the QOL subscales of EORTC QLQ-C30 and | |
| | QLQ-MY20 (except for disease symptoms subscale). | QLQ-MY20 (except for disease symptoms subscale). | |
| | Instead, the analysis of these endpoints will be descriptive | Instead, the analysis of these endpoints will be descriptive | |
| | only and considered exploratory. Details of the analyses and | only and considered exploratory. Details of the analyses and | |
| | the impact and handling of missing data in analyses will be | the impact and handling of missing data in analyses will be | |
| | addressed in the SAP. | addressed in the SAP. | |



Supplemental Clinical Study Report: 20130411

Date: 30 July 2019


# Section 14.5.3 (Safety Analysis)

The safety population will be used in all safety analyses (see Section 14.5.1.1). Results of safety analyses will be presented separately for Part 1 and Part 2 of the study. Part 1: Phase 1b Dose-Escalation and Dose-Expansion

Portions of the Study

For the Phase 1b portion of the study, safety data will be summarized for each cohort and for the pooled cohorts. Safety will be assessed through summaries of DLTs, AEs, changes in laboratory test results, ECGs, vital signs, and oprozomib, pomalidomide, and dexamethasone exposure. Part 2: Randomized Phase 3 Portion of the Study

For the Phase 3 portion of the study, safety data will be summarized grouped according to treatment actually received.

Treatment-emergent AEs are defined as AEs that start on or after the first day study treatment is administered and within 30 days of the last administration of study treatment or before start of subsequent anticancer treatment (whichever occurs first). Treatment-emergent AEs will be summarized by the number and percentage of subjects who experienced the event, according to system organ class and preferred term. A subject experiencing multiple instances of the same AE will be counted once within each system organ class and similarly counted once within each preferred term. Adverse event incidence rates may also be calculated based on other measures of subject exposure (e.g., total number of treatment cycles administered). Adverse events will also be summarized by NCI-CTCAE Version 4.03 severity grade and by relationship to each study drug. For AEs not adequately addressed by NCI-CTCAE Version 4.03, the severity grading described in Table 17 may be used. Additional summaries may also be provided for SAEs and events resulting in the permanent discontinuation of therapy. All AEs will be included in individual subject listings. Incidence, severity, and duration of specific signs and symptoms indicative of neuropathy and other neurotoxicities will be assessed. The appropriate terms in these categories

The safety population will be used in all safety analyses (see Section 14.5.1.1).

For this study, safety data will be summarized for each cohort and for the pooled cohorts. Safety will be assessed through summaries of DLTs, AEs, changes in laboratory test results, ECGs, vital signs, and oprozomib, pomalidomide, and dexamethasone exposure.

Removed Phase 3 text to reflect what data was collected for the study



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | will be codified and analyses performed to provide a subject incidence of those with the relevant events. | | |
| | Laboratory parameters will be summarized using descriptive statistics, by postdose shifts in toxicity grades of laboratory parameters relative to baseline, changes from baseline, and data listings of clinically significant abnormalities. The changes in hematology, chemistry, and other laboratory values will be summarized descriptively for each scheduled and unscheduled protocol assessment time point. Changes will be calculated relative to the values collected at baseline and on the first day of each cycle of treatment. The incidence of Grade 3 and 4 hematological toxicities (including neutropenia, thrombocytopenia, and anemia) will be provided by treatment cycle and across all treatment cycles. The use of blood transfusions (platelets, RBC) and/or growth factor support will be summarized. Subject listings of all laboratory data collected during the study will be presented. Laboratory values outside normal limits will be identified in the subject listings. | | |
| | Vital sign results (systolic and diastolic blood pressure, pulse, respiration, and temperature) and ECGs will be summarized descriptively. | | |
| Section 14.5.5<br>(Pharmacokinet | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study | The study is no longer |
| ic Analyses) | In the Phase 1b Dose-Escalation and Dose-Expansion portions of the study, blood samples will be collected from all subjects for determination of plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose) and 1 predose time point on Day 2 of Cycle 1 for both schedules. | In the Phase 1b-Dose-Escalation and Dose-Expansion portions of the study, blood samples will be collected from all subjects for determination of plasma concentrations of oprozomib at 1 predose time point and up to 7 postdose time points on Day 1 of Cycle 1 and Cycle 2 (0.25, 0.5, 1, 2, 3, 4, and 6 hours postdose) and 1 predose time point on Day 2 of Cycle 1 for both schedules. | divided into 2 parts |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Section 14.5.5<br>(Pharmacokinet<br>ic Analyses) | Part 2: Randomized Phase 3 Portion of the Study In Phase 3, population PK of oprozomib will be characterized in the OPomd regimen. The population modeling program will be used to fit a nonlinear mixed effects model to estimate PK parameters including C <sub>max</sub> , AUC, clearance, the inter- and intrasubject variability, and the population variability in the parameter estimates. The sparse sampling concentrations obtained from subjects in this study and results from other oprozomib studies with intensive sampling will be used in the development of a structural model. The best model will be evaluated by goodness-of-fit statistics and reduction in the objective function and posterior predictive checks. Subject characteristics such as age, gender, body weight, body surface area (BSA), and race will be included in the model to identify potential covariates affecting PK of oprozomib. Potential correlations of relevant PK parameters with dose, safety or efficacy outcomes, and other covariates may be explored. | Part 2: Randomized Phase 3 Portion of the Study In Phase 3, population PK of oprozomib will be characterized in the OPomd regimen. The population modeling program will be used to fit a nonlinear mixed effects model to estimate PK parameters including C <sub>max5</sub> AUC, clearance, the inter- and intrasubject variability, and the population variability in the parameter estimates. The sparse sampling concentrations obtained from subjects in this study and results from other oprozomib studies with intensive sampling will be used in the development of a structural model. The best model will be evaluated by goodness- of fit statistics and reduction in the objective function and posterior predictive checks. Subject characteristics such as age, gender, body weight, body surface area (BSA), and race will be included in the model to identify potential covariates affecting PK of oprozomib. Potential correlations of relevant PK parameters with dose, safety or efficacy outcomes, and other covariates may be explored. | Removed<br>Phase 3 text<br>to reflect<br>what data<br>was<br>collected<br>for the<br>study |
| Section 14.7<br>(Determination<br>of Sample Size) | Part 1: Phase 1b Dose-Escalation and Dose-Expansion Portions of the Study A total enrollment of approximately 82 subjects is planned for Part 1 of the study. During the Part 1 Phase 1b dose-escalation portion of the study, approximately 21 subjects are expected to be enrolled for each schedule. | A total enrollment of approximately 82 subjects is planned for this study. During the dose-escalation portion of the study, approximately 21 subjects are expected to be enrolled for each schedule. | The study is<br>no longer<br>divided into<br>2 parts |
| Section 14.7<br>(Determination<br>of Sample Size) | A minimum of 20 additional subjects are planned for enrollment and treatment for 1 or both schedules at the sponsor's discretion at the RP3D during the Phase 1b dose-expansion portion of Part 1 of the study. | A minimum of 20 additional subjects are planned for enrollment and treatment for 1 or both schedules at the sponsor's discretion at the RP3D during the <del>Phase 1b</del> dose-expansion portion of <del>Part 1</del> of the study. | The study is no longer divided into 2 parts |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | | Changed to | | Rationale | |
|---|---|---|---|---|---|---|
| Section 14.7<br>(Determination<br>of Sample Size) | For the Phase 3 portion of the study, 157 PFS events are required to detect a 45.7% reduction in the risk of PFS (HR = 0.543) with 95% power and a 1-sided significance level of 0.025. Enrollment of 270 subjects (2:1 OPomd versus Pomd, respectively) is consistent with reaching the required 157 events in approximately 14 months, assuming an enrollment rate of approximately 22 subjects per month, a 5% drop-out rate at 18 months, and a median PFS of 3.8 and 7 months for Pomd and OPomd, respectively. Therefore, the total planned enrollment will be | | | required to detect a 45.7% (HR = 0.543) with 95% p level of 0.025. Enrollmer versus Pomd, respectively required 157 events in app an enrollment rate of appr | Ethe study, 157 PFS events are breduction in the risk of PFS ower and a 1-sided significance at of 270 subjects (2:1-OPomd e) is consistent with reaching the proximately 14 months, assuming oximately 22 subjects per month, onths, and a median PFS of 3.8 and PFS of 3.8 and enrollment will be | |
| Appendix A1<br>(Schedule of<br>Study | Visit SPEP/UPEP/Serum | Long-term Follow-up | | Visit SPEP/UPEP/Serum | Long-term Follow-up **X | Provide<br>convenience<br>for those on |
| Assessments –<br>Long-term<br>Follow-up | FLC Immunofixation <sup>n</sup> Skeletal Survey <sup>o</sup> | X | | FLC Immunofixation <sup>n</sup> Skeletal Survey <sup>o</sup> | X | study<br>treatment as<br>study has |
| column) | Plasmacytoma<br>Evaluation <sup>p</sup> | X | | Plasmacytoma<br>Evaluation <sup>p</sup> | X | completed |
| Appendix A2 (Schedule of Study Assessments – Long-term Follow-up column) Appendix B1 (Schedule of Study Assessments – Long-term Follow-up column) | Bone Marrow Aspirate<br>and FISH Analyses <sup>q</sup> | X | | Bone Marrow Aspirate<br>and FISH Analyses <sup>q</sup> | ¥ | abbreviated<br>report |



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Study<br>Assessments –<br>Long-term<br>Follow-up<br>column) | | | |
| Appendix A1 (Schedule of Study Assessments – footnote b) Appendix A2 (Schedule of Study Assessments – footnote b) Appendix B1 (Schedule of Study Assessments – footnote b) Appendix B2 (Schedule of Study Assessments – footnote b) Appendix B2 (Schedule of Study Assessments – footnote b) | New text added | All other physical examinations will be limited physical examinations only if clinically indicated. | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |
| Appendix A1<br>(Schedule of<br>Study<br>Assessments –<br>footnote c)<br>Appendix A2<br>(Schedule of<br>Study<br>Assessments –<br>footnote c) | New text added | Neurological assessments (BPNS and if applicable record AEs with CTCAE grading) will be performed at Screening and on Day 1 of every cycle starting from Cycle 2 if clinically indicated and at the End of Study Treatment/Early Discontinuation (See Appendix M). | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Appendix B1<br>(Schedule of<br>Study<br>Assessments –<br>footnote c)<br>Appendix B2<br>(Schedule of<br>Study<br>Assessments –<br>footnote c) | | | |
| Appendix A1 (Schedule of Study Assessments – footnote f) Appendix A2 (Schedule of Study Assessments – footnote f) Appendix B1 (Schedule of Study Assessments – footnote f) Appendix B2 (Schedule of Study Assessments – footnote f) Appendix B2 (Schedule of Study Assessments – footnote f) | For Cycle 2, vital signs are required. For Cycles 3 and higher, vital signs are required | For Cycle 2, <b>if clinically indicated</b> , vital signs are required. For Cycles 3 and higher, <b>if clinically indicated</b> , vital signs are required | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |
| Appendix A1<br>(Schedule of<br>Study<br>Assessments –<br>footnote g) | New text added | Perform ECG approximately within 1 hour before (predose) and approximately 1 hour after (postdose) administration of oprozomib for Cycles 1, 2, 3, 4, 6, 8, 12, 18, 24 and then every 6 months <b>solely if clinically indicated</b> , until progression or unacceptable toxicity. Perform standard ECG | Provide<br>convenience<br>for those on<br>study<br>treatment as |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019 Page 277

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Appendix A2 (Schedule of Study Assessments – footnote g) Appendix B1 (Schedule of Study Assessments – footnote g) Appendix B2 (Schedule of Study Assessments – footnote g) | | assessment at Screening and End of Study Treatment/Early Discontinuation visit. | study has<br>completed<br>its<br>abbreviated<br>report |
| Appendix A1 (Schedule of Study Assessments – footnote i) Appendix A2 (Schedule of Study Assessments – footnote i) Appendix B1 (Schedule of Study Assessments – footnote i) Appendix B2 (Schedule of Study Assessments – footnote i) Appendix B2 (Schedule of Study Assessments – footnote i) | New text added | Full chemistry panel (sodium, potassium, calcium, alkaline phosphatase, blood urea nitrogen, uric acid, lactate dehydrogenase, creatinine, chloride, bicarbonate, glucose, total protein, albumin, total bilirubin, ALT, AST, phosphorous, and magnesium), done locally if clinically indicated. | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Appendix A1 (Schedule of Study Assessments – footnote j) Appendix A2 (Schedule of Study Assessments – footnote j) Appendix B1 (Schedule of Study Assessments – footnote j) Appendix B2 (Schedule of Study Assessments – footnote j Appendix B2 (Schedule of Study Assessments – footnote j) | New text added | Day 1 samples for laboratory analyses can be drawn within 72 hours prior to dosing on Day 1 for all subsequent cycles after Cycle 1 only if clinically indicated. | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |
| Appendix A1 (Schedule of Study Assessments – footnote I) Appendix A2 (Schedule of Study Assessments – footnote I) Appendix B1 (Schedule of Study Assessments – footnote I) | New text added | Coagulation tests, done locally <b>if clinically indicated</b> , and includes the following: Prothrombin time, activated partial thromboplastin time, and international normalized ratio. | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |



Supplemental Clinical Study Report: 20130411
Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets

**Product: Oprozomib** 


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Appendix B2<br>(Schedule of<br>Study<br>Assessments –<br>footnote l) | | | |
| Appendix A1 (Schedule of Study Assessments – footnote o) Appendix A2 (Schedule of Study Assessments – footnote o) Appendix B1 (Schedule of Study Assessments – footnote o) Appendix B2 (Schedule of Study Assessments – footnote o) Appendix B2 (Schedule of Study Assessments – footnote o) | For subjects who did not progress during treatment with bone lesions present at Baseline, skeletal survey will continue to be measured every 4 weeks as clinically indicated (every 28 days ± 4 days) until PD. During long-term follow-up, skeletal survey evaluation should be performed as clinically indicated. | P For subjects who did not progress during treatment with bone lesions present at Baseline, skeletal survey will <b>no longer be required</b> . During long-term follow-up, skeletal survey evaluation <b>will also no longer be required</b> . | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |
| Appendix A1<br>(Schedule of<br>Study<br>Assessments –<br>footnote p)<br>Appendix A2<br>(Schedule of<br>Study<br>Assessments –<br>footnote p) | For subjects with plasmacytoma at Baseline and did not progress during treatment, plasmacytoma will continue to be measured every 4 weeks as clinically indicated (every 28 days ± 4 days) until PD. During long-term follow-up, plasmacytoma evaluation should be performed as clinically indicated. | For subjects with plasmacytoma at Baseline and did not progress during treatment, plasmacytoma will <b>no longer be required</b> . During long-term follow-up, plasmacytoma evaluation will also no longer be required. | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |




Approved

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019 Page 280

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Appendix B1<br>(Schedule of<br>Study<br>Assessments –<br>footnote p)<br>Appendix B2<br>(Schedule of | | | |
| Study Assessments – footnote p) | | | |
| Appendix A1 (Schedule of Study Assessments – footnote q) Appendix A2 (Schedule of Study Assessments – footnote q) Appendix B1 (Schedule of Study Assessments – footnote q) Appendix B2 (Schedule of Study Assessments – footnote q) Appendix B2 (Schedule of Study Assessments – footnote q) | Bone marrow aspirate will also be collected at disease progression (may be collected at End of Study Treatment/Early Discontinuation due to PD or during Long-Term Follow-Up) for subjects who consent to optional genomic biomarker analysis. | Bone marrow aspirate will also be collected at disease progression if clinically indicated (may be collected at End of Study Treatment/Early Discontinuation due to PD; it will no longer be required during Long-term Follow-up) for subjects who consent to optional genomic biomarker analysis. | Provide<br>convenience<br>for those on<br>study<br>treatment as<br>study has<br>completed<br>its<br>abbreviated<br>report |



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets






**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411

Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets






**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| Appendix N (Example Electronic Serious Adverse Event Contingency Report Form) | | APPENDIX N Example Electronic Serious Adverse Event Contingency Report Form Appendix Serious Contingency Report Form | Provide updated adverse event reporting form. |
| | | CONTRACTOR (New York Contractor) (New York Contractor) (New York Contractor) (New York Contractor) (New York Contractor) | |



Supplemental Clinical Study Report: 20130411 Date: 30 July 2019

Onyx Therapeutics Oprozomib ER Tablets


| Section(s) | Changed from | Changed to | Rationale |
|---|---|---|---|
| | | Section 1 Sectio | |
| Appendix O<br>(Example<br>Amgen | | APPENDIX O EXAMPLE AMGEN PREGNA NOTIFICATION WORKSHEET | updated pregnancy |
| Pregnancy<br>Notification<br>Worksheet) | | ** See the American Company of the | reporting<br>worksheet. |
| | | Segment State of the control of the | |
| | | (Refer the Real C. (31) Page of 1 | |



**Product: Oprozomib** 

Supplemental Clinical Study Report: 20130411 Date: 30 July 2019


| Changed to | Rationale |
|---|---|
| APPENDIX P EXAMPLE AMGEN LACTATION NOTIFICATION WORKSHEET ********************************** | Provide<br>updated<br>lactation<br>reporting<br>worksheet. |
| | APPENDIX P EXAMPLE AMGEN LACTATION NOTIFICATION WORKSHEET ACTION WORKSHEET For Companying the continue to continue to management to the continue to |

Approved

